

# **CLINICAL INVESTIGATIONAL PLAN**

Prospe**C**tive, n**O**n-rando**M**ized, **M**ultic**EN**ter **C**linical evaluation of the **E**dwards Pericardial Aortic & Mitral Bioprostheses (Models 11000A & 11000M) with a new tissue treatment platform (COMMENCE #2012-02)

NCT01757665

March 03, 2021



# **Protocol Number 2012-02**

# **CLINICAL INVESTIGATIONAL PLAN Revision J** 03 March 2021

ProspeCtive, nOn-randoMized, MulticENter Clinical evaluation of the Edwards Pericardial Aortic & Mitral Bioprostheses (Models 11000A & 11000M) with a new tissue treatment platform (COMMENCE TRIAL)

# **Trial Sponsor:**

**Edwards Lifesciences LLC** One Edwards Lifesciences Way Irvine, CA 92614 USA

Edwards Lifesciences, the stylized E logo, Carpentier-Edwards, Magna Ease, PERIMOUNT, PERIMOUNT Magna, and ThermaFix are trademarks of Edwards Lifesciences Corporation

CONFIDENTIAL AND PROPRIETATARY DATA: This document and the information contained herein may not be reproduced, used, or disclosed without written permission from Edwards Lifesciences LLC Page 1 of 43

# 1.0 INVESTIGATOR SIGNATURE PAGE

| Trial Title: | Prospe <b>C</b> tive, n <b>O</b> n-rando <b>M</b> ized, <b>M</b> ultic <b>EN</b> ter <b>C</b> linical evaluation of the <b>E</b> dwards Pericardial Aortic & Mitral Bioprostheses(Models 11000A and 11000M) with a new tissue treatment platform (COMMENCE TRIAL) | | |
|---|---|---|---|
| Protocol Number: | | 2012-02 | |
| Version Number: | | Rev. J | |
| Date: | | 03 March 2021 | |
| Model 11000M sponsored be the trial shape of the tr | by Edwards Lifesciences LL<br>al protocol and in accordar<br>nd conditions imposed b<br>s Board. I agree to supervi | the clinical investigation of the C. I agree to conduct this investigation of the C. I agree to conduct this investige with Good Clinical Practice, by the reviewing Institutional I is all sub-investigators at my such and to ensure appropriate al. | atigation according to<br>applicable State and<br>Review Board/Ethics<br>ite as well as the use |
| INVESTIGATOR NAME | | INVESTIGATOR TITLE | |
| INVESTIGATOR SIGNATURE | | DATE | |

REVISION J: 03 MARCH 2021 

#### REV J: 03March2021

# 2.0 TRIAL CONTACT PERSONNEL

# 2.1 SPONSOR CONTACT

| TRIAL DIRECTOR | TRIAL LEAD / MONITORING |
|----------------|-------------------------|

# 2.2 TRIAL CONTACT

| NATIONAL PI | ECHOCARDIOGRAPHY CORE LAB |
|---------------------------|------------------------------|
| CLINICAL EVENTS COMMITTEE | GLYCEROL ASSESSMENT CORE LAB |
| DATA MONITORING COMMITTEE | |

REVISION J: 03 MARCH 2021 

# 3.0 PROTOCOL SYNOPSIS

| Title: | Prospe <b>C</b> tive, n <b>O</b> n-rando <b>M</b> ized, <b>M</b> ultic <b>EN</b> ter <b>C</b> linical evaluation of the <b>E</b> dwards Pericardial Aortic & Mitral Bioprostheses(Models 11000A and 11000M) with a new tissue treatment platform (COMMENCE TRIAL) |
|---|---|
| <b>Protocol Number</b> | 2012-02 |
| | Edwards Lifesciences |
| | One Edwards Way |
| Trial Sponsor: | Irvine, CA 92614 |

| Edwards Pericardial Aortic Bioprosthesis, Model 11000A |
|---|
| Edwards Pericardial Mitral Bioprosthesis, Model 11000M |
| The Edwards Pericardial Aortic Bioprosthesis, Model 11000A, is indicated for |
| patients who require replacement of their native or prosthetic aortic valve. |
| The Edwards Pericardial Mitral Bioprosthesis, Model 11000M, is indicated for |
| patients who require replacement of their native or prosthetic mitral valve. |
| The objective of this trial is to confirm that the modifications to tissu |
| processing, valve sterilization, and packaging of the FDA-approve |
| (P860057/S042) Carpentier-Edwards PERIMOUNT Magna Ease Pericardial Aorti |
| Bioprosthesis, Model 3300TFX, which will be designated as the Edward |
| Pericardial Aortic Bioprosthesis Model 11000A, and the Carpentier-Edwards |
| PERIMOUNT Magna Mitral Ease Pericardial Bioprosthesis, Model 7300TF |
| which will be designated as the Edwards Pericardial Mitral Bioprosthesis Model |
| 11000M do not raise any new questions of safety and effectiveness in subjects |
| who require replacement of their native or prosthetic aortic or mitral valve. Th |
| only differences between the Model 3300TFX and the Model 11000A an |
| between the Model 7300TFX and the Model 11000M are modifications in tissu |
| processing, valve sterilization, and packaging. |
| Multicenter, prospective, double arm trial – Up to seven hundred (700) aorti |
| valve replacement (AVR) subjects and up to one hundred seventy five (175 |
| mitral valve replacement (MVR) subjects at up to forty (40) clinical sites will b |
| enrolled. An enrollment rate of three (3) to four (4) subjects per site per mont |

is anticipated. At least eight (8) centers will implant and follow for at least 1 year,

REVISION J: 03 MARCH 2021 

PROTOCOL NUMBER: 2012-02

thirty (30) or more AVR or thirty (30) or more AVR/MVR subjects. Analysis for the aortic arm will be performed when at least three hundred (300) AVR subjects have completed the POD 390 follow-up visit and at least eight hundred (800) AVR patient-years of cumulative follow-up have been reached. Analysis for the mitral arm will be completed when at least three hundred (300) combined aortic and mitral subjects have completed the POD 390 follow-up visit and at least eight hundred (800) AVR and at least one hundred (100) MVR patient-years of cumulative follow-up have been reached. The tests for the trial endpoints were performed and the trial data was submitted to FDA for the PMA approval of the devices evaluated under the aortic and mitral arms. All IDE Subjects (aortic and mitral arms) who are currently enrolled and alive will be followed to 5 years. In an effort to obtain sufficient long-term data, approximately 250 Subjects implanted with the Model 11000A valve at up to 10 sites will be asked to consent for extended follow-up annually through 10 years post-procedure. In addition, approximately 25 Subjects implanted with the Model 11000M valve at select sites will be asked to consent for extended follow-up annually through 10 years post procedure.

#### **Trial Sites:**

Participating sites are chosen based on their experience in conducting clinical trials, their surgical experience implanting bioprosthetic valves, as well as their ability to maintain robust subject enrollment and follow-up. The investigational sites will be selected throughout the United States, Canada, Europe and Asia Pacific.

#### **Trial Duration:**

Total enrollment period for this trial is estimated to be 1095 days or 3 years. Subject duration in the trial is estimated to be no longer than 1825 days (5 years) or 3650 days (10 years) for those who have consented to continued follow-up. Overall duration of the trial is estimated to be 3833 days or 10.5 years, and will involve at least 800 AVR patient-years and at least 100 MVR patient-years of cumulative follow-up. The trial begins with the enrollment of the first subject and ends after the last subject is exited from the trial after completing the last follow-up visit at approximately postoperative day (POD) 3650, all subjects are fully monitored, all outstanding data queries are resolved and all trial sites are closed to follow-up.

| Visit | Visit Window (Days) | Timing from Implant (Day 0) |
|--------------------|---------------------|-----------------------------|
| Screening/Baseline | | Day -60 to Day 0 |

| | Discharge <sup>1</sup> | | Prior to Discharge |
|-----------------|------------------------|----------|--------------------|
| | POD 30 | -5/+10 | Day 25 to 40 |
| | POD 105 | - 15/+30 | Day 90 to 135 |
| | POD 390 (1 yr) | -25/+45 | Day 365 to 435 |
| | POD 730 (2 yr) | -25/+45 | Day 705 to 775 |
| Trial Follow-Up | POD 1095 (3 yr) | -25/+45 | Day 1070 to 1140 |
| Visits: | POD 1460 (4 yr) | -25/+45 | Day 1435 to 1505 |
| | POD 1825 (5 yr) | -25/+45 | Day 1800 to 1870 |
| | POD 2190 (6 yr)* | -55/+75 | Day 2135 to 2265 |
| | POD 2555 (7 yr)* | -55/+75 | Day 2500 to 2630 |
| | POD 2920 (8 yr)* | -55/+75 | Day 2865 to 2995 |
| | POD 3285 (9 yr)* | -55/+75 | Day 3230 to 3360 |
| | POD 3650 (10yr)* | -55/+75 | Day 3595 to 3725 |
| | 1 - 1 - 1 - 1 - 1 | | |

<sup>&</sup>lt;sup>1</sup> Subjects who are not discharged within 10 days post procedure must have an echocardiogram to assess performance of the trial valve. Those subjects will not require an additional echocardiogram at discharge.

# **Trial Endpoints:**

# Primary Safety Endpoint (up to 390 days post-implant):

The primary safety endpoint for the trial is the rate of implanted subjects that experience structural deterioration of the trial valve by the time of the POD 390 follow-up visit. The null hypothesis is that the rate of structural valve deterioration at one year is greater than 1%. The alternative hypothesis is that this rate is less than 1%.

## Primary Safety Endpoint (Continued follow-up):

For continued follow-up of Subjects, the primary safety endpoint for the trial is the rate of implanted subjects that experience structural deterioration of the trial valve as determined by a Clinical Events Committee (CEC).

### Secondary Safety Endpoints (Pre-approval):

Safety is established by comparing the occurrence of specific safety endpoints to the objective performance criteria (OPC) reported in Table R.1 in ISO 5840:2009, Annex R.1 as recommended by the FDA in the Draft Guidance involving Heart Valves – Investigational Device Exemption (IDE) and Premarket Approval (PMA) Applications (2010).

# Secondary Safety Endpoints (Continued follow-up):

REVISION J: 03 MARCH 2021 

<sup>\*</sup>Subjects who have consented to continued follow up with the Model 11000A or Model 11000M valve.

For continued follow-up of Subjects, linearized rates will be used to summarize the following safety endpoints for the late (>30 days) post-operative period.

- Thromboembolism
- Valve thrombosis
- All bleeding/hemorrhage
- Major bleeding/hemorrhage
- All paravalvular leak
- Major paravalvular leak
- Non-structural valve deterioration

- Endocarditis
- All-cause mortality
- Trial valve-related mortality
- Trial valve-related reoperation
- Explant
- Hemolysis

# **Effectiveness Endpoints:**

- Clinically acceptable hemodynamic performance confirmed by core lab evaluation of echocardiography
- New York Heart Association (NYHA) functional class compared to baseline
- Change in Quality of Life questionnaire Short Form 12 version 2 (SF-12v2)
   from baseline/screening to POD 390

# Additional Data in support of analysis:

Blood Data

# **Subject Enrollment:**

#### Inclusion Criteria:

# Each subject is required to meet all of the following inclusion criteria:

- 1. Is 18 years or older
- 2. Provides written informed consent prior to trial procedures
- 3. Agrees to attend all follow-up assessments for up to 5 years and is willing to comply with specified follow-up evaluations at clinical investigational sites that are participating in the COMMENCE trial and/or obtain the protocol-specified diagnostic tests at centers that are under the same IRB or the same healthcare system
- **4.** Diagnosed with aortic or mitral valve disease requiring valve replacement based on pre- operative evaluation
- **5**. Scheduled to undergo planned aortic or mitral valve replacement with or without concomitant bypass surgery
- **6.** Scheduled to undergo planned aortic valve replacement with or without resection and replacement of the ascending aorta from the sinotubular junction and without the need for circulatory arrest for hemi arch or arch replacement

REVISION J: 03 MARCH 2021 

#### Exclusion criteria: A subject meeting any of the following criteria shall be excluded:

- 1. Requires emergency surgery
- 2. Requires planned multiple valve replacement/ repair (with the exception of mitral valve replacement with tricuspid valve repair)
- **3.** Has prior valve surgery, which included implant of a bioprosthetic valve, mechanical valve, or annuloplasty ring that will remain *in situ*
- **4.** Requires a surgical procedure outside of the cardiac area (e.g. vascular bypass)
- 5. Requires surgical replacement of the aortic root
- **6.** Has active endocarditis/myocarditis or endocarditis/myocarditis within 3 months to the scheduled aortic or mitral valve replacement surgery
- 7. Has renal insufficiency as determined by creatinine (S-Cr) level ≥ 2.5 mg/dL or end-stage renal disease requiring chronic dialysis at screening visit
- **8.** Has MRI or CT scan confirmed stroke, cerebrovascular accident (CVA) or transient ischemic attack (TIA) within 6 months (180 days) prior to planned valve surgery
- **9.** Has acute myocardial infarction (MI) within 30 days prior to planned valve surgery
- Has presence of non-cardiac disease limiting life expectancy to less than 12 months
- 11. Diagnosed with hypertrophic obstructive cardiomyopathy (HOCM)
- 12. Diagnosed with abnormal calcium metabolism and hyperparathyroidism
- **13.** Exhibits left ventricular ejection fraction ≤ 20% as validated by diagnostic procedure prior to planned valve surgery
- **14.** Echocardiographic evidence of an intra-cardiac mass, thrombus, or vegetation
- **15.** Hemodynamic or respiratory instability requiring inotropic support, mechanical circulatory support, or mechanical ventilation within 30 days prior to planned valve surgery
- 16. Documented leukopenia (WBC <  $3.5 \times 10^3/\mu$ L), acute anemia (Hgb < 10.0 gm/dL or 6 mmol/L), or thrombocytopenia (platelet count <  $50 \times 10^3/\mu$ L) accompanied by history of bleeding diathesis or coagulopathy
- 17. Has prior organ transplant or is currently an organ transplant candidate
- **18.** Current or recent participation (within 6 weeks prior to surgery) in another drug or device trial
- 19. Was previously implanted with trial device (Model 11000A or Model 11000M)<sup>1</sup>
- **20.** Pregnant (female subject of childbearing potential only), lactating or planning to become pregnant during the duration of participation in trial
- 21. Currently incarcerated or unable to give voluntary informed consent
- **22.** Documented history of substance (drug or alcohol) abuse within the last 5 years prior to implant
- 23. Requires concomitant left ventricular assist device (LVAD) placement

REVISION J: 03 MARCH 2021


# 4.0 ABBREVIATIONS

| 400 | | 100 | |
|---|---|---|---|
| ACC | American College of Cardiology | IRB | Institutional Review Board |
| AE | Adverse Event | ISO | International Standardization Organization |
| AHA | American Heart Association | LVOT | Left Ventricular Outflow Tract |
| AS | Aortic Stenosis | MI | Myocardial Infarction |
| ASD | Atrial Septal Defect | MOF | Multi-system Organ Failure |
| AVR | Aortic Valve Replacement | MR | Magnetic Resonance |
| CABG | Coronary Artery Bypass Graft | MVR | Mitral Valve Replacement |
| CBC | Complete Blood Count | NSVD | Nonstructural Valve Dysfunction |
| CEC | Clinical Events Committee | NYHA | New York Heart Association |
| CFR | Code of Federal Regulations | OPC | Objective Performance Criteria |
| CO/CI | Cardiac Output/Cardiac Index | OUS | Outside United States |
| CRF | Case Report Form | PFO | Patent Foramen Ovale |
| CV | Critical Value | PMA | Premarket Approval |
| CVA | Cerebrovascular Accident | PO | Postoperative |
| DIC | Disseminated Intravascular Coagulation | POD | Postoperative Day |
| DMC | Data Monitoring Committee | PT | Prothrombin Time |
| EC | Ethics Committee | PTFE | Polytetrafluoroethylene |
| eCRF | Electronic Case Report Form | PTT | Partial Thromboplastin Time |
| ECG | Electrocardiogram | PVL | Paravalvular Leak |
| EDC | Electronic Data Capture | QOL | Quality of Life |
| EOA | Effective Orifice Area | RBC | Red Blood Cell |
| FDA | Food and Drug Administration | REB | Research Ethics Board |
| <b>FMEA</b> | Failure Modes and Effects Analysis | RGA | Returned Good Authorization |
| GCP | Good Clinical Practice | SAE | Serious Adverse Effect |
| GLP | Good Laboratory Practices | SAR | Specific Absorption Rate |
| HGB | Hemoglobin | SAVR | Surgical Aortic Valve Replacement |
| HIPAA | Health Insurance Portability & Accountability Act | SMVR | Surgical Mitral Valve Replacement |
| HCT | Hematocrit | SF-12 | Short Form 12 Health Survey |
| HIT | Heparin Induced Thrombocytopenia | SVD | Structural Valve Deterioration |
| HOCM | Hypertrophic Obstructive Cardiomyopathy | TAD | Tissue Annulus Diameter |
| ICF | Informed Consent Form | TEE | Transesophageal Echocardiography |
| ICU | Intensive Care Unit | TIA | Transient Ischemic Attack |
| ID | Identification | TTE | Transthoracic Echocardiography |
| IDE | Investigational Device Exemption | UADE | Unanticipated Adverse Device Effect |
| IE | Infective Endocarditis | WBC | White Blood Cell |
| IFU | Instructions for Use | | |
| INR | International Normalized Ratio | | |

REVISION J: 03 MARCH 2021 

# **Table of Contents**

| Section | n | | Page |
|---------|-----|-----------------------------------|------|
| 1.0 | INV | ESTIGATOR SIGNATURE PAGE | 2 |
| 2.0 | TRI | AL CONTACT PERSONNEL | 3 |
| | 2.1 | SPONSOR CONTACT | 3 |
| | 2.2 | TRIAL CONTACT | 3 |
| 3.0 | PRO | OTOCOL SYNOPSIS | 4 |
| 4.0 | ABE | BREVIATIONS | 9 |
| 5.0 | TRI | AL OVERVIEW | 13 |
| | 5.1 | INTRODUCTION AND BACKGROUND | 13 |
| | 5.2 | DEVICE DESCRIPTION | 14 |
| | 5.3 | REPORT OF PRIOR INVESTIGATIONS | 16 |
| 6.0 | BEN | NEFITS AND RISKS | 17 |
| | 6.1 | BENEFITS | 17 |
| | 6.2 | RISKS | 18 |
| | 6.3 | MINIMIZING SUBJECT RISK | 19 |
| 7.0 | TRI | AL DESIGN | 19 |
| | 7.1 | OBJECTIVE | 19 |
| | 7.2 | DESIGN | 20 |
| | 7.3 | ENDPOINTS | 20 |
| | 7.4 | ADDITIONAL CLINICAL MEASURES | 22 |
| | 7.5 | NUMBER OF SUBJECTS | 22 |
| | 7.6 | METHODS OF FOLLOW-UP | 23 |
| 8.0 | TRI | AL POPULATION | 24 |
| | 8.1 | SUBJECT INCLUSION CRITERIA | 24 |
| | 8.2 | SUBJECT EXCLUSION CRITERIA | 24 |
| | 8.3 | ENROLLED POPULATION | 26 |
| | 8.4 | INDEX VALVE POPULATION | 26 |
| | 8.5 | SUBJECT AND TRIAL DURATION | 26 |
| | 8.6 | SUBJECT TERMINATION OR WITHDRAWAL | 26 |
| 9.0 | STA | TISTICAL METHODS | 27 |
| | 9.1 | ANALYSIS POPULATION | 27 |
| | 9.2 | SAMPLE SIZE | 27 |
| | 9.3 | STATISTICAL ANALYSIS | 27 |

# CLINICAL INVESTIGATIONAL PLAN PROTOCOL NUMBER: 2012-02

| | 9.4 ADDITIONAL MEASURES | 30 |
|---|---|---|
| | 9.5 POOLABILITY | 31 |
| | 9.6 ANALYSIS OF COVARIATES | 31 |
| | 9.7 MISSING DATA | 31 |
| | 9.8 FOLLOW-UP AND COMPLIANCE DATA | 31 |
| 10.0 | TRIAL PROCEDURES | 32 |
| | 10.1 SUBJECT SCREENING | 32 |
| | 10.2 INFORMED CONSENT | 32 |
| | 10.3 BASELINE ASSESSMENT | 33 |
| | 10.4 VALVE REPLACEMENT PROCEDURE | 33 |
| | 10.5 POST INDEX VALVE IMPLANT | 34 |
| | 10.6 DISCHARGE | 34 |
| | 10.7 POST DISCHARGE FOLLOW-UP ASSESSMENTS | 35 |
| | 10.8 MISSED FOLLOW-UP | 36 |
| | 10.9 DEVICE REMOVAL OR EXPLANT | 37 |
| 11.0 | ADVERSE EVENTS | 37 |
| | 11.1 REPORTING | 37 |
| | 11.2 NOTIFICATION OF UADE AND/OR SERIOUS DEVICE RELATED ADVERSE EFFECTS | 38 |
| | 11.3 DEATH AND EXPLANTS | 38 |
| | 11.4 DATA MONITORING COMMITTEE | 39 |
| | 11.5 CLINICAL EVENTS COMMITTEE | 39 |
| 12.0 | TRIAL AND DATA MANAGEMENT | 40 |
| | 12.1 TRIAL CORE LABS | 40 |
| | 12.2 DEVICE ACCOUNTABILITY | 40 |
| | 12.3 PROTOCOL DEVIATIONS | 41 |
| | 12.4 TRIAL SITE INITIATION AND MONITORING PLAN | 42 |
| | 12.5 DOCUMENTATION REQUIREMENTS | 43 |
| | 12.6 DATA COLLECTION | 44 |
| | 12.7 DATA AND DOCUMENT RETENTION | 44 |
| | 12.8 TRIAL PROTOCOL AMENDMENTS | 45 |
| | 12.9 TRIAL COMPLETION | 45 |
| | 12.10 FUTURE PLANS | 45 |
| 13.0 | STATEMENTS OF COMPLIANCE, CONFIDENTIALITY AND RESPONSIBILITIES | 45 |
| | 13.1 GOOD CLINICAL PRACTICE STATEMENT | 45 |
| | 13.2 REGULATIONS AND GUIDELINES | 46 |

CLINICAL INVESTIGATIONAL PLAN PROTOCOL NUMBER: 2012-02

REV J: 03March2021

| | 13.3 INVESTIGATOR RESPONSIBILITIES | 46 |
|------|------------------------------------|----|
| | 13.4 SPONSOR RESPONSIBILITIES | 46 |
| 14.0 | PUBLICATIONS | 47 |
| 15.0 | REFERENCES | 47 |

# TRIAL PROTOCOL ATTACHMENTS

ATTACHMENT A: CLINICAL TRIAL SCHEME

ATTACHMENT B: INSTRUCTIONS FOR USE

ATTACHMENT C: INFORMED CONSENT FORM TEMPLATE

ATTACHMENT D: CASE REPORT FORMS

ATTACHMENT E: CORE LABORATORY PROCEDURE MANUAL

ATTACHMENT F: SERUM GLYCEROL SAMPLE COLLECTION MANUAL

ATTACHMENT G: QUALITY OF LIFE QUESTIONNAIRE (SF-12 V2)

ATTACHMENT H: ADVERSE EFFECT (CODES & DEFINITIONS)

ATTACHMENT J: RESPONSIBILITIES (INVESTIGATOR & SPONSOR)

ATTACHMENT K: SUBJECT IMPLANT CARD

ATTACHMENT L: PROTOCOL DEVIATION CODES

ATTACHMENT M: DEVICE DEFICIENCY CODES

ATTACHMENT N: CLINICAL TRIAL AGREEMENT

ATTACHMENT O: POWER SIMULATION CODE FOR PRIMARY SAFETY ENDPOINT

REVISION J: 03 MARCH 2021

# **5.0 TRIAL OVERVIEW**

#### 5.1 INTRODUCTION AND BACKGROUND

Valvular heart disease is a life-threatening disease that afflicts millions of people worldwide and leads to approximately 250,000 valve repairs and/or replacements each year. The number of subjects requiring aortic valve replacement (AVR) is increasing due to prolonged life expectancy. Many subjects are asymptomatic until the disease is well advanced and, once diagnosed, have poor prognosis depending on the severity of valve calcification and history of cardiac events<sup>1</sup>. Diseased heart valves can be treated by medication, surgical repair or surgical replacement.

#### 5.1.1 AORTIC AND MITRAL HEART DISEASE

Aortic valvular heart disease includes conditions involving any of the following – obstructions of the aortic heart valve or stenosis; leakage of the aortic valve, known as regurgitation, incompetence, or insufficiency, and combinations of the two, sometimes referred to as mixed disease or combined lesions. Valvular heart disease may be caused by any number of factors, including congenital abnormalities, infection by various micro-organisms, degenerative calcification and rheumatic heart disease. When subjects become symptomatic, angina, syncope, and congestive heart failure (CHF) are the primary clinical signs observed. Studies report that among symptomatic subjects with medically treated moderate-to-severe AS, mortality rates after the onset of symptoms are approximately 25% at one year and 50% at two years. Other studies show that subjects with symptomatic AS have a life expectancy of 2 – 4 years. Neither aortic stenosis nor aortic insufficiency can be effectively treated medically; however, the symptoms of aortic valve disease can be managed medically.

Stenosis of the mitral valve is the narrowing of the valve opening that causes lower blood flow through the valve. In over 99% of stenotic mitral valves, the etiology is rheumatic disease.<sup>3</sup> Other rare causes of mitral stenosis include congenital malformed valves, active infective endocarditis, massive annular calcium, and metabolic or enzymatic abnormalities.<sup>3</sup> Regurgitation of the mitral valve occurs when blood flows back into the valve as the leaflets close or leaks through the leaflets after they are closed. Mitral regurgitation has multiple etiologies including: floppy mitral valves, active or healed infective endocarditis, papillary muscle dysfunction, annular calcium, idiopathic chordae tendineae rupture, rheumatic disease, dilated and hypertrophic cardiomyopathies, endocardial fibrosis, and collagenvascular disorders (lupus, scleroderma), or Marfan's or Marfan-like disorders. Edward et al reviewed data collected from 1648 patients between January 1990 and December 1999 in northern New England, and noted that mitral valve replacements and repair procedures have substantially increased and indications for these procedures have expanded to also include older and sicker patients with less rheumatic and more degenerative and coronary artery-related mitral valve problems.<sup>4</sup> As the incidence of rheumatic mitral stenosis and regurgitation has decreased, mitral regurgitation caused by degenerative disease of

REVISION J: 03 MARCH 2021 

REV J: 03March2021

CLINICAL INVESTIGATIONAL PLAN


the mitral apparatus and caused by the left ventricular dysfunction associated with coronary artery

disease has become the predominant hemodynamic lesion of the mitral valve.<sup>5</sup>

5.1.2 TREATMENT OF AORTIC AND MITRAL VALVULAR HEART DISEASE

Aortic stenosis and insufficiency can be treated by surgical intervention, including balloon valvuloplasty,

valve repair, and valve replacement. Balloon valvuloplasty, a treatment option for aortic stenosis, utilizes

a balloon-tipped catheter to stretch open the narrowed valve. Valvuloplasty is predominately used to

treat children or adults who are poor surgical candidates. Valve repair techniques include annuloplasty

for dilated valve disease, patching leaflet perforations, resected vegetations, or tears, and leaflet

extension.<sup>6,7</sup> Aortic valve repair for stenosis does not show good clinical results.<sup>8</sup> Replacement of the

aortic valve is indicated for symptomatic subjects and asymptomatic subjects with left ventricular

dysfunction.

Diseased mitral valves can be treated by medication, surgical repair and surgical replacement. Repairing

the native valve is generally preferred over replacing it. Surgical repair can involve modifying the valve

tissue or underlying structures. This procedure can be performed with or without implantation of an

annuloplasty ring that provides support to the native valve so that it closes completely and functions

normally. If the native valve cannot be repaired, it is replaced by either a mechanical valve (constructed

from synthetic material) or a tissue bioprosthetic valve (made primarily from animal tissue including

bovine pericardium, or human valves from cadavers.

**BIOPROSTHETIC HEART VALVES** 

Bioprosthetic heart valves are indicated for use in subjects suffering from valvular heart disease. These

tissue valves are used particularly in those subjects for whom long-term anticoagulation therapy is

contraindicated or who may be difficult to maintain on anticoagulation therapy.

5.2 **DEVICE DESCRIPTION** 

**Edwards Pericardial Aortic Bioprosthesis** 

The Edwards Pericardial Aortic Bioprosthesis, Model 11000A (also referred to as the Model 11000A) is a

bioprosthesis comprised of bovine pericardium. It is based on the same design as the Carpentier-Edwards

PERIMOUNT Magna Ease Pericardial Aortic Bioprosthesis, Model 3300TFX, which was approved under

P860057/S042 on 07 May 2009.

The physical structure and design of the Model 11000A is identical to the Model 3300TFX, except for tissue

processing, sterilization and packaging. The Edwards Pericardial Aortic Bioprosthesis, Model 11000A, is a

trileaflet bioprosthesis comprised of treated bovine pericardium that is mounted on a flexible frame. It is

available in sizes 19, 21, 23, 25, 27, and 29 mm. The bioprosthesis is stored in non-aqueous packaging,

and does not require rinsing prior to implantation.

REVISION J: 03 MARCH 2021  CLINICAL INVESTIGATIONAL PLAN


The wireform is made of a cobalt-chromium alloy and is covered with a woven polyester fabric. A cobalt-

REV J: 03March2021

chromium alloy/polyester film laminate band surrounds the base of the wireform frame. A silicone sewing

ring that is covered with a porous polytetrafluoroethylene (PTFE) cloth is attached to the wireform frame.

The sewing ring has three, equally spaced black silk suture markers at the cusp centers to aid in

bioprosthesis orientation and suture placement.

The Model 11000A valve is treated with a new tissue process that builds on Edwards' existing tissue

process, ThermaFix (TFX). The new process allows the valve to be stored in non-aqueous packaging and

the valve is ethylene oxide sterilized.

**Edwards Pericardial Mitral Bioprosthesis** 

The Edwards Pericardial Mitral Bioprosthesis, Model 11000M is a bioprosthesis comprised of bovine

pericardium. It is based on the same design as the Carpentier-Edwards PERIMOUNT Magna Mitral Ease

Pericardial Bioprosthesis, Model 7300TFX, which was approved under P860057/S068 on 24 June 2010.

The physical structure and design of the Model 11000M is identical to the Model 7300TFX, except for

tissue processing, sterilization and packaging. The Edwards Pericardial Mitral Bioprosthesis, Model

11000M, is a trileaflet bioprosthesis comprised of treated bovine pericardium that is mounted on a flexible

frame. It is available in sizes 25, 27, 29, 31, and 33 mm. The bioprosthesis is stored in non-aqueous

packaging, and does not require rinsing prior to implantation.

The wireform is made of a cobalt-chromium alloy and is covered with a woven polyester fabric. A cobalt

chromium alloy/polyester film laminate band surrounds the base of the wireform frame. A waffled silicone

sewing ring that is covered with a porous polytetrafluoroethylene (PTFE) cloth is attached to the wireform

frame. The sewing ring is scalloped along its anterior portion. Black silk suture markers on the anterior

portion facilitate the orientation of the bioprosthesis and help avoid obstruction of the left ventricular

outflow tract by a strut. A black silk suture guide line circles the sewing ring.

The Model 11000M valve is treated with a new tissue process that builds on Edwards' existing tissue

process, ThermaFix (TFX). The new process allows the valve to be stored in non-aqueous packaging and

the valve is ethylene oxide sterilized.

5.2.1 DEVICE INDICATION FOR USE

The Edwards Pericardial Aortic Bioprosthesis, Model 11000A, is indicated for patients who require

replacement of their native or prosthetic aortic valve. The device is contraindicated only if the implanting

surgeon decides the anatomy and pathology pose unwarranted risk.

The Edwards Pericardial Mitral Bioprosthesis, Model 11000M, is indicated for patients who require

replacement of their native or prosthetic mitral valve. The device is contraindicated only if the implanting

surgeon decides the anatomy and pathology pose unwarranted risk.

REVISION J: 03 March 2021 


#### 5.2.2 DEVICE TRAINING

Training on the Model 11000A and Model 11000M will be per the Instructions for Use (IFUs) provided in *Attachment B*. The implant technique for the Model 11000A and Model 11000M is the same as other supraannular bioprosthetic valves. The only usage difference in Model 11000A and Model 11000M from other tissue valves is that Models 11000A and 11000M do not require rinsing prior to implantation. If the bioprosthesis is rinsed prior to implantation, the valve must then be kept hydrated with sterile physiological saline irrigation on both sides of the leaflets until the heart is closed.

### 5.3 REPORT OF PRIOR INVESTIGATIONS

A clinical trial (Protocol Number 2010-03) initiated in Europe in July 2011 is underway to gather data on the Model 11000A. This is a prospective, non-randomized clinical trial of the investigational valve for subjects undergoing aortic valve replacement (AVR). This trial is an observational, confirmatory trial and not powered for statistical analysis. To date, the trial has enrolled one hundred thirty three (133) subjects at two (2) investigational sites in Poland. There are three (3) early deaths, of which two (2) deaths were adjudicated by the CEC as not related to the valve, and one (1) death was adjudicated as valve related.

There are sixteen (16) late deaths, of which three (3) have been adjudicated as valve related. One (1) incident of late study valve related mortality was adjudicated to be due to valve thrombosis, one (1) was adjudicated as to be due to nonspecific/unknown cause, and one (1) valve-related late death was adjudicated to be due to cardiac arrest. As of 7 April 2017, 100% of the eligible subjects completed the discharge, 99.2% completed the 3 month, 97.6% completed the 1 year follow-up, 92.5% completed the 2 year follow-up, 93.8% completed the 3 year follow-up, 92.7% of eligible subjects completed the 4 year follow-up, and 100% completed the 5 year follow up visits. At the time of this interim report there are no occurrences of study valve related bleeding, hemolysis, structural valve deterioration or unanticipated adverse device effects.

REVISION J: 03 MARCH 2021 

# Clinical Follow-up

Clinical follow-up endpoints are listed in Table 1 for the first 133 subjects implanted.

Table 1: Safety endpoints Events (2010-03 Cohort)

| | Early Events<br>(≤30 POD)<br>N = 133 | Late Events<br>(>30 POD)<br>Late pt-yrs = 495.29 | |
|---|---|---|---|
| Safety Endpoint | % (n) | %/pt-yr (m) | 95% CL |
| Mortality | 2.3 (3) | 3.2 (16) | 4.8 |
| Valve-related mortality | 0.8 (1) | 0.6 (3) | 1.4 |
| Thromboembolism | 2.3 (3) | 0.2 (1) | 0.8 |
| Valve thrombosis | 0.0 (0) | 0.2 (1) | 0.8 |
| Major bleeding events | 6.8 (9) | 0.4 (2) | 1.1 |
| Major paravalvular leakage <sup>§</sup> | 0.8 (1) | 0 (0) | 0.5 |
| Endocarditis | 0.0 (0) | 0.2 (1) | 0.8 |
| Structural valve deterioration | 0.0 (0) | 0 (0) | 0.5 |
| Hemolysis | 0.0 (0) | 0 (0) | 0.5 |
| Nonstructural valve dysfunction | 0.0 (0) | 0.2 (1) | 0.8 |
| Reoperation (trial valve) | 0.0 (0) | 0.2 (1) | 0.8 |
| Explant (trial valve) | 0.0 (0) | 0.2 (1) | 0.8 |

<sup>&#</sup>x27;n' is the number of subjects who experienced the event; 'm' is the number of events observed.

The investigational valve, Model 11000 is the same design as Model 11000A, and was later renamed as Model 11000A.

# 6.0 BENEFITS AND RISKS

#### 6.1 BENEFITS

The benefits of the Models 11000A and 11000M are the same as other bioprosthetic valves including improved valvular function, acute alleviation of symptoms related to valve stenosis or insufficiency, and/or improved morbidity and mortality.

The anticipated additional benefits of aortic valve Model 11000A, and mitral valve Model 11000M are to eliminate the need for rinsing the bioprosthesis prior to implantation, less exposure to the risks of glutaraldehyde, and elimination of hazardous waste requiring special disposal.

REVISION J: 03 March 2021 

Early event rates are described as simple proportions (n/N); late event rates utilize linearized rates (m/ late pt-yrs).

One-sided upper 95% confidence limit for the linearized rate (CI: Confidence Interval).

<sup>&</sup>lt;sup>5</sup>Major paravalvular leak is defined as paravalvular leak graded as +3 Moderate or +4 Severe by the Echo Core Lab or any paravalvular leak requiring intervention. Previous report included one late major PVL (+3) and one early minor PVL (+2) in Subject 201003-330 which was reassessed by the Core Lab to be minor late PVL (+2) and no early PVL (0/None).


#### 6.2 RISKS

As with all prosthetic heart valves, serious complications, sometimes leading to death may be associated with the use of tissue valves. Complications due to individual subject reaction to an implanted device, or to physical or chemical changes in the components, particularly those of biological origin, may occur at varying intervals (hours or days) necessitating reoperation and replacement of the prosthetic device. Some or all of the risks listed below could require a reoperation or explant, and/or they may lead to permanent disability or death.

# Known/potential risks associated with stented bioprosthetic heart valves include but not limited to:

- Angina
- Bleeding diatheses (coagulopathy) related to anticoagulant therapy
- Cardiac arrhythmias
- Cardiac failure
- Coronary ostial blockage
- Endocarditis
- Hemolysis/Hemolytic anemia
- Hemorrhage
- Immunological response
- Leaflet entrapment (impingement)
- Myocardial infarction
- Nonstructural valve dysfunction
- Paravalvular/Perivalvular leak

- Malfunctions of valve due to distortion at implant, fracture of wireform, physical and or chemical deterioration of valve components
- Patient prosthetic mismatch (PPM)
- Regurgitation/insufficiency
- Stenosis
- Thromboembolism/stroke
- Tissue deterioration including infection, calcification, thickening, perforation, degeneration, suture abrasion, instrument trauma, and or leaflet detachment
- Transient ischemic attack (TIA)
- Valve pannus
- Valve thrombosis

## Potential risks associated with aortic valve replacement surgery include but not limited to:

- Allergic reaction
- Annular dissection
- Aortic dissection
- Arterial dissection
- Bleeding, anticoagulant related
- Bleeding, procedural
- Bleeding, post-procedural
- Cardiac arrest
- Cardiogenic shock
- Disseminated intravascular coagulation (DIC)
- Esophageal rupture
- Heart failure

- Hypoxemia
- Infection, local or wound
- Infection, systemic (septicemia)
- Myocardial infarction
- Multi-system organ failure (MOF)
- Pericardial effusion
- Pericardial tamponade
- Pleural effusion
- Pulmonary edema
- Pneumonia
- Renal dysfunction
- Respiratory failure

REVISION J: 03 March 2021 

CLINICAL INVESTIGATIONAL PLAN


Hematoma

Heparin induced thrombocytopenia (HITs)

Hypotension

Hypertension

Thromboembolism

Venous, peripheral or central

REV J: 03March2021

Arterial, peripheral or central

- Pulmonary, thrombus or other

Risks associated with Models 11000A and 11000M are anticipated to be the same as those listed above for other aortic or mitral bioprosthetic valves and valve replacement surgery. Based on pre-clinical testing, it is not anticipated that any new risks associated with the Model 11000A and Model 11000M tissue process, sterilization method, or packaging will be observed.

# 6.3 MINIMIZING SUBJECT RISK

Several safeguards are incorporated into the trial to minimize subject risk. The pre-clinical device testing for the implantable valve was performed in accordance with FDA guidance, ISO 5840:2009 and recognized product standards. All test results met or passed the required specifications supporting reasonable safety for this investigational product.

This clinical trial is conducted under the direction of qualified physicians experienced with cardiac surgery including aortic and mitral valve repair/replacement and the use of investigational devices. All participating investigators and sites are screened and qualified. They must be experienced in conducting clinical research and have adequate personnel to assure compliance to the trial protocol. No special training is required to implant the Models 11000A and 11000M. The Instructions for Use (*Attachment B*) provide detailed instructions on the proper handling and implantation of these investigational valves.

#### 7.0 TRIAL DESIGN

This trial design methodology is based on a one year structural valve deterioration primary endpoint, as discussed in Sections 7.3.1 and 9.0. Based on the results of a pre-clinical assessment and OUS clinical trial, the use of the investigational valve is justified.

# 7.1 OBJECTIVE

The objective of this trial is to confirm that the modifications to tissue processing, valve sterilization, and packaging of the FDA-approved (P860057/S042) Carpentier-Edwards PERIMOUNT Magna Ease Pericardial Aortic Bioprosthesis, Model 3300TFX, which will be designated as the Edwards Pericardial Aortic Bioprosthesis Model 11000A, and the Carpentier-Edwards PERIMOUNT Magna Mitral Pericardial Bioprosthesis, Model 7300TFX, which will be designated as the Edwards Pericardial Mitral Bioprosthesis Model 11000M do not raise any new questions of safety and effectiveness in subjects who require replacement of their native or prosthetic aortic or mitral valve. The only differences between the Model 3300TFX and Model 11000A, and Model 7300TFX and 11000M are modifications in tissue processing,

REVISION J: 03 MARCH 2021 

CLINICAL INVESTIGATIONAL PLAN


valve sterilization, and packaging. The primary safety hypothesis to be accepted or rejected by statistical data is provided in **Statistical Methods Section 9.0**.

REV J: 03March2021

#### 7.2 DESIGN

The trial is a multicenter, prospective, double arm trial to be conducted throughout the United States, Canada, Europe and Asia Pacific. It will include subjects with valve stenosis or insufficiency, or stenosis plus insufficiency requiring a planned valve replacement of their native or prosthetic valve. Final analysis for the aortic arm will be performed when at least three hundred (300) AVR subjects have completed the POD 390 follow-up visit, and at least 800 AVR patient-years of cumulative follow-up have been reached. Analysis for the mitral arm will be completed when at least three hundred (300) combined aortic and mitral subjects have completed the POD 390 follow-up visit and at least eight hundred (800) AVR and at least one hundred (100) MVR patient-years of cumulative follow-up have been reached. The tests for the trial endpoints were performed and the trial data was submitted to FDA for the PMA approval of the devices evaluated under the aortic and mitral arms. All IDE Subjects (aortic and mitral arms) who are currently enrolled and alive will be followed to 5 years. In an effort to obtain sufficient long-term data, approximately 250 Subjects implanted with the Model 11000A valve at up to 10 sites will be asked to consent for extended follow-up annually through 10 years post-procedure. In addition, approximately 25 Subjects implanted with the Model 11000M valve at select sites will be asked to consent for extended follow-up annually through 10 years post-procedure.

# 7.3 ENDPOINTS

All safety and effectiveness data for the Model 11000A and Model 11000M valves will be compared to control data published in articles in the prosthetic heart valve literature.

REVISION J: 03 MARCH 2021 

**7.3.1 SAFETY** 

Primary Safety Endpoint (up to 390 days post-implant):

The primary safety endpoint for the trial is the rate of implanted subjects that experience structural deterioration of the trial valve by the time of the POD 390 follow-up visit. The null hypothesis is that the

rate of structural valve deterioration at one year is greater than 1%. The alternative hypothesis is that this

rate is less than 1%.

Primary Safety Endpoint (Continued follow-up):

For continued follow-up of Subjects, the primary safety endpoint for the trial is the rate of implanted

subjects that experience structural deterioration of the trial valve as determined by a Clinical Events

Committee (CEC).

Secondary Safety Endpoints (Pre-approval):

Safety will be established by comparing the occurrence of specific safety endpoints to the objective

performance criteria (OPC) reported in Table R.1 in ISO 5840:2009, Annex R.1 as recommended by the

FDA in the Draft Guidance involving Heart Valves – Investigational Device Exemption (IDE) and Premarket

Approval (PMA) Applications issued January 20, 2010.

Secondary Safety Endpoints (Continued follow-up):

For continued follow-up of Subjects, linearized rates will be used to summarize the following safety

endpoints for the late (>30 days) post-operative period.

Thromboembolism

Valve thrombosis

All bleeding/hemorrhage

Major bleeding/hemorrhage

All paravalvular leak

Major paravalvular leak

Non-structural valve deterioration

Endocarditis

All-cause mortality

Trial valve-related mortality

Trial valve-related reoperation

Explant

Hemolysis

The Data Monitoring Committee (DMC) will review aggregate safety and hemodynamic data to determine if the trial is being conducted safely and in accordance to the protocol. The DMC will decide if the clinical

investigation should be modified, suspended and or stopped.

The Clinical Events Committee (CEC) evaluates the adverse events that are endpoint related as well as those resulting in death. The CEC adjudicates early and late events for their relatedness to the

investigational device and/or the surgical procedure.

Adverse event categories are provided in **Section 11.0** and definitions are provided in **Attachment H** –

REVISION J: 03 March 2021 


# Adverse Effect (Codes and Definitions).

#### 7.3.2 EFFECTIVENESS

Effectiveness endpoints include the following:

 Clinically acceptable hemodynamic performance confirmed by echocardiography and core lab evaluation which will include the following parameters:

Mean gradient

Peak gradient

Effective orifice area [EOA]

EOA index

Performance index

- Cardiac Output [CO]
- Cardiac index
- Valvular regurgitation including

paravalvular leak

- New York Heart Association (NYHA) functional class compared to baseline
- Change in Quality of Life assessment Short Form 12 version 2 (SF-12v2) score from baseline to POD 390.

#### 7.4 ADDITIONAL CLINICAL MEASURES

# Additional Data in support of analysis:

- Blood Data
  - White Blood Cell Count
  - Red Blood Cell Count
  - Hemoglobin
  - Hematocrit
  - Platelet Count
  - Plasma free hemoglobin or haptoglobin or serum LDH
  - Coagulation profile (If collected per standard of care dependent on anticoagulation regimen)
  - Serum Glycerol (See Section 10.4.1 for details)

#### 7.5 NUMBER OF SUBJECTS

Up to seven hundred (700) aortic valve replacement (AVR) subjects and up to one hundred seventy five (175) mitral valve replacement (MVR) subjects at up to forty (40) clinical sites will be enrolled. At least eight (8) centers will implant thirty (30) or more AVR or thirty (30) or more AVR/MVR subjects with one year follow-up. An enrollment rate of three (3) to four (4) subjects per site per month is anticipated. Sites with less than ten (10) subjects enrolled will have data combined and reported. Enrollment period completion is anticipated within 1095 days or three (3) years.

REVISION J: 03 MARCH 2021 


REV J: 03March2021 CLINICAL INVESTIGATIONAL PLAN

#### 7.6 **METHODS OF FOLLOW-UP**

Following informed consent and determination of eligibility, subjects undergo a pre-operative echocardiogram to document the function of their current valve prior to surgery. Evaluation of the echocardiogram (echo) is performed by a qualified cardiologist/sonographer at the site and over read by an independent core lab. Other baseline exams include physical assessment, recording of pertinent medical history, electrocardiogram (ECG), NYHA classification, Canadian Cardiovascular Society (CCS) Angina classification, quality of life (QOL) assessment, and selected hematological variables.

During the procedure, a transesophageal echo (TEE) and blood collection (if applicable, see Section 10.4.1) will be completed, and a post-operative ECG/rhythm strip will be conducted upon admission to the intensive care unit. In addition, follow-up will occur at or prior to hospital discharge where physical assessment, NYHA classification, CCS Angina classification, ECG, echo and evaluation of selected hematological variables will occur. A post-op echocardiogram must be completed on or prior to postoperative Day 10. At POD 30, a phone follow-up will assess NYHA classification and information on any adverse events that have occurred since discharge. At POD 105 follow-up visit, a physical assessment, NYHA classification, ECG, echocardiogram, and selected hematological variables will be evaluated. The subsequent follow-up visits will be made at POD 390, and annually thereafter up to POD 1825 or 3650. **Table 2** lists the follow-up visit time points and visit windows.

Adverse events and anti-thromboembolic therapy/medications are collected from the time of the index procedure until the subject exits the clinical trial.

REVISION J: 03 MARCH 2021 

Table 2. Visit Follow-Up Schedule

| Visit | Visit Window (Days) | Timing from Implant (Day 0) |
|------------------------|---------------------|-----------------------------|
| Screening/Baseline | | Day -60 to Day 0 |
| Discharge <sup>1</sup> | | Prior to Discharge |
| POD 30 | -5/+10 | Day 25 to 40 |
| POD 105 | -15/+30 | Day 90 to 135 |
| POD 390 (1 yr) | -25/+45 | Day 365 to 435 |
| POD 730 (2 yr) | -25/+45 | Day 705 to 775 |
| POD 1095 (3 yr) | -25/+45 | Day 1070 to 1140 |
| POD 1460 (4 yr) | -25/+45 | Day 1435 to 1505 |
| POD 1825 (5 yr) | -25/+45 | Day 1800 to 1870 |
| POD 2190 (6 yr)* | -55/+75 | Day 2135 to 2265 |
| POD 2555 (7 yr)* | -55/+75 | Day 2500 to 2630 |
| POD 2920 (8 yr)* | -55/+75 | Day 2865 to 2995 |
| POD 3285 (9 yr)* | -55/+75 | Day 3230 to 3360 |
| POD 3650 (10yr)* | -55/+75 | Day 3595 to 3725 |

<sup>&</sup>lt;sup>1</sup> Subjects who are not discharged within 10 days post procedure must have an echocardiogram to assess performance of the trial valve. Those subjects will not require an additional echocardiogram at discharge.

# 8.0 TRIAL POPULATION

#### 8.1 SUBJECT INCLUSION CRITERIA

A subject who meets all of the following criteria potentially may be included in the trial:

- Is 18 years or older
- 2. Provides written informed consent prior to trial procedures
- 3. Agrees to attend follow-up assessments for up to 5 years and is willing to comply with specified follow-up evaluations at clinical investigational sites that are participating in the COMMENCE trial and/or obtain the protocol-specified diagnostic tests at centers that are under the same IRB or the same healthcare system
- 4. Diagnosed with aortic or mitral valve disease requiring valve replacement based on pre- operative evaluation
- 5. Scheduled to undergo planned aortic or mitral valve replacement with or without concomitant bypass surgery
- Scheduled to undergo planned aortic valve replacement with or without resection and replacement of the ascending aorta from the sinotubular junction and without the need for circulatory arrest for hemi arch or arch replacement

# 8.2 SUBJECT EXCLUSION CRITERIA

A subject who meets *any of the following criteria will not be included* in the trial:

- 1. Requires emergency surgery
- 2. Requires planned multiple valve replacement/repair (with the exception of mitral valve replacement with tricuspid valve repair)
- 3. Has prior valve surgery, which included implant of a bioprosthetic valve, mechanical valve, or annuloplasty ring that will remain *in situ*

REVISION J: 03 March 2021 

<sup>\*</sup>Subjects who have consented to continued follow up with the Model 11000A or Model 11000M valve.

- 4. Requires a surgical procedure outside of the cardiac area (e.g. vascular bypass)
- 5. Requires surgical replacement of the aortic root
- 6. Has active endocarditis/myocarditis or endocarditis/myocarditis within 3 months to the scheduled aortic or mitral valve replacement surgery
- 7. Has renal insufficiency as determined by creatinine (S-Cr) level ≥ 2.5 mg/dL or end-stage renal disease requiring chronic dialysis at screening visit
- 8. Has MRI or CT scan confirmed stroke, cerebrovascular accident (CVA) or transient ischemic attack (TIA) within 6 months (180 days) prior to planned valve surgery
- 9. Has acute myocardial infarction (MI) within 30 days prior to planned valve surgery
- 10. Has presence of non-cardiac disease limiting life expectancy to less than 12 months
- 11. Diagnosed with hypertrophic obstructive cardiomyopathy (HOCM)
- 12. Diagnosed with abnormal calcium metabolism and hyperparathyroidism
- 13. Exhibits left ventricular ejection fraction ≤ 20% as validated by diagnostic procedure prior to planned valve surgery
- 14. Echocardiographic evidence of an intra-cardiac mass, thrombus, or vegetation
- 15. Hemodynamic or respiratory instability requiring inotropic support, mechanical circulatory support, or mechanical ventilation within 30 days prior to planned valve surgery
- 16. Documented leukopenia (WBC <  $3.5 \times 10^3/\mu$ L), acute anemia (Hgb < 10.0 gm/dL or 6 mmol/L), or thrombocytopenia (platelet count <  $50 \times 10^3/\mu$ L) accompanied by history of bleeding diathesis or coagulopathy
- 17. Has prior organ transplant or is currently an organ transplant candidate
- 18. Current or recent participation (within 6 weeks prior to surgery) in another drug or device trial
- 19. Was previously implanted with investigational device (Model 11000A or Model 11000M)<sup>2</sup>
- 20. Pregnant (female subject of childbearing potential only), lactating or planning to become pregnant during the duration of participation in trial
- 21. Currently incarcerated or unable to give voluntary informed consent
- 22. Documented history of substance (drug or alcohol) abuse within the last 5 years prior to implant
- 23. Requires concomitant left ventricular assist device (LVAD) placement

CONFIDENTIAL AND PROPRIETATARY DATA: This document and the information contained herein may not be reproduced, used, or disclosed without written permission from Edwards Lifesciences LLC

REVISION J: 03 MARCH 2021


<sup>&</sup>lt;sup>2</sup> Note: Previously implanted means that the index valve replacement procedure was completed. The procedure is complete when the surgeon takes the subject off cardiopulmonary bypass and restarts the heart.

# 8.3 ENROLLED POPULATION

Subjects will be included in the enrolled population after meeting all the enrollment criteria, signing the informed consent, and after the surgeon assesses the subject's anatomy, sizes the annulus, and determines that the trial valve can be implanted. If the surgeon is unable to complete the implant procedure, the subject is considered "intent to treat" and will be followed for safety (adverse event collection) for 30 days or until any adverse events experienced by subject are resolved. No protocol-specified tests during this period will be required.

Each investigator screens subjects for potential inclusion into the trial. Screening results are used to make a final determination as to subject suitability for enrollment. Early and late results from this trial (i.e., immediate post-operative and up to one year) serve as the basis for determining the safety and effectiveness of the Edwards Pericardial Aortic Bioprosthesis, Model 11000A and the Edwards Pericardial Mitral Bioprosthesis, Model 11000M. Subjects must meet all applicable inclusion criteria and no preoperative exclusion criteria at the time of enrollment evaluation in order to participate.

#### 8.4 INDEX VALVE POPULATION

The investigational valve population includes all enrolled subjects that receive and retain the index valve. The analysis of the effectiveness endpoints and of the primary safety endpoint will be based on the investigational valve population.

#### 8.5 SUBJECT AND TRIAL DURATION

Total enrollment period for this trial is estimated to be 1095 days or 3 years. Subject duration in the trial is estimated to be no longer than 1825 days (5 years) or 3650 days (10 years) for those who have consented to continued follow-up. Overall duration of the trial is estimated to be 3833 days or 10.5 years, and will involve at least eight hundred (800) AVR patient-years and at least one hundred (100) mitral valve replacement (MVR) patient-years of follow-up. Trial begins with the enrollment of the first subject and ends after the last subject is exited from the trial after completing the last follow-up visit at approximately POD 3650, all subjects are fully monitored, all outstanding data queries are resolved and all trial sites are closed to follow-up.

#### 8.6 SUBJECT TERMINATION OR WITHDRAWAL

Once enrolled, subjects may discontinue participation at any time by withdrawing informed consent or meeting the requirement for termination. Participation in the trial is entirely voluntary. Subject participation for any patient requiring explant or valve-in-valve (ViV) procedure will be terminated at either 30 days post-explant/ViV (followed for safety only) or when all post-explant/ViV adverse events are resolved (whichever comes last). If the surgeon is unable to complete the implant procedure, those subjects are considered enrolled as "intent to treat" and will be followed for safety (adverse event

REVISION J: 03 March 2021 

collection) for 30 days or until any adverse events experienced by this cohort are resolved and then will be exited from the trial.

# 9.0 STATISTICAL METHODS

#### 9.1 ANALYSIS POPULATION

The analysis populations will include the enrolled population and the index valve population. The index valve population will include all subjects who meet enrollment criteria, provide written informed consent, those deemed able to implant in the operating room and who receive the index valve. The enrolled population will include the index valve population and the "intent to treat" population. For the enrolled population, the number of patients enrolled per site will be reported. Summaries of baseline and procedural data will be based on the enrolled population. The analysis of mortality and all safety data, including the primary endpoint, shall in general be based on the index valve population; however, the analysis will also be provided using the enrolled cohort. For the investigational valve population, the number of subjects implanted per site will be reported, stratified by implant position and valve size within each position.

#### 9.2 SAMPLE SIZE

The sample size for this study follows the recommendation from the FDA in the Draft Guidance involving Heart Valves – Investigational Device Exemption (IDE) and Premarket (PMA) Applications (2010).

Assuming the Poisson distribution and the true rate being equal to its OPC, and with probabilities of Type I error of 0.05 and Type II error of 0.20, the amount of data necessary to achieve the smallest OPC of 1.2% per patient-year (excluding the OPCs for valve thrombosis, major hemorrhage, and major paravalvular leak, which are all less than 1.2% per patient-year) is 800 patient-years.

# 9.3 STATISTICAL ANALYSIS

# 9.3.1 SAFETY ANALYSIS

# 9.3.1.1 Primary Safety Endpoint (up to 390 days post-implant)

The primary safety endpoint for the trial is the rate of structural deterioration of the study valve at the time of the POD 390 visit. If we let p denote the probability that an implanted subject will experience structural valve deterioration by the time of the POD 390 visit, then the null and alternative hypotheses for the primary safety endpoint are:

REVISION J: 03 March 2021 

<sup>&</sup>lt;sup>3</sup> If the surgeon is unable to complete the implant procedure, those subjects are considered enrolled as "intent to treat" and will be followed for 30 days or until any adverse events experienced by this cohort are resolved and then will be exited from the trial.


*H*<sub>0</sub>: *p* ≥ 1%

REV J: 03March2021

 $H_a$ : p < 1%

The statistical test of the null hypothesis for the primary safety endpoint is based on a one-sided, upper 95% confidence interval calculated by the method of Clopper and Pearson<sup>9</sup>:

$$B(0.95; x + 1, n - x)$$

Here x is the number of structural valve deteriorations occurring by the POD 390 visit, n is the number of patients completing the POD 390 visit, and B(0.95; x + 1, n - x) is the 95% upper quantile of the Beta distribution with parameters x + 1 and n - x. If the confidence interval above is less than 1%, then it will be concluded with 95% confidence that p is less than 1% and the acceptance criterion for the primary safety endpoint will be met. For the purposes of this hypothesis test, both aortic and mitral patients will be combined; however, results for the primary safety endpoint also will be reported separately for each implant position.

Based on a simulation, the power of the confidence interval above to reject the null hypothesis is greater than 80% for the sample size of 300 patients receiving the POD 390 visit. The simulation assumed for the purposes of power calculation a rate of SVD at the POD 390 visit of 0.05%; if a smaller rate is assumed, the power of the statistical test would of course be higher. The code for this simulation has been provided to FDA and is included in *Attachment O*.

# 9.3.1.2 PRIMARY SAFETY ENDPOINT (CONTINUED FOLLOW-UP):

For continued follow-up of Subjects, the primary safety endpoint for the trial is the rate of implanted subjects that experience structural deterioration of the trial valve as determined by a Clinical Events Committee (CEC). The linearized rate will be calculated as the number of late events divided by the total number of late-subject years. These results will be reported for both implant positions combined and separately for each position.

# 9.3.1.3 Secondary Safety Endpoints (Pre-approval)

The secondary safety endpoints listed in **Section 7.3.1** will be analyzed using the enrolled population. Early adverse events within 30 days of procedure will be reported as the number of events divided by the number of enrolled subjects. Linearized rates will be used to summarize adverse events for the late (>30 days) post-operative period. The linearized rates will be calculated as the number of late events divided by the total number of late-subject years. In addition, a one-sided upper 95% confidence limit will be calculated for the linearized rate.

The hypotheses for the secondary safety endpoints are:

REVISION J: 03 MARCH 2021 

DWARDS LIFESCIENCES LLC REV J: 03March2021


$$H_0: p \ge 2 \times OPC$$
 vs.  $H_A: p < 2 \times OPC$ 

where p is the complication rate for a given valve-related event. If the one-sided sided upper 95% confidence limit for p for a given secondary endpoint is less than  $2 \times OPC$  then the trial will be considered a success with regards to that secondary endpoint. These hypotheses will be tested based on the combined aortic and mitral populations; however the results will also be reported separately for each implant position.

Percentages for the early events and linearized rates for the late events also will be calculated for all other complications observed in the trial, including structural deterioration. These results will be reported for both implant positions combined and separately for each position.

Actuarial rates based on the method of Kaplan - Meier will be calculated for SVD and for each of the safety events in Section 7.3.1 at each of the follow-up time points; the number of subjects at risk for the event will be reported at each of these intervals. These results will be reported for both implant positions combined and separately for each position.

# 9.3.1.4 SECONDARY SAFETY ENDPOINTS (CONTINUED FOLLOW-UP):

For continued follow-up of Subjects, percentages for the early events and linearized rates for the late events also will be calculated for all other complications observed in the trial, including structural deterioration.

Actuarial rates based on the method of Kaplan - Meier will be calculated for SVD and for each of the safety events in Section 7.3.1 at each of the follow-up time points; the number of subjects at risk for the event will be reported at each of these intervals. These results will be reported for both implant positions combined and separately for each position.

#### 9.3.2 EFFECTIVENESS ANALYSIS

The following effectiveness endpoints will be analyzed using the investigational valve population. The analysis for valve performance will be performed separately for each implant position, and the analyses for NYHA Class and Quality of Life will be performed for both implant positions combined, separately for each position, and for isolated mitral valve replacement and mitral valve replacement with concomitant tricuspid valve repair.

# 9.3.2.1 VALVE PERFORMANCE

The following parameters will be summarized at baseline and at each follow-up visit for all subjects in the investigational valve population

CLINICAL INVESTIGATIONAL PLAN


Peak pressure gradient

Mean pressure gradient

Effective orifice area

Valvular regurgitation

Effective orifice area index

REV J: 03March2021

Performance index

Cardiac output

Cardiac index

Valvular regurgitation will be summarized by the number and percentage of subjects in each level of regurgitation. All other parameters will be summarized by N, mean, and standard deviation, and a 95% confidence interval. These summaries will be stratified by valve size.

9.3.2.2 NYHA CLASS

A comparison of preoperative and postoperative NYHA functional class (presented as the percentage of subjects in each class at baseline, at each follow-up time-point, and as the percentage of subjects at each follow-up time-point who improved, worsened, or did not change in class) will be presented. This comparison will be based on the investigational valve population. Additionally, a cross-tabulation of baseline vs. POD 390 NYHA will be presented for all subjects in the investigational valve population with both baseline and POD 390 NYHA data.

9.3.2.3 QUALITY OF LIFE

The N, mean and standard deviation for the SF-12 physical and mental health summary measures (PCS-12 and MCS-12, respectively) will be calculated for baseline and POD 390. In addition, the N and mean for the change from baseline to POD 390 in PCS-12 and MCS-12 will be presented with a 95% confidence interval. These summaries will be based on the investigational valve population.

9.4 ADDITIONAL MEASURES

9.4.1.1 BLOOD DATA

For all measured blood parameters, individual results will be compared to documented normal ranges. The Investigator will determine for each parameter that is out-of-range whether the value is not clinically significant and summary statistics will be provided.

Summary statistics (N, mean, and standard deviation) will be calculated preoperatively and postoperatively. In addition, the percentage of patient within the normal range preoperatively and postoperatively will be calculated. The percentage of patients within the normal range post-operatively will be reported separately for patients within and without the normal range preoperatively and for all patients combined.

Analyses of blood data will be performed for both implant positions combined and separately for each position.

#### 9.5 POOLABILITY

Subject baseline risk will be statistically compared between the regions (US, Canada, Europe and Asia Pacific) and among centers for the implanted population. Chi-square tests will be used to compare categorical risk factors while analysis of variance will be used to compare continuous risk factors. Comparisons will be based on the following demographic and pre-operative variables: age, sex, etiology, pre-operative NYHA, and concomitant CABG procedures, and any other baseline risk factors as deemed appropriate.

One-year Kaplan Meier estimates for the implanted population will be compared between the regions (US, Canada, Europe and Asia Pacific) and among sites for the following events: thromboembolism, valve thrombosis, major bleeding/ hemorrhage, all paravalvular leak, endocarditis, explant, and death. Estimates will be compared via a log-rank test. The primary safety endpoint will not be compared between regions or sites as it is expected that no structural valve deteriorations will be observed within the first year at any site or within any region.

#### 9.6 ANALYSIS OF COVARIATES

A hazard regression analysis will be performed to test for the effect of gender, age at implant, preoperative NYHA functional classification, previous valve surgery, concomitant coronary artery bypass surgery, implant position, and implant size on survival. This analysis will be performed by using a Cox proportional hazards model and will be based on the implanted population. Additionally, one-year Kaplan Meier estimates for each of the adverse events listed in the **Safety Endpoints Section 7.3.1** will be compared between the genders via a log-rank test.

Finally, the effect of gender on each of the following effectiveness endpoints at POD 390 (1 year) will be investigated with a linear regression model: peak gradient, mean gradient, effective orifice area (EOA) index. These linear regression models will be adjusted by BSA (to adjust for the effect of body size), implant position, and by valve size. The effect of gender on all valvular regurgitation at POD 390 (1 year) will be investigated via an ordinal logistic regression; this model also will be adjusted by BSA, implant position, and by valve size. All analyses will be based on the implanted population.

#### 9.7 MISSING DATA

All statistical tests on the effectiveness endpoints will be performed using only those subjects with available data required for endpoint analysis. No missing value imputation will be performed.

#### 9.8 FOLLOW-UP AND COMPLIANCE DATA

The number of valve population subjects followed to 390 days post-implant will be reported stratified by site and valve size; follow-up duration information, including mean follow-up, standard deviation and range of follow-up, and cumulative follow-up in subject-years will be reported for the valve population.

REVISION J: 03 MARCH 2021 

CLINICAL INVESTIGATIONAL PLAN


Subject compliance will be calculated and reported as the following four percentages: the number of

subjects a) having completed follow-up visits; b) with NYHA functional classification data; c) with

echocardiographic data; and d) with clinical laboratory results at each follow-up time-point, divided by

the total number of implanted subjects available (i.e., who have not died or had their valve explanted)

and eligible (i.e., who have reached the given time-point) for follow-up at that particular time-point.

Compliance will be reported for each follow-up visit and will be based on the investigational valve

population.

**10.0 TRIAL PROCEDURES** 

10.1 SUBJECT SCREENING

All subjects diagnosed with aortic or mitral stenosis, insufficiency or stenosis-insufficiency requiring valve

replacement as assessed by cardiac surgeons participating in this clinical trial, should be screened for

eligibility. All subjects who may meet eligibility requirements will be asked to participate.

A "Screening Log" is provided to the investigational sites to maintain a cumulative log of all screened

subjects. For subjects who are ineligible for participation in the clinical investigation, a reason supporting

the disqualification of the subject must be entered on the Screening Log. Sites are not required to enter

data into the EDC system for any preoperative or intraoperative screen failures. Any subject deemed

ineligible due to active or recent endocarditis/myocarditis, recent myocardial infarction, pregnancy or

lactation, or participation in another clinical investigation may be re-screened later. Re-screened subjects

must be re-entered on the Screening Log.

**10.2 INFORMED CONSENT** 

Written informed consent, in accordance with applicable international standards and trial center

regulations, shall be obtained from each subject, prior to the trial procedures. The investigator retains a

copy of the signed informed consent document in each subject's record, and provides a copy to the

subject.

The Investigator must obtain the written informed consent of all subjects, and must not allow any subject

to participate in the investigation prior to obtaining governing institutional review board (IRB), research

ethics board (REB) approval, or Ethics Committee (EC) approval. Before starting the trial, the investigator

provides trial Sponsor with a copy of the sample Informed Consent document approved by the IRB, REB,

or EC with documented evidence that the IRB, REB, or EC approved the protocol and the informed

consent.

Attachment C provides an example of a consent form submitted to each IRB, REB, or EC. The example

form contains the minimal consent language content that must be incorporated into the Informed

REVISION J: 03 MARCH 2021


REV J: 03March2021

Consent document. Other elements may be added or minor language changes may be made for clarity by the investigator or by the IRB/REB/EC, but substantial content may not be deleted.

#### 10.3 BASELINE ASSESSMENT

After a written informed consent is obtained from the subject, the following baseline data is obtained as noted in Table 3 below. This data includes physical assessment, demographic and medical history, 12-lead electrocardiogram (ECG), transthoracic echocardiogram (TTE) or transesophageal echocardiogram (TEE) per protocol, blood studies, an assessment of NYHA Functional Classification, CCS Angina Classification, an assessment of quality of life (QoL), and coagulation profile (via INR or PTT). Test results conducted within 60 days before planned valve surgery may be used for this trial if all values are available and are no significant changes in the subject's condition would invalidate the test results.

Table 3. Baseline Assessment

| Clinical/Physical Assessmen | t | Blood Studies | Echocardiography |
|---|---|---|---|
| Date of Assessment | Anti-thromboembolic | Blood Draw Date | Date of Exam |
| Date of Birth | Therapy | White Blood Cell Count | |
| Sex/Gender | (medications) | Red Blood Cell Count | |
| Height | Cardiovascular Risk Factors | Hemoglobin | REFER TO ECHO |
| Weight | Cardiovascular Conditions | Hematocrit | MANUAL |
| Heart Rate | Previous Procedures / | Platelet Count | |
| Blood Pressure | Interventions | Plasma Free Hemoglobin or | |
| Cardiac Rhythm (12-lead | Non-Cardiovascular | haptoglobin or serum LDH | |
| ECG) | Conditions | Serum Creatinine | |
| NYHA Classification | Pregnancy Test | Coagulation Profile | |
| CCS Angina Classification | | | |
| Quality of Life (SF-12) | | | |

#### 10.4 VALVE REPLACEMENT PROCEDURE

All procedures are performed in an operating room, or a surgical suite having cardiac surgery and anesthesia services. The surgical approach used is at the discretion of the Investigator's routine surgical practice. At the time of valve replacement, transesophageal echocardiography (TEE) is recommended to assess the subject's anatomy. After performing the aortotomy, the native valve and surrounding anatomy will be examined for compatibility with the investigational device.

**Note:** The Edwards Pericardial Bioprostheses, Models 11000A and 11000M do not require rinsing prior to implant. **Note:** If the valve is rinsed prior to implant, it must be kept hydrated with sterile physiological solution throughout the remainder of the surgical procedure. Rinsing every 1-2 minutes is recommended. **Caution:** Contact of the leaflet tissue with any articles or sources of particulate matter should be avoided.

Transesophageal echocardiography (TEE) should be performed within 1 hour after the bioprosthesis is implanted (from cross-clamp removal) to assess placement and bioprosthesis function. The echocardiography requirements may be found in *Attachment E*. A post-operative ECG or rhythm strip should also be performed upon arrival to the intensive care unit (ICU).

REVISION J: 03 MARCH 2021 

#### 10.4.1 SERUM GLYCEROL ANALYSIS

In order to obtain serum glycerol levels in a minimum of 100 subjects, the first 15 subjects enrolled at each of 8 sites will be evaluated. Two (2) blood samples for this assay will be collected from each of these subjects, one (1) pre-operatively (post-heparinization) and one (1) between 60 and 120 minutes after the heart has been restarted. The time that each sample is drawn will be recorded, as will the time the heart was restarted.

Samples will be appropriately labeled, frozen and shipped to the Glycerol Assessment Core Laboratory following the instructions provided in the Serum Glycerol Sample Collection Manual (*Attachment F*). Any subject who becomes an intra-operative screen failure will be replaced with next consecutively enrolled subject until up to 15 subject samples are achieved at each of the 8 sites.

Procedural information, findings, results and device identification information to be recorded are identified in Table 4.

Table 4. Procedural Information

| General Information | Clinical Information | Device Information |
|---|---|---|
| Date of Admission Date of Procedure Implanting Surgeon Type of Operation | Etiology Diagnosis for Replacement Valve Implant/ Valve Position Sizing Condition of the Native Valve | Valve Size and Serial Number Valve Performance Post-operative TEE (within 1 hour) REFER TO ECHO MANUAL |
| | Concomitant Procedures Intra-operative Adverse Events Post-operative Cardiac Rhythm upon arrival to ICU | |
| | *Blood collection for Glycerol Analysis<br>(See Section 10.4.1) REFER TO SERUM<br>GLYCEROL SAMPLE COLLECTION<br>MANUAL | |

#### 10.5 POST INDEX VALVE IMPLANT

At the discretion of the investigator, bioprosthetic heart valve recipients should be maintained on anticoagulant therapy (except when contraindicated) during the initial healing stage after implant, in accordance with the ACC/AHA 2006 Guidelines for the Management of Subjects with Valvular Heart Disease. However, the appropriate anticoagulation therapy must be determined by the physician on an individual basis.

# 10.6 DISCHARGE

The medical information and clinical evaluation of trial subjects prior to discharge is identified in Table 5. Subjects not discharged within 10 days post procedure, must have an echocardiogram to assess placement and performance of the index valve. This echocardiogram is required to complete the evaluation of short-term valve function. Those subjects will not require an additional echocardiogram at

REVISION J: 03 March 2021 


discharge.

Table 5. Discharge Information

| Clinical/Physical Assessment | Blood Studies | Echocardiography (TTE) |
|---|---|---|
| Date of Discharge | Blood Draw Date | Date of Exam |
| Weight | White Blood Cell Count | |
| Heart Rate | Red Blood Cell Count | REFER TO ECHO MANUAL |
| Blood Pressure | Hemoglobin | |
| Cardiac Rhythm (12-lead ECG) | Hematocrit | |
| Anti-thromboembolic Therapy | Platelet Count | |
| (medications) | Plasma Free Hemoglobin or | |
| Adverse Events | haptoglobin or serum LDH | |
| | Coagulation Profile | |

### 10.7 POST DISCHARGE FOLLOW-UP ASSESSMENTS

A summary of the tests and measurements to be conducted at screening, operatively, prior to discharge, and during follow-up are illustrated in the Clinical Trial Scheme in *Attachment A*.

A telephone follow-up visit is conducted at POD 30 (-5/+10 days) to document anti-thromboembolic therapy (medications), adverse events and determine NYHA and CCS Angina functional classification.

Post-procedure clinical evaluation is performed on all trial subjects at the investigational site. Information to be recorded at scheduled visits is further detailed in **Table 6**.

During each postoperative follow-up visit, the investigator(s) will determine the subject's availability for future follow-up visits. If any subject needs to be seen at a time other than a regularly scheduled follow-up visit, and the data will be recorded as an interim visit, and any applicable data pertinent to the visit will be collected. Coagulation profile is only required if collected per standard of care dependent on anticoagulation regimen (i.e. non-Vitamin K oral anticoagulants (NOAC's) do not require monitoring of coagulation profile).

Table 6. Follow-Up Information at all Post-Discharge Visits

| Clinical/Physical Assessment | Blood Studies | Echocardiography (TTE) |
|---|---|---|
| Date of Discharge | Blood Draw Date | Date of Exam |
| Weight | White Blood Cell Count | |
| Heart Rate | Red Blood Cell Count | REFER TO ECHO MANUAL |
| Blood Pressure | Hemoglobin | |
| Cardiac Rhythm (12-lead ECG) | Hematocrit | |
| NYHA Classification | Platelet Count | |
| CCS Angina Classification | Plasma Free Hemoglobin or | |
| Quality of Life (SF-12)* | haptoglobin or serum LDH | |
| Anti-thromboembolic Therapy | | |
| (medications) | Coagulation Profile** | |
| Adverse Events | | |

<sup>\*</sup>Conducted only at the POD 390 visit \*\*Only required if collected per standard of care dependent on anticoagulation regimen

REVISION J: 03 March 2021 
EDWARDS LIFESCIENCES LLC REV J: 03March2021

CLINICAL INVESTIGATIONAL PLAN


All efforts should be taken by the Investigator and the research staff to encourage subjects to return for required follow-up visits. If a subject cannot return for follow-up visits, all attempts will be made to collect the protocol-specified data from outside hospitals or clinics. For echocardiography exams performed outside of the trial site, a copy of the Core Laboratory Procedure Manual is provided in **Attachment E** to

ensure compliance with the echocardiography requirements.

10.8 MISSED FOLLOW-UP

The Investigator(s) will make every attempt to follow the subjects. All subjects will be encouraged by the Investigator(s) to report any address or telephone number changes to the trial site. They are informed of

the importance of returning for scheduled follow-up visits even if they are not having any medical issues.

If a subject cannot be reached for a follow-up visit, the Investigator will document on the CRF, the efforts undertaken to contact the subject or the subject's primary health care provider. These efforts should include three (3) attempts of telephone contact at separate dates and times, and a registered letter sent before the end of the follow-up window (telephone attempts may include a family member if available). If a subject cannot be reached for a follow-up visit, or misses a scheduled visit, the visit will be recorded as a missed visit on the date of last attempted contact. Subjects who miss a visit will not be considered withdrawn. At the next visit interval, the Investigator and/or designee will make three (3) attempts of telephone contact at separate dates and times, and a registered letter sent before the end of the follow-up window (telephone attempts may include a family member if available). Subjects who miss two (2) sequential follow-up visits will be considered lost to follow-up at the second missed visit and exempt from

further trial follow-up. After the subject is terminated from the trial, the Investigator will attempt to

determine if the subject is alive, including searching national mortality registries as permitted by local

laws.

Trial Subjects exit the trial when no additional follow-up visits, procedures, or data collection are required. A subject is exited from the trial in the following instances:

· Fails enrollment criteria after written consent

• Is Lost-to-follow-up (LTFU)

Voluntarily withdraws from the trial

Death

• Explant or valve-in-valve (ViV) intervention (after 30 days for safety endpoints only; or after adverse events from explant/ViV are resolved, whichever comes later)

• Does not retain trial valve after attempt to implant (after 30 days for safety endpoints only; or after adverse events from explant are resolved, whichever comes later)

Completes last trial follow-up visit (at POD 1825 or POD 3650 for Continued Follow-Up Subjects)

Investigator withdraws the subject from the trial

# 10.9 DEVICE REMOVAL OR EXPLANT

Index valve 'removal' is the excision of the investigational valve, before implant of the investigational valve is complete, i.e., the subject does not leave the OR with the investigational valve. If the surgeon is unable to satisfactorily position or sew in the index valve, it will be removed and returned to the trial Sponsor who will provide a return valve kit. If the subject leaves the OR with the investigational valve in place, the valve will be considered implanted and if removal is required from this point forward, it will be considered an explant.

In the event a valve is explanted/ requires a valve-in-valve intervention, a copy of the procedure report must be provided to the trial Sponsor. Information on the cause of explant and its relationship to the valve will be provided by the investigator(s). Explanted valves must be returned to the trial Sponsor for analysis. Return kits for devices will be provided by the trial Sponsor.

# 11.0 ADVERSE EVENTS

# 11.1 REPORTING

Adverse event information is reported throughout the clinical investigation. Adverse events are followed until they are adequately resolved. A list of potential adverse events, which may result from the trial procedure, are included in the Risk Section 6.2, the Instructions for Use (IFU) in **Attachment C**, and further defined in **Attachment G**.

# 11.1.1 UNANTICIPATED ADVERSE DEVICE EFFECT

An *unanticipated adverse device effect (UADE)* is any serious adverse effect on health or safety or any life threatening problem or death caused by or associated with the device, if that effect, problem, or death was not previously identified in nature, severity, degree of incidence in this Investigational Plan. Additionally, an unanticipated adverse event includes any other unanticipated serious problem associated with the device that relates to the rights, safety, or welfare of subjects.

Investigator(s) are required to submit to the reviewing IRB/REB/EC and the trial Sponsor a report of any *unanticipated adverse device effect (UADE)* occurring during this investigation as soon as possible, but in no event later than two (2) business days after the investigator(s) first learns of the effect (21CFR 812.150(a)(I)). The trial Sponsor must immediately conduct an evaluation of an UADE, and must report the results of the evaluation to FDA, all reviewing IRB/REB/ECs, and participating investigators within ten (10) business days after the trial Sponsor first receives notice of the effect (21CFR 812.46(b), 812.150(b)(I)).

If it is determined that an UADE occurred, the trial Sponsor will notify the Data Monitoring Committee (DMC) within five (5) business days after the trial Sponsor or its designee first receives notice of the event. If the trial Sponsor and/or the DMC determines an event or event rate presents an unreasonable risk to a

REVISION J: 03 March 2021 

**EDWARDS LIFESCIENCES LLC** 

CLINICAL INVESTIGATIONAL PLAN


subject, all investigations or parts of investigations presenting that risk are terminated, as soon as

REV J: 03March2021

possible. Termination of the investigation shall occur no later than five (5) working days after the trial

Sponsor makes this determination and no later than fifteen (15) days after trial Sponsor or its designee

first receives notice of the event.

11.1.2 ADVERSE DEVICE EFFECTS

An adverse event is any undesirable experience associated with the use of a medical product in a patient.

The event is serious and should be reported to FDA (and other relevant regulatory agencies) when the

subject outcome is/led to:

Death

Life-threatening

Hospitalization or prolonged hospitalization

Disability or permanent damage

• Congenital Anomaly or birth defect

• Intervention to prevent permanent impairment or damage

Other serious or important medical events – medical or surgical intervention to prevent one of

the above outcomes

.

Investigational sites report all applicable serious adverse events in accordance with the reviewing

IRB/REB/EC committee's requirements.

Trial Sponsor or its designee determines reportability of applicable adverse events according to its

responsibilities for European vigilance reporting.

11.2 NOTIFICATION OF UADE AND/OR SERIOUS DEVICE RELATED ADVERSE EFFECTS

Notification of UADE and serious device related adverse effects should be done via email to

<u>HVTClinicalResearch@edwards.com</u> or faxed to 949-809-5610.

11.3 DEATH AND EXPLANTS

In the event of subject death, every effort should be made to obtain a copy of the autopsy report and/or

death summary. Information on the cause of death and its relationship to the device used in this clinical

trial will be determined by the investigator(s). Copies of an autopsy report, if available, and/or a death

summary are to be sent to the trial Sponsor.

If a device is explanted during autopsy, the device should be returned to the trial Sponsor for analysis.

Return kits for devices will be provided by the trial Sponsor.

REVISION J: 03 March 2021 


REV J: 03March2021

11.4 DATA MONITORING COMMITTEE

The trial Sponsor will appoint a Data Monitoring Committee (DMC) composed of two or more independent

physicians including a cardiothoracic surgeon and a cardiologist, and a statistician. Members of the DMC

will not have scientific, financial, or other conflict of interest related to the trial Sponsor or the

Investigators. Curricula Vitae for the DMC members are maintained by the trial Sponsor, and are available

for regulatory review. These individuals may not participate in this trial as investigators, and may not hold

significant material, financial or other interests, which create a potential conflict with respect to this role.

DMC members must sign a non-conflict-of-interest statement in this regard.

The primary purpose of the DMC is to ensure a consistent, independent review of events and their clinical

significance using standardized criteria and definitions. The DMC will be tasked with identifying any issues

such as higher than expected AE and/or death rates, UADEs or hemodynamic performance that is

substantially worse than expected, to determine if the trial should be stopped, suspended, or modified at

any time. The DMC will establish guideline criteria for recommending trial termination.

The DMC will meet at least yearly or more often as determined by the Chairperson and possibly on an ad

hoc basis to evaluate trial progress and results during the enrollment phase. The Chairperson of the DMC

will be informed of all UADEs within five (5) business days of these events being reported to the trial

Sponsor or its designee. This requirement, in addition to the guideline criteria for recommending trial

termination, will be incorporated into the DMC charter.

11.5 CLINICAL EVENTS COMMITTEE

The Clinical Events Committee (CEC) evaluates adverse events that are endpoint related. The CEC

adjudicates events for their relatedness to the investigational device and/or the surgical procedure. The

CEC will be composed of physicians familiar with the treatment of valvular heart disease and cardiac

surgery and who are not participating in the investigational trial.

The trial Sponsor will provide the CEC completed case report forms and any relevant source

documentation/subject information as provided by the clinical site investigators. The trial Sponsor will

insure that all information is de-identified before presenting to the committee. The CEC documents its

findings or rulings on each event. All meeting minutes and supporting documentation are maintained by

the CEC administrator with a copy provided to the trial Sponsor.

REVISION J: 03 MARCH 2021 

# 12.0 TRIAL AND DATA MANAGEMENT

# 12.1 TRIAL CORE LABS

# 12.1.1 ECHOCARDIOGRAPHY CORE LAB

The Echocardiography Core Lab is responsible for independently evaluating echocardiograms submitted preoperatively and postoperatively by trial sites, and for reporting of hemodynamic and other valvular function results. The purpose of the Echocardiography Core Lab is to ensure unbiased, timely and consistent analysis of the diagnostic data, and for evaluating changes in subject status over the course of the trial based on serial echocardiographic studies conducted on the same subject.

Personnel at the Echocardiography Core Lab must demonstrate appropriate training and experience for analyzing Doppler Echocardiography data. The trial Sponsor or its designee periodically will audit the Echocardiography Core Lab. Echocardiograms will be sent directly from the investigational sites to the Echocardiography Core Lab. The Echocardiography Core Lab reviews the Doppler echocardiograms upon receipt, and promptly notifies the site and the trial Sponsor if the quality of the echocardiograph is insufficient for analysis. The Echocardiography Core Lab will enter the data into the eCRF. See Attachment **E** for the Core Laboratory Procedure Manual.

# 12.1.2 GLYCEROL ASSESSMENT CORE LAB

The Glycerol Assessment Core Lab is responsible for independently analyzing all blood samples collected for measurement of serum glycerol. The purpose is to ensure unbiased, timely and consistent analysis of the data. See **Attachment F** for the Serum Glycerol Sample Collection Manual.

# 12.2 DEVICE ACCOUNTABILITY

An initial set of Edwards Pericardial Bioprostheses Models 11000A and/or 11000M, is shipped to the clinical site once the following conditions are met: the site obtained regulatory approval (Institutional Review Board, Ethics Committee approval or Research Ethics Board), a signed Clinical Trial Agreement is in place, and the Site Initiation Visit, including Principal Investigator training, is complete. Additional devices are sent to the clinical site as devices are used or as needed.

# 12.2.1 INVENTORY AND ACCOUNTABILITY RECORDS

A Device Accountability Log is maintained by the Investigator noting all investigational devices received for use during this clinical trial. The log is kept with the documents for the clinical trial and is available for review during trial Sponsor monitoring visits.

All device shipments include inventory and shipment records (packing slip). The Principal Investigator or designee will take inventory of the product, note the condition of the device, and attest to accuracy of the valve shipment by signing the packing slip. Both the investigational site and the trial Sponsor retain copies of the packing slips and the Device Accountability Log.

REVISION J: 03 MARCH 2021  12.2.2 DEVICE STORAGE

The device inventory is to be stored in a locked, controlled, cool, dry and clean area. This storage area

shall be accessible only to the Principal Investigator(s), Co-Investigator(s) or approved designee(s). Only

cardiac surgeons identified in the Clinical Trial Agreement and/or on the Delegation of Authority form on

file may implant the investigational device.

12.2.3 DEVICE RETURN

The Principal Investigator(s) is notified in writing upon termination of the clinical trial. All unused devices

in original package and/or those in opened packages will be returned upon receipt of this notice as

described in the IFU. The Investigator's copy of the Device Accountability Log must document any unused

devices that are returned. The trial Sponsor will provide shipping instructions.

12.3 PROTOCOL DEVIATIONS

A protocol deviation is defined as an event where the Investigator or trial personnel did not conduct the

trial according to the clinical protocol or the Clinical Trial Agreement.

Deviations shall be reported to the trial Sponsor regardless of whether medically justifiable or taken to

protect the subject in an emergency. Subject specific deviations and non-subject specific deviations, (e.g.

unauthorized use of a trial device outside the trial, unauthorized use of a trial device by a physician who

is not listed in the Clinical Trial Agreement, etc.) will be reported in writing. Investigators will adhere to

procedures for reporting trial deviations to the IRB/EC/REB in accordance with their specific reporting

policies and procedures.

For reporting purposes, deviations are classified as major or minor:

• Major deviations – will be reported to the trial Sponsor within 48 hours but no later than 3 business

days of awareness of the major deviation and document on the appropriate case report form

provided; and to the IRB/REB/EC per their guidelines

Any deviation from subject inclusion and exclusion criteria

Any deviation from subject informed consent procedures

Unauthorized use of an investigational device outside the trial

Unauthorized use of an investigational device by a physician who is not listed in the Clinical Trial

Agreement

• Minor deviations – will be reported to the trial Sponsor in writing on the appropriate form provided

Deviation from a protocol requirement such as incomplete/inadequate testing procedures;

Follow-up performed outside specified time windows in the protocol

NOTE: Information that is not essential to the trial endpoints is not considered a deviation if absent.

REVISION J: 03 MARCH 2021 

# 12.4 TRIAL SITE INITIATION AND MONITORING PLAN

## 12.4.1 SITE INITIATION AND TRAINING

Site staff will be trained and experienced to perform their delegated tasks. Training may be in person, webinar, read and review, or other methods as deemed appropriate.

REV J: 03March2021

Training is documented on a "Training Log". A "Delegation of Authority Form" is completed at each site designating which individuals are allowed to perform specific clinical trial related tasks. The delegated tasks will determine what the training requirements are for each member of the trial support staff.

New research staff members may be trained by previously trained personnel on the Delegation of Authority Form.

## 12.4.2 MONITORING

Written procedures have been established by the trial Sponsor for monitoring clinical investigations, to assure the quality of the trial and to assure that each person involved in the monitoring process carries out his or her duties. Standardized written procedures, sufficiently detailed to cover the general aspects of clinical investigations, will be used as a basic monitoring plan and will be supplemented by more specific / additional procedures specific to this clinical investigation.

A pre-trial monitoring visit or meeting will be conducted to ensure that the Investigator clearly understands and accepts the obligations incurred in undertaking the clinical investigation as listed in **Table** 7 (Regulations and Guidelines), and that the facilities are acceptable. Periodic monitoring visits will be conducted with adequate frequency to ensure that the Investigator's obligations as set forth in 21 CFR Part 56 and 21 CFR Part 812 are being fulfilled and that the facilities continue to be acceptable.

The trial Sponsor will assign a monitor to oversee the progress of the clinical investigation at each investigational center. The monitor will remain in close contact with each investigational center throughout the duration of the investigation to provide any needed materials, (i.e., investigation forms) and answer any questions. The monitor will be responsible for verifying that the subject signed the consent, reviewing all data recorded on the eCRFs, and visiting each investigational center periodically to observe trial progress and compliance with clinical protocol and regulations applicable to this clinical investigation. Additionally, the monitor will provide assurance that complete records are being maintained, appropriate timely reports are made to the trial Sponsor and IRB/REB/EC, device inventory is controlled, and that the Investigator is carrying out all agreed upon activities. Any personnel changes must be reported to the monitor immediately and a training program must be scheduled and documented. A trial termination monitoring visit will be conducted at the completion of the clinical trial to ensure that all data are properly documented and reported.

REVISION J: 03 March 2021 

REV J: 03March2021

CLINICAL INVESTIGATIONAL PLAN


Site Termination: If a clinical monitor becomes aware that an Investigator is not complying with the signed

Investigator's Agreement, the Investigational Plan, the requirements of applicable health authority

regulations, or any conditions of approval imposed by the reviewing IRB/REB/EC or health authority, trial

Sponsor will immediately either secure compliance or terminate the Investigator's participation in the

trial. The final action will be taken with the goal of assuring the rights, safety and welfare of the patients.

12.5 DOCUMENTATION REQUIREMENTS

12.5.1 SOURCE DOCUMENTS

Clinical regulations require that Investigators maintain information in the clinical trial subject's medical

records that corroborate data collected on the eCRF. Some examples of critical information to be

maintained for review by the regulatory inspectors and trial Sponsor monitors are:

Medical history and physical condition of the clinical trial subject before involvement in the clinical

trial sufficient to verify protocol entry criteria

Dated and signed notes in the subject's medical record on the day of entry into the clinical trial

Dated and signed notes, laboratory records, and test reports, from each clinical subject visit with

reference to the eCRF for further information, if appropriate (for specific results of procedures

and exams).

Notations on abnormal lab results, adverse events reported and their resolution

Notes regarding concomitant anticoagulant/antithrombotic medications taken during the clinical

trial

Subject's condition upon completion of or withdrawal from the clinical trial.

To protect subject confidentiality, the subject's name must not appear anywhere on the imaging media

sent to trial Sponsor e.g. for reporting serious adverse device effects (SADE), or prepared for evaluation

by the core lab. Each page should be identified with the subject's unique trial ID number. All other subject

identifiers (i.e. medical record number, personal number) are to be obscured. Original copies of all data

must be kept at the site.

Site monitoring will include 100% primary source verification of events contributing to the safety and

effectiveness endpoints and unanticipated adverse device effects (UADE).

12.5.2 TRIAL DOCUMENTS

The trial Sponsor will provide pre-printed forms to each trial site for documentation of:

Investigator and site training to the protocol (Training Log)

Authorized trial site personnel (Delegation of Authority)


EDWARDS LIFESCIENCES LLC

CLINICAL INVESTIGATIONAL PLAN


Subject consent and screening (Screening and Enrollment Log)

Monitoring visit tracking (Site Visit Log)

Investigational Device Accountability (Investigational Device Accountability Log)

The site visit is recorded on the appropriate site visit report. All tasks and action items noted during the visit should be documented with detailed findings and comments provided as appropriate. The monitor provides a visit follow-up letter to the investigator and other appropriate trial staff briefly summarizing the visit and specifically addressing any outstanding issues and/or action items from the visit, any incidents of noncompliance with the protocol or applicable regulations noted during the visit, and any necessary corrective actions.

REV J: 03March2021

During the course of the clinical trial, all correspondence (letters, records of telephone calls, emails and faxes) regarding the trial must be maintained in the regulatory binder provided by the trial Sponsor. This binder must be made available for monitoring visits and audits.

12.6 DATA COLLECTION

All required data for this trial are to be collected with standardized Case Report Forms (CRF) for individual subjects; the eCRF outline is included in *Attachment D*. Electronic CRF (eCRF) will be utilized for this trial. Each eCRF must be signed electronically by the Principal Investigator listed in the Clinical Trial Agreement and Delegation of Authority Log. If for any reason an eCRF is unavailable and/or inaccessible, a paper CRF will be provided by the trial Sponsor to be completed, signed by the Principal Investigator or designee and submitted to the trial Sponsor.

Case Report Form Instructions will be provided to assist the Investigator(s) and appropriate trial staff with the completion of each required eCRF.

The Sponsor's data management group is responsible for database development, validation, control and management of input from each monitored CRF, issuance and resolution of queries, database maintenance, and statistical support. Data Management personnel will employ a full-featured relational Oracle database application (or equivalent) on a central server that is 21 CFR Part 11 compliant. The application provides the capability of data collection remotely through the Internet so the participating site personnel may log on to the system securely and enter the data. Other data management programming and/or data analyses will be done in the database system through the trial Sponsor's internal network.

12.7 DATA AND DOCUMENT RETENTION

Trial-related correspondence, subject records, consent forms, records of device implant, and source document worksheets are to be maintained on file by the trial site. The trial Sponsor requires that it be notified in writing if the Principal Investigator wishes to relinquish ownership of the data and information

REVISION J: 03 MARCH 2021 

**EDWARDS LIFESCIENCES LLC** 

CLINICAL INVESTIGATIONAL PLAN


so that mutually agreed upon arrangements can be made for transfer of ownership to a qualified entity.

REV J: 03March2021

Per FDA regulation 21 CFR 812.140, records of each subject's participation in the trial must be maintained

for a period of two (2) years after trial closure and submission of the final report to the IRB/REB/EC.

12.8 TRIAL PROTOCOL AMENDMENTS

Changes in the protocol are made only by written amendment agreed upon by the trial Sponsor, the

applicable regulatory agency, including the United States Food and Drug Administration, and if pertinent,

the IRB/REB/EC. As appropriate, the trial Sponsor will submit changes in the protocol to the applicable

regulatory agencies, including the United States Food and Drug Administration and investigators to obtain

IRB/REB/EC re-approval. A report of withdrawal of IRB, REB or EC approval must be submitted to the trial

Sponsor within five (5) business days. Any revisions to the protocol, including the Informed Consent Form

and the Case Report Forms, other than very minor revisions must be approved by trial Sponsor, the

IRB/EC/REB and the FDA and/or other regulatory agencies.

12.9 TRIAL COMPLETION

The principal investigator will be notified in writing upon termination/conclusion of the clinical trial. The

trial Sponsor retains the right to suspend or terminate this clinical trial at any time.

A final clinical report shall be compiled once data collection is complete. Such reports include all

information required and outlined in this protocol. The final report will be provided to regulatory agencies

and/or institutional review boards/independent ethics committees and other regulatory agencies as per

applicable laws. The final clinical report will be filed in the clinical trial master file.

**12.10 FUTURE PLANS** 

No changes are planned at this time.

13.0 STATEMENTS OF COMPLIANCE, CONFIDENTIALITY AND RESPONSIBILITIES

13.1 GOOD CLINICAL PRACTICE STATEMENT

This trial will be conducted in compliance with all applicable US Federal regulations pertaining to

investigational devices including but not limited to: 21 CFR Part 50, Part 54, Part 56, Part 812, Good Clinical

Practice (GCP) standards, and Health and Insurance Portability and Accountability Act (HIPAA). The

protocol and supporting documents for this trial will be reviewed and approved by an appropriately

constituted IRB, REB or EC prior to trial initiation. All reviews and approvals will be in accordance with

Good Clinical Practice (GCP) and all other applicable standards, regulations (local and national), guidelines

and institutional policies.

REVISION J: 03 March 2021 

#### REV J: 03MARCH2021

# 13.1.1 PROTECTION OF SUBJECT CONFIDENTIALITY

Subject confidentiality will be maintained in accordance with GCP, the HIPAA and all other applicable standards, regulations (local and national), guidelines and institutional policies.

# 13.2 REGULATIONS AND GUIDELINES

The regulations listed in **Table 7** must be observed to comply with the trial Sponsor's policy for conduct of clinical studies; they represent good clinical practice. It is the responsibility of the investigator(s) to comply with the requirements set forth in their country specific regulations.

Table 7. Regulations and Guidelines

| Country or Region | Regulation / Guideline |
|---|---|
| US | <ul> <li>Investigational Device Exemption (IDE), 21 CFR Part 812</li> <li>Institutional Review Board (IRB), 21 CFR Part 56</li> <li>Protection of Human Subjects, 21 CFR Part 50</li> <li>Financial Disclosure, 21 CFR part 54</li> <li>Draft Guidance for Industry and FDA Staff - Heart Valves – Investigational Device Exemption (IDE) and Premarket Approval (PMA) Applications, January 20, 2010</li> </ul> |
| Europe | <ul> <li>93/42/EEC European Medical Device Directive (MDD)</li> <li>ISO 14155:2011 (Clinical Investigation of Medical Devices for Human Subjects)</li> <li>ISO 5840:2009 (Cardiovascular implants-Cardiac valve prostheses)</li> <li>Declaration of Helsinki (2008)</li> </ul> |
| Canada | <ul> <li>Canadian Medical Device Regulations (CMDR)</li> <li>Canadian Investigational Testing Authorization as defined in the Medical Devices<br/>Regulation, May 1998</li> </ul> |
| Asia<br>Pacific | - Regional requirements will be added in an Appendix as required. |

# 13.3 INVESTIGATOR RESPONSIBILITIES

The trial Investigator(s) will adhere to the trial protocol, Good Clinical Practice, HIPAA, and compliance with applicable government and institutional regulations. The trial Investigator(s) is responsible for obtaining proper regulatory approvals, and reporting to regulatory authorities per all applicable regulations. *Attachment J* provides a comprehensive list of Investigator(s) responsibilities.

# 13.4 SPONSOR RESPONSIBILITIES

The trial Sponsor will adhere to the trial protocol, Good Clinical Practice, HIPAA, and compliance with applicable government and institutional regulations. The trial Sponsor is responsible for obtaining proper regulatory approvals, and reporting to regulatory authorities per all applicable regulations. *Attachment J* provides a comprehensive list of trial Sponsor responsibilities.

REVISION J: 03 March 2021 

# 14.0 PUBLICATIONS

Edwards Lifesciences, as the trial Sponsor of record, has a proprietary interest in this trial. Authorship and manuscript composition will reflect cooperation between multiple investigators and sites, core laboratories, and Edwards Lifesciences. Authorship will be established prior to writing of the manuscript. No individual publications will be allowed prior to the completion of the final report for this trial and as agreed in writing by Edwards Lifesciences.

# 15.0 REFERENCES

- 1. Rosenhek R, Binder R, Porenta G et al. Predictors of outcome in severe asymptomatic aortic stenosis. *N Engl J Med* 2000; 343(9): 611-7.
- 2. Waller BF, Howard J, Fess S. Pathology of mitral valve stenosis and pure mitral regurgitation, part I. *Clin Cardiol* 1994; 17:330.
- 3. Waller BF, Howard J, Fess S. Pathology of mitral valve stenosis and pure mitral regurgitation, part II. *Clin Cardiol* 1994; 17:395.
- 4. Edward NR et al. Mitral valve repair and replacement in northern New England. *American Heart Journal* 2003; 145(6): 1058-1062.
- 5. Horstkotte D, Loogen F. The natural history of aortic valve stenosis. *Eur Heart J Supp E* 1998; 57-64.
- 6. Carpentier A. Cardiac valve surgery. The French Correction. *J Thorac Cardiovasc Surg* 1983; 86: 323-37.
- 7. Carpentier A. Carpentier's Reconstructive Valve Surgery. Maryland Heights: Saunders, 2010.
- 8. Craver JM. Aortic valve debridement by ultrasonic surgical aspirator: A word of caution. *Ann Thorac Surg* 1990; 49: 746-52.
- 9. Clopper, C.; Pearson, E. S. (1934). "The use of confidence or fiducial limits illustrated in the case of the binomial". *Biometrika* **26**: 404–413.

REVISION J: 03 March 2021 

EDWARDS LIFESCIENCES LLC
CLINICAL INVESTIGATIONAL PLAN


**ATTACHMENTS** 

# ATTACHMENT A - CLINICAL TRIAL SCHEME

REVISION J: 03 MARCH 2021

# **CLINICAL TRIAL SCHEME**

| Schedule of Tests: | Baseline | Procedure<br>(Day 0) | Discharge | 30 Days<br>(Phone) | 105 Days | 390 Days | 730-3650<br>Days <sup>7</sup> |
|---|---|---|---|---|---|---|---|
| Signed Informed Consent | Х | | | | | | |
| Physical Exam <sup>1</sup> | Х | | Х | | Х | Х | Χ |
| Medical History <sup>2</sup> | Х | | | | | | |
| Blood Labs <sup>3</sup> | Х | Х | Х | | Х | Х | Х |
| ECG | Х | Х | Х | | Х | Х | Χ |
| Echocardiogram <sup>4</sup> | Х | Х | Х | | Х | Х | Χ |
| NYHA Class/ CCS Angina Class | Х | | | Х | Х | Х | Χ |
| QOL Questionnaire (SF-12 v2) | Х | | | | | Х | |
| Coagulation Profile <sup>5</sup> | Х | | Х | | Х | х | Χ |
| Anti-thromboembolic<br>Therapy & Medications | х | | x | Х | Х | Х | Х |
| Pregnancy Test <sup>6</sup> | Х | | | | | | |
| Adverse Events | | Х | Х | Х | Х | Х | Х |

<sup>&</sup>lt;sup>1</sup> Physical exam: height, weight and vital signs [BP, HR].

Serum glycerol is only required at the procedure interval (See Section 10.4.1).

- <sup>4</sup> TTE will be the standard echocardiography assessment for the aortic or mitral valve. TEE intra-operatively or within 1 hour (from cross clamp removal) to confirm placement of the device and confirm initial function of the valve.
- <sup>5</sup> Coagulation profile will be determined for subjects on anticoagulant therapy only, where coagulation profile is collected per standard of care. Non-Vitamin K oral anticoagulants (NOACs) that do not require monitoring of coagulation profile, for example, will not require collection/reporting of coagulation profile.
- <sup>6</sup> Applicable only to females of child bearing age.
- All IDE subjects to be followed to POD 1825 (5 yrs). All Subjects implanted with the Model 11000A or Model 11000M valve who have consented to continued follow-up will be followed annually through 10 years post-procedure.

<sup>&</sup>lt;sup>2</sup> Includes cardiovascular & non-cardiovascular conditions, prior cardiac interventions and surgeries.

<sup>&</sup>lt;sup>3</sup> Blood labs: CBC [RBC, WBC, Hgb, HCT, PLT], plasma free hemoglobin or haptoglobin or serum LDH; Serum creatinine is required only at baseline.

**EDWARDS LIFESCIENCES LLC**CLINICAL INVESTIGATIONAL PLAN

# **ATTACHMENT B – INSTRUCTIONS FOR USE**

REVISION J: 03 MARCH 2021

| DIRECTORY | |
|-----------|----|
| English | 1 |
| Français | 13 |
| Polski | 26 |

#### English

# Edwards Pericardial Aortic Bioprosthesis, Model 11000A

# Instructions for use

CAUTION: Investigational device. Limited by Federal (United States) law to investigational use.

CAUTION: Investigational device. Exclusively for Clinical Investigations.

Caution: Investigational Device. Limited to Investigational Use. To be used by Qualified Investigators (Physicians).

#### 1. Device and Accessories Description

#### 1.1 Device Description

The Edwards Pericardial Aortic Bioprosthesis, Model 11000A, is a trileaflet bioprosthesis comprised of treated bovine pericardium that is mounted on a flexible frame. It is available in sizes 19, 21, 23, 25, 27, and 29 mm (Table 1). The bioprosthesis is stored in non-aqueous packaging, and does not require rinsing prior to implantation.

| Table 1. Nominal Dimensions | | | | | | |
|---|---|---|---|---|---|---|
| A HVT48 | | | | | | |
| Size | 19 21 23 25 27 29<br>Size mm mm mm mm mm mm mm | | | | | |
| A. Tissue Annulus Diameter<br>(Stent Diameter, mm) | 19 | 21 | 23 | 25 | 27 | 29 |
| B. Internal Diameter<br>(Stent ID, mm) | 18 | 20 | 22 | 24 | 26 | 28 |
| C. Profile Height (mm) | 13 | 14 | 15 | 16 | 17 | 18 |
| D. External Sewing Ring<br>Diameter (mm) | 24 | 26 | 28 | 30 | 32 | 34 |
| Geometric Orifice Area (mm²) | 235 | 289 | 354 | 420 | 499 | 570 |

The wireform is made of a cobalt-chromium alloy and is covered with a woven polyester fabric. A cobalt-chromium alloy/polyester film laminate band surrounds the base of the wireform frame

A silicone sewing ring that is covered with a porous polytetrafluoroethylene (PTFE) doth is attached to the wireform frame. The sewing ring has three, equally spaced black silk suture markers at the cusp centers to aid in bioprosthesis orientation and suture placement.

A holder is attached to the bioprosthesis by means of sutures to facilitate handling and suturing the bioprosthesis during implantation. The holder is easily detached by the surgeon. (See 10.4 Device Implantation)

#### 1.2 Accessories Description

#### Sizers and Trav

The use of a sizing instrument facilitates selection of the correct size bioprosthesis for implantation. The translucent Model 1133 sizers permit direct observation of their fit within the annulus. Each sizer consists of a handle with a different sizing configuration at each end (Figure 1a). On one side of the handle is a cylindrical end with an integrated lip that reflects the bioprosthesis sewing ring geometry (Figure 1b). On the other side of the handle is a bioprosthesis replica end that reflects the bioprosthesis sewing ring geometry as well as the height and location of the stent posts (Figure 1c). A sizer is available for each size of the Model 11000A bioprosthesis (19, 21, 23, 25, 27, and 29 mm). The complete set of sizers is housed in a tray, Model TRAY1133, which can be reused and resterilized.

Edwards Lifesciences, the stylized E logo, Edwards, Carpentier-Edwards, ThermaFix, TFX, PERIMOUNT, PERIMOUNT Magna and Magna Ease are trademarks of Edwards Lifesciences Corporation.

Figure 1a. Aortic Sizer



Figure 1b. Cylindrical End

Figure 1c. Replica End



#### **Bioprosthesis Holder and Handle**

The handle/holder assembly consists of two components: an integral disposable part that is physically mounted to the bioprosthesis by the manufacturer and a malleable handle (reusable Model 1111 or disposable Model 1126 for single use) that is attached to the holder at the time of surgery (Figures 2a and 2b).

Figure 2a. Model 1111 Handle



Figure 2b. Model 1126 Handle



#### 2. Indications for Use

The Edwards Pericardial Aortic Bioprosthesis, Model 11000A, is indicated for patients who require replacement of their native or prosthetic aortic valve.

#### 3. Contraindications

Do not use the bioprosthesis if the surgeon believes use is contrary to the best interests of the patient. The decision for or against use of this bioprosthesis remains with the surgeon who must evaluate all the various risks involved, including the anatomy and pathology observed at the time of surgery.

#### 4. Warnings

FOR SINGLE USE ONLY. This device is designed, intended, and distributed for single use only. Do not resterilize or reuse this device. There are no data to support the sterility, non-pyrogenicity, and functionality of the device after sterile reprocessing.

DO NOT FREEZE OR EXPOSE THE BIOPROSTHESIS TO EXTREME HEAT. Exposure of the bioprosthesis to extreme temperatures will render the device unfit for use.

#### DO NOT USE the bioprosthesis:

- If the foil pouch, sealed trays, or lids are opened, damaged, or stained
- If the expiration date has elapsed, or
- If it is dropped, damaged, or mishandled in any way. Should a bioprosthesis be damaged during insertion, do not attempt repair.

DO NOT EXPOSE the bioprosthesis to any solutions, chemicals, antibiotics, etc., except for sterile physiological saline solution. Irreparable damage to the leaflet tissue, which may not be apparent under visual inspection, may result.

DO NOT GRASP the leaflet tissue of the bioprosthesis with instruments or cause any damage to the bioprosthesis. Even the most minor leaflet tissue perforation may enlarge in time to produce significant impairment of bioprosthesis function.

DO NOT OVERSIZE. Oversizing may cause bioprosthesis damage or localized mechanical stresses, which may in turn injure the heart or result in leaflet tissue failure, stent distortion and regurgitation.

As with any implanted medical device, there is a potential for patient immunological response. Some components of the model 11000A are a metal alloy that contains cobalt, thoronium, nickel, molybdenum, manganese, carbon, beryllium and iron. Care should be exercised in patients with hypersensitivities to these materials. This device was manufactured without latex, but may have been produced in a latex-containing environment.

#### Adverse Events

#### 5.1 Observed Adverse Events

As with all prosthetic heart valves, serious adverse events, sometimes leading to death, may be associated with the use of tissue valves. In addition, adverse events due to individual patient reaction to an implanted device or to physical or chemical changes to the components, particularly those of biological origin, may occur at varying intervals (hours or days) necessitating reoperation and replacement of the prosthetic device.

The Edwards Pericardial Aortic Bioprosthesis, Model 11000A is similar in design to the Carpentier-Edwards PERIMOUNT Magna Ease Pericardial Bioprostheses, Model 3300TFX.

Adverse events associated with the use of Carpentier-Edwards PERIMOUNT pericardial bioprostheses compiled from the literature and from reports received through the product surveillance system in accordance with the United States (Federal) regulations establishing Good Manufacturing Practices, section 820.198, include stenosis, regurgitation through an incompetent valve. perivalvular leak, endocarditis, hemolysis, thromboembolism, thrombotic obstruction, bleeding diatheses related to the use of anticoagulation therapy. and malfunctions of the valve due to distortion at implant, fracture of the wireform, or physical or chemical deterioration of valve components. Types of tissue deterioration include infection, calcification, thickening, perforation, degeneration, suture abrasion, instrument trauma, and leaflet detachment from the valve stent posts. These complications may present clinically as abnormal heart murmur, shortness of breath, exercise intolerance, dyspnea, orthopnea, anemia, fever, arrhythmia, hemorrhage, transient ischemic attack, stroke, paralysis, low cardiac output, pulmonary edema, congestive heart failure. cardiac failure, and myocardial infarction.

Note: Based on reports in the literature on tissue valves (Refs. 6, 7, 8, 9 & 10), there appears to be an increased incidence of leaflet calcification in patients under the age of 20. In this regard, animal research studies (Ref. 11) show that a high systemic calcium level can lead to early calcification. Furthermore, at least one published report describes a potential relationship between the consumption of daily calcium supplements and early leaflet calcification in an adult (Ref. 13). When feasible, repeated intravenous injections containing calcium should be avoided during the postoperative period; and excessive milk or dairy product consumption should be avoided in children. There are no clinical data demonstrating increased resistance of the Edwards Pericardial Aortic Bioprosthesis Model 11000A to calcification as compared to other commercially available bioprostheses.

#### 5.2 Potential Adverse Events

Adverse events potentially associated with the use of bioprosthetic heart valves include:

- Angina
- Bleeding diatheses (coagulopathy) related to anticoagulant therapy
- Cardiac arrhythmias
- · Coronary ostial blockage
- Endocarditis
- Heart failure
- Hemolysis
- Hemolytic anemia
- Hemorrhage
- Local and/or systemic infection
- Mvocardial infarction
- Patient prosthetic mismatch (PPM)
- Prosthesis leaflet entrapment (Impingement)
- · Prosthesis nonstructural dysfunction
- Prosthesis pannus
- Prosthesis perivalvular leak
- Prosthesis regurgitation
- · Prosthesis structural deterioration
- Prosthesis thrombosis
- Stroke
- Thromboembolism
- Transient ischemic attack (TIA)

It is possible that these complications may lead to:

- Reoperation
- Explantation
- · Permanent disability
- Death

#### 6. Clinical Studies

#### **Pre-Approval Patient Cohort**

Clinical data, available on 719 patients requiring isolated aortic valve replacement (AVR) with the model 2700 Carpentier-Edwards PERIMOUNT pericardial bioprosthesis with mean follow-up of 3.9 years, indicate overall actuarial survival rate at 6 years of 73.7% ± 2.0%. Clinical data, available on 70 patients requiring double valve replacement (DVR) with mean follow-up of 3.7 years, indicate overall actuarial survival rate at 6 years of 67.2% ± 6.5%. These pre-approval patient cohort data were collected from the period between August 1981 to January 1989.

In the isolated AVR population, there were a total of 455 (63.3%) males and 264 (36.7%) females with a mean age at implant ( $\pm$  standard deviation) of 64 ( $\pm$  12.4) years and a range of 18 to 90 years. The indications for valve replacement were stenosis (63.4%), regurgitation (16.3%), mixed disease (15.3%) and previous prosthetic aortic valve dysfunction (5.0%).

In the DVR population, there were a total of 24 (34.3%) males and 46 (65.7%) females with a mean age (± standard deviation) of 62.9 (± 12.7) years and a range of 31 to 94 years. The indications for valve replacement were stenosis (45.7%), regurgitation (25.7%), mixed disease (21.4%) and previous prosthetic aortic valve dysfunction (7.4%).

The follow-up methods included hospital visits, office visits and contact by telephone or letter with either the patient, the patient's family or local doctor.

Table 2 summarizes the operative and postoperative complication rates for the isolated AVR and DVR populations. The operative rates are based on 719 patients for the isolated AVR population and on 70 patients for the DVR population. The postoperative rates are based on 2767.9 and 255.8 years of follow-up occurring > 30 days after implant for the isolated AVR and DVR populations, respectively.

Table 3 presents, by valve size, the postoperative echocardiography results of patients in this study population.

Information on preoperative and postoperative NYHA Functional Class was gathered for the isolated AVR population. The NYHA Functional Class was not reported in 220 patients (171 patients expired and 49 patients not available). Of the 499 patients with reported preoperative and postoperative NYHA Functional Class at the last available follow up, 10 patients, (2.0%) got worse, 59 patients (11.8%) remained the same and 430 patients (86.2%) improved.

Table 4 presents data comparing preoperative NYHA Functional Class to postoperative NYHA Functional Class at the last available follow up.

#### Post-Approval Patient Cohort

Edwards has followed a post-approval cohort of 267 patients with isolated valve replacements (AVR) (model 2700) from four centers of the original clinical trial for the Carpentier-Edwards PERIMOUNT pericardial bioprosthesis since November 1981. The population is comprised of 171 (64%) males and 96 (36%) females. The mean age ( $\pm$  standard deviation) of these patients at the time of implant was 64.9  $\pm$  11.8 years and ranged from 21 to 86 years. A total of 2,407 patient years of data were available for analysis (2,386 late patient years). Mean follow-up was 9.0  $\pm$  5.5 years, with a maximum of 20.3 years. A total of 189 deaths occurred between 1981 and 1994. Forty-eight (25.3%) of the 189 deaths were determined to be valve-related. The follow-up methods used at each clinic included hospital visits, office visits, and contact by telephone or letter with either the patient, the patient's family, or local doctor.

Table 5 summarizes the freedom from complication rates at 20 years. Patient status as of the last follow-up interval included 189 expired (70.8%), 10 alive (3.8%), 46 explanted (17.2%), and 22 lost to follow-up (8.2%).

There were a total of 48 valve-related expirations in this patient population; 1 valve-related expiration occurred in the operative period and consisted of bleeding. Twenty-eight postoperative valve-related expirations included 5 due to thromboembolism, 4 due to endocarditis/sepsis, 3 due to structural valve deterioration and 1 due to bleeding. There were 15 other expirations that were considered to be valve-related because of lack of information or because the expiration was classified as valve-related by the investigator. The actuarial freedom from valve-related expiration was 67.9  $\pm$  6.6% at 20 years. Nineteen additional expirations were due to either unknown causes or sudden death and might have been valve related. These deaths were conservatively classified as valve related; accordingly, the resulting actuarial freedom from valve-related expiration was 55.4  $\pm$  6.4% at 20 years.

Improvement in NYHA functional classification also was demonstrated postoperatively. As of the latest follow-up evaluation, 108 patients (44.8%) were in NYHA Functional Class I

These data were compiled from a multi-center clinical trial conducted by Edwards Lifesciences. For additional information on this trial, please contact Edwards Lifesciences LLC, Heart Valve Therapy Marketing Department, One Edwards Way, Irvine, CA 92614-5686.

#### **Confirmatory Study**

From August 2003 through January 2004, 60 patients requiring aortic valve replacement (AVR) were implanted with the Carpentier-Edwards PERIMOUNT Magna aortic bioprosthesis, model 3000, from five institutions (two European and three Canadian). Shortly thereafter, the clinical protocol was amended to allow implantation with the Carpentier-Edwards PERIMOUNT Magna aortic bioprosthesis, model 3000TFX, and to add three US institutions. Subsequently, 193 additional patients were implanted with the model 3000TFX from December 2004 through December 2006. The model 3000TFX differs from the model 3000 in that the model 3000TFX is treated with the ThermaFix process.

In the model 3000TFX population, there were a total of 116 males (60.1%) and 77 females (39.9%) with a mean age at implant of 72.0 (± 8.59 SD) years and an age range from 26 to 89 years. The main indication for valve replacement was stenosis (78.2%) followed by mixed disease (14.5%), and regurgitation (7.3%).

In the combined models 3000 and 3000TFX population, there were a total of 150 males (59.3%) and 103 females (40.7%) with a mean age at implant of 72.2 (± 8.31 5D) years and an age range from 26 to 89 years. Again the major indication for valve replacement was stenosis (77.5%), mixed disease (15.4%), and requiridation (7.1%).

Patients were evaluated preoperatively, intraoperatively, at discharge, at 3 to 6 months, at 1 year, and annually thereafter. The cumulative follow-up for the model 3000TFX was 167 patient-years, with a mean follow-up of 0.9 years (SD = 0.42, range = 0.0 to 2.1 years); and the cumulative follow-up for both models 3000 and 3000TFX combined was 232 patient-years with a mean follow-up of 0.9 years (SD = 0.42, range = 0.0 to 2.1 years).

Table 6 summarizes early ( $\leq$  30 days) and late postoperative (> 30 days) valve-related adverse event rates for the model 3000TFX and the combined models 3000/3000TFX populations, respectively.

Table 7 illustrates, by valve size, hemodynamic variables reported in echocardiograms at one year performed on patients in the model 3000TFX and the combined model 3000/3000TFX studies

Table 8 presents the change in NYHA Functional Class from baseline assessment to the 1-year visit. It should be noted that there was a 56.5% improvement in functional class at the 1-year visit for model 3000TFX. For the model 3000/3000TFX combined population, there was a 60.9% improvement in functional class at the 1-year visit.

Several published clinical studies demonstrate the long-term durability of Carpentier-Edwards PERIMOUNT pericardial aortic bioprostheses, the foundation

on which the Carpentier-Edwards PERIMOUNT Magna and Magna Ease pericardial aortic bioprostheses are designed (Refs. 14, 15, 16 & 17). Additionally, published data show the PERIMOUNT Magna aortic bioprosthesis demonstrates exceptional hemodynamic performance, with a very low risk of patient-prosthesis mismatch (Refs. 18, 19, 20, 21, 22 & 23).

#### 7. Individualization of Treatment

Bioprosthetic heart valve recipients should be maintained on anticoagulation therapy, except where contraindicated, during the initial stages after implantation as determined by the physician on an individual basis. Long-term anticoagulation and/or antiplatelet therapy should be considered for patients with risk factors for thromboembolism.

The ultimate judgment regarding care of a particular patient must be made by the healthcare provider and patient in light of all the circumstances presented by that patient (Ref. 12). A bioprosthesis is recommended for AVR in patients of any age who will not take warfarin or who have major medical contraindications to warfarin therapy. Patient preference is a reasonable consideration in the selection of aortic valve operation and valve prosthesis. A mechanical prosthesis is reasonable for AVR in patients under 65 years of age who do not have a contraindication to anticoagulation. A bioprosthesis is reasonable for AVR in patients under 65 years of age who elect to receive this valve for lifestyle considerations after detailed discussions of the risks of anticoagulation versus the likelihood that a second AVR may be necessary (Ref. 12).

#### 7.1 Specific Patient Populations

The safety and effectiveness of the Model 11000A bioprosthesis has not been established for the following specific populations because it has not been studied in these populations:

- patients who are pregnant;
- · nursing mothers:
- patients with abnormal calcium metabolism (e.g., chronic renal failure, hyperparathyroidism);
- patients with aneurysmal aortic degenerative conditions (e.g., cystic medial necrosis. Marfan's syndrome):
- children, adolescents, and young adults

Caution: Based on reports in the literature on tissue valves (Refs. 6, 7, 8, 9 & 10), there appears to be an increased incidence of leaflet calcification in patients under the age of 20. When feasible, repeated intravenous injections containing calcium should be avoided during the postoperative period, and excessive milk or dairy product consumption should be avoided in children. Animal research studies (Ref. 11) show that a high systemic calcium level can lead to early calcification.

# 8. Patient Counseling Information

Careful and continued medical follow up (at least by an annual visit to the physician) is advised so that bioprosthesis-related complications, particularly those related to material failure, can be diagnosed and properly managed. Patients with bioprostheses are at risk from bacteremia (e.g., undergoing dental procedures) and should be advised about prophylactic antibiotic therapy. Patients should be encouraged to carry their Patient Identification Card at all times and to inform their healthcare providers that they have an implant when seeking care.

### 9. How Supplied

#### 9.1 Packaging

The Edwards Pericardial Aortic Bioprosthesis, Model 11000A, is provided sterile and non-pyrogenic, in a double barrier tray package. The double tray package is in a foil pouch, which is in a carton.

Each bioprosthesis is contained in a carton with a temperature indicator displayed through a window on the side panel. The temperature indicator is intended to identify products that were exposed to transient temperature extremes. Upon receipt of the bioprosthesis, immediately inspect the indicator and refer to the carton label to confirm a "Use" condition. If the "Use" condition is not apparent, do not use the bioprosthesis and contact the local supplier or Edwards Lifesciences representative to make arrangements for return authorization and replacement.

Warning: Carefully inspect the bioprosthesis before implantation for evidence of extreme temperature exposure or other damage.

#### 9.2 Storage

The Edwards Pericardial Aortic Bioprosthesis, Model 11000A, should be stored at  $10\,^{\circ}$ C to  $25\,^{\circ}$ C (50-77  $^{\circ}$ F), in the foil pouch and shelf carton.

#### 10. Directions for Use

#### 10.1 Physician Training

The techniques for implanting this bioprosthesis are similar to those used for supra-annular placement of any stented aortic bioprosthesis. No special training is required to implant the Edwards Pericardial Aortic Bioprosthesis, Model 11000A.

#### 10.2 Sizing

Verify that the accessories have been sterilized according to the recommended instructions provided with the reusable accessories.

#### Supra-annular sizing

For supra-annular implantation, the sewing ring of the bioprosthesis is placed above the annulus, thereby maximizing valve orifice area. When sizing for supra-annular implantation, the sizer should be parallel with the plane of the annulus and the following sizing technique should be used:

| Step | Procedure |
|---|---|
| 1 | Using the Model 1133 sizer, select the cylindrical end of the<br>largest diameter sizer that comfortably fits in the patient's<br>annulus. |
| | HVT21 |

# 2 Once the appropriate cylindrical end is verified, use the replica end of the same sizer to verify that the sewing ring will fit comfortably on top of the annulus. Ensure that the coronary ostia are not obstructed and that the stent posts of the replica end do not interfere with the aortic wall at the sinotubular junction. If satisfied with the fit of the replica end, choose this size of the bioprosthesis for implant. HVT37

#### 10.3 Handling and Preparation Instructions

Procedure

Step

In-service training is recommended prior to handling and preparing the Edwards Pericardial Aortic Bioprosthesis, Model 11000A.

Caution: Do not onen the Edwards Pericardial Aortic

| ' | Bioprosthesis, Model 11000A package until implantation is certain. |
|---|---|
| | Warning: Do not open foil pouch into sterile field. Foil<br>pouch is protective cover only. Only the innermost<br>package tray may be introduced into the sterile field. |
| | Once the appropriate size bioprosthesis is chosen, remove the foil pouch from the carton in the non-sterile field. Before opening, examine the package for evidence of damage and broken or missing seals. |
| 2 | Near the sterile field, hold the base of the outer tray and peel the lid from the outer tray. |
| 3 | The inner tray and contents are sterile. Transfer the inner tray to the sterile field. The contents of the inner tray must be handled using a sterile surgical technique to prevent contamination. |
| | HVIZ6 |

| Step | Procedure |
|---|---|
| 4 | Caution: Do not open the inner package until implantation is certain and the surgeon is ready to place the valve. Caution: The bioprosthesis is not secured to the inner tray. Care should be taken while peeling the lid and opening the plastic tab. |
| | Before opening, examine the inner tray and lid for evidence of damage, stains, and broken or missing seals. Hold the base of the inner tray and peel the lid from the inner tray. |
| 5 | To access the bioprosthesis, pull up on the plastic tab with the arrow. |
| | HVT28<br>Pull up on Tab with Arrow |
| | НИТ29 |
| | HVT30 |

| Step | Procedure |
|---|---|
| 6 | Attach the handle, Model 1111 or Model 1126, to the bioprosthesis holder while the bioprosthesis is still in the tray. To attach, insert the handle into the holder and turn the handle clockwise until resistance is felt. |
| | Caution: Do not grasp the bioprosthesis with hands or surgical instruments. |
| | Caution: Do not push the bioprosthesis off the dip while attaching the handle to the holder. |
| | Caution: The handle/holder assembly is required for implantation and should not be removed until the bioprosthesis is sutured to the annulus. |
| | Caution: Care should be taken to avoid entangling the serial tag in the handle during attachment. |
| | HVT31<br>Handle Holder |
| 7 | Once the handle is attached, remove the bioprosthesis and clip from the inner tray. |
| | HVT32 |

| Step | Procedure |
|---|---|
| 8 | To remove the clip from the bioprosthesis, grasp the clip and pull away from the handle/holder assembly. HVT33 |
| | Case is the second seco |
| | HVT34 |
| | The second secon |
| 9 | A serial number tag is attached to the sewing ring of each bioprosthesis by a suture. This serial number should be confirmed with the number on the bioprosthesis package and bioprosthesis implant data card. This tag should not be detached from the bioprosthesis until implantation is certain. |
| | Caution: If any difference in serial number is noted, the bioprosthesis should be returned unused. |
| | Caution: Care should be exercised to avoid cutting or<br>tearing the sewing ring cloth during removal of the<br>serial number tag. |
| | Caution: To prevent damage to the sewing ring cloth, avoid pulling the knot of the serial tag suture through the sewing ring. |

| Step | Procedure |
|---|---|
| 10 | The Edwards Pericardial Aortic Bioprosthesis, Model 11000A, DOES NOT REQUIRE RINSING prior to implantation. |
| | Caution: If the bioprosthesis is rinsed prior to<br>implantation, it must then be kept hydrated with<br>sterile physiological saline irrigation on both sides of<br>the leaflet tissue throughout the remainder of the<br>surgical procedure. Rinsing every one to two minutes<br>is recommended. |
| | Caution: Avoid contact of the leaflet tissue with towels, linens, or other sources of particulate matter that may be transferred to the leaflet tissue. |

| is recommended. Caution: Avoid contact of the leaflet tissue with towels linens, or other sources of particulate matter that may be transferred to the leaflet tissue. | |
|---|---|
| 10.4 Device Implantation The Edwards Pericardial Aortic Bioprosthesis, Model 11000A, is designed for supra-annular implant. | |
| Step | Procedure |
| 1 | The surgeon should be familiar with the recommendations for proper sizing and placement in the supra-annular position (See 10.2 Sizing). |
| | Because of the complexity and variation of cardiac valve replacement surgery, the choice of surgical technique, appropriately modified in accordance with the previously described <b>Warnings</b> , is left to the discretion of the individual surgeon. In general, the following steps should be employed: |
| | Surgically remove the diseased or damaged valve leaflets<br>and all associated structures deemed necessary. |
| | <ol><li>Surgically remove any calcium from the annulus to ensure<br/>proper seating of the sewing ring of the bioprosthesis to<br/>avoid damage to the delicate leaflet tissue.</li></ol> |
| | <ol> <li>Measure the annulus using only the Carpentier-Edwards<br/>aortic sizers, Model 1133 (Figures 1a-1c).</li> </ol> |
| | Caution: When choosing a bioprosthesis for a given patient, the size, age, and physical condition of the patient in relation to the size of the bioprosthesis must be taken into consideration to minimize the possibility of obtaining a suboptimal hemodynamic result. The selection of a bioprosthesis, however, must ultimately be made by the physician on an individual basis after carefully weighing all of the risks and benefits to the patient. |
| | Caution: Do not use other manufacturer's prosthesis sizers, or sizers for other Edwards Lifesciences bioprostheses, to size the Edwards Pericardial Aortic Bioprosthesis, Model 11000A. |
| | Caution: Examine sizers for signs of wear, such as dullness, cracking or crazing. Replace sizer if any deterioration is observed. |
| | Warning: Fragments of handles and sizers are not<br>radio-opaque and cannot be located by means of an<br>external imaging device. |

#### Step Procedure

A suture technique resulting in supra-annular placement of the bioprosthesis, such as a non-everting horizontal mattress technique, should be employed. When placing sutures through the sewing ring of the Edwards Pericardial Aortic Bioprosthesis, Model 11000A, it is recommended that the sutures pass through the sewing ring as close as possible to the frame of the bioprosthesis.

Once the sutures are completely tied, it is important to cut the sutures close to the knots to ensure that exposed suture tails will not come into contact with the leaflet tissue of the bioprosthesis.

HVT35



The integral holder and attached handle are removed as a unit at the completion of the suturing procedure.

 Using a scalpel, cut each of the three exposed sutures that are on the top of the holder.

HVT36



Caution: Avoid cutting or damaging the stent or delicate leaflet tissue when cutting the sutures.

- After all three holder sutures are cut, remove the handle/ holder assembly, along with the holder sutures, from the bioprosthesis as a unit.
- Remove the handle from the holder and discard the holder.

#### 10.5 Accessory Cleaning and Sterilization

The accessories for the Edwards Pericardial Aortic Bioprosthesis, Model 11000A, are packaged separately. The model 1126 handle is provided sterile and is intended for single use only. The model 1111 handle and model 1133 sizers are supplied nonsterile and must be sterilized before using. The handle, sizers, tray base and tray lid must be cleaned and resterilized prior to each use. Refer to the Instructions for Use supplied with the reusable accessories for cleaning and sterilization instructions.

#### 10.6 Return of Bioprostheses

Edwards Lifesciences is interested in obtaining recovered clinical specimens of the Edwards Pericardial Aortic Bioprosthesis, Model 11000A, for analysis. Contact the local representative for return of recovered bioprostheses.

- Unopened Package with Sterile Barrier Intact: If the foil pouch or trays have not been opened, return the bioprosthesis in its original packaging.
- Package Opened but Bioprosthesis Not Implanted: If the tray is opened, the bioprosthesis is no longer sterile. If the bioprosthesis is not implanted, it should be placed into a suitable histological fixative such as 10% formalin or 2% glutaraldehyde and returned to the company. Refrigeration is not necessary under these circumstances.
- Explanted Bioprosthesis: The explanted bioprosthesis should be placed into a suitable histological fixative such as 10% formalin or 2% glutaraldehyde and returned to the company. Refrigeration is not necessary under these circumstances.

# 11. Safety in the Magnetic Resonance (MR) Environment



#### MR Conditional

Non-clinical testing has demonstrated that the Edwards Pericardial Aortic Bioprosthesis, Model 11000A, is MR Conditional. A patient with the model 11000A valve can be scanned safely, immediately after placement of this implant under the following conditions:

- Static magnetic field of 1.5 tesla or 3.0 tesla.
- Maximum spatial magnetic gradient field of 2670 gauss/cm.
- Maximum MR system-reported whole-body averaged specific absorption rate (SAR) of 2.0 W/kg in the normal operating mode for 15 minutes of scanning per sequence.

In non-clinical testing, the Edwards Pericardial Aortic Bioprosthesis, Model 11000A, produced an estimated maximum in vivo temperature rise of less than or equal to 1.8 °C at a maximum MR system reported, whole-body-averaged special to absorption rate (SAR) of 2.0 W/kg, for 15 minutes of MR scanning in a GE Signa 64 MHz (1.5 T) RF coil and a GE Signa HDx (3 T) MR system with Software Version 15 UX/MR Software release 15.0.M4.0910.a.

Image artifact was measured non-clinically in a GE Signa 3T HDx MR system according to ASTM F2119-07 using the spin echo and gradient echo sequences specified therein. The spin echo images exhibited light and dark artifacts that extended as far as 40 mm from the implant and partially to fully obscured the lumen. The gradient echo images exhibited opaque dark or light and dark triangular shaped artifacts that extended as far as 40 mm from the implant and totally obscured the lumen. Reduction in artifact may be possible with sequences designed for reduction of metal artifact.

#### 12. Patient Information

#### 12.1 Study Identification Card

A Study Identification Card is provided to each subject implanted with the Edwards Pericardial Aortic Bioprosthesis, Model 11000A.

#### 12.2 Patient Information Materials

Patient information materials may be obtained from Edwards or an Edwards clinical sales specialist.

#### 13. References

- Carpentier, A., et al. Biological Factors Affecting Long Term Results of Valvular Heterografts. J Thorac Cardiovasc Surg 1969, 58:467-483.
- 2. Carpentier, A., et al. Six Year Follow-up of Glutaraldehyde Preserved Heterografts. *J Thorac Cardiovasc Surg* 1974, 68:771-782.
- Reis, Robert L., et al. The Flexible Stent. A New Concept in the Fabrication of Tissue Heart Valve Prostheses. J Thorac Cardiovasc Surg 1971, 62(5):683-689 and 693-695.
- Barratt-Boyes, B.G. and A.H.G. Roche. A Review of Aortic Valve Homografts Over a Six and One-half Year Period. Ann Surg 1969, 170:483-492.
- Brewer, R.J., et al. The Dynamic Aortic Root. Its Role in Aortic Valve Function. J Thorac Cardiovasc Surg 1976, 72:413-417.
- Jamieson, W.R.E., et al. Carpentier-Edwards Standard Porcine Bioprosthesis: Primary Tissue Failure (Structural Valve Deterioration) by Age Groups. Ann Thorac Sura 1988. 46:155-162.
- Odell, J.A. Calcification of Porcine Bioprostheses in Children. In Cohn, L. and V. Gallucci (eds): Cardiac Bioprostheses. Yorke Medical Books. New York, 1982, pp 231-237.
- Reul, G.J., et al. Valve Failure with the lonescu-Shiley Bovine Pericardial Bioprosthesis: Analysis of 2680 Patients. J Vasc Surg 1985, 2(1):192-204.
- Sanders, S.P., et al. Use of Hancock Porcine Xenografts in Children and Adolescents. Am J Cardiol 1980, 46(3):429-438.
- Silver, M.M., et al. Calcification in Porcine Xenograft Valves in Children. Am J Cardiol 1980, 45:685-689.
- Carpentier, A., et al. Continuing Improvements in Valvular Bioprostheses. *J Thorac Cardiovasc Sura* 1982, 83(1):27-42.
- Bonow R.O., et al. ACC/AHA Guidelines for the Management of Patients with Valvular Heart Disease: A Report of the American College of Cardiology/ American Heart Association Task Force on Practice Guidelines (Committee on Management of Patients With Valvular Heart Disease). J Am Coll Cardiol 2006. 48:e1-148.
- Moront, M.G. and N.M. Katz. Early Degeneration of a Porcine Aortic Valve Bioprosthesis in the Mitral Valve Position in an Elderly Woman and its Association with Long-Term Calcium Carbonate Therapy. Am J Cardiol 1987, 59:1006-1007.
- Aupart, M.R., et al. Perimount Pericardial Bioprosthesis for Aortic Calcified Stenosis: 18-Year Experience with 1,133 Patients. J Heart Valve Dis 2006, 15:768-776.
- Dellgren, G., et al. Late Hemodynamic and Clinical Outcomes of Aortic Valve Replacement with the Carpentier-Edwards Perimount Pericardial Bioprosthesis. J Thorac Cardiovasc Sura 2002. 124:146-154.

- Frater, R.W.M., et al. Long-Term Durability and Patient Functional Status of the Carpentier-Edwards Perimount Pericardial Bioprosthesis in the Aortic Position. J Heart Valve Dis 1998, 7:48-53.
- Jamieson, W.R.E., et al. 15-Year Comparison of Supra-Annular Porcine and PERIMOUNT Aortic Bioprostheses. Asian Cardiovasc Thorac Ann 2006, 14:200-205
- Borger, M.A., et al. Carpentier-Edwards Perimount Magna Valve Versus Medtronic Hancock II: A Matched Hemodynamic Comparison. Ann Thorac Surg 2007; 83:2054-2058.
- Botzenhardt, F., et al. Hemodynamic Comparison of Bioprostheses for Complete Supra-Annular Position in Patients With Small Aortic Annulus. J Am Coll Cardiol 2005. 45:2054-2060.
- Botzenhardt, F., et al. Hemodynamic Performance and Incidence of Patient-Prosthesis Mismatch of the Complete Supraanular Perimount Magna Bioprosthesis in the Aortic Position. *Thorac Cardiov Surg* 2005, 53:226–230.
- Dalmau, M.J., et al. The Carpentier-Edwards Perimount Magna Aortic Xenograft: A New Design with an Improved Hemodynamic Performance. Interact Cardiovasc Thorac Surg 2006, 5:263-267.
- Totaro, P., et al. Carpentier-Edwards PERIMOUNT Magna Bioprosthesis: A Stented Valve with Stentless Performance? J Thorac Cardiovasc Surg 2005, 130:1668-1674.
- Wagner, I.M., et al. Influence of Completely Supra-annular Placement of Bioprostheses on Exercise Hemodynamics in Patients With a Small Aortic Annulus. J Thorac Cardiovascular Surg 2007; 133:1234-1241.

This product is manufactured and distributed under at least one or more of the following U.S. Patents: US-Patent Nos. 5,928,281; 5,931,969; 5,961,549; 6,102,944; 6,245,105; 6,413,275; 6,561,970; 6,585,766; 6,837,902; 6,945,997; 7,214,344; 7,972,376; 8,007,992; 8,357,387; 8,366,769; 8,632,608; and RE 40570; and corresponding foreign patents. Likewise, additional patents pending.

Refer to the symbol legend at the end of this document.

Table 2. Summary of Complication Rates, Model 2700

| | ls | olated AVR Pop | ulation | | ion | |
|---|---|---|---|---|---|---|
| Complication | Operative<br>% of Pts. | Post-<br>Operative<br>% Per Pt. Yr. | % Event-Free<br>at Six Years<br>(Standard Error) | Operative<br>% of Pts. | Post-<br>Operative<br>% Per Pt. Yr. | % Event-Free<br>at Six Years<br>(Standard Error) |
| Death | 4.7 | 4.6 | 73.5 (2.0) | 12.9 | 4.2 | 67.2 (6.5) |
| Explant | 0 | 0.3 | 98.5 (1.0) | 0 | 0.8 | NA * |
| Valve Related Reoperation | 0.7 | 0.1 | 99.8 (0.4) | 0 | 0 | NA * |
| All Reoperation | 22.4 | 1.8 | 75.4 (1.8) | 34.3 | 2.3 | NA * |
| Valve Related Thromboembolism | 3.1 | 1.5 | 91.4 (1.1) | 1.4 | 5.1 | NA * |
| All Thromboembolism | 5.0 | 2.4 | 84.9 (1.6) | 5.7 | 6.6 | NA * |
| Endocarditis | 0.6 | 0.8 | 95.8 (0.9) | 1.4 | 1.5 | NA * |
| Valve Dysfunction | 0.1 | 0.7 | 96.0 (1.1) | 0 | 0.4 | NA * |
| Perivalvular Leak | 0.1 | 0.3 | 98.8 (0.5) | 0 | 1.2 | NA * |
| Hemorrhagic Anticoagulation Complication | 1.4 | 0.4 | 96.4 (1.1) | 4.3 | 2.3 | NA * |
| Hemolysis | 0 | 0.2 | 99.1 (0.4) | 0 | 0.4 | NA * |
| Valve Thrombosis | 0 | 0 | 100.0 (0) | 0 | 0.4 | NA* |

<sup>\*</sup> NA = Not Applicable

Table 3. Postoperative Echocardiography Results, Model 2700

| | Valve Size | | | | | | |
|---|---|---|---|---|---|---|---|
| | 19 mm | 21 mm | 23 mm | 25 mm | 27 mm | 29 mm | Total |
| Total N | 12 | 22 | 15 | 8 | 3 | 3 | 63 |
| Avg. Months Postoperative | $28.6\pm7.2$ | $34.9 \pm 8.6$ | $36.9 \pm 9.2$ | $39.9 \pm 7.6$ | $31.4 \pm 15.9$ | $15.3 \pm 12.2$ | $34.6 \pm 9.2$ |
| Velocity (M/sec) | | | | | | | |
| $mean \pm S.D.$ | $2.80\pm0.49$ | $2.56\pm0.46$ | $2.36 \pm 0.42$ | $2.15\pm0.56$ | $2.09 \pm 0.27$ | $2.08\pm0.1$ | $2.46\pm0.50$ |
| n = | 12 | 21 | 15 | 7 | 3 | 3 | 61 |
| range | 1.90 - 3.60 | 1.90 - 3.90 | 1.39 - 2.86 | 1.00 - 2.60 | 1.90 - 2.40 | 2.05 - 2.10 | 1.00 - 3.90 |
| Peak Instantaneous<br>Gradient (mmHg) | | | | | | | |
| $mean \pm S.D.$ | $32.22 \pm 11.08$ | $27.04 \pm 10.49$ | $23.00 \pm 7.30$ | $19.50 \pm 8.16$ | $17.60 \pm 4.70$ | $14.4 \pm 0.58$ | 25.67 ± 10.14 |
| $\mathbf{n} =$ | 12 | 21 | 15 | 7 | 3 | 3 | 61 |
| range | 14.40 - 51.80 | 14.40 - 60.80 | 7.70 - 32.70 | 4.00 - 27.00 | 14.40 - 23.00 | 13.95 - 15.06 | 4.00 - 60.80 |

Table 4. Effectiveness Outcomes, NYHA Functional Class, Model 2700

| Preoperative<br>NYHA Functional Class | | | | erative<br>ctional Class | | |
|---|---|---|---|---|---|---|
| | 1 | II | III | IV | Expiration | Not<br>Available |
| I | 18 | 19 | | | 9 | |
| II | 140 | 37 | | | 35 | 15 |
| III | 181 | 48 | 4 | 1 | 72 | 24 |
| IV | 43 | 16 | 2 | | 53 | 2 |
| Not Available | 5 | 1 | | | 2 | 2 |

Table 5. Freedom from Complication Rates at 20 years (N = 267), Model 2700

| Freedom from Complications at 20 Years | Actual | Actuarial | Linearized (%/ptyr) |
|---|---|---|---|
| Valve-Related Expirations | $85.8 \pm 2.5\%$ | $67.9 \pm 6.6\%$ | 1.2 |
| Thromboembolism/Thrombosis | $82.4 \pm 2.6\%$ | $68.2 \pm 6.8\%$ | 1.7 |
| Bleeding | $94.0 \pm 1.5\%$ | $91.7 \pm 2.2\%$ | 0.4 |
| Endocarditis/Sepsis | 91.7 ± 1.7% | $89.3 \pm 2.4\%$ | 0.8 |
| Explant due to SVD | | | |
| ≥ 60 | $92.6 \pm 2.0\%$ | $77.1 \pm 7.2\%$ | n.r.* |
| ≥ 65 | $96.3 \pm 1.6\%$ | $81.5 \pm 9.6\%$ | |
| > 70 | $96.0\pm2.3\%$ | $69.9 \pm 20.5\%$ | |

<sup>\*</sup> Not relevant. SVD does not occur as a constant hazard function; consequently, linearized rates are not meaningful.

Table 6. Summary of Valve-Related Adverse Events, Models 3000 and 3000TFX

| | ≤ 30 Days Po | ost-Operative | > 30 Days Po | ost-Operative |
|---|---|---|---|---|
| Adverse Events | 3000TFX (N = 193)<br># of events (% of Pts) | 3000/3000TFX<br>(N = 253)<br># of events (% of Pts) | 3000TFX (N = 193)<br># of events (% of Pts) | 3000/3000TFX<br>(N = 253)<br># of events (% of Pts) |
| Valve-Related Thromboembolism | 6 (3.1) | 7 (2.8) | 3 (2.0) | 3 (1.4) |
| Non-Structural Valve Dysfunction (PVL) | 3 (1.5) | 4 (1.6) | 3 (2.0) | 3 (1.4) |
| Explant (NSVD) | 2 (1.0) | 2 (0.8) | 0 (0.0) | 0 (0.0) |
| Death (Cardiac Arrest, Bleeding Event, CVA) | 1 (0.5) | 1 (0.4) | 3 (2.0) | 3 (1.4) |
| Reoperation | 1 (0.5) | 1 (0.4) | 1 (0.7) | 1 (0.5) |
| Hemolysis | 1 (0.5) | 1 (0.4) | 3 (2.0) | 3 (1.4) |
| AC related Bleeding | 0 (0.0) | 0 (0.0) | 2 (1.4) | 2 (1.0) |
| Endocarditis | 0 (0.0) | 0 (0.0) | 0 (0.0) | 0 (0.0) |
| Structural Valve Deterioration | 0 (0.0) | 0 (0.0) | 0 (0.0) | 0 (0.0) |
| Valve Thrombosis | 0 (0.0) | 0 (0.0) | 0 (0.0) | 0 (0.0) |
| Other (Tear In Aorta) | 1 (0.5) | 1 (0.4) | 0 (0.0) | 0 (0.0) |

Table 7. Hemodynamic Variables at 1-Year Follow-Up Echo Assessment, Models 3000 and 3000TFX

| Valve Type | Variable | 19 mm<br>Mean ± SD (N) | 21 mm<br>Mean ± SD (N) | 23 mm<br>Mean ± SD (N) | 25 mm<br>Mean ± SD (N) | 27 mm<br>Mean ± SD (N) | 29 mm<br>Mean ± SD (N) |
|---|---|---|---|---|---|---|---|
| 3000TFX | Mean Systolic | 16.7 ± 4.7 | 15.8 ± 4.4 | 11.3 ± 3.7 | 11.1 ± 4.1 | 9.4 ± 4.3 | 9.0 ± 0.0 |
| | Gradient (mmHg) | (10) | (18) | (45) | (37) | (12) | (2) |
| | Ejection | 65.8 ± 10.4 | 62.7 ± 9.4 | 60.6 ± 11.3 | 61.4 ± 11.2 | 59.5 ± 10.7 | 55.0 ±14.1 |
| | Fraction (%) | (10) | (19) | (48) | (38) | (12) | (2) |
| | Aortic EOA | 1.2 ± 0.4 | 1.5 ± 0.4 | 1.8 ± 0.6 | 1.8 ± 0.5 | 2.1 ± 0.6 | 2.1 ± 0.1 |
| | (cm²) | (10) | (18) | (44) | (36) | (12) | (2) |
| 3000/ | Mean Systolic | 16.7 ± 4.2 | 13.8 ± 4.8 | 11.7 ± 4.7 | 11.0 ± 3.8 | 9.5 ± 4.1 | 9.0 ± 0.0 |
| 3000TFX | Gradient (mmHg) | (16) | (34) | (56) | (47) | (14) | (2) |
| | Ejection | 62.1 ± 15.1 | 58.6 ± 11.6 | 60.2 ± 11.2 | 60.2 ± 11.5 | 58.5 ± 10.5 | 55.0 ± 14.1 |
| | Fraction (%) | (16) | (34) | (59) | (47) | (14) | (2) |
| | Aortic EOA | 1.3 ± 0.5 | 1.5 ± 0.4 | 1.8 ± 0.6 | 1.8 ± 0.6 | 2.1 ± 0.6 | 2.1 ± 0.1 |
| | (cm²) | (16) | (32) | (55) | (46) | (14) | (2) |

Table 8. NYHA Functional Class: Change From Baseline To 1-Year Visit, Models 3000 and 3000TFX

| | | | | Baseline | | |
|---|---|---|---|---|---|---|
| Valve Type | Follow-Up NYHA Class | Class I | Class II | Class III | Class IV | N/A |
| | Class I | 10 | 33 | 51 | 10 | 3 |
| | Class II | 2 | 8 | 13 | 2 | 1 |
| | Class III | - | - | 3 | - | - |
| 3000TFX<br>N = 193 | Class IV | - | - | - | 1 | - |
| N = 195 | Expiration | - | 3 | 16 | 1 | - |
| | Explant | - | - | 3 | - | - |
| | N/A | 2 | 6 | 21 | 4 | - |
| | Class I | 12 | 40 | 71 | 11 | 3 |
| | Class II | 2 | 14 | 29 | 3 | 1 |
| 3000/ | Class III | - | - | 3 | - | - |
| 3000TFX | Class IV | - | - | 1 | 1 | - |
| N = 253 | Expiration | - | 3 | 19 | 2 | - |
| | Explant | - | - | 3 | - | - |
| | N/A | 2 | 7 | 22 | 4 | - |

## NYHA Functional Class: Change From Baseline To 1-Year Visit

| Valve Type | Improve<br>N (%) | Same<br>N (%) | Worse<br>N (%) | N/A<br>N (%) |
|---|---|---|---|---|
| 3000TFX (N = 193) | 109 (56.5) | 22 (11.4) | 2 (1.0) | 60 (31.1) |
| 3000/3000TFX (N = 253) | 154 (60.9) | 30 (11.9) | 3 (1.2) | 66 (26.1) |

# Bioprothèse aortique péricardique d'Edwards, modèle 11000A

# Mode d'emploi

AVERTISSEMENT: dispositif expérimental. Limité à une utilisation expérimentale par les lois fédérales (États-Unis).

AVERTISSEMENT: dispositif expérimental. Exclusivement à des fins de recherche clinique.

Avertissement: dispositif expérimental. Utilisation limitée à la recherche. Pour une utilisation par des (médecins) chercheurs qualifiés uniquement.

#### Description du dispositif et des accessoires

#### 1.1 Description du dispositif

La bioprothèse aortique péricardique d'Edwards, modèle 11000A, est une bioprothèse trivalve composée d'un péricarde bovin installé sur une structure flexible. Elle est disponible en plusieurs tailles: 19, 21, 23, 25, 27 et 29 mm (tableau 1). Elle est conservée dans un emballage non aqueux et ne nécessite aucune poussée avant l'implantation.

Tableau 1 - Dimensions nominales HVT48 19 21 23 25 27 29 Taille mm mm mm mm mm mm A. Diamètre de l'annulus du tissu (diamètre de 19 21 23 25 27 29 l'endoprothèse, en mm) B. Diamètre interne (D.I. de 18 20 22 24 28 26 l'endoprothèse, en mm) 13 15 17 18 C. Hauteur du profil (en mm) 14 16 D. Diamètre de l'anneau de 24 26 28 30 32 34 suture externe (en mm) Surface de l'orifice (en mm<sup>2</sup>) 235 289 354 420 499 570

Le fil métallique est fabriqué avec un alliage de chrome-cobalt et est recouvert d'un matériau tissé en polyester. Une bande laminée en alliage en chrome-cobalt/film en polyester entoure la base de la structure en fil métallique.

Edwards Lifesciences, le logo E stylisé, Edwards, Carpentier-Edwards, ThermaFix, TFX, PERIMOUNT, PERIMOUNT Magna et Magna Ease sont des marques de commerce d'Edwards Lifesciences Corporation. Un anneau de suture en silicone, qui est couvert d'un tissu poreux en polytétrafluoroéthylène (PTFE), est attaché à la structure en fil métallique. L'anneau de suture possède trois marqueurs de suture en soie noire et à distance égale aux centres de la valve pour aider à l'orientation de la bioprothèse et au placement des sutures.

Un support est attaché à la bioprothèse par suture afin de faciliter la manipulation et la suture de la bioprothèse lors de l'implantation. Le chirurgien peut facilement détacher le support (voir la section 10.4 Implantation du dispositif).

#### 1.2 Description des accessoires

#### Calibreurs et plateau

L'utilisation d'un instrument de mesure permet de sélectionner facilement la bioprothèse de taille appropriée pour l'implantation. Les calibreurs translucides, modèle 1133, permettent une observation directe du placement dans l'annulus. Chaque calibreur comprend une poignée dotée d'une configuration de mesure différente à chaque extrémité (figure 1a). Sur l'une des extrémités de la poignée se trouve un embout cylindrique doté d'une lèvre reprenant la forme géométrique de l'anneau de suture de la bioprothèse (figure 1b). Sur l'autre extrémité se trouve un embout de réplique de la bioprothèse qui reprend la forme de l'anneau de suture de la bioprothèse ainsi que la hauteur et l'emplacement des montants de l'endoprothèse (figure 1c). Un calibreur est disponible pour chaque taille de la bioprothèse de modèle 11000A (19, 21, 23, 25, 27 et 29 mm). La trousse complète de calibreurs se trouve dans un plateau, modèle 1RAY1133, qui peut être réutilisé et restérilisé.

Figure 1a. Calibreur aortique



Figure 1b. Embout cylindrique Figure 1c. Embout de réplique



#### Poignée et support de la bioprothèse

L'assemblage poignée/support est constitué de deux composants : une partie jetable intégrable qui est installée sur la bioprothèse par le fabricant et une poignée malléable (modèle 1111 réutilisable ou modèle 1126 jetable pour utilisation unique) qui est attachée au suppor au moment de la chirurgie (figures 2a et 2b).

Figure 2a. Poignée du modèle 1111



Figure 2b. Poignée du modèle 1126



#### Mode d'emploi

La bioprothèse aortique péricardique d'Edwards, modèle 11000A, est destinée aux patients nécessitant le remplacement de leur valve aortique d'origine ou prothétique.

#### 3. Contre-indications

Ne pas utiliser la bioprothèse si le chirurgien estime que son utilisation est contraire à l'intérêt du patient. La décision concernant cette bioprothèse relève du chirurgien qui doit évaluer tous les risques impliqués, y compris l'anatomie et la pathologie observées au moment de l'opération chirurgicale.

#### Mises en garde

POUR UTILISATION UNIQUE SEULEMENT. Ce dispositif est conçu, destiné et distribué pour une utilisation unique seulement. Ne pas restériliser ou réutiliser ce dispositif. Aucune donnée n'existe pour corroborer le caractère stérile, la non-pyrogénicité et la fonctionnalité du dispositif après le processus de restérilisation.

NE PAS CONGELER NI EXPOSER LA BIOPROTHÈSE À UNE CHALEUR EXTRÊME. L'exposition de la bioprothèse à des températures extrêmes rendra le dispositif inutilisable.

#### NE PAS UTILISER la bioprothèse :

- si le sachet métallisé, les plateaux scellés ou les lèvres sont ouverts, endommagés ou tachés ;
- si la date d'expiration est passée ;
- si elle est tombée, endommagée ou mal manipulée de quelque façon que ce soit. Si une bioprothèse est endommagée lors de l'insertion, ne pas tenter de la réparer.

NE PAS EXPOSER la bioprothèse à des solutions, des produits chimiques, des antibiotiques, etc., à l'exception de solutions salines physiologiques. Des dommages irréparables, qui ne semblent peut-être pas apparents lors d'une inspection visuelle, peuvent avoir lieu sur le tissu de la valve.

NE PAS SAISIR le tissu de la valve de la bioprothèse avec des instruments ni endommager la bioprothèse. Même la plus petite perforation du tissu de la valve peut s'agrandir à terme et compromettre gravement le fonctionnement de la bioprothèse.

NE PAS CHOISIR UNE TAILLE SUPÉRIEURE. Le choix d'une taille supérieure peut entraîner des dommages à la bioprothèse ou un stress mécanique localisé, susceptible de blesser le cœur ou de causer une panne du tissu de la valve, une distorsion de l'endoprothèse ou une régurgitation du tissu de la valve.

Comme pour tout dispositif médical implanté, il existe un risque de réponse d'immunisation de la part du patient. Certains composants du modèle 11000A sont en alliage contenant du cobalt, du chrome, du nickel, du molybdène, du manganèse, du carbone, du béryllium et du fer. Il faut prendre des précautions avec les patients souffrant d'hypersensibilité à ces matières. Ce dispositif ne contient pas de latex mais peut avoir été fabriqué dans un environnement qui en contient.

#### Événements indésirables

#### 5.1 Événements indésirables observés

Comme pour toutes les valvules cardiaques prothétiques, des événements indésirables graves pouvant parfois aller jusqu'au décès peuvent être associés à l'utilisation de valvules tissulaires. En outre, des événements indésirables découlant de la réaction du patient au dispositif implanté ou encore d'une modification physique ou chimique de ses composants, plus particulièrement de ceux dont l'origine est biologique, peuvent survenir à des intervalles variables (allant de plusieurs heures à plusieurs jours) et nécessitent une nouvelle opération pour remplacer la prothèse.

La conception de la bioprothèse aortique péricardique d'Edwards, modèle 11000A, est similaire à celle des bioprothèses péricardiques PERIMOUNT Magna Ease du modèle 3300TFX de Carpentier-Edwards.

Les événements indésirables associés à l'utilisation de bioprothèses péricardiques PERIMOUNT de Carpentier-Edwards et compilés à partir de documentation et de rapports provenant du système de surveillance du produit. conformément aux dispositions réglementaires américaines (fédérales) régissant les bonnes pratiques de fabrication (Good Manufacturing Practices. section 820.198), incluent la sténose, la régurgitation par une valve insuffisante. la fuite périvalvulaire, l'endocardite, l'hémolyse, la thrombo-embolie, l'obstruction thrombotique, la diathèse hémorragique associée à l'utilisation d'une anticoagulothérapie et la dysfonction de la valvule découlant d'une déformation de l'implant, d'une rupture du fil métallique ou d'une détérioration physique ou chimique des éléments de la valvule. Les types de détérioration des tissus pouvant survenir sont l'infection, la calcification, l'amincissement, la perforation, la dégénérescence, l'abrasion de la suture, le trauma causé par un instrument et le détachement de la valve des montants de l'endoprothèse. Ces complications peuvent se manifester de facon clinique, sous forme, par exemple, de souffle cardiaque anormal, d'essoufflement, d'intolérance à l'exercice, de dyspnée, d'orthopnée, d'anémie, de fièvre, d'arythmie, d'hémorragie, d'accident ischémique transitoire, d'accident vasculaire cérébral, de paralysie, de débit cardiaque faible, d'œdème pulmonaire, d'insuffisance cardiaque congestive, d'insuffisance cardiaque et d'infarctus du myocarde.

Remarque: selon des rapports issus de documentation sur des valvules tissulaires (téfs. 6, 7, 8, 9 et 10), la fréquence des calcifications de la valve serait supérieure chez les patients de moins de 20 ans. À cet égard, les recherches effectuées sur les animaux (téf. 11) démontrent qu'un niveau élevé de calcium dans le système peut entraîner une calcification précoce. En outre, au moins un rapport publié décrit la relation possible entre la consommation quotidienne de compléments de calcium et la calcification précoce de la valve chez l'adulte (réf. 13). Lorsque cela est possible, il faut éviter les injections intraveineuses répétées contenant du calcium pendant la période postopératoire. Parallèlement, la consommation excessive de lait ou de produits laitiers doit être évitée chez l'enfant. Il n'existe aucune donnée clinique démontrant la résistance accrue de la bioprothèse aortique péricardique d'Edwards, modèle 11000A, à la calcification, par rapport aux autres bioprothèses du marché.

#### 5.2 Événements indésirables potentiels

Les événements indésirables potentiels associés à l'utilisation de biovalvules cardiagues prothétiques sont les suivants :

- · Angine de poitrine
- · Diathèse hémorragique (coaqulopathie) en lien avec l'anticoaqulothérapie
- · Arythmie cardiague
- Blocage de la valvule ostiale coronaire
- Endocardite
- Insuffisance cardiague
- Hémolyse
- Anémie hémolytique
- Hémorragie
- · Infection locale et systémique
- Infarctus du mvocarde
- Inadaptation de la prothèse au patient
- · Enclavement de la valve prothétique (coincement)
- · Dysfonction non structurelle de la prothèse
- Pannus de la prothèse
- Fuite périvalvulaire de la prothèse
- Régurgitation de la prothèse
- Détérioration de la structure de la prothèse
- · Thrombose prothétique
- Accident vasculaire cérébral
- · Thrombo-embolie
- · Insuffisance cardiague congestive

Ces complications peuvent avoir les conséquences suivantes :

- Nouvelle opération chirurgicale
- Explantation
- Handicap permanent
- Décès

# 6. Études cliniques

# Cohorte de patients avec approbation préalable

Des données cliniques sur 719 patients ayant besoin isolément d'un remplacement de la valvule aortique (RVA) par la bioprothèse péricardique PERIMOUNT de Carpentier-Edwards, modèle 2700, avec suivi moyen de 3,9 années, indiquent un taux de survie global (calcul actuariel) de 73,7 % ± 2 % à la 6e année. Les données cliniques provenant de 70 patients ayant besoin d'un remplacement double de la valvule (RDV) avec suivi moyen de 3,7 années, indiquent un taux de survie global (calcul actuariel) de 67,2 % ± 6,5 % à la 6e année. Ces données sur une cohorte de patients avec approbation préalable ont été recueillies dans la période allant d'août 1981 à janvier 1989.

La population ayant subi isolément un RVA comprenait un total de 455 hommes (63,3 %) et de 264 femmes (36,7 %). Leur âge moyen ( $\pm$  l'écart-type) au moment de l'implantation était de 64 ans ( $\pm$  12,4), et ils étaient âgés de 18 à 90 ans. Les

indications pour le remplacement de la valvule étaient la sténose (63,4%), la régurgitation (16,3%), des maladies mixes (15,3%) et une dysfonction de la valvule aortique prothétique (5%).

La population ayant subi un RDV comprenait un total de 24 hommes (34,3 %) et de 46 femmes (65,7 %). L'âge moyen ( $\pm$  l'écart-type) était de 62,9 ans ( $\pm$  12,7), et ils étaient âgés de 31 à 94 ans. Les indications pour le remplacement de la valvule étaient la sténose (45,7 %), la régurgitation (25,7 %), des maladies mixes (21,4 %) et une dysfonction de la valvule aortique prothétique (7,4 %).

Les méthodes de suivi incluaient des visites à l'hôpital, des visites au cabinet et des communications par téléphone ou par lettre avec le patient, sa famille ou le médecin.

Le tableau 2 récapitule les taux de complications opératoires et postopératoires pour la population avec RVA isolé et pour la population ayant subi un RDV. Les taux de complications opératoires proviennent de 719 patients de la population ayant subi un RVA isolé et de 70 patients de la population ayant subi un RDV. Les taux de complications postopératoires se basent sur un suivi de 2767,9 et 255,8 années ayant eu lieu plus de 30 jours après les implantations chez la population ayant subi un RDV, respectivement.

Le tableau 3 présente les résultats de l'échocardiographie postopératoire des patients de la population de cette étude, par taille de valvule.

Les données sur la classification fonctionnelle préopératoire et postopératoire de la NYHA ont été recueillies pour la population ayant subi isolément un RVA. La classification fonctionnelle de la NYHA n'a pas été mentionnée pour 220 patients (171 patients décédés et 49 patients non disponibles). En ce qui concerne les 499 patients pour lesquels la classification fonctionnelle préopératoire et postopératoire de la NYHA a été mentionnée lors du dernier suivi disponible, la situation s'était empirée pour 10 d'entre eux (2 %), était inchangée pour 59 d'entre eux (11,8 %) et s'était améliorée pour 430 d'entre eux (86,2 %).

Le tableau 4 présente une comparaison des données de la classification fonctionnelle préopératoire de la NYHA avec celles de la classification postopératoire lors du dernier suivi.

#### Cohorte de patients avec approbation postérieure

Depuis novembre 1981, Edwards a suivi une cohorte approuvée postérieurement de 267 patients ayant subi un remplacement de la valvule (RVA) (modèle 2700), provenant de quatre centres de l'étude clinique d'origine de la bioprothèse péricardique PERIMOUNT de Carpentier-Edwards. Cette population était constituée de 171 hommes (64 %) et de 96 femmes (36 %). Leur âge moyen (± écart-type) au moment de l'implantation était de 64,9 ans ± 11,8 ans, et ils étaient âgés de 21 à 86 ans. En tout, 2407 années-patient de données étaient disponibles pour l'analyse (2386 d'années-patient tardives). Le suivi moyen était de 9 ± 5,5 ans, avec un maximum de 20,3 ans. En tout, on compte 189 décès entre 1981 et 1994, dont 48 (25,3 %) en lien établi avec la valvule. Les méthodes de suivi utilisées par chaque clinique incluaient des visites à l'hôpital, des visites au cabinet et des communications par téléphone ou par lettre avec le patient, sa famille ou le médecin.

Le tableau 5 résume la latitude découlant des taux de complications après 20 ans. La situation des patients à partir du dernier intervalle de suivi incluait 189 décédés (70,8 %), 10 vivants (3,8 %), 46 ayant subi une explantation (17,2 %) et 22 ayant quitir le suivi (8,2 %).

Cette population comptait 48 décès en lien avec la valvule. Un décès en lien avec la valvule est survenu au cours de la période de l'opération, par saignement. Sur les 28 décès postopératoires en lien avec la valvule, 5 découlaient de thromboembolie, 4 d'endocarditré/sepsie, 3 de détérioration de la structure de la valvule et 1 de saignement. Quinze autres décès ont été associés à la valvule à cause du manque d'information, ou parce qu'ils ont été dassés ainsi par le chercheur. Le calcul actuariel de la latitude des décès liés à la valvule donne  $67.9 \pm 6.6\%$  après 20 ans. Enfin, 19 autres décès sont reliés à une cause inconnue ou à une

mort subite, et pourraient avoir un lien avec la valvule. Par prudence, ces décès sont associés à la valvule. Par conséquent, la latitude actuarielle qui en découle pour les décès en lien avec la valvule sont de 55,4 ± 6,4 % après 20 ans.

Une amélioration dans la classification fonctionnelle de la NYHA a également été démontrée dans la période postopératoire. Jusqu'à l'évaluation du dernier suivi, 108 patients (44.8 %) faisaient partie de la classe fonctionnelle I de la NYHA.

Ces données sont été compilées à partir d'un essai clinique multicentre effectué par Edwards Lifesciences. Pour en savoir plus sur cet essai, communiquez avec Edwards Lifesciences S.A.R.L., Heart Valve Therapy Marketing Department, One Edwards Way. Irvine. CA 92614-5686.

#### Étude de confirmation

Entre les mois d'août 2003 et janvier 2004, 60 patients ayant besoin d'un remplacement de la valvule aortique (RVA) se sont vus implanter la bioprothèse aortique Magna PERIMOUNT de Carpentier-Edwards (modèle 3000) dans cinq établissements (deux en Europe et trois au Canada). Peu de temps après, le protocole a été modifié en vue d'autoriser l'implantation de la bioprothèse aortique Magna PERIMOUNT de Carpentier-Edwards (modèle 3000TFX), et d'ajouter trois établissements américains. Par la suite, 193 autres patients se sont vus implanter le modèle 3000TFX entre décembre 2004 et décembre 2006. À la différence du modèle 3000, le modèle 3000TFX est traité par le biais du processus ThermaFix.

La population ayant reçu le modèle 3000TFX comprenait un total de 116 hommes (60,1 %) et de 77 femmes (39,9 %). L'âge moyen au moment de l'implantation était de 72 ans (écart-type de ± 8,59) et ils étaient âgés de 26 à 89 ans. La principale indication pour le remplacement de la valvule était la sténose (78,2 %), suivie des maladies mixtes (14,5 %) et de la régurditation (7,3 %).

La population ayant reçu les modèles 3000 et 3000TFX comprenait un total de 150 hommes (59,3 %) et de 103 femmes (40,7 %). L'âge moyen au moment de l'implantation était de 72,2 ans (écart-type de ± 8,31) et ils étaient âgés de 26 à 89 ans. Ici encore, la principale indication pour le remplacement de la valvule était la sténose (77,5 %), suivie des maladies mixtes (15,4 %) et de la réquirditation (7,1 %).

Les patients étaient évalués avant l'opération, pendant l'opération, lors de la sortie, entre 3 et 6 mois, après un an, et chaque année par la suite. Le suivi cumulatif pour le modèle 3000TFX était de 167 années-patient, pour un suivi moyen de 0,9 année (écart-type = 0,42, plage = 0 à 2,1 années). Le suivi cumulatif pour les modèles 3000 et 3000TFX combinés était de 232 années-patient, avec un suivi moyen de 0,9 année (écart-type = 0,42, plage = 0 à 2,1 années).

Le tableau 6 récapitule les taux d'événements indésirables en lien avec la valvule et survenus au début (< 30) jours) et à la fin (> 30 jours) de la période postopératoire dans les populations ayant reçu le modèle 3000TFX et les modèles 3000 et 3000TFX combinés, respectivement.

Le tableau 7 illustre, par taille de valvule, les variables hémodynamiques signalées dans les échocardiogrammes effectués après un an chez les patients des études sur le modèle 3000TFX et sur les modèles 3000 et 3000TFX combinés.

Le tableau 8 présente le changement de classe fonctionnelle de la NYHA par rapport à l'évaluation de base de la visite après un an. Il convient de remarquer qu'une amélioration de 56,5 % a été signalée lors de la visite de un an dans la classification fonctionnelle de la population portant le modèle 3000TFX. En ce qui concerne les modèles 3000 et 3000TFX combinés, on constate une amélioration de 60,9 % dans la classification fonctionnelle au bout d'un an

Plusieurs études cliniques ayant été publiées démontrent la durabilité à long terme des bioprothèses aortiques péricardiques PERIMOUNT de Carpentier-Edwards, qui constituent la base sur laquelle les bioprothèses aortiques péricardiques Magna et Magna Ease PERIMOUNT de Carpentier-Edwards sont conçues (réfs. 14, 15, 16 & 17). De plus, des données publiées prouvent que la bioprothèse aortique Magna PERIMOUNT a un

rendement hémodynamique exceptionnel et ne présente qu'un risque très réduit d'inadaptation de la prothèse au patient (réfs. 18, 19, 20, 21, 22 & 23).

#### 7. Individualisation du traitement

Sauf indication contraire, les destinataires de la valvule bioprothétique doivent suivre une anticoagulothérapie pendant les premiers stades suivant l'implantation, selon les consignes données à chacun par le médecin. Une anticoagulothérapie ou un traitement antiplaquettaire doit être envisagé pour les patients montrant des facteurs de risque de thrombo-embolie.

Le jugement final concernant les soins pour un patient donné doit être pris par le fournisseur de santé et le patient à la lumière de l'ensemble de la situation que présente ce dernier (réf. 12). Il est recommandé de poser une bioprothèse en cas de RVA sur des patients de tous âges qui ne prennent pas de warfarine ou pour lesquels il existe une contre-indication importante à la thérapie à base de warfarine. Les préférences du patient sont également à prendre en compte dans une mesure raisonnable lors du choix de l'opération de la valvule aortique et de la valve prothétique. Il est raisonnable d'envisager l'implantation d'une prothèse mécanique pour un RVA de patients de moins de 65 ans pour lesquels l'anticoagulation n'est pas contre-indiquée. Il est également raisonnable d'envisager l'implantation d'une bioprothèse pour un RVA de patients de moins de 65 ans qui ont fait ce choix pour des raisons de mode de vie après avoir été informés dans les détails des risques de l'anticoagulation par rapport à l'éventuelle nécessité d'un deuxième RVA (réf. 12).

#### 7.1 Populations de patients spécifiques

L'innocuité et l'efficacité de la bioprothèse 11000A n'ont pas été établies pour les populations suivantes, sur lesquelles elles n'ont pas été étudiées :

- · patientes enceintes;
- · mères qui allaitent :
- patients métabolisant le calcium de manière anormale (p. ex., insuffisance rénale, hyperparathyroïdisme);
- patients présentant une insuffisance dégénérative anévrismale de l'aorte (p. ex.. nécrose médiale kystique, syndrome de Marfan);
- · enfants, adolescents et ieunes adultes.

Avertissement : selon des rapports issus de documentation sur des valvules tissulaires (réfs. 6, 7, 8, 9 et 10), la fréquence des calcifications de la valve serait supérieure chez les patients de moins de 20 ans. Lorsque cela est possible, il faut éviter les injections intraveineuses répétées contenant du calcium pendant la période postopératoire. Parallèlement, la consommation excessive de lait ou de produits laitiers doit être évitée chez l'enfant. À cet égard, les recherches effectuées sur les animaux (réf. 11) démontrent qu'un niveau élevé de calcium dans le système peut entraîner une calcification précoce.

# 8. Informations et conseils au patient

Il est conseillé de procéder à un suivi sérieux et continu (au moins par une visite annuelle chez le médecin) afin que les complications liées à la bioprothèse, et plus particulièrement aux problèmes de matériau, puissent faire l'objet d'un diagnostic et d'un traitement adaptés. Les patients porteurs de bioprothèses sont vulnérables à la bactériémie (p. ex., lors de procédures dentaires) et doivent recevoir des conseils concernant l'antibioprophylaxie. Enfin, il faut encourager les patients à porter en permanence leur carte d'identification et d'informer les fournisseurs dont ils sollicitent des soins qu'ils possèdent un implant.

#### 9. Présentation

#### 9.1 Conditionnement

La bioprothèse aortique péricardique d'Edwards, modèle 11000A, est fournie stérile et non pyrogène. Elle est livrée dans un emballage de plateau à double barrière placé dans un sachet métallisé, se trouvant lui-même dans un carton.

Chaque bioprothèse se trouve dans un carton avec un indicateur de température visible à travers une fenêtre sur le panneau latéral. Cet indicateur vise à repérer les produits exposés à des températures extrêmes transitoires. À la réception de la bioprothèse, inspecter immédiatement l'indicateur et consulter l'étiquette du carton pour confirmer l'état « Utiliser ». Si l'état « Utiliser » n'est pas apparent, ne pas se servir de la bioprothèse et contacter le fournisseur local ou le représentant d'Edwards Lifesciences pour prendre des arrangements en vue d'une autorisation de retour et d'un remplacement.

Mise en garde : inspecter soigneusement la bioprothèse avant l'implantation pour trouver des traces d'exposition à des températures extrêmes ou d'autres dégâts.

#### 9.2 Stockage

La bioprothèse aortique péricardique d'Edwards, modèle 11000A, doit être entreposée à une température comprise entre 10 °C et 25 °C (50 °F et 77 °F), dans son sachet métallisé et son carton de rangement.

#### 10. Directives d'utilisation

#### 10.1 Formation du médecin

Les techniques d'implantation de cette bioprothèse sont semblables à celles du placement supra-annulaire de n'importe quelle bioprothèse aortique avec endoprothèse. Aucune formation particulière n'est nécessaire pour implanter la bioprothèse aortique péricardique d'Edwards, modèle 11000A.

#### 10.2 Choix de la taille

Vérifier que les accessoires ont été stérilisés conformément aux recommandations fournies avec les articles réutilisables.

#### Mesure supra-annulaire

Pour l'implantation supra-annulaire, l'anneau de suture de la bioprothèse est placé au-dessus de l'annulus, maximisant ainsi la zone de l'orifice de la valve. Lors de la mesure pour une implantation supra-annulaire, le calibreur doit être placé parallèlement au plan de l'annulus et il faut utiliser la technique de mesure suivante:

| Étape | Procédure |
|---|---|
| 1 | À l'aide du calibreur de modèle 1133, sélectionner l'embout<br>cylindrique du calibreur ayant le diamètre le plus large qui<br>s'adapte confortablement dans l'annulus du patient. |
| | HVT21 |

| Étape Procédure | |
|---|---|
| 2 | Une fois que l'embout cylindrique approprié a été vérifié, utiliser l'embout de réplique du même calibreur afin de vérifier que l'anneau de suture s'adapte bien sur le dessus de l'annulus. S'assurer que l'ostium coronaire n'est pas bloqué et que les montants de l'endoprothèse du bout de réplique n'interfèrent pas avec la paroi aortique à la jonction sinotubulaire. Si l'embout de réplique convient. Choisir cette taille de |
| | bioprothèse pour l'implantation. |

HVT37



#### 10.3 Instructions de manipulation et de préparation

Il est conseillé de suivre une formation sur le tas avant de manipuler et de préparer la bioprothèse aortique péricardique d'Edwards, modèle 11000A.

| Étape | Procédure |
|---|---|
| 1 | Avertissement : ne pas ouvrir pas l'emballage du<br>modèle 11000A de la bioprothèse aortique péricardique<br>d'Edwards avant d'avoir l'assurance que l'implantation<br>aura lieu. |
| | Mise en garde : Ne pas ouvrir le sachet métallisé dans une<br>zone stérile. Ce sachet ne sert qu'à protéger la<br>bioprothèse. Seul l'emballage le plus à l'intérieur peut<br>pénétrer dans la zone stérile. |
| | Une fois que la bonne taille de bioprothèse a été choisie, retirer le<br>sachet métallisé du carton dans la zone non stérile. Avant<br>d'ouvrir, examiner l'emballage pour vérifier s'il y a des<br>dommages et des scellés cassés ou manquants. |
| 2 | Près de la zone stérile, tenir la base du plateau extérieur et retirer son couvercle. |

| Étape | Procédure |
|---|---|
| 3 | Le plateau intérieur et son contenu sont stériles. Transférer le<br>plateau interne sur la zone stérile. Le contenu du plateau<br>intérieur doit être manipulé en utilisant une technique<br>chirurgicale stérile afin d'empêcher la contamination. |
| | HVT26 |
| 4 | Avertissement : ne pas ouvrir pas l'emballage intérieur<br>avant d'avoir l'assurance que l'implantation aura lieu et<br>que le chirurgien est prêt à mettre la valvule en place. |
| | Avertissement : la bioprothèse n'est pas fixée sur le<br>plateau intérieur. Il faut faire attention en ouvrant le<br>couvercle et en tirant sur la languette en plastique. |
| | Avant d'ouvrir, examiner le plateau intérieur et le couvercle<br>pour vérifier s'il y a des dommages, des tâches et des scellés<br>cassés ou manquants. Tenir la base du plateau intérieur et<br>retirer son couvercle. |



# Étape Procédure Étape Procédure Fixer la poignée (modèle 1111 ou 1126) au support de la Pour retirer le clip de la bioprothèse, saisir le clip et le retirer de bioprothèse alors que cette dernière se trouve toujours dans le l'assemblage poignée/support. plateau. Pour la fixer, insérer la poignée sur le support et la HVT33 tourner vers la droite jusqu'à sentir une résistance. Avertissement : ne pas saisir la bioprothèse avec les mains ou des instruments chirurgicaux. Avertissement : ne pas retirer la bioprothèse du dip lorsque la poignée est fixée au support. Avertissement : l'assemblage poignée/support est nécessaire à l'implantation et ne doit pas être retiré jusqu'à ce que la bioprothèse soit suturée sur l'annulus. Avertissement : il faut éviter d'enchevêtrer l'étiquette avec le numéro de série dans la poignée lors de la fixation. HVT31 Poignée Support HVT34 Une fois la poignée fixée, retirer la bioprothèse et le clip du plateau intérieur. HVT32 Une étiquette avec le numéro de série est fixée à l'anneau de suture de chaque bioprothèse par une suture. Ce numéro de série doit être comparé avec le numéro se trouvant sur l'emballage de la bioprothèse et sur la carte de données d'implantation de la bioprothèse. L'étiquette ne doit pas être détachée de la bioprothèse jusqu'à ce que l'implantation soit sûre. Avertissement : si les numéros de série sont différents, la bioprothèse doit être renvoyée sans avoir été utilisée. Avertissement : il faut faire attention en coupant ou déchirant le tissu de l'anneau de suture lorsque l'étiquette du numéro de série est retirée. Avertissement : pour éviter d'endommager le tissu de

l'anneau de suture, ne pas tirer sur la suture à travers

l'anneau.

| Étape | Procédure |
|---|---|
| 10 | IL EST INUTILE DE RINCER la bioprothèse aortique<br>péricardique d'Edwards, modèle 11000A, avant l'implantation. |
| | Avertissement : si la bioprothèse est rincée avant<br>l'implantation, elle doit être ensuite conservée<br>hydratée à l'aide d'une irrigation saline physiologique<br>stérile sur les deux côtés du tissu de la valve pendant<br>toute la durée de la procédure chirurgicale. Il est<br>recommandé de la rincer toutes les une à deux minutes.<br>Avertissement : éviter que le tissu de la valve entre en<br>contact avec des serviettes, des linges ou d'autres |
| | sources de particules susceptibles de s'y transférer. |

#### 10.4 Implantation du dispositif

| a bioprothèse aortique péricardique d'Edwards, modèle 11000A, est conçue<br>our une implantation supra-annulaire. | |
|---|---|
| Étape | Procédure |
| 1 | Le chirurgien doit être familier avec les recommandations<br>concernant la mesure et le positionnement supra-annulaire<br>(voir la section <b>10.2 Choix de la taille.</b> ) |
| | À cause de la complexité et de la variété du remplacement<br>chirurgical de la valve cardiaque, le choix de la technique<br>chirurgicale, correctement modifiée selon les <b>mises en garde</b><br>décrites précédemment, est à la discrétion du chirurgien<br>individuel. En général, les étapes suivantes doivent être suivies : |
| | Retirer par chirurgie les valves malades ou endommagées<br>ainsi que toutes les structures associées au besoin. |
| | Retirer par chirurgie le calcium de l'annulus afin d'assurer un<br>bon positionnement de l'anneau de suture de la bioprothèse<br>pour éviter d'endommager le tissu délicat de la valve. |
| | <ol> <li>Mesurer l'annulus à l'aide des calibreurs aortiques<br/>Carpentier-Edwards de modèle 1133 (figures 1a-1c).</li> </ol> |
| | Avertissement: lors d'un choix d'une bioprothèse, il faut<br>prendre en compte la taille, l'âge et l'état physique par<br>rapport à la taille de la bioprothèse, afin de minimiser le<br>risque d'hémodynamique sous-optimale. Toutefois, le<br>choix final revient au médedn individuellement après<br>l'évaluation des risques et des avantages pour le patient. |
| | Avertissement: ne pas utiliser les calibreurs de prothèse d'autres fabricants ou des calibreurs de toute autre bioprothèse Edwards Lifesciences pour mesurer la bioprothèse aortique péricardique d'Edwards, modèle 11000A. |
| | Avertissement : vérifier si les calibreurs contiennent des<br>traces d'eau, telles que des ternissures, des fissurations<br>ou des craquelures. Remplacer le calibreur si des<br>détériorations sont observées. |
| | Mise en garde : les fragments des poignées et des<br>calibreurs ne sont pas radio-opaques et ne peuvent pas<br>ètre trouvés par un imageur externe. |

#### Étape Procédure

Il faut utiliser une technique de suture pour l'emplacement de l'annulus supérieur de la bioprothèse, telle que la technique du matelas horizontal à point simple interrompu. En cas de suture dans l'anneau de suture de la bioprothèse aortique péricardique d'Edwards, modèle 11000A, il est recommandé que les sutures passent dans l'anneau de suture aussi près que possible de la structure de la bioprothèse.

Une fois que les sutures sont entièrement nouées, il est important de couper les sutures près des nœuds pour s'assurer que les fils de suture exposés n'entrent pas en contact avec le tissu de la valve de la bioprothèse.

HVT35



- 3 Le support intégral et la poignée attachée sont retirés comme une unité à la fin de la procédure de suture.
  - À l'aide d'un scalpel, couper chacune des trois sutures exposées qui se trouvent sur le dessus du support.

HVT36



Avertissement : éviter de couper ou d'endommager l'endoprothèse ou le tissu délicat de la valve lorsque les sutures sont coupées.

- 2. Après avoir coupé les trois sutures du support, retirer ensemble l'assemblage poignée/support, ainsi que les sutures du support, de la bioprothèse.
- 3. Retirer la poignée du support et jeter ce dernier.

#### 10.5 Nettoyage et stérilisation des accessoires

Les accessoires de la bioprothèse aortique péricardique d'Edwards, modèle 11000A, sont emballés à part. La poignée du modèle 1126 est stérile et est destinée à un usage unique. La poignée du modèle 1111 et les calibreurs du modèle 1133 ne sont pas stériles et doivent être stérilisés avant l'utilisation. Les poignées, les calibreurs, la base et le couvercle du plateau doivent être nettoyés et restérilisés avant chaque utilisation. Consulter le mode d'emploi fourni avec les accessoires réutilisables pour connaître les consignes de nettovage et de stérilisation.

#### 10.6 Retour de la bioprothèse

Edwards Lifesciences est intéressé à obtenir des échantillons cliniques recouverts de la bioprothèse aortique péricardique d'Edwards, modèle 11000A, à des fins d'analyse. Pour retourner des bioprothèses recouvertes, contacter votre représentant.

- Emballage non ouvert avec la barrière stérile intacte: si le sachet métallisé ou les plateaux n'ont pas été ouverts, retourner la bioprothèse dans son emballage d'origine.
- Emballage ouvert, mais avec la bioprothèse non implantée: si le plateau est ouvert, la bioprothèse n'est plus stérile. Si la bioprothèse n'est pas implantée, elle doit être placée dans un fixateur histologique adapté comme di formaldéhyde à 10 % ou du glutaraldéhyde à 2 %, puis retournée à l'entreprise. La réfrigération n'est pas nécessaire dans ces circonstances.
- Bioprothèse explantée: la bioprothèse explantée doit être placée dans un fixateur histologique adapté comme di formaldéhyde à 10 % ou du glutaraldéhyde à 2 %, puis retournée à l'entreprise. La réfrigération n'est pas nécessaire dans ces dirconstances.

# Sécurité dans l'environnement de résonance magnétique (RM)



#### Condition RM

Des tests non cliniques ont montré que la bioprothèse aortique péricardique d'Edwards, modèle 11000A, est conforme à la condition RM. Un patient la possédant peut subir un balayage sans danger immédiatement après l'implantation, dans les conditions suivantes :

- Champ magnétique statique de 1,5 ou 3 tesla.
- Gradient de champ magnétique spatial maximum de 2670 gauss/cm.
- Taux d'absorption spécifique moyen signalé par le système RM pour tout le corps de 2 W/kg en mode de fonctionnement normal pour un balayage de 15 par séquence.

En essai non clinique, la bioprothèse aortique péricardique d'Edwards, modèle 11000A, a produit une élévation maximale estimée de température in vivo inférieure ou égale à 1,8 °C a un taux d'absorption spécifique moyen signalé par le système RM pour tout le corps de 2 W/kg en mode de fonctionnement normal pour un balayage de 15 par séquence, dans un circuit RF Signa de GE de 64 MHz (1,5 T) et un système MR Signa HDx de GE (3 T) équipé de la version logicielle 15\LX\MR, édition 15.0.\Mc.0910.a.

L'artéfact d'image a été mesuré de manière non dinique dans un système RM Signa HDx de GE (3T) conformément à la norme ASTM F2119-07, à l'aide d' un écho de spin et des séquences d'écho de gradient indiquées dans ce document. Les images d'écho de spin montraient des artéfacts clairs et foncés allant jusqu'à 40 mm de l'implant et bouchant la lumière de manière partielle à complète. Les images d'écho de gradient montraient des artéfacts opaques clairs et foncés et des artéfacts triangulaires foncés allant jusqu'à 40 mm de l'implant et bouchant la lumière de manière partielle à complète. Il est possible de procéder à une réduction dans l'artéfact à l'aide de séquences conçues pour réduire les artéfacts de métal.

#### 12. Informations du patient

#### 12.1 Carte d'identification de la recherche

Une carte d'identification de la recherche est donnée à chaque sujet sur qui a été implantée la bioprothèse aortique péricardique d'Edwards, modèle 11000A.

#### 12.2 Documents d'informations du patient

Il est possible d'obtenir des documents d'informations du patient d'Edwards ou de l'un de ses spécialistes des ventes cliniques.

#### 13. Références

- Carpentier, A., et al. Biological Factors Affecting Long Term Results of Valvular Heterografts. J Thorac Cardiovasc Surg 1969, 58:467-483.
- Carpentier, A., et al. Six Year Follow-up of Glutaraldehyde Preserved Heterografts. J Thorac Cardiovasc Surg 1974, 68:771-782.
- Reis, Robert L., et al. The Flexible Stent. A New Concept in the Fabrication of Tissue Heart Valve Prostheses. J Thorac Cardiovasc Surg 1971, 62(5):683-689 and 693-695.
- Barratt-Boyes, B.G. and A.H.G. Roche. A Review of Aortic Valve Homografts Over a Six and One-half Year Period. Ann Surg 1969, 170:483-492.
- Brewer, R.J., et al. The Dynamic Aortic Root. Its Role in Aortic Valve Function. J Thorac Cardiovasc Surg 1976, 72:413-417.
- Jamieson, W.R.E., et al. Carpentier-Edwards Standard Porcine Bioprosthesis: Primary Tissue Failure (Structural Valve Deterioration) by Age Groups. Ann Thorac Sura 1988. 46:155-162.
- Odell, J.A. Calcification of Porcine Bioprostheses in Children. In Cohn, L. and V. Gallucci (eds): Cardiac Bioprostheses. Yorke Medical Books. New York, 1982, pp 231-237.
- Reul, G.J., et al. Valve Failure with the lonescu-Shiley Bovine Pericardial Bioprosthesis: Analysis of 2680 Patients. J Vasc Surq 1985, 2(1):192-204.
- Sanders, S.P., et al. Use of Hancock Porcine Xenografts in Children and Adolescents. Am J Cardiol 1980, 46(3):429-438.
- Silver, M.M., et al. Calcification in Porcine Xenograft Valves in Children. Am J Cardiol 1980, 45:685-689.
- Carpentier, A., et al. Continuing Improvements in Valvular Bioprostheses. *J Thorac Cardiovasc Sura* 1982, 83(1):27-42.
- Bonow R.O., et al. ACC/AHA Guidelines for the Management of Patients with Valvular Heart Disease: A Report of the American College of Cardiology/ American Heart Association Task Force on Practice Guidelines (Committee on Management of Patients With Valvular Heart Disease). J Am Coll Cardiol 2006, 48:e1-148.
- Moront, M.G. and N.M. Katz. Early Degeneration of a Porcine Aortic Valve Bioprosthesis in the Mitral Valve Position in an Elderly Woman and its Association with Long-Term Calcium Carbonate Therapy. Am J Cardiol 1987, 59:1006–1007.
- Aupart, M.R., et al. Perimount Pericardial Bioprosthesis for Aortic Calcified Stenosis: 18-Year Experience with 1,133 Patients. J Heart Valve Dis 2006, 15:768-776.
- Dellgren, G., et al. Late Hemodynamic and Clinical Outcomes of Aortic Valve Replacement with the Carpentier-Edwards Perimount Pericardial Bioprosthesis. J Thorac Cardiovasc Surg 2002, 124:146-154.
- Frater, R.W.M., et al. Long-Term Durability and Patient Functional Status of the Carpentier-Edwards Perimount Pericardial Bioprosthesis in the Aortic Position. J Heart Valve Dis 1998, 7:48-53.
- Jamieson, W.R.E., et al. 15-Year Comparison of Supra-Annular Porcine and PERIMOUNT Aortic Bioprostheses. Asian Cardiovasc Thorac Ann 2006, 14:200-205
- Borger, M.A., et al. Carpentier-Edwards Perimount Magna Valve Versus Medtronic Hancock II: A Matched Hemodynamic Comparison. Ann Thorac Surg 2007; 83:2054-2058.
- Botzenhardt, F., et al. Hemodynamic Comparison of Bioprostheses for Complete Supra-Annular Position in Patients With Small Aortic Annulus. JAm Coll Cardiol 2005. 45:2054-2060.
- Botzenhardt, F., et al. Hemodynamic Performance and Incidence of Patient-Prosthesis Mismatch of the Complete Supraanular Perimount Magna Bioprosthesis in the Aortic Position. *Thorac Cardiov Surg* 2005, 53:226–230.
- Dalmau, M.J., et al. The Carpentier-Edwards Perimount Magna Aortic Xenograft: A New Design with an Improved Hemodynamic Performance. Interact Cardiovasc Thorac Surg 2006, 5:263-267.
- Totaro, P., et al. Carpentier-Edwards PERIMOUNT Magna Bioprosthesis: A Stented Valve with Stentless Performance? J Thorac Cardiovasc Surg 2005, 130:1668-1674.
- Wagner, I.M., et al. Influence of Completely Supra-annular Placement of Bioprostheses on Exercise Hemodynamics in Patients With a Small Aortic Annulus. J Thorac Cardiovascular Surg 2007; 133:1234-1241.

Ce produit est fabriqué et distribué selon au moins un des brevets américains suivants: Nos de brevets américains 5,928,281; 5,931,969; 5,961,549; 6,102,944; 6,245,105; 6,413,275; 6,561,970; 6,585,766; 6,837,902; 6,945,997; 7,214,344; 7,972,376; 8,007,992; 8,357,387; 8,366,769; 8,632,608; et RE 40570; ainsi que les brevets étrangers correspondants. De plus, des brevets supplémentaires sont en attente.

Se référer à la légende des symboles à la fin du document.

Tableau 2 - Récapitulation des taux de complications, modèle 2700

| | Population ayant subi isolémentun RVA | | | Рори | Population ayant subi un RDV | |
|---|---|---|---|---|---|---|
| Complication | Opératoires<br>% de pt | Post<br>Opératoires<br>% par année-<br>patient | % sans<br>événement<br>après 6 ans<br>(écart-type) | Opératoires<br>% de pt | Post<br>Opératoires<br>% par année-<br>patient | % sans<br>événement<br>après 6 ans<br>(écart-type) |
| Décès | 4,7 | 4,6 | 73,5 (2,0) | 12,9 | 4,2 | 67,2 (6,5) |
| Explantation | 0 | 0,3 | 98,5 (1,0) | 0 | 0,8 | S.O.* |
| Nouvelle opération en lien avec la valvule | 0,7 | 0,1 | 99,8 (0,4) | 0 | 0 | S.O.* |
| Toutes les nouvelles opérations | 22,4 | 1,8 | 75,4 (1,8) | 34,3 | 2,3 | S.O.* |
| Thrombo-embolie en lien avec la valvule | 3,1 | 1,5 | 91,4 (1,1) | 1,4 | 5,1 | S.O.* |
| Toutes les thrombo-embolies | 5,0 | 2,4 | 84,9 (1,6) | 5,7 | 6,6 | S.O.* |
| Endocardite | 0,6 | 0,8 | 95,8 (0,9) | 1,4 | 1,5 | S.O.* |
| Dysfonction de la valvule | 0,1 | 0,7 | 96,0 (1,1) | 0 | 0,4 | S.O.* |
| Fuite périvalvulaire | 0,1 | 0,3 | 98,8 (0,5) | 0 | 1,2 | S.O.* |
| Complication hémorragique anticoagulation | 1,4 | 0,4 | 96,4 (1,1) | 4,3 | 2,3 | S.O.* |
| Hémolyse | 0 | 0,2 | 99,1 (0,4) | 0 | 0,4 | S.O.* |
| Thrombose de la valvule | 0 | 0 | 100,0 (0) | 0 | 0,4 | S.O.* |

<sup>\*</sup> S.O. = sans objet

Tableau 3 - Résultats de l'échocardiographie postopératoire, modèle 2700

| | Taille de la valvule | | | | | | |
|---|---|---|---|---|---|---|---|
| | 19 mm | 21 mm | 23 mm | 25 mm | 27 mm | 29 mm | Total |
| Total N | 12 | 22 | 15 | 8 | 3 | 3 | 63 |
| Moyenne des mois<br>après l'opération | 28,6 ± 7,2 | 34,9 ± 8,6 | 36,9 ± 9,2 | 39,9 ± 7,6 | 31,4 ± 15,9 | 15,3 ± 12,2 | 34,6 ± 9,2 |
| Vélocité (M/s) | | | | | | | |
| moyen $\pm$ ET. | $2,80 \pm 0,49$ | $2,\!56\pm0,\!46$ | $2,36 \pm 0,42$ | $2,15\pm0,56$ | $2,09 \pm 0,27$ | $2,08 \pm 0,1$ | $2,46 \pm 0,50$ |
| n = | 12 | 21 | 15 | 7 | 3 | 3 | 61 |
| Plage | 1,90 - 3,60 | 1,90 - 3,90 | 1,39 - 2,86 | 1,00 - 2,60 | 1,90 - 2,40 | 2,05 - 2,10 | 1,00 - 3,90 |
| Gradient instantané<br>de crête (mmHg) | | | | | | | |
| moyen $\pm$ ET. | $32,22 \pm 11,08$ | $27,04 \pm 10,49$ | $23,00 \pm 7,30$ | $19,50 \pm 8,16$ | $17,60 \pm 4,70$ | $14,4 \pm 0,58$ | 25,67 ± 10,14 |
| n = | 12 | 21 | 15 | 7 | 3 | 3 | 61 |
| Plage | 14,40 - 51,80 | 14,40 - 60,80 | 7,70 - 32,70 | 4,00 - 27,00 | 14,40 - 23,00 | 13,95 - 15,06 | 4,00 - 60,80 |

Tableau 4 - Résultats en matière d'efficacité, classification fonctionnelle de la NYHA, modèle 2700

| Préopératoire Classification<br>fonctionnelle de la NYHA | | postopératoire<br>Classification fonctionnelle de la NYHA | | | | |
|---|---|---|---|---|---|---|
| | I | II | III | IV | Décès | Non disponible |
| I | 18 | 19 | | | 9 | |
| II | 140 | 37 | | | 35 | 15 |
| III | 181 | 48 | 4 | 1 | 72 | 24 |
| IV | 43 | 16 | 2 | | 53 | 2 |
| Non disponible | 5 | 1 | | | 2 | 2 |

Tableau 5 - Latitude concernant les taux de complications après 20 ans (N = 267), modèle 2700

| Réelle | Actuarielle | Linéarisée<br>(%/année-patient) |
|---|---|---|
| 85,8 ± 2,5% | 67,9 ± 6,6% | 1,2 |
| $82,4 \pm 2,6\%$ | $68,2 \pm 6,8\%$ | 1,7 |
| $94,0 \pm 1,5\%$ | 91,7 ± 2,2% | 0,4 |
| 91,7 ± 1,7% | 89,3 ± 2,4% | 0,8 |
| $92,6 \pm 2,0\%$ | 77,1 ± 7,2% | n.p.* |
| $96,3 \pm 1,6\%$ | $81,5 \pm 9,6\%$ | |
| $96.0 \pm 2.3\%$ | $69,9 \pm 20,5\%$ | |
| | $85,8 \pm 2,5\%$<br>$82,4 \pm 2,6\%$<br>$94,0 \pm 1,5\%$<br>$91,7 \pm 1,7\%$<br>$92,6 \pm 2,0\%$<br>$96,3 \pm 1,6\%$ | $85,8 \pm 2,5\%$ $67,9 \pm 6,6\%$ $82,4 \pm 2,6\%$ $68,2 \pm 6,8\%$ $94,0 \pm 1,5\%$ $91,7 \pm 2,2\%$ $91,7 \pm 1,7\%$ $89,3 \pm 2,4\%$ $92,6 \pm 2,0\%$ $77,1 \pm 7,2\%$ $96,3 \pm 1,6\%$ $81,5 \pm 9,6\%$ |

<sup>\*</sup> Non pertinent. La DSV ne relève pas d'une fonction de risque constante. Par conséquent, les taux linéarisés ne sont pas significatifs.

Tableau 6 - Résumé des événements indésirables en lien avec la valvule, modèles 3000 et 3000TFX

| | ≤ 30 jours après l'opération | | > 30 jours ap | rès l'opération |
|---|---|---|---|---|
| Événements indésirables | 3000TFX<br>(N = 193)<br>Nbre d'événements<br>(% de patients) | 3000/3000TFX<br>(N = 253)<br>Nbre d'événements<br>(% de patients) | 3000TFX<br>(N = 193)<br>Nbre d'événements<br>(% de patients) | 3000/3000TFX<br>(N = 253)<br>Nbre d'événements<br>(% de patients) |
| Thrombo-embolies en lien avec la valvule | 6 (3,1) | 7 (2,8) | 3 (2,0) | 3 (1,4) |
| Dysfonction non structurelle de la valvule (PVL) | 3 (1,5) | 4 (1,6) | 3 (2,0) | 3 (1,4) |
| Explantation (DNSV) | 2 (1,0) | 2 (0,8) | 0 (0,0) | 0 (0,0) |
| Décès (arrêt cardiaque, saignement, AVC) | 1 (0,5) | 1 (0,4) | 3 (2,0) | 3 (1,4) |
| Nouvelle opération chirurgicale | 1 (0,5) | 1 (0,4) | 1 (0,7) | 1 (0,5) |
| Hémolyse | 1 (0,5) | 1 (0,4) | 3 (2,0) | 3 (1,4) |
| Saignement en lien avec l'AC | 0 (0,0) | 0 (0,0) | 2 (1,4) | 2 (1,0) |
| Endocardite | 0 (0,0) | 0 (0,0) | 0 (0,0) | 0 (0,0) |
| Détérioration de la structure de la valvule | 0 (0,0) | 0 (0,0) | 0 (0,0) | 0 (0,0) |
| Thrombose de la valvule | 0 (0,0) | 0 (0,0) | 0 (0,0) | 0 (0,0) |
| Autre (déchirure de l'aorte) | 1 (0,5) | 1 (0,4) | 0 (0,0) | 0 (0,0) |

Tableau 7 - Variables hémodynamiques à l'évaluation échographique du suivi d'un an, modèles 3000 et 3000TFX

| Type de valvule | Variable | 19 mm<br>Moyenne ±<br>écart-type (N) | 21 mm<br>Moyenne ±<br>écart-type (N) | 23 mm<br>Moyenne ±<br>écart-type (N) | 25 mm<br>Moyenne ±<br>écart-type (N) | 27 mm<br>Moyenne ±<br>écart-type (N) | 29 mm<br>Moyenne ±<br>écart-type (N) |
|---|---|---|---|---|---|---|---|
| 3000TFX | Gradient systolique | 16,7 ± 4,7 | 15,8 ± 4,4 | 11,3 ± 3,7 | 11,1 ± 4,1 | 9,4 ± 4,3 | 9,0 ± 0,0 |
| | moyen (mmHg) | (10) | (18) | (45) | (37) | (12) | (2) |
| | Fraction | 65,8 ± 10,4 | 62,7 ± 9,4 | 60,6 ± 11,3 | 61,4 ± 11,2 | 59,5 ± 10,7 | 55,0 ±14,1 |
| | d'éjection (%) | (10) | (19) | (48) | (38) | (12) | (2) |
| | Aire valvulaire efficace | 1,2 ± 0,4 | 1,5 ± 0,4 | 1,8 ± 0,6 | 1,8 ± 0,5 | 2,1 ± 0,6 | 2,1 ± 0,1 |
| | de l'aorte (cm²) | (10) | (18) | (44) | (36) | (12) | (2) |
| 3000/ | Gradient systolique | 16,7 ± 4,2 | 13,8 ± 4,8 | 11,7 ± 4,7 | 11,0 ± 3,8 | 9,5 ± 4,1 | 9,0 ± 0,0 |
| 3000TFX | moyen (mmHg) | (16) | (34) | (56) | (47) | (14) | (2) |
| | Fraction | 62,1 ± 15,1 | 58,6 ± 11,6 | 60,2 ± 11,2 | 60,2 ± 11,5 | 58,5 ± 10,5 | 55,0 ± 14,1 |
| | d'éjection (%) | (16) | (34) | (59) | (47) | (14) | (2) |
| | Aire valvulaire efficace | 1,3 ± 0,5 | 1,5 ± 0,4 | 1,8 ± 0,6 | 1,8 ± 0,6 | 2,1 ± 0,6 | 2,1 ± 0,1 |
| | de l'aorte (cm²) | (16) | (32) | (55) | (46) | (14) | (2) |

Tableau 8 - Classe fonctionnelle de la NYHA : changement par rapport à l'évaluation de base lors de la visite de un an, modèles 3000 et 3000TFX

| | | | | -Évaluation de base- | | |
|---|---|---|---|---|---|---|
| Type de valvule | Suivi de la<br>classification NYHA | Classe I | Classe II | Classe III | Classe IV | S.O. |
| | Classe I | 10 | 33 | 51 | 10 | 3 |
| | Classe II | 2 | 8 | 13 | 2 | 1 |
| 2000 | Classe III | - | - | 3 | - | - |
| 3000TFX | Classe IV | - | - | - | 1 | - |
| N = 193 | Décès | - | 3 | 16 | 1 | - |
| | Explantation | - | - | 3 | - | - |
| | S.O. | 2 | 6 | 21 | 4 | - |
| | Classe I | 12 | 40 | 71 | 11 | 3 |
| | Classe II | 2 | 14 | 29 | 3 | 1 |
| 3000/ | Classe III | - | - | 3 | - | - |
| 3000TFX | Classe IV | - | - | 1 | 1 | - |
| N = 253 | Décès | - | 3 | 19 | 2 | - |
| | Explantation | - | - | 3 | - | - |
| | S.O. | 2 | 7 | 22 | 4 | - |

#### Classe de fonctionnement de la NYHA : changement par rapport à l'évaluation de base lors de la visite de un an

| Type de valvule | Amélioration<br>N (%) | ldentique<br>N (%) | Aggravation<br>N (%) | S.O.<br>N (%) |
|---|---|---|---|---|
| 3000TFX (N = 193) | 109 (56,5) | 22 (11,4) | 2 (1,0) | 60 (31,1) |
| 3000/3000TFX (N = 253) | 154 (60,9) | 30 (11,9) | 3 (1,2) | 66 (26,1) |

# Osierdziowa bioproteza aortalna Edwards model 11000A

# Instrukcja użytkowania

PRZESTROGA: Urządzenie badawcze. Prawo federalne. (Stanów Zjednoczonych Ameryki) ogranicza użytkowanie tego przyrządu do celów badawczych.

PRZESTROGA: Urządzenie badawcze. Wyłącznie do badań klinicznych.

Przestroga: Urządzenie badawcze. Przeznaczone wyłącznie do celów badawczych. Do stosowania wyłącznie przez wykwalifikowanych badaczy (lekarzy).

#### Opis urządzenia i akcesoriów

#### 1.1 Opis urządzenia

Osierdziowa bioproteza aortalna Edwards model 11000A jest trójpłatkową bioprotezą wykonaną z odpowiednio przygotowanego wołowego osierdzia, umocowaną na elavycznej ramie. Bioproteza jest dostępna w rozmiarach 19, 21, 23, 25, 27 i 29 mm (tabela 1). Bioproteza jest przechowywana w opakowaniu niewodnym i nie wymaga przemywania przed wszczepieniem.



Edwards Lifesciences, logo stylizowanej litery E, Carpentier-Edwards, ThermaFix, TFX, PERIMOUNT, PERIMOUNT Magna i Magna Ease to znaki towarowe firmy Edwards Lifesciences Corporation. Prowadnica druciana jest wykonana ze stopu kobaltowo-chromowego i jest pokryta tkaniną poliestrową. Stop kobaltowo-chromowy/warstwa laminatu poliestrowego otacza podstawe ramy prowadnicy drucianej.

Silikonowy pierścień do wszywania pokryty porowatym politetrafluoroetylenem (PTFE) jest przymocowany do ramy prowadnicy drucianej. Pierścień do wszywania ma trzy czarne jedwabne oznaczenia szwów rozmieszczone w równych odległościach w środku zastawki w celu ułatwienia ustawienia bioprotezy i założenia szwów.

Uchwyt jest dołączony do bioprotezy za pomocą szwów w celu ułatwienia obchodzenia się z bioprotezą i jej wszycia w trakcie implantacji. Uchwyt może zostać łatwo odłaczony przez chirurga. (Patrz 10.4 Implantacja urzadzenia)

#### 1.2 Opis akcesoriów

#### Kalibratory i taca

Zastosowanie kalibratora ułatwia wybór prawidłowego rozmiaru bioprotezy do implantacji. Półprzezroczysty model kalibratorów 1133 umożliwia bezpośrednią obserwację ich dopasowania w obrębie pierścienia. Każdy kalibrator składa się z rekojeści z różną konfiguracją narzędzi pomiarowych na każdym zakończeniu (Rysunek 1a). Na jednym końcu rękojeści znajduje się zakończenie cylindryczne z wchodzącą w jego skład krawędzią, która odzwierciedla geometrię pierścienia do wszywania bioprotezy (Rysunek 1b). Na jej drugim końcu znajduje się zakończenie replikujące bioprotezy, które odzwierciedla zarówno geometrię pierścienia do wszywania, jak i wysokość oraz lokalizację wsporników stentu (Rysunek 1c). Kalibrator jest dostępny dla każdego rozmiaru bioprotezy model 11000A (19, 21, 23, 25, 27 i 29 mm). Kompletny zestaw kalibratorów jest umieszczony na tacy model TRAY1133, która może zostać ponownie wykorzystana i wysterylizowana.

Rysunek 1a. Kalibrator aortalny

Rysunek 1b.



Zakończenie cylindryczne Zakończenie replikujące

HVT17

HVT18

Rysunek 1c.

#### Uchwyt i rękojeść bioprotezy

Zespół uchwyt/rękojeść składa się z dwóch części: integralnej, jednorazowej części, fizycznie przymocowanej do bioprotezy przez producenta oraz giętkiej rękojeści (model 1111 do wielokrotnego użytku lub jednorazowy model 1126), dołączanej do uchwytu w czasie operacji (Rysunki Za i 2b).

#### Rysunek 2a. Rękojeść model 1111



Rysunek 2b. Rękojeść model 1126



#### 2. Wskazania do stosowania

Osierdziowa bioproteza aortalna Edwards model 11000A jest przeznaczona dla pacjentów wymagających wymiany naturalnej lub protetycznej zastawki aortalnej.

#### 3. Przeciwwskazania

Nie stosować bioprotezy, jeżeli chirurg uzna jej użycie za sprzeczne z najlepiej pojętym interesem pacjenta. To chirurg powinien podjąć decyzję dotyczącą zastosowania tej bioprotezy lub zrezygnowania z jej użycia, ponieważ może ocenić różne czynniki ryzyka związane z jej wszczepieniem, w tym również budowę anatomiczna pacienta oraz zmiany patologiczne widoczne podczas operacii.

#### 4. Ostrzeżenia

WYŁĄCZNIE DO JEDNORAZOWEGO UŻYTKU. Opisywane urządzenie jest zaprojektowane i rozprowadzane wyłącznie z zamiarem jednorazowego użytku i takie jest jego przeznaczenie. Niniejszego produktu nie wolno ponownie sterylizować/używać. Nie istnieją żadne dane potwierdzające jałowość, niepirogenność i sprawność produktu po ponownej sterylizacji.

NIE WOL NO ZAMRAŻAĆ BIOPROTEZY ANI PODDAWAĆ DZIAŁANIU SKRAJNIE WYSOKIEJ TEMPERATURY. Narażenie bioprotezy na skrajne temperatury uczyni urządzenie niezdatnym do użycia.

Protezy biologicznej NIE NALEŻY UŻYWAĆ:

- jeśli torebka foliowa, zapieczętowane tace lub pokrywy są otwarte, uszkodzone lub zabrudzone
- · jeśli minął termin ważności lub
- jeśli bioproteza została upuszczona, zniszczona lub postępowano z nią w niewłaściwy sposób. Jeśli podczas wszczepiania bioproteza ulegnie uszkodzeniu, nie należy podejmować próby jej naprawy.

NIE NALEŻY NARAŻAĆ bioprotezy na działanie jakichkolwiek roztworów, środków chemicznych, antybiotyków itp., z wyjątkiem jałowego roztworu soli fizjologicznej. Może nastąpić nienaprawialne uszkodzenie tkanki płatków, które może nie być widoczne godym okiem.

NIE WOL NO CHWYTAĆ tkanki płatków bioprotezy narzędziami ani w żaden sposób uszkadzać bioprotezy. Nawet najmniejsza perforaga ktanki płatków może z czasem ulec powiększeniu, powodując znaczne upośledzenie czynność bioprotezy.

NIE NALEŻY STOSOWAĆ ZBYT DUŻEGO ROZMIARU. Stosowanie zbyt dużego rozmiaru może spowodować uszkodzenie bioprotezy lub miejscowe naprężenia mechaniczne, których efektem może być zranienie serca, zniszczenie tkanki płatków, zniekształcenie stentu i przepływ fali zwrotnej. Podobnie jak w przypadku każdego implantowanego przyrządu medycznego, istnieje rzysko odpowiedzi immunologicznej u pacjenta. Do składników modelu 11000A należy stop metalu, który zawiera kobalt, chrom, nikiel, molibden, mangan, węgiel, beryl oraz żelazo. Należy zachować ostrożność u pacjentów z nadwrażliwościami na te materiały. Urządzenie zostało wytworzone bez lateksu, ale mogło być produkowane w środowisku zawierającym lateks.

#### 5. Zdarzenia niepożądane

#### 5.1 Zaobserwowane zdarzenia niepożądane

Podobnie jak w przypadku wszystkich sztucznych zastawek serca, stosowanie zastawek tkankowych może wiązać się z poważnymi zdarzeniami niepożądanymi, niekiedy prowadzącymi do zgonu. Ponadto po upływie różnych okresów czasu (godzin lub dni) mogą występować zdarzenia niepożądane wynikające z indywidualnej reakcji pacjenta na wszczepione urządzenie lub fizycznych i chemicznych zmian jego komponentów, zwłaszcza pochodzenia biologicznego; mogą one powodować konieczność ponownej operacji i wymiany protezy.

Osierdziowa bioproteza aortalna Edwards model 11000 A jest podobna w konstrukcji do bioprotez osierdziowych Carpentier-Edwards PERIMOUNT Magna Ease model 3300TFX.

Do zdarzeń niepożądanych związanych z zastosowaniem bioprotez osierdziowych Carpentier-Edwards PERIMOUNT według zestawienia na podstawie źródeł literaturowych i doniesień otrzymanych z systemu nadzoru nad produktem, zgodnie z przepisami prawa federalnego USA ustalającymi dobrą praktykę produkcyjna, rozdział 820.198, zalicza się: zweżenie, niedomykalność niewydolnej zastawki, nieszczelność wokół zastawki, zapalenie wsierdzia, hemolize, zaburzenia zakrzepowo-zatorowe, zaburzenia przepływu spowodowane przez zakrzep, skazy krwotoczne zwiazane z leczeniem przeciwzakrzepowym, a także wadliwe funkcjonowanie zastawki wskutek zniekształcenia implantu, złamania prowadnicy drucianej albo zmian fizycznych lub chemicznych komponentów zastawki. Do rodzajów uszkodzenia tkankowego należy zakażenie, zwapnienie, pogrubienie, perforacia, degeneracia, przetarcie szwu, uraz narzedziem oraz odłaczenie płatka od wsporników stentu zastawki. Manifestacją kliniczną tych powikłań mogą być nieprawidłowe szmery serca, duszności, nietolerancia wysiłku, duszność, ortopnoe, niedokrwistość, goraczka, arytmia, krwotok, przejściowe ataki niedokrwienne, udar mózgu, niedowład, niska pojemność minutowa serca, obrzęk płuc, zastoinowa niewydolność serca, niewydolność serca i zawał mięśnia sercowego.

Uwaga: Na podstawie doniesień w piśmiennictwie na temat zastawek tkankowych (poz. 6, 7, 8, 9 i 10) wydaje się występować zwiększony odsetek zwapnienia listków u pacjentów w wieku poniżej 20 lat. Badsania na zwierzętach prowadzone w tym zakresie (poz. 11) wykazują, że wysoki poziom wapnia w krążeniu ustrojowym może prowadzić do wczesnego wapnienia. Ponadto przynajmniej jedno z opublikowanych doniesień opisuje potencjalną zależność pomiędzy codziennym spożywaniem preparatów wapnia i wczesnym wapnieniem płatków zastawek u osób dorosłych (poz. 13). Jeśli jest to możliwe, należy unikać powtarzanych dożylnych wstrzyknięć preparatów zawierających wapń w okresie pooperacyjnym, a dzieci powinny także unikać nadmiernego spożycia mleka oraz nabiału. Brak danych klinicznych wskazujących na zwiększoną odporność osierdziowej bioprotezy aortalnej Edwards model 11000A na zwapnienie w porównaniu do innych dostępnych na rynku bioprotez.

#### 5.2 Możliwe zdarzenia niepożądane

Zdarzenia niepożądane potencjalnie związane z zastosowaniem bioprotez zastawek serca to:

- Dławica piersiowa
- Skazy krwotoczne związane z leczeniem przeciwzakrzepowym (koagulopatia)
- Zaburzenia rytmu serca

- · Zablokowanie ujścia wieńcowego
- Zapalenie wsierdzia
- Niewydolność serca
- Hemoliza
- Niedokrwistość hemolityczna
- Krwotok
- Mieiscowe i/lub uogólnione zakażenie
- Zawał mięśnia sercowego
- Niedopasowanie protezy do pacjenta (PPM)
- · Usidlenie płatka zastawki (wklinowanie)
- Niestrukturalna dysfunkcja protezy
- Wytworzenie łuszczki
- Przeciek okołozastawkowy
- Niedomykalność protezy
- · Strukturalne uszkodzenie protezy
- Zakrzepica protezy
- Udar mózgu
- Zaburzenia zakrzepowo-zatorowe
- Przemijające niedokrwienie mózgu (TIA)

Wymienione powikłania mogą prowadzić do:

- powtórnego zabiegu operacyjnego
- · usunięcia zastawki
- trwałej niepełnosprawności
- zaonu

#### Badania kliniczne

#### Kohorta pacjentów przed zatwierdzeniem produktu

Dostępne dane kliniczne 719 pacjentów wymagających operacji wymiany jednej zastawki aortalnej (aortic valve replacement, AVR) na model bioprotezy osierdziowej 2700 Carpentier-Edwards PERIMOUNT, ze średnim okresem obserwacji wynoszącym 3,9 roku, wskazują na ogólny aktuarialny wskaźnik przeżycia 73,7% ± 2,0% w okresie 6 lat. Dostępne dane kliniczne 70 pacjentów wymagających operacji wymiany dwóch zastawek (double valve replacement, DVR), ze średnim okresem obserwacji wynoszącym 3,7 roku, wskazują na ogólny aktuarialny wskaźnik przeżycia 67,2% ± 6,5% w okresie 6 lat. Te dane dla grupy kontrolnej pacjentów przed zatwierdzeniem produktu zgromadzono w okresie od sierpnia 1981 do stycznia 1989 roku.

W populacji wymagającej pojedynczego zabiegu AVR znajdowało się ogółem 455 mężczyzn (63,3%) i 264 kobiety (36,7%), zaś średni wiek pacjentów podczas wszczepienia (± odchylenie standardowe) wynosił 64 lata (± 12,4) przy zakresie wieku od 18 do 90 lat. Wskazaniami do wymiany zastawki były zwężenie (63,4%), niedomykalność (16,3%), wada mieszana (15,3%) oraz dysfunkcja poprzedniej prostetycznej zastawki aortalnej (5,0%).

W populacji wymagającej zabiegu DVR znajdowało się ogółem 24 mężczyzn (34,3%) i 46 kobiet (65,7%), zaś średni wiek pacjentów podczas wszczepienie dz odchylenie standardowe) wynosił 62,9 lat (± 12,7) przy zakresie wieku od 31 do 94 lat. Wskazaniami do wymiany zastawki były: zwężenie (45,7%),

niedomykalność (25,7%), wada mieszana (21,4%) oraz dysfunkcja poprzedniej protezy zastawki aorty (7,4%).

Metody obserwacji obejmowały wizyty w szpitalu, wizyty w gabinetach oraz kontakt telefoniczny lub listowny z pacjentem, jego rodziną lub miejscowym lekarzem.

Tabela 2 zawiera zestawienie współczynników powikłań operacyjnych i pooperacyjnych dla izolowanych populacji AVR i DVR. Obliczenia wskaźników z okresu operacji oparto na grupie 719 pacjentów przechodzących zabieg AVR i 70 pacjentów w grupie poddanej zabiegowi DVR. Wskaźniki pooperacyjne obliczono na podstawie obserwacji wynoszącej 2767,9 i 255,8 pacjentolat, odpowiednio dla grup poddanych zabiegom AVR i DVR, mającej miejsce > 30 dni po implantacji.

Tabela 3 przedstawia, według rozmiaru zastawki, wyniki echokardiografii w okresie pooperacyjnym dla tej populacji badania.

Zebrano informacje dotyczące przynależności pacjentów poddanych zabiegowi izolowanej AVR do poszczególnych klas czynnościowych NYHA przed i po operacji. Klasy czynnościowej NYHA nie podawano w przypadku 220 pacjentów (171 pacjentów zmarło, a 49 pacjentów nie było dostępnych). Spośród 499 pacjentów, u których podano klasę czynnościową NYHA przed i po operacji (z ostatniej dostępnej wizyty kontrolnej), 10 pacjentów (2,0%) wykazywało pogorszenie, stan 59 pacjentów (11,8%) pozostawał bez zmian, zaś u 430 pacjentów (86,2%) stwierdzono poprawe.

W tabeli 4 przedstawiono dane wynikające z porównania klasy czynnościowej NYHA sprzed operacji i po operacji z ostatniej wizyty kontrolnej.

#### Kohorta pacjentów po zatwierdzeniu produktu

Firma Edwards od listopada 1981 r. kontynuuje badania kontrolne zatwierdzonej kohorty 267 pacjentów, którzy przeszli zabieg wymiany wyłącznie jednej zastawki (AVR) (model 2700) z czterech ośrodków z oryginalnego badania klinicznego nad osierdziową bioprotezą Carpentier-Edwards PERIMOUNT. Ta grupa składa się ze 171 (64%) mężczyzn 196 (36%) kobiet. Średni wiek tych pacjentów w chwili implantacji (± odchylenie standardowe) wynosił 64,9 ± 11,8 roku przy zakresie wieku od 21 do 86 lat. Łączna liczba danych w ilości 2407 pacjentolat była dostępna do analizy (2386 późnych pacjentolat). Średni czas obserwacji kontrolnej wynosił 9,0 ± 5,5 lat, a maksymalnie 20,3 lat. W okresie od 1981 r. do 1994 r. doszło łącznie do 189 zgonów. Czterdzieści osiem (25,3%) z tych 189 zgonów zostało uznane za powiązane z zastawkami. Metody obserwacji wykorzystywane w każdej klinice obejmowały wizyty w szpitalu, wizyty w gabinetach oraz kontakt telefoniczny lub listowny z pacjentem, jego rodziną lub miejsrowym lekarzem.

Tabela 5 podsumowuje współczynniki wolności od powikłań po 20 latach. Stan pacjentów na ostatni okres obserwacji to 189 osób zmarłych (70,8%), 10 osób zyjących (3,8%), 46 osób poddanych zabiegowi usunięcia zastawki (17,2%) i 22 osoby, z którymi utracono kontakt podczas okresu obserwacji (8,2%).

W tei grupie pacientów odnotowano 48 zgonów powiazanych z zastawka: do

1 zgónu powiązanego z zastawką doszło w okresie operacyjnym i wynikał on z krwawienia. Do dwudziestu ośmiu zgonów związanych z zastawką w okresie pooperacyjnym zaliczono 5 spowodowanych zaburzeniami zakrzepowo-zatorowymi, 4 spowodowane zapaleniem wsierdzia/posocznicą, 3 spowodowane strukturalnym uszkodzeniem protezy i 1 spowodowany krwawieniem. Wystąpiło 15 innych zgonów, które rozpatrywano jako związane zastawką ze względu na brak danych lub w związku z tym, że zgon został zaklasyfikowany jako powiązany z zastawką przez badacza. Wolność aktuarialna od zgonu powiązanego z zastawką wynosiła 67,9 ± 6,6% po 20 latach. Dziewiętnaście dodatkowych zgonów były spowodowanych nieznanymi przyczynami lub nagłą śmiercią i mogło mieć związek z zastawką. Te zgony zaklasyfikowano w sposób zachowawczy jako powiązane z zastawką; odpowiednio, wynikająca aktuarialna wolność od zgonu powiązanego z zastawką wnosiła 55,4 ± 6,4% po 20 latach.

Wykazano także poprawę klasy czynnościowej NYHA w okresie pooperacyjnym. Zgodnie z ostatnimi wynikami obserwacji 108 pacjentów (44,8%) znajdowało sie w I klasie czynnościowej NYHA.

Niniejsze dane zostały skompilowane na podstawie wieloośrodkowego badania klinicznego prowadzonego przez firmę Edwards Lifesciences. W celu uzyskania dodatkowych informacji na temat tego badania należy skontaktować się z Edwards Lifesciences LLC, Heart Valve Therapy Marketing Department, One Edwards Wav. Irvine. CA 92614-5686.

#### Badanie potwierdzające

W okresie od sierpnia 2003 r. do stycznia 2004 r. 60 pacjentom z pięciu ośrodków (dwóch europejskich i trzech kanadyjskich), wymagającym wymiany zastawki aortalnej (AVR) wszczepiono bioprotezę aortalną Carpentier-Edwards PERIMOUNT Magna, model 3000. Wkrótce potem wprowadzono do protokołu klinicznego poprawki pozwalające na implantację bioprotezy aortalnej Carpentier-Edwards PERIMOUNT Magna, model 3000TFX, oraz dodanie trzech ośrodków amerykańskich. Następnie, w okresie od grudnia 2004 r. do grudnia 2006 r., 193 dodatkowym pacjentom wszczepiono model 3000TFX. Model 3000TFX różni się od modelu 3000 tym, że model 3000TFX jest poddawany procesowi ThermaFix.

W grupie modelu 3000TFX znajdowało się łącznie 116 mężczyzn (60,1%) i 77 kobiet (39,9%) o średniej wieku w momencie wszczepienia rzędu 72,0 (± 8,59 SD) lat i zakresie wieku od 26 do 89 lat. Głównym wskazaniem do wymiany zastawki było zwężenie (78,2%), a w dalszej kolejności wada mieszana (14.5%) oraz niedomykalność (7.3%).

W połączonej grupie modeli 3000 i 3000TFX znajdowało się łącznie 150 mężczyzn (59,3%) i 103 kobiety (40,7%) o średniej wieku w momencie wszczepienia rzędu 72,2 (± 8,31 SD) lata i zakresie wieku od 26 do 89 lat. Ponownie głównym wskazaniem do wymiany zastawki było zwężenie (77,5%), wada mieszana (15,4%) o raz niedomykalność (7,1%).

Stan pacjentów oceniano przedoperacyjnie, śródoperacyjnie, przy wypisywaniu ze szpitala, po 3 do 6 miesiącach, po 1 roku i następnie corocznie. Skumulowana obserwacja dla modelu 3000TFX wynosiła 167 pacjentolat, ze średnim okresem obserwacji wynoszącym 0,9 roku (SD = 0,42, zakres = 0,0 do 2,1 roku); a skumulowana obserwacja dla obu modeli 3000 i 3000TFX łącznie wynosiła 232 pacjentolat ze średnim okresem obserwacji wynoszącym 0,9 roku (SD = 0,42, zakres = 0,0 do 2,1 roku).

Tabela 6 podsumowuje wczesne (≤ 30 dni) oraz późne pooperacyjne (> 30 dni) współczynniki zdarzeń niepożądanych związanych z zastawką dla, odpowiednio, grup modelu 3000TFX i połączonych modeli 3000/3000TFX.

Ta bela 7 ilustruje, według modelu zastawki, zmienne hemodynamiczne odnotowywane w elektrokardiogramach po jednym roku, wykonywanych na pacjentach w badaniach modelu 3000TFX. i połaczonych modeli 3000/3000TFX.

Tabela 8 prezentuję zmianę w klasie czynnościowej NYHA od oceny dokonywanej w momencie wyjściowym do wizyty po 1 roku. Należy zwrócić uwagę na fakt, że w przypadku modelu 3000TFX odnotowano poprawę klasy czynnościowej na poziomie 56,5% dla wizyty po 1 roku. Dla modelu grupy łączonej 3000/3000TFX odnotowano 60,9% poprawę klasy czynnościowej dla wizyty po 1 roku.

Kilka opublikowanych badań klinicznych demonstruje długoterminową trwałość osierdziowych bioprotez aortalnych Carpentier-Edwards PERIMOUNT, na podstawie których konstruowano osierdziowe bioprotezy aortalne Carpentier-Edwards PERIMOUNT Magna oraz Magna Ease (poz. 14, 15, 16 & 17). Ponadto opublikowane dane pokazują, że bioproteza aortalna PERIMOUNT Magna wykazuje wyjątkowe parametry hemodynamiczne, z bardzo niskim ryzykiem niedopasowania pacjenta i protezy (poz. 18, 19, 20, 21, 22 & 23).

#### 7. Indywidualizacja leczenia

We wszystkich przypadkach bez przeciwwskazań pacjenci z wszczepionymi bioprotezami zastawek serca powinni otrzymywać leczenie przeciwzakrzepowe podczas wstępnych etapów po implantacji indywidualnie, według zaleceń lekarza. Długoterminowe leczenie przeciwzakrzepowe i/lub przeciwpłytkowe należy rozważyć u pacjentów z czynnikami ryzyka zaburzeń zakrzepowo-zatorowych.

Ostateczną decyzję w sprawie opieki nad konkretnym pacjentem powinien podjąć personel medyczny oraz pacjent, w świetle wszystkich okoliczności dotyczących tego pacjenta (poz. 12). Bioproteza jest zalecana do AVR u pacjentów w każdym wieku, który nie będą przyjmować warfaryny lub mają poważne przeciwwskazania medyczne do leczenia warfaryną. Preferencje pacjenta to racjonalne kryterium przy wyborze operacji wymianz zastawki aortalnej oraz wyborze protezy aortalnej. Mechaniczna bioproteza jest rosządnym wyborem do AVR u pacjentów poniżej 65 roku życia, którzy nie mają przeciwskazania do leczenia przeciwzakrzepowego. Bioproteza jest rosządnym wyborem do AVR u pacjentów poniżej 65 roku życia, którzy wybrali wymianę zastawki ze względów związanych ze stylem życia po szczegółowych omówieniach ryzyka leczenia przeciwzakrzepowego względem prawdopodobieństwa konieczności przeprowadzenia kolejnego zabiegu AVR (poz. 12).

#### 7.1 Szczególne grupy pacjentów

Nie potwierdzono bezpieczeństwa ani skuteczności stosowania modelu bioprotez 11000A w następujących szczególnych populacjach, ponieważ nie przebadano ich w takich grupach:

- · kobiety ciężarne;
- matki karmiące;
- pacjenci z nieprawidłowym metabolizmem wapnia (np. z przewlekłą niewydolnością nerek lub nadczynnością przytarczyc);
- pacjenci ze schorzeniami zwyrodnieniowymi aorty powodującymi powstawanie tętniaków (np. martwica torbielowata błony środkowej, zespół Marfana):
- · dzieci, młodzież lub młode osoby dorosłe.

Przestroga: Na podstawie doniesień w piśmiennictwie na temat zastawek tkankowych (poz. 6, 7, 8, 9 i 10) wydaje się występować zwiększony odsetek zwapnienia listków u pacjentów w wieku poniżej 20 lat. W miarę możliwości należy unikać podawania w okresie pooperacyjnym wielokrotnych wstrzyknięć dożylnych zawierających wapń oraz unikać spożywania przez dzieci nadmiernych ilości mleka lub nabiału. Wyniki badań prowadzonych na zwierzętach (poz. 11) wskazują, że wysoki poziom wapnia w organizmie może prowadzić do wczesnego powstawania zwapnień.

# 8. Informacja dla pacjenta

Po operacji zaleca się uważną i stałą obserwację lekarską (przynajmniej jedna wizyta rocznie), aby umożliwić rozpoznanie i właściwe leczenie powikłań związanych z bioprotezą, szczególnie wynikających z uszkodzenia materiału. Pacjentom z bioprotezą, którzy są w grupie podwyższonego ryzyka bakteriemii (np. poddawanym zabiegom stomatologicznym), warto doradzić profilaktyczną terapię antybiotykową. Pacjentom należy doradzać, aby zawsze nosili przy sobie Kartę danych wszczepu oraz informowali pracowników slużby zdrowia o posiadanym implancie przy zasięganiu porady lekarskiej.

#### 9. Sposób dostarczania

#### 9.1 Opakowanie

Osierdziowa bioproteza aortalna Edwards model 11000A jest dostarczana w postaci jałowej i niepirogennej w opakowaniu tacowym z podwójną ochroną. Opakowanie tacowe z podwójną ochroną mieści się w torebce foliowej, która znaidule się w kartonie.

Każda bioproteza umieszczona jest w kartonie ze wskaźnikiem temperatury widocznym przez okienko na panelu bocznym. Wskaźnik temperatury przeznaczony jest do identyfikacji produktów narażonych na przejściowe skrajne warunki temperaturowe. W chwili otrzymania bioprotezy należy niezwłocznie sprawdzić wskaźnik i zapoznać się z etykietą kartonu, aby potwierdzić stan "Do wykorzystania". Jeśli stan "Do wykorzystania" nie jest oczywisty, nie należy używać bioprotezy i skontaktować się z lokalnym dostawcą lub przedstawicielem firmy Edwards Lifesciences v celu dokonania ustaleń dotyczacych potwierdzenia zwrotu i wymiany.

Ostrzeżenie: Dokładnie sprawdzić bioprotezę przed implantacją pod kątem dowodów ekspozycji na skrajne temperatury lub innych uszkodzeń.

#### 9.2 Przechowywanie

Osierdziową bioprotezę aortalną Edwards model 11000A należy przechowywać w temperaturze 10°C do 25°C (50-77°F), w torebce foliowej i na półce kartonowej.

#### 10. Wskazówki dotyczace użycia

#### 10.1 Szkolenia lekarzy

Techniki implantacji niniejszej bioprotezy są podobne do stosowanych podczas wszczepiania ponad pierścieniem jakichkolwiek stentowych protez biologicznych zastawki aorty. Przeszkolenie lekarzy nie jest konieczne do wykonywania implantacji osierdziowej bioprotezy aortalnej Edwards model 11000A.

#### 10.2 Kalibrowanie

Sprawdzić, czy akcesoria zostały wyjałowione zgodnie z zalecanymi instrukcjami dostarczonymi z akcesoriami wielorazowymi.

#### Kalibrowanie w implantacji nadpierścieniowej

W celu przeprowadzenia implantacji nadpierścieniowej pierścień do wszywania bioprotezy należy umieścić nad pierścieniem włóknistym, maksymalnie powiększając w ten sposób otwór zastawki. Podczas dobierania rozmiaru do implantacji nadpierścieniowej kalibrator powinien być ułożony równolegle do płaszczyzny pierścienia; należy zastosować następującą technikę kalibracji:

| Krok | Postępowanie |
|---|---|
| 1 | Używając kalibratora model 1133, wybrać cylindryczne<br>zakończenie kalibratora o największej średnicy, które można<br>bez trudu dopasować do pierścienia włóknistego pacjenta. |
| | HVT21 |

#### Krok Postępowanie

2

Po zweryfikowaniu odpowiedniego zakończenia cylindrycznego należy użyć zakończenia replikującego w tym samym rozmiarze, aby sprawdzić, czy pierścień do wszywania będzie dobrze dopasowany do górnej części pierścienia włóknistego. Należy zwrócić szczególną uwagę na to, czy ujścia naczyń wieńcowych nie są zablokowane i czy wsporniki stentu zakończenia replikującego nie kolidują ze ścianą aorty przy połączeniu opuszkowo-komorowym. Jeśli dopasowanie zakończenia replikującego jest satysfakcjonujące, do implantacji należy wybrać ten rozmiar bioprotezy.

HVT37



#### 10.3 Instrukcje dotyczące manipulacji i przygotowania

Doctonowania

Vuole

Zaleca się przeprowadzenie szkolenia w miejscu pracy przed rozpoczęciem manipulowania i przygotowania osierdziowej bioprotezy aortalnej Edwards, model 11000A.

| Postępowanie |
|---|
| Przestroga: Nie otwierać opakowania osierdziowej<br>bioprotezy aortalnej Edwards, model 11000A przed<br>upewnieniem się, że dojdzie do implantacji. |
| Ostrzeżenie: Nie otwierać torebki foliowej w polu<br>jałowym. Torebka foliowa stanowi jedynie osłonę<br>zabezpieczającą. Jedynie najbardziej wewnętrzne<br>opakowanie tacowe można wprowadzać do pola<br>jałowego. |
| Po wyborze odpowiedniego rozmiaru bioprotezy należy, poza<br>polem jałowym, wyjąć z kartonu torebkę foliową. Przed<br>otwarciem należy sprawdzić, czy opakowanie nie jest<br>uszkodzone i czy nie brakuje pieczęci lub czy nie są one<br>uszkodzone. |
| Należy przytrzymać podstawę tacy zewnętrznej w pobliżu pola<br>jałowego i oderwać pokrywę tacy zewnętrznej. |

| Krok | Postępowanie |
|---|---|
| 3 | Taca wewnętrzna i jej zawartość są jałowe. Należy przełożyć tacę wewnętrzną do pola jałowego. Przy postępowaniu z wewnętrzną tacą należy stosować jałowe techniki chirurgiczne w celu uniknięcia skażenia. HVT26 |
| 4 | Przestroga: Nie otwierać wewnętrznego opakowania<br>przed upewnieniem się, że dojdzie do implantacji, i zanim<br>chirurg nie przygotuje się do umieszczenia zastawki. |
| | Przestroga: Bioproteza nie jest przymocowana do tacy<br>wewnętrznej. Należy ostrożnie odrywać pokrywę i<br>otwierać plastikowy języczek. |
| | Przed otwarciem należy sprawdzić, czy taca i pokrywa nie są<br>uszkodzone i czy nie brakuje pieczęci lub czy nie są one<br>uszkodzone. Należy przytrzymać podstawę tacy wewnętrznej w<br>pobliżu pola sterylnego i oderwać pokrywę tacy wewnętrznej. |
| 5 | W celu uzyskania dostępu do bioprotezy należy pociągnąć w<br>górę plastikowy języczek ze strzałką. |
| | HVT28<br>Pociągnąć za języczek ze strzałką |
| | HVT29 |



| Krok | Postępowanie |
|---|---|
| 7 | Po przymocowaniu rękojeści należy usunąć bioprotezę i zaczep z tacy wewnętrznej. HVT32 |
| 8 | W celu usunięcia zaczepu z bioprotezy należy chwycić zaczep i odciągnąć go od zespołu rękojeść/uchwyt. MYT33 |
| | HVT34 |

| 9 | Do każdego pierścienia do wszywania protezy biologicznej dołączona jest etykieta z numerem seryjnym. Należy sprawdzić, czy numer seryjny jest zgodny z numerem na opakowaniu bioprotezy i kartą danych implantacji bioprotezy. Etykiety nie należy odrywać od bioprotezy przed upewnieniem się, że dojdzie do wszczepienia. |
|---|---|
| | Przestroga: W przypadku zauważenia jakiejkolwiek<br>różnicy w numerze seryjnym należy zwrócić nieużywaną<br>bioprotezę. |
| | Przestroga: Należy zwrócić szczególną uwagę na to, aby<br>podczas usuwania etykiety z numerem seryjnym uniknąć<br>nacięcia lub rozerwania tkaniny pierścienia do<br>wszywania. |
| | Przestroga: By uniknąć uszkodzenia tkaniny pierścienia<br>do wszywania, nie należy przeciągać supła szwu z etykietą<br>z numerem seryjnym przez pierścień do wszywania. |
| 10 | Osierdziowa bioproteza aortalna Edwards model 11000A NIE<br>WYMAGA PŁUKANIA przed implantacją. |
| | Przestroga: Jeśli bioproteza zostanie wypłukana przed<br>implantacją, należy ją utrzymywać w stanie<br>nawodnienia jałowym roztworem soli fizjologicznej po<br>obu stronach tkanki płatka przez pozostały czas trwania<br>zabiegu chirurgicznego. Zaleca się przepłukiwanie co<br>1 lub 2 minuty. |
| | Przestroga: Należy unikać kontaktu tkanki płatka z<br>ręcznikami, płótnem i innymi źródłami materii pylastej,<br>która może zostać przeniesiona na tkankę płatka. |

## 10.4 Implantacja urządzenia

Krok

Postępowanie

Osierdziowa bioproteza aortalna Edwards model 11000A jest przeznaczona do implantacji nadpierścieniowej.

| ширансасун | raupiers demowej. |
|---|---|
| Krok | Postępowanie |
| 1 | Chirurg powinien znać zalecenia dotyczące doboru rozmiarów oraz umiejscowienia protezy ponad pierścieniem (Patrz 10.2 Kalibrowanie). |
| | Ze względu na złożoność i rodzaje operacji wymiany zastawki<br>serca, wybór techniki chirurgicznej, odpowiednio zmodyfikowan<br>zgodnie z wcześniej opisanymi <b>Ostrzeżeniami</b> , zależy od decyz<br>chirurga. Zasadniczo należy wykonać następujące kroki: |
| | Chirurgicznie usunąć zmienione chorobowo lub uszkodzone<br>płatki zastawki i wszystkie związane z nią struktury<br>konieczne do usunięcia. |
| | <ol> <li>Chirurgicznie usunąć wapń z pierścienia w celu zapewnienia<br/>odpowiedniego umieszczenia pierścienia do wszywania<br/>bioprotezy i niedopuszczenia do uszkodzenia delikatnej<br/>tkanki platka.</li> </ol> |
| | <ol> <li>Należy zmierzyć pierścień włóknisty, używając kalibratorów<br/>aortalnych Carpentier-Edwards model 1133 (Rysunki 1a-1c).</li> </ol> |

#### Krok Postepowanie

Przestroga: Podczas doboru wymiarów bioprotezy dla danego pacjenta należy wziąć pod uwagę jego wymiary anatomiczne, wiek i kondycję fizyczną, aby zmniejszyć do minimum możliwość uzyskania suboptymalnego wyniku hemodynamicznego. Jednak ostatecznego doboru bioprotezy w poszczególnych przypadkach powinien dokonać lekarz po starannym rozważeniu wszystkich zagrożeń i korzyści dla określonego pacjenta.

Przestroga: Nie należy stosować kalibratorów protez innych producentów lub kalibratorów przeznaczonych do innych bioprotez Edwards Lifesciences w celu określenia rozmiaru osierdziowej bioprotezy aortalnej Edwards model 11000A.

Przestroga: Sprawdzić kalibratory pod kątem zużycia, takiego jak stępienie, popękanie lub spękanie włoskowate. Wymienić kalibrator, jeśli widoczne są oznaki zniszczenia.

Ostrzeżenie: Fragmenty rękojeści i kalibratorów nie są radiologicznie nieprzezroczyste i nie można ich lokalizowaćza pomocą zewnętrznego urządzenia obrazującego.

Należy zastosować technikę szycia pozwalająca na nadpierścieniowe umieszczenie bioprotezy, taką jak przerywany poziomy ścieg materacowy. Podczas zakładania szwów przez pierścień do przyszywania osierdziowej bioprotezy aortalnej Edwards model 11000A zaleca się, by szwy przechodziły przez pierścień do przyszywania jak najbliżej ramy bioprotezy.

> Kiedy szwy zostaną założone, należy je przyciąć blisko węzłów, by zapobiec kontaktowi końcówek szwu z tkanką płatka bioprotezy.

> > HVT35



#### Krok Postępowanie

3 Uchwyt z dołączoną do niego rękojeścią zostają usunięte jako całość po zakończeniu procedury zakładania szwów.

 Za pomocą skalpela należy obciąć każdy z trzech wyeksponowanych szwów znajdujących się na górze uchwytu.

HVI:



Przestroga: Należy uniknąć przedęcia lub uszkodzenia stentu lub delikatnej tkanki płatków podczas przecinania szwów.

- Po odcięciu wszystkich trzech szwów przy uchwycie należy usunąć z bioprotezy zespół rękojeść/uchwyt, w całości, wraz ze szwami przy uchwycie.
- Należy wyjąć rękojeść z uchwytu i wyrzucić uchwyt.

#### 10.5 Czyszczenie i sterylizacja

Akcesoria do osierdziowej bioprotezy aortalnej Edwards, model 11000A są pakowane oddzielnie. Rękojeść model 1126 dostarczana jest jalowa i przeznaczona wyłącznie do jednorazowego użytku. Rękojeść model 1111 oraz kalibratory model 1133 dostarczane są jako niejałowe i muszą być wysterylizowane przed użyciem. Należy wyczyścić i ponownie wysterylizować rękojeści, kalibratory, podstawę i pokrywę tacy przed każdym użyciem. Instrukcje dotyczące mycia i wyjaławiania zawiera instrukcja stosowania dostarczana z akcesoriami wielorazowymi.

#### 10.6 Zwrot bioprotez

Firma Edwards Lifesciences jest zainteresowania otrzymaniem odzyskanych klinicznych egzemplarzy osierdziowej bioprotezy aortalnej model 11000A do analizy. W celu zwrotu odzyskanych bioprotez należy skontaktować się z lokalnym przedstawicielem firmy.

- Nieotwarte opakowanie z nienaruszoną barierą jałową: Jeśli torebka foliowa ani tace nie zostały otwarte, bioprotezę należy zwrócić w oryginalnym opakowaniu.
- Otwarte opakowanie, lecz bioproteza nie została wszczepiona: Jeśli taca została otwarta, bioproteza nie jest już jałowa. Jeśli bioproteza nie zostanie wszczepiona, należy ją umieścić w odpowiednim utrwalaczu histologicznym takim jak 10% formalina lub 2% aldehyd glutarowy i zwrócić do firmy. W takich okolicznościach schłodzenie nie jest konieczne.
- Eksplantowana bioproteza: Eksplantowane bioprotezy należy umieścić w odpowiednim utrwalaczu histologicznym, takim jak 10% formalina lub 2% glutaraldehyd, i zwrócić do firmy. W takich okolicznościach schłodzenie nie jest konieczne.

## Zasady bezpieczeństwa w środowisku rezonansu magnetycznego (MR)



#### Warunki w badaniu MR

Badania pozakliniczne wykazały, że osierdziowa bioproteza aortalna Edwards model 11000A może być warunkowo stosowana w środowisku MR. Badanie pacjenta bezpośrednio po wszczepieniu zastawki model 11000A można wykonać bezpiecznie po umieszczeniu tego implantu w następujących warunkach:

- Statyczne pole magnetyczne o indukcji równej 1,5 tesli (T) lub 3 tesli.
- Maksymalny gradient przestrzenny pola magnetycznego 2670 gausów/cm.
- Maksymalny średni specyficzny współczynnik wchłaniania zgłoszony dla systemu rezonansu magnetycznego dla całego ciała (SAR) na poziomie 2,0 W/kg w normalnym trybie działania przez 15 minut skanowania jednej sekwencji.

W badaniach pozaklinicznych, osierdziowa bioproteza aortalna Edwards, model 11000A, dawała szacowany maksymalny wzrost temperatury in vivo mniejszy niż lub równy 1,8°C dla maksymalnego zgłoszonego systemu rezonansu magnetycznego, średni specyficzny współczynnik wchłaniania dla całego ciała (SAR) na poziomie 2,0 W/kg, przez 15 minut skanowania MR w systemie rezonansu magnetycznego cewki RF GE Signa 64 MHz (1,5 T) oraz GE Signa HDx (3 T) z wersją oprogramowania 15 UX/MR Software wersją 15.0.M4.0910.a.

Artefakty obrazu mierzono pozaklinicznie w systemie rezonansu magnetycznego 6E Signa 3T HDx MR według ASTM F2119-07, stosując określone dla tego systemu sekwencje echa spinowego i gradientu. Obrazy echa spinowego wykazywały jasne i ciemne artefakty, które rozciągały się tak daleko, jak 40 mm od implantu, oraz częściowo lub całkowicie przesłaniały światło. Obrazy gradientu echa wykazywały nieprzezorczyste ciemne lub jasne i ciemne artefakty o trójkątnym kształcie, które rozciągały się tak daleko, jak 40 mm od implantu i całkowicie przesłaniały światło. Możliwa jest redukcja ilości artefaktów przy użyciu sekwencji przeznaczonych do redukcji artefaktów metalu.

#### 12. Informacje dla pacjentów

#### 12.1 Karta identyfikacyjna badania

Karta identyfikacyjna badania jest przekazywana każdemu pacjentowi ze wszczepioną osierdziową protezą aortalną Edwards model 11000A.

#### 12.2 Materialy informacyine dla pacienta

Materiały informacyjne dla pacjenta można uzyskać w firmie Edwards lub u przedstawiciela klinicznego firmy Edwards.

#### 13. Piśmiennictwo

- Carpentier, A., et al. Biological Factors Affecting Long Term Results of Valvular Heterografts. J Thorac Cardiovasc Surg 1969, 58:467-483.
- Carpentier, A., et al. Six Year Follow-up of Glutaraldehyde Preserved Heterografts. J Thorac Cardiovasc Sura 1974, 68:771-782.
- Reis, Robert L., et al. The Flexible Stent. A New Concept in the Fabrication of Tissue Heart Valve Prostheses. J Thorac Cardiovasc Surg 1971, 62(5):683-689 and 693-695.
- Barratt-Boyes, B.G. and A.H.G. Roche. A Review of Aortic Valve Homografts Over a Six and One-half Year Period. Ann Surg 1969, 170:483-492.
- Brewer, R.J., et al. The Dynamic Aortic Root. Its Role in Aortic Valve Function. J Thorac Cardiovasc Surg 1976, 72:413-417.

- Jamieson, W.R.E., et al. Carpentier-Edwards Standard Porcine Bioprosthesis: Primary Tissue Failure (Structural Valve Deterioration) by Age Groups. Ann Thorac Surg 1988, 46:155-162.
- Odell, J.A. Calcification of Porcine Bioprostheses in Children. In Cohn, L. and V. Gallucci (eds): Cardiac Bioprostheses. Yorke Medical Books. New York, 1982, pp 231-237.
- Reul, G.J., et al. Valve Failure with the lonescu-Shiley Bovine Pericardial Bioprosthesis: Analysis of 2680 Patients. J Vasc Surq 1985, 2(1):192-204.
- Sanders, S.P., et al. Use of Hancock Porcine Xenografts in Children and Adolescents. Am J Cardiol 1980. 46(3):429-438.
- Silver, M.M., et al. Calcification in Porcine Xenograft Valves in Children. Am J Cardiol 1980, 45:685-689.
- Carpentier, A., et al. Continuing Improvements in Valvular Bioprostheses. *J Thorac Cardiovasc Surg* 1982, 83(1):27-42.
- Bonow R.O., et al. ACC/AHA Guidelines for the Management of Patients with Valvular Heart Disease: A Report of the American College of Cardiology/ American Heart Association Task Force on Practice Guidelines (Committee on Management of Patients With Valvular Heart Disease). J Am Coll Cardiol 2006. 48:e1-148.
- Moront, M.G. and N.M. Katz. Early Degeneration of a Porcine Aortic Valve Bioprosthesis in the Mitral Valve Position in an Elderly Woman and its Association with Long-Term Calcium Carbonate Therapy. Am J Cardiol 1987, 59:1006-1007.
- Aupart, M.R., et al. Perimount Pericardial Bioprosthesis for Aortic Calcified Stenosis: 18-Year Experience with 1,133 Patients. J Heart Valve Dis 2006, 15:768-776.
- Dellgren, G., et al. Late Hemodynamic and Clinical Outcomes of Aortic Valve Replacement with the Carpentier-Edwards Perimount Pericardial Bioprosthesis. J Thorac Cardiovasc Surg 2002, 124:146-154.
- Frater, R.W.M., et al. Long-Term Durability and Patient Functional Status of the Carpentier-Edwards Perimount Pericardial Bioprosthesis in the Aortic Position. J Heart Valve Dis 1998, 7:48-53.
- Jamieson, W.R.E., et al. 15-Year Comparison of Supra-Annular Porcine and PERIMOUNT Aortic Bioprostheses. Asian Cardiovasc Thorac Ann 2006, 14:200-205.
- Borger, M.A., et al. Carpentier-Edwards Perimount Magna Valve Versus Medtronic Hancock II: A Matched Hemodynamic Comparison. Ann Thorac Surg 2007; 83:2054-2058.
- Botzenhardt, F., et al. Hemodynamic Comparison of Bioprostheses for Complete Supra-Annular Position in Patients With Small Aortic Annulus. J Am Coll Cardiol 2005, 45:2054-2060.
- Botzenhardt, F., et al. Hemodynamic Performance and Incidence of Patient-Prosthesis Mismatch of the Complete Supraanular Perimount Magna Bioprosthesis in the Aortic Position. Thorac Cardiov Surg 2005, 53:226-230.
- Dalmau, M.J., et al. The Carpentier-Edwards Perimount Magna Aortic Xenograft: A New Design with an Improved Hemodynamic Performance. Interact Cardiovasc Thorac Surg 2006, 5:263-267.
- Totaro, P., et al. Carpentier-Edwards PERIMOUNT Magna Bioprosthesis: A Stented Valve with Stentless Performance? JThorac Cardiovasc Surg 2005, 130:1668-1674.

 Wagner, I.M., et al. Influence of Completely Supra-annular Placement of Bioprostheses on Exercise Hemodynamics in Patients With a Small Aortic Annulus. J Thorac Cardiovascular Surg 2007; 133:1234-1241.

Niniejszy produkt jest wytwarzany i sprzedawany zgodnie z co najmniej jednym spośród następujących patentów amerykańskich: patenty amerykańskie nr: 5,928,281; 5,931,969; 5,961,549; 6,102,944; 6,245,105; 6,413,275; 6,561,970; 6,585,766; 6,837,902; 6,945,997; 7,214,344; 7,972,376; 8,007,992; 8,357,387; 8,366,769; 8,632,608; IRE 40570; oraz odpowiadające patenty zagraniczne. Ponadto trwa uzyskiwanie innych patentów.

Należy zapoznać się z objaśnieniami symboli, umieszczonymi na końcu niniejszego dokumentu.

Tabela 2. Zestawienie współczynników powikłań, model 2700

| | 0 | irupa po izolowa | nej AVR | Populacja DVR | | |
|---|---|---|---|---|---|---|
| Powikłanie | pooperacyjny<br>% pacjentów | Okres<br>pooperacyjny<br>% na<br>pacjentorok | % wolności<br>od zdarzeń po<br>sześciu latach<br>(błąd standardowy) | pooperacyjny<br>% pacjentów | Okres<br>pooperacyjny<br>% na<br>pacjentorok | % wolności<br>od zdarzeń po<br>sześciu latach<br>(błąd standardowy) |
| Zgon | 4,7 | 4,6 | 73,5 (2,0) | 12,9 | 4,2 | 67,2 (6,5) |
| Eksplantacja | 0 | 0,3 | 98,5 (1,0) | 0 | 0,8 | N/D * |
| Powtórny zabieg operacyjny<br>związany z zastawką | 0,7 | 0,1 | 99,8 (0,4) | 0 | 0 | N/D* |
| Wszystkie przypadki<br>powtórnej operacji | 22,4 | 1,8 | 75,4 (1,8) | 34,3 | 2,3 | N/D* |
| Zaburzenia zakrzepowo-zatorowe<br>związane z zastawką | 3,1 | 1,5 | 91,4 (1,1) | 1,4 | 5,1 | N/D* |
| Wszystkie zdarzenia<br>zakrzepowo-zatorowe | 5,0 | 2,4 | 84,9 (1,6) | 5,7 | 6,6 | N/D* |
| Zapalenie wsierdzia | 0,6 | 0,8 | 95,8 (0,9) | 1,4 | 1,5 | N/D * |
| Dysfunkcja zastawki | 0,1 | 0,7 | 96,0 (1,1) | 0 | 0,4 | N/D * |
| Przeciek okołoza-stawkowy | 0,1 | 0,3 | 98,8 (0,5) | 0 | 1,2 | N/D * |
| Powikłania krwotoczne leczenia | 1,4 | 0,4 | 96,4 (1,1) | 4,3 | 2,3 | N/D * |
| Hemoliza | 0 | 0,2 | 99,1 (0,4) | 0 | 0,4 | N/D * |
| Zakrzepica zastawki | 0 | 0 | 100,0 (0) | 0 | 0,4 | N/D * |

| | Rozmiar zastawki | | | | | | |
|---|---|---|---|---|---|---|---|
| | 19 mm | 21 mm | 23 mm | 25 mm | 27 mm | 29 mm | Całkowita |
| Ogółem N | 12 | 22 | 15 | 8 | 3 | 3 | 63 |
| Śr. liczba miesięcy po operacji | $28,6 \pm 7,2$ | $34,9 \pm 8,6$ | $36,9 \pm 9,2$ | $39,9 \pm 7,6$ | $31,4 \pm 15,9$ | $15,3 \pm 12,2$ | $34,6 \pm 9,2$ |
| Prędkość przepływu (m/sek.) | ) | | | | | | |
| $srednia \pm S.D.$ | $2,80 \pm 0,49$ | $2,56 \pm 0,46$ | $2,36 \pm 0,42$ | $2,15 \pm 0,56$ | $2,09 \pm 0,27$ | $2,08 \pm 0,1$ | $2,46 \pm 0,50$ |
| n = | 12 | 21 | 15 | 7 | 3 | 3 | 61 |
| zakres | 1,90 - 3,60 | 1,90 - 3,90 | 1,39 - 2,86 | 1,00 - 2,60 | 1,90 - 2,40 | 2,05 - 2,10 | 1,00 - 3,90 |
| Chwilowa wartość szczytowa<br>gradientu (mmHg) | 1 | | | | | | |
| $srednia \pm S.D.$ | $32,22 \pm 11,08$ | $27,04 \pm 10,49$ | $23,00 \pm 7,30$ | $19,50 \pm 8,16$ | $17,60 \pm 4,70$ | $14,4 \pm 0,58$ | $25,67 \pm 10,14$ |
| n = | 12 | 21 | 15 | 7 | 3 | 3 | 61 |
| zakres | 14,40 - 51,80 | 14,40 - 60,80 | 7,70 - 32,70 | 4,00 - 27,00 | 14,40 - 23,00 | 13,95 - 15,06 | 4,00 - 60,80 |

Tabela 4. Wyniki skuteczności, klasa czynnościowa NYHA, model 2700

| Okres przedoperacyjny Klasa<br>czynnościowa NYHA | Okres pooperacyjny<br>Klasa czynnościowa NYHA | | | | | |
|---|---|---|---|---|---|---|
| | ı | II | III | IV | Zgon | Brak dostępnych<br>danych |
| ı | 18 | 19 | | | 9 | |
| II | 140 | 37 | | | 35 | 15 |
| III | 181 | 48 | 4 | 1 | 72 | 24 |
| IV | 43 | 16 | 2 | | 53 | 2 |
| Niedostępne | 5 | 1 | | | 2 | 2 |

Tabela 5. Współczynniki wolności od powikłań po 20 latach (n = 267), model 2700

| Wolność od powikłań po 20 latach | Faktyczna | Aktuarialna | Liniowa (%/pacjentorok |
|---|---|---|---|
| Zgony związane z zastawką | 85,8 ± 2,5% | 67,9 ± 6,6% | 1,2 |
| Zaburzenia zakrzepowo-zatorowe/zakrzepica | $82,4 \pm 2,6\%$ | $68,2 \pm 6,8\%$ | 1,7 |
| Krwawienie | $94,0 \pm 1,5\%$ | $91,7 \pm 2,2\%$ | 0,4 |
| Zapalenie wsierdzia/posocznica | 91,7 ± 1,7% | $89,3 \pm 2,4\%$ | 0,8 |
| Eksplantacja spowodowana SVD | | | |
| ≥ 60 | $92,6 \pm 2,0\%$ | $77,1 \pm 7,2\%$ | b/z* |
| ≥ 65 | $96,3 \pm 1,6\%$ | $81,5 \pm 9,6\%$ | |
| > 70 | $96.0 \pm 2.3\%$ | $69,9 \pm 20,5\%$ | |

<sup>\*</sup> Bez znaczenia. SVD nie występuje jako stała funkcja ryzyka; w rezultacie liniowe współczynniki nie są istotne.

Tabela 6. Podsumowanie zdarzeń niepożądanych związanych z zastawką, modele 3000 oraz 3000TFX

| | ≤ 30 dni <sub>l</sub> | po operacji | > 30 dni p | oo operacji |
|---|---|---|---|---|
| Zdarzenia niepożądane | 3000TFX<br>(N = 193)<br>liczba zdarzeń<br>(% pacjentów) | 3000/3000TFX<br>(N = 253)<br>liczba zdarzeń<br>(% pacjentów) | 3000TFX<br>(N = 193)<br>liczba zdarzeń<br>(% pacjentów) | 3000/3000TFX<br>(N = 253)<br>liczba zdarzeń<br>(% pacjentów) |
| Zaburzenia zakrzepowo-zatorowe związane z zastawką | 6 (3,1) | 7 (2,8) | 3 (2,0) | 3 (1,4) |
| Niestrukturalna dysfunkcja zastawki (PVL) | 3 (1,5) | 4 (1,6) | 3 (2,0) | 3 (1,4) |
| Eksplantacja (NSVD) | 2 (1,0) | 2 (0,8) | 0 (0,0) | 0 (0,0) |
| Zgon (zatrzymanie akcji serca, zdarzenie typu krwawienie, CVA) | 1 (0,5) | 1 (0,4) | 3 (2,0) | 3 (1,4) |
| Powtórny zabieg operacyjny | 1 (0,5) | 1 (0,4) | 1 (0,7) | 1 (0,5) |
| Hemoliza | 1 (0,5) | 1 (0,4) | 3 (2,0) | 3 (1,4) |
| Krwawienie związane z AC | 0 (0,0) | 0 (0,0) | 2 (1,4) | 2 (1,0) |
| Zapalenie wsierdzia | 0 (0,0) | 0 (0,0) | 0 (0,0) | 0 (0,0) |
| Strukturalne pogorszenie stanu zastawki | 0 (0,0) | 0 (0,0) | 0 (0,0) | 0 (0,0) |
| Zakrzepica zastawki | 0 (0,0) | 0 (0,0) | 0 (0,0) | 0 (0,0) |
| Inne (rozdarcie aorty) | 1 (0,5) | 1 (0,4) | 0 (0,0) | 0 (0,0) |

Tabela 7. Zmienne hemodynamiczne w elektrokardiogramach dla kontroli po 1 roku, modele 3000 i 3000TFX

| Rodzaj<br>zastawki | Parametr | 19 mm<br>Średnia ± SD<br>(n) | 21 mm<br>Średnia ± SD<br>(n) | 23 mm<br>Średnia ± SD<br>(n) | 25 mm<br>Średnia ± SD<br>(n) | 27 mm<br>Średnia ± SD<br>(n) | 29 mm<br>Średnia ± SD<br>(n) |
|---|---|---|---|---|---|---|---|
| 3000TFX | Średni gradient ciśnienia | 16,7 ± 4,7 | 15,8 ± 4,4 | 11,3 ± 3,7 | 11,1 ± 4,1 | 9,4 ± 4,3 | 9,0 ± 0,0 |
| | skurczowego (mmHg) | (10) | (18) | (45) | (37) | (12) | (2) |
| | Frakcja | 65,8 ± 10,4 | 62,7 ± 9,4 | 60,6 ± 11,3 | 61,4 ± 11,2 | 59,5 ± 10,7 | 55,0 ±14,1 |
| | wyrzutowa (%) | (10) | (19) | (48) | (38) | (12) | (2) |
| | EOA aorty | 1,2 ± 0,4 | 1,5 ± 0,4 | 1,8 ± 0,6 | 1,8 ± 0,5 | 2,1 ± 0,6 | 2,1 ± 0,1 |
| | (cm²) | (10) | (18) | (44) | (36) | (12) | (2) |
| 3000/ | Średni gradient ciśnienia | 16,7 ± 4,2 | 13,8 ± 4,8 | 11,7 ± 4,7 | 11,0 ± 3,8 | 9,5 ± 4,1 | 9,0 ± 0,0 |
| 3000TFX | skurczowego (mmHg) | (16) | (34) | (56) | (47) | (14) | (2) |
| | Frakcja | 62,1 ± 15,1 | 58,6 ± 11,6 | 60,2 ± 11,2 | 60,2 ± 11,5 | 58,5 ± 10,5 | 55,0 ± 14,1 |
| | wyrzutowa (%) | (16) | (34) | (59) | (47) | (14) | (2) |
| | EOA aorty | 1,3 ± 0,5 | 1,5 ± 0,4 | 1,8 ± 0,6 | 1,8 ± 0,6 | 2,1 ± 0,6 | 2,1 ± 0,1 |
| | (cm²) | (16) | (32) | (55) | (46) | (14) | (2) |

Tabela 8. Klasa czynnościowa NYHA: Zmiana wzgledem wartości wyiściowych dla wizyty kontrolnej po 1 roku, modele 3000 i 3000TFX

| | | Wartości wyjściowe | | | | |
|---|---|---|---|---|---|---|
| Rodzaj zastawki | Klasa NYHA w<br>okresie obserwacji | Klasa I | Klasa II | Klasa III | Klasa IV | Nie dotyczy |
| | Klasa I | 10 | 33 | 51 | 10 | 3 |
| | Klasa II | 2 | 8 | 13 | 2 | 1 |
| 2000TFV | Klasa III | - | - | 3 | - | - |
| 3000TFX<br>N = 193 | Klasa IV | - | - | - | 1 | - |
| N = 195 | Zgon | - | 3 | 16 | 1 | - |
| | Eksplantacja | - | - | 3 | - | - |
| | Nie dotyczy | 2 | 6 | 21 | 4 | - |
| | Klasa I | 12 | 40 | 71 | 11 | 3 |
| | Klasa II | 2 | 14 | 29 | 3 | 1 |
| 3000/ | Klasa III | - | - | 3 | - | - |
| 3000TFX | Klasa IV | - | - | 1 | 1 | - |
| N = 253 | Zgon | - | 3 | 19 | 2 | - |
| | Eksplantacja | - | - | 3 | - | - |
| | Nie dotyczy | 2 | 7 | 22 | 4 | - |

#### Klasa czynnościowa NYHA: Zmiana względem wartości wyjściowych dla wizyty kontrolnej po 1 roku

| Rodzaj zastawki | Poprawa<br>N (%) | Bez zmian<br>N (%) | Pogorszenie<br>N (%) | Nie dotyczy<br>N (%) |
|---|---|---|---|---|
| 3000TFX (N = 193) | 109 (56,5) | 22 (11,4) | 2 (1,0) | 60 (31,1) |
| 3000/3000TFX (N = 253) 154 (60,9) | | 30 (11,9) | 3 (1,2) | 66 (26,1) |

# Symbol Legend • Légende des symboles • Legenda Symboli

| | English | Français | Polski | Г | | English | Français | Polski |
|---|---|---|---|---|---|---|---|---|
| REF | Catalogue<br>Number | Numéro de<br>référence | Numer<br>Katalogowy | | STER <b>I</b> LE EO | Ethylene<br>Oxide<br>Sterilized | Stérilisé<br>à l'oxyde<br>d'éthylène | Wysterylizowano<br>Przy Użyciu<br>Tlenku Etylenu |
| <u>^</u> | Caution | Attention | Przestroga | | | Do not use | Ne pas utiliser | Nie używać, |
| (li | Consult<br>instructions<br>for use | Consulter<br>le mode<br>d'emploi | Zapoznać się<br>z instrukcją<br>użycia | | 8 | if package<br>is opened or<br>damaged. | si l'emballage<br>est ouvert ou<br>endommagé. | jeśli opakowanie<br>jest otwarte<br>lub uszkodzone. |
| 2 | Single Use | À usage<br>unique | Do<br>jednorazowego<br>użytku | | EC REP | European<br>Authorized<br>Representative | Mandataire<br>européen | Autoryzowany<br>przedstawiciel<br>w Europie |
| # | Quantity | Quantité | llość | | | Contents<br>sterile and | Contenu stérile et<br>apyrogène si le | Zawartość<br>sterylna i |
| $\square$ | Use By | Utiliser avant | Zużyć Do | | STER <b>IL</b> E 388 | nonpyrogenic<br>if package is<br>unopened or | conditionnement<br>n'est ni ouvert ni<br>endommagé. | niepirogenna, o ile<br>opakowanie nie<br>zostało otwarte |
| SN | Serial<br>Number | Numéro<br>de série | Numer<br>Serii | | | undamaged. | | ani uszkodzone. |
| ш | Manufacturer | Fabricant | Producent | | <b>}</b> 25 ℃ | Do not freeze -<br>Store between | Ne pas<br>congeler - | Nie zamrażać -<br>Przechowywać w |
| SZ | Size | Taille | Rozmiar | | 10-7 | 10 °C and 25 °C | Conserver entre<br>10°C et 25°C | temperaturze od<br>10 °C do 25 °C |

Note: Not all symbols may be included in the labeling of this product. • Remarque: il est possible que certains symboles n'apparaissent pas sur les étiquettes de ce produit. • Uwaga: Nie wszystkie symbole muszą być użyte na etykietach niniejszego produktu.

GLX3SL5x7.1



EC REP

Germany

Edwards Lifesciences Services GmbH Edisonstr. 6 85716 Unterschleissheim

©Copyright 2014, Edwards Lifesciences LLC All rights reserved.

Manufacturer Edwards Lifes dences LLC
One Edwards Way
Irvine, CA 92614-5688 USA
Made in USA

Telephone 949.250.2500 800.424.3278 FAX 949.250.2525



2/14 156983003 A

# Vendor: Do Not Print this page. For Internal Edwards Lifesciences Use Only.

| | Title: IFU, 11000A, IDE, E, F, P | | | |
|---|---|---|---|---|
| | Part Number: 15698 | 33003 Rev.: A | Page 41 of 41 | ECR: 118875 |
| Edwards<br>Irvine, CA 92614 | Graphic Artist: Gleni | n Getler | | Date: 2/24/14 |
| First<br>Proofer: Lee Vi | ibber | Date: 2/25/14 | Second<br>Proofer: See below | Date: |
| Full<br>Proof | Proofed<br>Against<br>Redline | Docuproof X | Full X Proofed Against X Docuproof | |
| First<br>Proofer: n/a | | Date: n/a | Second<br>Proofer: Theresa Menchaca | Date: 2/28/14 |
| Pages: <b>n/a</b> | | | Pages: 1 - 25 | |
| First proofer: n/a Date: n/a | | | Second Proofer: Lenore Dunn Date: 2/28 | |
| Pages: n/a | | | Pages: 26 - 41 | |

# NOTE

1. ALL ART PRINTS 100% BLACK UNLESS OTHERWISE NOTED.

<u>INK</u> Black

# DIRECTORY English 1 Français 20 Polski 39

### English

# Edwards Pericardial Mitral Bioprosthesis, Model 11000M

#### Instructions for use

CAUTION: Investigational Device. Limited by Federal (United States) law to Investigational Use.

CAUTION: Investigational device. Exclusively for Clinical Investigations.

Caution: Investigational Device. Limited to Investigational Use. To be used by Qualified Investigators (Physicians).

#### 1. Device and Accessories Description

#### 1.1 Device Description

The Edwards Pericardial Mitral Bioprosthesis, Model 11000M, is a trileaflet bioprosthesis comprised of treated bovine pericardium that is mounted on a flexible frame. It is available in sizes 25, 27, 29, 31, and 33 mm (Table 1). The bioprosthesis is stored in non-aqueous packaging, and does not require rinsing prior to implantation.

The wireform is made of a cobalt chromium alloy covered with a woven polyester fabric. A cobalt-chromium alloy/polyester film laminate band surrounds the base of the wireform frame.

A waffled silicone sewing ring that is covered with a porous polytetrafluoroethylene (PTFE) doth is attached to the wireform frame. The sewing ring is scalloped along its anterior portion. Black silk suture markers on the anterior portion facilitate the orientation of the bioprosthesis and help avoid obstruction of the left ventricular outflow tract by a strut.

A black silk suture guide line circles the sewing ring. Placing sutures through the sewing ring and in the region from the suture guide line to the outer portion of the sewing ring eases needle penetration and provides variable compliance. The waffle has wider cells along the posterior portion, where calcifications or irregularities of the native mitral annulus are more frequent (Ref. 6).

Edwards Lifesciences, the stylized E logo, Edwards, Carpentier-Edwards, Tricentrix, PERIMOUNT, PERIMOUNT Magna, PERIMOUNT Plus, TFX and Magna Mitral Ease are trademarks of Edwards Lifesciences Corporation.



#### 1.2 Accessories Description

Accessories available for use with the 11000M bioprosthesis are:

- Tricentrix holder system
- Replica Sizer 1173R
- Barrel Sizer 1173B
- Sterilization Tray provided in model SET1173
- Handle models 1111, 1117, 1173, and 1126 (single use)

All accessories are supplied non-sterile, except for the Tricentrix holder system that is supplied sterile attached to the sterile bioprosthesis, and the handle 1126 that is supplied sterile and is for single use only.

#### Sizers and Tray

Only sizers model 1173B (Figure 1a) or 1173R (Figure 1b) may be used with the 11000M bioprosthesis.

Caution: Do not use other manufacturer's valve sizers, or sizers for other Edwards Lifesciences valve prostheses to size the 11000M bioprosthesis.

Use only the sizers model 1173B or 1173R to determine the appropriate 11000M bioprosthesis size. Sizers model 1173B and 1173R permit direct observation of their fit within the annulus and are provided for each available 11000M bioprosthesis size. The barrel of the sizers model 1173B and 1173R indicate the

external stent diameter at the base. The lip of the replica sizer 1173R replicates the sewing ring of the bioprosthesis, with its scalloped anterior portion and black markings, to determine the outcomes of specific suture or subvalvular apparatus preservation techniques.

The sizers 1173B and 1173R are labeled with the bioprosthesis size. The complete set of sizers is housed in a tray, model SET1173, which can be reused and resterilized



#### **Tricentrix Holder System and Handles**

The holder/handle assembly consists of two components: the Tricentrix holder system (Figure 2) that is mounted to the 11000M bioprosthesis, and a handle (1111, 1117, 1173, or 1126) that is attached to the Tricentrix holder system at the time of surgery.





The following handles (Table 2) may be used with the 11000M Bioprosthesis:

| Table 2. Accessory Handles | | | | |
|---|---|---|---|---|
| | | Overall | Overall Length | |
| Model | Shaft Material | inch | cm | Reusable |
| 1111 | Stainless steel | 7.0 | 17.8 | Yes |
| 1117 | Nitinol | 9.1 | 23.2 | Yes |
| 1126 | Stainless steel | 11.5 | 29.2 | No |
| 1173 | Nitinol | 11.3 | 28.6 | Yes |

Handles with a nitinol shaft are more flexible than stainless steel. With each sterilization cycle, they return to their original straight shape for easier attachment to the holder.

#### 2. Indications for Use

The Edwards Pericardial Mitral Bioprosthesis, Model 11000M is indicated for patients who require replacement of their native or prosthetic mitral valve.

#### 3. Contraindications

Do not use if the surgeon believes such would be contrary to the best interests of the patient. The actual decision for or against the use of this bioprosthesis must remain with the surgeon who can evaluate all the various risks involved, including the anatomy and pathology observed at the time of surgery.

#### 4. Warnings

FOR SINGLE USE ONLY. This device is designed, intended, and distributed for single use only. Do not re-sterilize or reuse this device. There are no data to support the sterility, nonpyrogenicity, and functionality of the device after sterile reprocessing. Exposure of the bioprosthesis or package to irradiation, steam, ethylene oxide, or other chemical sterilants will render the bioprosthesis unfit for use.

DO NOT FREEZE OR EXPOSE THE BIOPROSTHESIS TO EXTREME HEAT. Exposure of the bioprosthesis to extreme temperatures will render the device unfit for use.

#### DO NOT USE the bioprosthesis:

- If the foil pouch, sealed trays, or lids are opened, damaged, or stained
- If the expiration date has elapsed, or
- If it has been dropped, damaged, or mishandled in any way. Should a bioprosthesis be damaged during insertion, do not attempt repair.

DO NOT EXPOSE the bioprosthesis to any solutions, chemicals, antibiotics, etc., except for sterile physiological saline solution. Irreparable damage to the leaflet tissue, which may not be apparent under visual inspection, may result.

DO NOT GRASP the leaflet tissue of the bioprosthesis with instruments or cause any damage to the bioprosthesis. Even the most minor leaflet tissue perforation may enlarge in time to produce significant impairment of valve function.

DO NOT OVERSIZE. Oversizing may cause bioprosthesis damage or localized mechanical stresses, which may in turn injure the heart or result in leaflet tissue failure, stent distortion and valve regurgitation.

DO NOT PASS CATHETERS, transvenous pacing leads, or any surgical instrument across the bioprosthesis with the exception of a surgical mirror used to examine struts and suture placement. Other surgical devices may cause leaflet tissue damage.

As with any implanted medical device, there is a potential for patient immunological response. Some components of the model 11000M are a metal alloy that contains cobalt, chromium, nickel, molybdenum, manganese, carbon, beryllium and iron. Care should be exercised in patients with hypersensitivities to these materials. This device was manufactured without latex, but may have been produced in a latex-containing environment.

#### 5. Adverse Events

#### 5.1 Observed Adverse Events

As with all prosthetic heart valves, serious adverse events, sometimes leading to death, may be associated with the use of tissue valves. In addition, adverse events due to individual patient reaction to an implanted device or to physical or chemical changes to the components, particularly those of biological origin, may occur at varying intervals (hours or days) necessitating reoperation and replacement of the prosthetic device.

The Edwards Pericardial Mitral Bioprosthesis Model 11000M is similar in design to the Carpentier-Edwards PERIMOUNT Magna Mitral Ease pericardial bioprostheses model 7300TFX.

Three (3) multi-center, non-randomized, prospective non-US clinical studies were conducted with the mitral pericardial bioprosthesis model 6900. Three hundred one (301) patients had isolated mitral valve replacement (MVR) and 62 patients had double valve replacement (DVR), where the aortic valve was replaced with a Carpentier-Edwards PERIMOUNT pericardial bioprosthesis aortic model.

In the first study, bioprostheses were implanted between 1984 and 1986; in the second study, bioprostheses were implanted between 1989 and 1994; and in the third study, bioprostheses were implanted between 1996 and 1997. Patients were evaluated preoperatively, intraoperatively, at discharge, at 1 year, and annually thereafter. Adverse events were captured throughout the postoperative period.

Table 3 presents the observed rates for early events ( $\leq$  30 days for valve-related adverse events), the linearized rates for late events (> 30 days postoperatively), and the actuarial adverse event rates at 1, 5, and 8 years postoperatively for model 6900. The adverse event rates were based on 363 patients at nine centers. The cumulative follow-up was 1100 patient-years with a mean follow-up of 3.0 years (SD = 2.4 years, range = 0 to 8.2 years). Preoperative and operative patient demographics are presented in Tables 5 and 7. Effectiveness results are orsesnted in Tables 9 and 11.

One (1) multi-center, non-randomized, prospective international clinical study was conducted with patients implanted with the Carpentier-Edwards PERIMOUNT Plus pericardial bioprosthesis model 6900P mitral. One hundred seventy five (175) patients had isolated mitral replacement (MVR) and 34 patients had double valve replacement (DVR), where the aortic valve was replaced with a Carpentier-Edwards PERIMOUNT pericardial bioprosthesis aortic model. In this study, patients were implanted between 1999 and 2007. Patients were evaluated preoperatively, intraoperatively at discharge, at 1 year, and annually thereafter. Adverse events were captured throughout the postoperative period. Table 4 presents the observed rates for early events ( $\leq$  30 days for valve related adverse events), the linearized rates for late events (> 30 days postoperatively), and the actuarial adverse event rates at 1- and 5-years postoperatively for model 6900P. The adverse event rates were based on two hundred nine (209) patients at seven centers. The cumulative follow-up was 873.18 patient-years with a mean follow-up of 4.2 years (SD = 2.3 years, range = 0 to 8.2 years). Preoperative and operative patient demographics are presented in Tables 6 and 8. Effectiveness results are presented in Tables 10 and 12.

#### 5.2 Potential Adverse Events

Adverse events potentially associated with the use of bioprosthetic heart valves include:

- Angina
- Bleeding diatheses (coagulopathy) related to anticoagulant therapy
- Cardiac arrhythmias
- Coronary ostial blockage
- Endocarditis
- Heart failure
- · Hemolysis
- · Hemolytic anemia
- Hemorrhage
- · Local and/or systemic infection
- Mvocardial infarction
- · Patient prosthetic mismatch (PPM)
- · Prosthesis leaflet entrapment (Impingement)
- Prosthesis nonstructural dysfunction
- · Prosthesis pannus
- Prosthesis perivalvular leak
- Prosthesis regurgitation
- Prosthesis structural deterioration
- Prosthesis thrombosis
- Stroke
- Thromboembolism
- · Transient ischemic attack (TIA)

It is possible that these complications could lead to:

- Reoperation
- Explantation
- · Permanent disability
- Death

Other adverse events associated with the use of Carpentier-Edwards PERIMOUNT mittal pericardial bioprostheses model 6900 compiled from the literature and from reports received through the Edwards Lifesciences compilant handling system include: stenosis, regurgitation through an incompetent valve, ventricular perforation by stent posts, malfunctions of the valve due to distortion at implant, and fracture of the wireform frame.

#### 6. Clinical Studies

The safety endpoints captured in the prospective studies were adverse events; blood analyses were used to confirm the absence or presence of certain adverse events. The safety results for model 6900 are provided in Table 3 and for model 6900P in Table 4. Preoperative patient demographics for model 6900 are provided in Table 5 and for model 6900P in Table 6. Operative patient demographics for model 6900P are provided in Table 7 and for model 6900P in Table 8. Effectiveness endpoints were New York Heart Association (NYHA) functional classification summarized in Table 9 for model 6900 and Table 10 for

model 6900P and echocardiographic assessments summarized in Table 11 for model 6900 and Table 12 for model 6900P.

There are no clinical data presently available demonstrating increased resistance of the Edwards Pericardial Mitral Bioprosthesis Model 11000M to calcification as compared to other commercially available bioprostheses.

#### 7. Individualization of Treatment

Bioprosthetic heart valve recipients should be maintained on anticoagulant therapy, except where contraindicated, during the initial stages after implantation, as determined by the physician on an individual basis. Long-term anticoagulant and/or antiplatelet therapy should be considered for patients with risk factors for thromboembolism.

The ultimate judgment regarding care of a particular patient must be made by the healthcare provider and patient in light of all the circumstances presented by that patient (Ref. 7). A bioprosthesis is recommended for MVR in patients of any age who will not take warfarin or who have major medical contraindications to warfarin therapy. Patient preference is a reasonable consideration in the selection of mitral valve operation and valve prosthesis. A mechanical prosthesis is reasonable for MVR in patients under 65 years of age who do not have a contraindication to anticoagulation. A bioprosthesis is reasonable for MVR in patients under 65 years of age who elect to receive this valve for lifestyle considerations after detailed discussions of the risks of anticoagulation versus the likelihood that a second MVR may be necessary (Ref. 7).

#### 7.1 Specific Patient Populations

The safety and effectiveness of the Model 11000M bioprosthesis has not been established for the following specific populations because it has not been studied in these populations:

- · patients who are pregnant;
- nursing mothers:
- patients with abnormal calcium metabolism (e.g., chronic renal failure, hyperparathyroidism);
- patients with aneurysmal aortic degenerative conditions (e.g., cystic medial necrosis, Marfan's syndrome);
- · children, adolescents, and young adults

Caution: Based on reports in the literature on tissue valves (Refs. 9, 10, 11, 12 & 13), there appears to be an increased incidence of leaflet calcification in patients under the age of 20. When feasible, repeated intravenous injections containing calcium should be avoided uning the postoperative period, and excessive milk or dairy product consumption should be avoided in children. Animal research studies (Ref. 14) show that a high systemic calcium level can lead to early calcification.

#### 8. Patient Counseling Information

Careful and continued medical follow-up (at least by an annual visit to the physician) is advised so that bioprosthesis-related complications, particularly those related to material failure, can be diagnosed and properly managed. Patients with bioprostheses are at risk from bacteremia (e.g., undergoing dental procedures) and should be advised about prophylactic antibiotic therapy. Patients should be encouraged to carry their Patient Identification Card at all times and to inform their healthcare providers that they have an implant when seeking care.

#### 9. How Supplied

#### 9.1 Packaging

The Edwards Pericardial Mitral Bioprosthesis, Model 11000M, is provided sterile and non-pyrogenic, in a double barrier tray package. The double tray package is in a foil pouch, which is in a carton.

Each bioprosthesis is contained in a carton with a temperature indicator displayed through a window on the side panel. The temperature indicator is intended to identify products which have been exposed to transient temperature extremes. Upon receipt of the bioprosthesis, immediately inspect the indicator and refer to the carton label to confirm a "Use" condition. If the "Use" condition is not apparent, do not use the bioprosthesis and contact the local supplier or Edwards Lifesciences representative to make arrangements for return authorization and reolacement.

Warning: Carefully inspect the bioprosthesis before implantation for evidence of extreme temperature exposure or other damage.

#### 9.2 Storage

The Edwards Pericardial Mitral Bioprosthesis, Model 11000M, should be stored at  $10^{\circ}$ C to  $25^{\circ}$ C (50- $77^{\circ}$ F), in the foil pouch and shelf carton.

#### 10. Directions for Use

#### 10.1 Physician Training

The techniques for implanting this bioprosthesis are similar to those for implanting any stented mitral bioprosthesis. No special training is required to implant the Edwards Pericardial Mitral Bioprosthesis. Model 11000M.

#### 10.2 Sizing

Caution: Do not use other manufacturer's valve sizers, or sizers for other Edwards Lifesciences valve prostheses to size the 11000M bioprosthesis.

Caution: Examine sizers and handles for signs of wear, such as dullness, cracking or crazing. Replace sizer or handle if any deterioration is observed.

Warning: Fragments of handles and sizers are not radiopaque and cannot be located by means of an external imaging device.

Verify that the accessories have been sterilized according to the recommended instructions provided with the reusable accessories.

The black marks on the lip replicate the black suture markers on the sewing ring. They delimit the anterior portion of the bioprosthesis sewing ring which should be positioned across the anterior intercommissural portion of the native annulus, in order to straddle the left ventricular outflow tract area. The height and location of the stent posts are marked on the replica sizer 1173R to aid in assessing optimal alignment and seating.

The sizers include pre-attached handles with increased handle length for improved access in the case of a difficult exposure, a deep thoracic cage or minimally invasive access. The posterior handle attachment to the sizer allows an unobstructed view through the barrel into the ventricle for assessment of subvalvular structures. The sizers 1173B and 1173R are labeled with the bioprosthesis size.

| Step | Procedure |
|---|---|
| 1 | Sizing with barrel sizer 1173B: To size with barrel sizer 1173B, pass the barrel portion of the sizer through the mitral annulus. Ensure the barrel portion is directly in plane of the mitral annulus. HVT60 |
| 2 | Sizing with replica sizer 1173R: To size with replica sizer 1173R, pass the barrel portion of the replica sizer through the mitral annulus so that the tip of the sizer, which simulates the sewing ring portion of the bioprosthesis, rests on the superior aspect of the annulus. HVT61 |

Some techniques such as use of pledgets, leaflet reefing, or mitral subvalvular apparatus preservation may further reduce the size of the mitral annulus which can result in the need for a smaller bioprosthesis to be implanted (Ref. 8). When using these techniques, it is recommended to re-size the annulus to avoid oversizing of the bioprosthesis. The consistent performance of the Edwards Pericardial Mitral Bioprostheses, Model 11000M makes oversizing unnecessary to achieve the desired hemodynamic performance in most patients (Table 11 and 12).

Due to the elastic nature of a chord, it may be extended by the Tricentrix holder system during implantation but retract back around the post once the holder is removed, entrapping leaflets and impairing function. Sizers 1173B and 1173R are made of a transparent material to allow visualization of the subvalvular apparatus during sizing. Make sure no chord will be in the way of the struts.

Caution: Exercise special care when using subvalvular apparatus preservation techniques to avoid chordae entrapment by a strut.

Warning: Avoid oversizing the bioprosthesis. Oversizing may cause bioprosthesis damage or localized mechanical stresses, which may in turn injure the heart or result in leaflet tissue failure, stent distortion and requrgitation.

#### 10.3 Handling and Preparation Instructions

In-service training is recommended prior to handling and preparing the Edwards Pericardial Mitral Bioprosthesis. Model 11000M.

| | reardiar mittar bioprostricsis, model 11000m. |
|---|---|
| Step | Procedure |
| 1 | Caution: Do not open the Edwards Pericardial Mitral<br>Bioprosthesis, Model 11000M package until<br>implantation is certain. |
| | Warning: Do not open foil pouch into sterile field. Foil<br>pouch is protective cover only. Only the innermost<br>package tray may be introduced into the sterile field. |
| | Once the appropriate size bioprosthesis is chosen, remove the foil pouch from the carton in the non-sterile field. Before opening, examine the package for evidence of damage and broken or missing seals. |
| 2 | Near the sterile field, hold the base of the outer tray and peel the lid from the outer tray. |
| 3 | The inner tray and contents are sterile. Transfer the inner tray to the sterile field. The contents of the inner tray must be handled using a sterile surgical technique to prevent contamination. HYIZ6 |
| 4 | Caution: Do not open the inner package until implantation is certain and the surgeon is ready to place the valve. |
| | Caution: The bioprosthesis is not secured to the inner tray. Care should be taken while peeling the lid and removing the plastic cover. |
| | Before opening, examine the inner tray and lid for evidence of damage, stains, and broken or missing seals. Hold the base of the inner tray and peel the lid from the inner tray. |

#### Step Procedure

5

To access the bioprosthesis, remove the plastic cover by pulling up on both tabs. Discard the plastic cover.

VID6



HVT54



6 Attach the handle to the Tricentrix holder system while the bioprosthesis is still in the tray. To attach, insert the handle into the holder and turn it clockwise until a positive resistance is felt.

HVT52



Caution: Do not grasp the bioprosthesis with hands or surgical instruments.

Caution: Care should be taken to avoid entangling the serial tag in the handle during attachment.

Caution: The handle/holder assembly is required for implantation and should not be removed until the bioprosthesis is sutured to the annulus.

#### Step Procedure

Once the handle is attached, remove the whole assembly (i.e., plastic sleeve, clip, the Tricentrix holder system and bioprosthesis) from the tray. The plastic sleeve is loosely fitted to the clip and may remain in the tray. This will not affect deployment.

HVT53

CP1089-23



Grasping the plastic sleeve or clip continue the rotation to overcome the resistance until the white holder post reaches the unlock position.

Or CP1089-6



| Step | Procedure | Step | Procedure |
|---|---|---|---|
| 8 | Apply the required push force on the handle until the white holder post slides across the leaflets and snaps into its fully deployed position. An audible click may be heard as the deployed position is reached. OP 1089-24 | 11 | Remove the clip by sliding it off the holder in a sideways direction. |
| 9 | Caution: If an adequate push force is not applied to the<br>handle when deploying the Tricentrix holder system,<br>the tenting system will not be secured and will not be<br>able to minimize the potential for suture entrapment. | | Both sleeve and clip should be discarded. |
| | Always check for proper deployment. There should be no more space between the blue adapter and the grey holder. The handle/post assembly should no longer be able to slide. The white holder post should protrude through the leaflets while the three commissures should deflect slightly towards the center of the bioprosthesis. The leaflets will temporarily be wrinkled by the deployed white holder post. When the holder is removed following implantation, the leaflets will return to their normal position. HVT56 | 12 | A serial number tag is attached to the sewing ring of each bioprosthesis by a suture. This serial number should be confirmed with the number on the bioprosthesis package and bioprosthesis implant data card. This tag should not be detached from the bioprosthesis until implantation is certain. Caution: If any difference in serial number is noted, the bioprosthesis should be returned unused. Caution: Care should be exercised to avoid cutting or tearing the sewing ring cloth during removal of the serial number tag. Caution: To prevent damage to the sewing ring cloth, avoid pulling the knot of the serial tag suture through the sewing ring. |
| 10 | | 13 | The Edwards Pericardial Mittal Bioprosthesis, Model 11000M, DOES NOT REQUIRE RINSING prior to implantation. Caution: If the bioprosthesis is rinsed prior to implantation, it must then be kept hydrated with sterile physiological saline irrigation on both sides of the leaflet tissue throughout the remainder of the surgical procedure. Rinsing every one to two minutes is recommended. |
| 10 | After deployment, remove the sleeve (if attached) by holding the handle and pulling the sleeve off the dip. (P1089-25 | | Caution: Avoid contact of the leaflet tissue with towels, linens, or other sources of particulate matter that may be transferred to the leaflet tissue. |

#### 10.4 Device Implantation

# Step Procedure

1

The surgeon should be familiar with the recommendations for proper sizing and placement in the supra-annular position (See 10.2 Sizing).

Because of the complexity and variation of cardiac valve replacement surgery, the choice of surgical technique, appropriately modified in accordance with the previously described **Warnings**, is left to the discretion of the individual surgeon. In general, the following steps should be employed:

- Surgically remove the diseased or damaged valve leaflets and all associated structures deemed necessary.
- Surgically remove any calcium from the annulus to ensure proper seating of the sewing ring of the bioprosthesis to avoid damage to the delicate leaflet tissue.
- 3. Proper sizing. Measure the annulus using only the mitral sizer models 1173B and 1173B (Figures 1a-1b).
- 4. Proper seating of the prosthesis;
- 5. Tying sutures with the holder in place to minimize the potential for suture looping or chordal entrapment;
- Examination of the bioprosthetic leaflets for distortion or leak during tying.

Caution: When choosing a bioprosthesis for a given patient, the size, age, and physical condition of the patient in relation to the size of the bioprosthesis must be taken into consideration to minimize the possibility of obtaining a suboptimal hemodynamic result. The selection of a bioprosthesis, however, must ultimately be made by the physician on an individual basis after carefully weighing all of the risks and benefits to the patient.

Caution: Adequate removal of calcium deposits from the patient's annulus must be performed before implantation to avoid damage to the delicate bioprosthesis leaflet tissue as a result of contact with calcium deposits. Insert the sizer into the mitral annulus. The barrel of the sizer should always fit comfortably in the annulus.

Caution: Use only sizers 1173B or 1173R during the selection of the bioprosthesis size; other sizers may result in improper valve selection (see 1.2 Accessory Description). Like other mitral bioprostheses, the Edwards Pericardial Mitral Bioprosthesis, Model 11000M is usually implanted using pledgeted mattress sutures. It is recommended to size the annulus after the sutures have been placed, as sutures may decrease the size of the bioprosthesis that can be implanted.

#### Step Procedure

2 Proper orientation of the bioprosthesis:

Caution: The wireform frame of the Model 11000M bioprosthesis is symmetrical, and the three commissure supports (struts) are equally spaced. However, the sewing ring is designed for a specific orientation of the bioprosthesis. The scalloped part of the sewing ring, between the two silicone protrusions, should be placed across the intercommissural anterior portion of the annulus and straddle the left ventricular outflow tract.

The contrasting suture markers in the sewing ring are intended to aid in proper orientation and denote a typical intercommissural distance. However, this distance may vary for each individual patient. On the left side, two close black sutures indicate where the first stitch should be placed and correspond to the anterior commissure. On the right side, only one black suture indicates the approximate location of the posterior commissure. Using these orientation aids, the third post should naturally fall in place in or around the middle of the posterior leafler location.

Caution: Special care must be exercised to avoid placing a strut in front of the left ventricular outflow tract, as it may impair the long-term hemodynamic performance.

#### 3 Suture Placement:

A black suture guide line circles the sewing ring. When placing sutures through the sewing ring, sliding drag forces are reduced when sutures are placed straight through the sewing ring and in the region from the suture guide line to the outer portion of the sewing ring.

Firm tension must be maintained on the sutures as the bioprosthesis is lowered into the annulus; this minimizes the potential for formation of suture loops that might entrap a leaflet. This, when combined with the fully retracted stent posts when the Tricentrix holder system is in place, helps guide the sutures into their correct position behind the struts and onto the sewing ring.

Remove the handle prior to tying the sutures. The handle and blue adapter must be removed as an assembly. Maintain the bioprosthesis placement in the annulus by gently placing forceps or gloved hands onto the holder and cutting the green thread on the blue adapter. Remove the blue adapter and handle assembly as one unit.

CP1089-27



#### Step Procedure

Caution: Avoid looping or catching a suture around the open cages, free struts, or commissure supports of the bioprosthesis, which would interfere with proper valvular function. To minimize the potential for suture looping, it is essential to leave the deployed holder in place until all knots are tied.

However, if leaving the holder in place obstructs the surgeon's view, all the sutures adjacent to each of the three frame struts must be tied down before cutting the three green holder attachment threads to remove the holder.

Caution: If the deployed holder attachment threads are cut before these adjacent sutures are tied down, the holder will no longer minimize the potential for suture looping around the frame struts.

Special attention must be given to avoid tying the sutures on top of the corners of the holder's grey legs. Before tying each suture, examine the leaflets while holding the two strands of the suture under tension. Distortion or movement of the leaflets during this maneuver suggests that the suture is looped around a strut. At no point before or after holder removal should tension on the sutures be released as this may facilitate formation of loops in the sutures and possible entrapment. It is recommended to place a surgical mirror through the leaflets after the holder removal in order to examine each strut and proper suture placement.

Caution: When using interrupted sutures, it is important to cut the sutures close to the knots and to ensure that exposed suture tails will not come into contact with the leaflet tissue (Ref. 8).

The Tricentrix holder system is removed as a unit at the completion of the suturing procedure as follows:

CP1089-14



- Cut each of the three (3) exposed green sutures using a scalpel
  or scissor placed only in the cutting channel. Never attempt to
  cut a suture below a partially separated holder as a part of the
  attaching suture may fall in the ventricle. Avoid cutting or
  damaging the stent or leaflet tissue when cutting the sutures.
- When all three (3) attaching sutures have been properly cut, remove the Tricentrix holder system from the bioprosthesis as a unit, along with attaching sutures, using sterile gloved hands or protected forceps.
- Following implant, remove the holder and discard.

#### 10.5 Accessory Cleaning and Sterilization

The accessories for the Edwards Pericardial Mitral Bioprosthesis, Model 11000M, are packaged separately. Handle model 1126 is provided sterile and is intended for single use only. Handle models 1111, 1117 and 1173 and sizer models 1173B and 1173R are supplied nonsterile and must be cleaned and sterilized before use. The handles, sizers, tray base and tray lid must be cleaned and resterilized prior to each use. Refer to the Instructions for Use supplied with the reusable accessories for cleaning and sterilization instructions.

#### 10.6 Return of Bioprostheses

Edwards Lifesciences is interested in obtaining recovered clinical specimens of the Edwards Pericardial Mitral Bioprosthesis, Model 11000M, for analysis. Contact the local representative for return of recovered bioprostheses.

- Unopened Package with Sterile Barrier Intact: If the foil pouch or trays have not been opened, return the bioprosthesis in its original packaging.
- Package Opened but Bioprosthesis Not Implanted: If the tray is opened, the bioprosthesis is no longer sterile. If the bioprosthesis is not implanted, it should be placed into a suitable histological fixative such as 10% formalin or 2% glutaraldehyde and returned to the company. Refrigeration is not necessary under these circumstances.
- Explanted Bioprosthesis: The explanted bioprosthesis should be placed into a suitable histological fixative such as 10% formalin or 2% glutaraldehyde and returned to the company. Refrigeration is not necessary under these circumstances.

# 11. Safety in the Magnetic Resonance (MR) Environment



#### MR Conditional

Non-clinical testing has demonstrated that the Edwards Pericardial Mitral Bioprosthesis, Model 11000M is MR Conditional. A patient with the model 11000M bioprosthesis can be scanned safely, immediately after placement of this implant under the following conditions:

- Static magnetic field of 3 tesla or less.
- Maximum Spatial gradient field of 720 gauss/cm.
- Maximum MR system-reported whole-body-averaged specific absorption rate (SAR) of 3W/kg for 15 minutes of scanning.

In non-clinical testing, the Edwards Pericardial Mitral Bioprosthesis, Model 11000M, produced a temperature rise of less than or equal to 0.5 °C at a maximum MR system reported whole-body-averaged specific absorption rate (SAR) of 3W/kg for 15 minutes of MR scanning in a 3 tesla MR system (Excite, Software 63.0-052B, General Electric Healthcare).

MR image quality may be compromised if the area of interest is in the same area or relatively close to the position of the Model 11000M bioprosthesis. Optimization of MR imaging parameters is recommended.

#### 12. Patient Information

#### 12.1 Study Identification Card

A Study Identification Card is provided to each subject implanted with the Edwards Pericardial Mitral Bioprosthesis, Model 11000M.

#### 12.2 Patient Information Materials

Patient information materials may be obtained from Edwards or an Edwards clinical sales specialist.

#### 13. References

- Marchand MA., et al. Fifteen-year Experience with the Mitral Carpentier-Edwards PERIMOUNT Pericardial Bioprosthesis. Ann Thorac Surg. 2001; 71:5236-9.
- Liao K., et al. Bovine Pericardium versus Porcine Aortic Valve: Comparison of Tissue Biological Properties As Prosthetic Valves; Artificial Organs. 1992:16(4):361-5.
- Vesely I., et al. Comparison of the Compressive Buckling of Porcine Aortic Valve Cusps and Bovine Pericardium. J. Heart Valve Dis. January 1998; 7(1):34-9.
- Carpentier A. From Valvular Xenograft to Valvular Bioprosthesis (1965-1977). Med. Instrum. 1977; 11(2):98-101.
- Carpentier A., et al. Continuing Improvements in Valvular Bioprostheses. J. Thorac. Cardiovasc. Surg. 1982; 83(1):27-42.
- Arounlangsy P., et al. Histopathogenesis of early stage mitral annular calcification. J. Med Dent Sci. 2004; 51(1):35-44.
- Bonow RO., et al. ACC/AHA Guidelines for the Management of Patients With Valvular Heart Disease: A Report of the American College of Cardiology/ American Heart Association Task Force on Practice Guidelines (Committee on Management of Patients with Valvular Heart Disease). J. Am Coll Cardiol. 2006; 48:e1–148.
- Aagaard J., et al. Mitral valve replacement with total preservation of native valves and subvalvular apparatus. J. Heart Valve Dis. May 1997; 6(3):274-8; discussion 279-80.
- Jamieson, W.R.E., et al. Carpentier-Edwards Standard Porcine Bioprosthesis: Primary Tissue Failure (Structural Valve Deterioration) by Age Groups. Ann Thorac Surg 1988, 46:155-162.
- Odell, J.A. Calcification of Porcine Bioprostheses in Children. In Cohn, L. and V. Gallucci (eds): Cardiac Bioprostheses. Yorke Medical Books. New York, 1982, pp 231-237.
- Reul, G.J., et al. Valve Failure with the lonescu-Shiley Bovine Pericardial Bioprosthesis: Analysis of 2680 Patients. J. Vasc Surg 1985, 2(1):192-204.
- Sanders, S.P., et al. Use of Hancock Porcine Xenografts in Children and Adolescents. Am J. Cardiol 1980, 46(3):429-438.
- Silver, M.M., et al. Calcification in Porcine Xenograft Valves in Children. Am J. Cardiol 1980, 45:685-689.
- 14. Carpentier, A., et al. Continuing Improvements in Valvular Bioprostheses.

  J. Thorac Cardiovasc Sura 1982, 83(1):27-42.

Prices subject to change without notice. This product is manufactured and distributed under at least one or more of the following U.S. Patents: US-Patent Nos. 5,928,281; 5,931,969; 5,961,549; 6,102,944; 6,245,105; 6,413,275; 6,416,547; 6,561,970; 6,585,766; 6,837,902; 6,945,997; 6,966,925; RE 40570; 7,214,344; 7,658,763; 7,682,391; 7,972,376; 8,007,992; 8,357,387; and 8,632,608; and corresponding foreign patents. Likewise, additional patents pending.

Refer to the symbol legend at the end of this document.

#### Table 3: Observed Adverse Event Rates for MVR and DVR (Model 6900)

All patients analyzed: N = 363

Cumulative follow-up: 1100 patient-years

| | Early | Events | Late Events <sup>1</sup> | | Freedom from Event (%) [95% CI] <sup>2</sup> | | |
|---|---|---|---|---|---|---|---|
| Complication | n <sup>3</sup> | % | n | %/ptyr. | 1 year (n = 287) | 5 years (n = 141) | 8 years (n = 18) |
| Mortality (all) | 34 | 9.4 | 50 | 4.7 | 85.5 [81.8, 89.2] | 75.4 [70.3, 80.6] | 65.4 [57.6, 73.2] |
| Valve-related events | | | | | | | |
| Mortality (valve-related) | 0 | 0 | 16 | 1.5 | 97.7 [96.0, 99.4] | 95.3 [92.8, 97.8] | 91.9 [87.5, 96.4] |
| Explants | 0 | 0 | 8 | 0.7 | 98.7 [98.0, 99.3] | 96.7 [95.3, 98.0] | 95.6 [93.9, 97.3] |
| Reoperations | 2 | 0.6 | 12 | 1.1 | 97.1 [96.2, 98.1] | 95.1 [93.6, 96.6] | 93.0 [90.9, 95.1] |
| Anticoagulant-related<br>hemorrhage | 2 | 0.6 | 9 | 0.8 | 97.1 [95.2, 99.0] | 97.1 [95.2, 99.0] | 94.1 [88.2, 100] |
| Endocarditis | 1 | 0.3 | 3 | 0.3 | 99.0 [97.9, 100] | 98.7 [97.4, 98.9] | 98.7 [97.4, 98.9] |
| Hemolysis | 0 | 0.0 | 1 | 0.1 | 99.7 [99.0, 100] | 99.7 [99.0, 100] | 99.7 [99.0, 100] |
| Nonstructural dysfunction | 0 | 0.0 | 3 | 0.3 | 100 [100, 100] | 99.3 [98.0, 100] | 98.3 [95.9, 100] |
| Perivalvular leak (all) | 1 | 0.3 | 5 | 0.5 | 98.4 [97.0, 99.8] | 98.4 [97.0, 99.8] | 97.3 [94.9, 99.8] |
| Structural valve deterioration | 0 | 0.0 | 5 | 0.5 | 100.0 [100, 100] | 97.6 [95.2, 100] | 92.8 [85.3, 100] |
| Thromboembolism | 5 | 1.4 | 8 | 0.7 | 97.5 [95.8, 99.2] | 96.1 [93.8, 98.5] | 96.1 [93.8, 98.5] |
| Thrombosis | 0 | 0.0 | 0 | 0.0 | 100.0 [100, 100] | 100.0 [100, 100] | 100.0 [100, 100] |

#### Notes:

- Late event rates were calculated as linearized rates (%/pt-yr) based on 1072.5 late patient-years (> 30 days postoperatively).
- Freedom from event rates were calculated using the Kaplan-Meier method. Greenwood's formula was used for calculation of the standard errors of these estimates.
- n = number of events.

Table 4: Observed Adverse Event Rates (Model 6900P)

All patients analyzed: N = 209

Cumulative follow-up: 873.18 total pt-vrs.

| | , | iii paueiii: | anaryzeu. | . H — 209 | Cullidiative follow-up. 673. 16 total pt-yis | ). |
|---|---|---|---|---|---|---|
| | Early | Events | Late | e Events1 | Freedom from Event (%) [95% CI] <sup>2</sup> | |
| Complication | n <sup>3</sup> | % | n | %/pt-yr | 1 year | 5 years |
| Mortality (all) | 3 | 1.4 | 45 | 5.3 | 93.2 [88.8, 95.9] | 74.4 [66.9, 80.5] |
| Valve-related events | | | | | | |
| Mortality (valve-related) | 1 | 0.5 | 12 | 1.4 | 98.5 [95.5, 99.5] | 92.0 [86.2, 95.5] |
| Explants | 1 | 0.5 | 8 | 0.9 | 97.5 [94.0, 98.9] | 96.5 [92.2, 98.5] |
| Reoperations | 0 | 0.0 | 0 | 0.0 | 100.0 [100, 100] | 100.0 [100, 100] |
| Bleeding Events | 5 | 2.4 | 13 | 1.5 | 96.1 [92.3, 98.0] | 91.9 [86.5, 95.2] |
| Endocarditis | 1 | 0.5 | 3 | 0.4 | 99.5 [96.6, 99.9] | 97.1 [92.1, 98.9] |
| Nonstructural dysfunction | 0 | 0.0 | 1 | 0.1 | 99.5 [96.4, 99.9] | 99.5 [96.4, 99.9] |
| Perivalvular leak (all) | 1 | 0.5 | 2 | 0.2 | 99.5 [96.7, 99.9] | 98.4 [95.2, 99.5] |
| Structural valve deterioration | 0 | 0.0 | 2 | 0.2 | 100.0 [100, 100] | 99.0 [93.2, 99.9] |
| Thromboembolism | 4 | 1.9 | 12 | 1.4 | 97.0 [93.5, 98.7] | 91.3 [85.8, 94.7] |
| Thrombosis | 0 | 0.0 | 0 | 0.0 | 100.0 [100, 100] | 100.0 [100, 100] |

#### Notes:

- Late event rates were calculated as linearized rates (%/pt-yr) based on 856.24 late patient-years (> 30 days postoperatively).
- Freedom from event rates were calculated using the Kaplan-Meier method. Greenwood's formula was used for calculation of the standard errors of these estimates.
- n = number of events.

Table 5: Preoperative Patient Demographics (Model 6900)

| | | Study Characteristics (N = 363; 1100 total pt-yrs.) | |
|---|---|---|---|
| Variable | Category | n % (n/N) <sup>1</sup> | |
| Age at implant (N = 363) | Mean ± SD | 66.1 ± 10.7 | |
| Gender | Female/Male | 212/151 58.4%/41.6% | |
| | None | 30 | 8.3% |
| Diamonia/Féinlean | Stenosis | 91 | 25.1% |
| Diagnosis/Etiology | Regurgitation | 184 | 50.7% |
| | Mixed Disease | 58 | 16.0% |

#### Note:

1. n = number of patients in each category; N = total number of study patients.

#### Table 6: Preoperative Patient Demographics (Model 6900P)

| | | Study Characteristics (N = 209; 873.18 total pt-yrs.) | |
|---|---|---|---|
| Variable | Category | n % (n/N) <sup>1</sup> | |
| Age at implant (N = 209) | Mean ± SD | 71.4 ± 9.4 | |
| Gender | Female/Male | 138/71 | 66.0%/34.0% |
| | Mixed Disease | 48 | 23.0% |
| Diagnosis/Etiology | Regurgitation | 121 | 57.9% |
| | Stenosis | 32 | 15.3% |
| | Valve Dysfunction | 8 | 3.8% |

#### Note:

<sup>1.</sup> n = number of patients in each category; N = total number of study patients.

Table 7: Operative Patient Demographics (Model 6900)

| Variable Category n % (n/N)¹ Rheumatic heart disease 135 37.2% Calcification 82 22.6% Degeneration 50 13.8% Etiology² Endocarditis 39 10.7% Failed Bioprosthesis 15 4.1% Ischemic Heart Disease 14 3.9% Congenital Abnormalities 8 2.2% Other 44 12.1% None 200 55.1% CABG³ 78 21.5% Tricuspid Repair 61 16.8% Intra-aortic balloon pump 17 4.7% Pacemaker⁴ 6 1.7% Aneurysm Repair 4 1.1% Aneurysm Repair 4 1.1% Other 31 8.5% Pre-existing Conditions² 72 19.8% Hypertension 61 16.8% Hypertension 61 16.8% Previous MI6 45 12.4% Cere | | | aracteristics<br>00 total pt-yrs.) | |
|---|---|---|---|---|
| Calcification 82 22.6% Degeneration 50 13.8% Endocarditis 39 10.7% Failed Bioprosthesis 15 4.1% Ischemic Heart Disease 14 3.9% Congenital Abnormalities 8 2.2% Other 44 12.1% None 200 55.1% CABG³ 78 21.5% Tricuspid Repair 61 16.8% Intra-aortic balloon pump 17 4.7% Pacemaker⁴ 6 1.7% Aortic repair/replacement 5 1.4% Aneurysm Repair 4 1.1% Other 31 8.5% None 122 33.6% CAD5/CABG 72 19.8% Hypertension 61 16.8% Hypertension 61 16.8% Previous MI6 45 12.4% Cerebrovascular Disease 36 9.9% Other 234 64.5% 25 22 6.1% | Variable | Category | n | % (n/N) <sup>1</sup> |
| Degeneration 50 13.8% | | Rheumatic heart disease | 135 | 37.2% |
| Etiology2 Endocarditis 39 10.7% Failed Bioprosthesis 15 4.1% Ischemic Heart Disease 14 3.9% Congenital Abnormalities 8 2.2% Other 44 12.1% None 200 55.1% CABG³ 78 21.5% Tricuspid Repair 61 16.8% Intra-aortic balloon pump 17 4.7% Pacemaker⁴ 6 1.7% Aortic repair/replacement 5 1.4% Aneurysm Repair 4 1.1% Other 31 8.5% None 122 33.6% CAD⁵/CABG 72 19.8% Hypertension 61 16.8% Pre-existing Conditions² Atrial Fibrillation 53 14.6% Previous MI6 45 12.4% Cerebrovascular Disease 36 9.9% Other 234 64.5% 25 22 6.1% | | Calcification | 82 | 22.6% |
| Failed Bioprosthesis 15 | | Degeneration | 50 | 13.8% |
| Failed Bioprostnesis 15 | Fr. 1 | Endocarditis | 39 | 10.7% |
| Congenital Abnormalities 8 2.2% | Etiology <sup>2</sup> | Failed Bioprosthesis | 15 | 4.1% |
| Other 44 12.1% None 200 55.1% CABG³ 78 21.5% Tricuspid Repair 61 16.8% Intra-aortic balloon pump 17 4.7% Pacemaker⁴ 6 1.7% Aortic repair/replacement 5 1.4% Aneurysm Repair 4 1.1% Other 31 8.5% None 122 33.6% CAD⁵/CABG 72 19.8% Hypertension 61 16.8% Pre-existing Conditions² Atrial Fibrillation 53 14.6% Previous MI6 45 12.4% Cerebrovascular Disease 36 9.9% Other 234 64.5% 25 22 6.1% | | Ischemic Heart Disease | 14 | 3.9% |
| None | | Congenital Abnormalities | 8 | 2.2% |
| CaBG <sup>3</sup> 78 21.5% Tricuspid Repair 61 16.8% Intra-aortic balloon pump 17 4.7% Pacemaker <sup>4</sup> 6 1.7% Aortic repair/replacement 5 1.4% Aneurysm Repair 4 1.1% Other 31 8.5% None 122 33.6% CAD <sup>5</sup> /CABG 72 19.8% Hypertension 61 16.8% Pre-existing Conditions <sup>2</sup> Atrial Fibrillation 53 14.6% Previous MI <sup>6</sup> 45 12.4% Cerebrovascular Disease 36 9.9% Other 234 64.5% | | Other | 44 | 12.1% |
| Tricuspid Repair 61 16.8% Intra-aortic balloon pump 17 4.7% Pacemaker <sup>4</sup> 6 1.7% Aortic repair/replacement 5 1.4% Aneurysm Repair 4 1.1% Other 31 8.5% None 122 33.6% CAD <sup>5</sup> /CABG 72 19.8% Hypertension 61 16.8% Pre-existing Conditions <sup>2</sup> Atrial Fibrillation 53 14.6% Previous MI <sup>6</sup> 45 12.4% Cerebrovascular Disease 36 9.9% Other 234 64.5% 25 22 6.1% | | None | 200 | 55.1% |
| Intra-aortic balloon pump 17 4.7% | | CABG <sup>3</sup> | 78 | 21.5% |
| Pacemaker4 | Concomitant Procedures <sup>2</sup> | Tricuspid Repair | 61 | 16.8% |
| Pacemaker4 | | Intra-aortic balloon pump | 17 | 4.7% |
| Aneurysm Repair 4 1.1% Other 31 8.5% None 122 33.6% CAD <sup>5</sup> /CABG 72 19.8% Hypertension 61 16.8% Pre-existing Conditions <sup>2</sup> Atrial Fibrillation 53 14.6% Previous MI <sup>6</sup> 45 12.4% Cerebrovascular Disease 36 9.9% Other 234 64.5% 25 22 6.1% | | Pacemaker <sup>4</sup> | 6 | 1.7% |
| Other 31 8.5% None 122 33.6% CAD <sup>5</sup> /CABG 72 19.8% Hypertension 61 16.8% Pre-existing Conditions <sup>2</sup> Atrial Fibrillation 53 14.6% Previous MI6 45 12.4% Cerebrovascular Disease 36 9.9% Other 234 64.5% 25 22 6.1% | | Aortic repair/replacement | 5 | 1.4% |
| None | | Aneurysm Repair | 4 | 1.1% |
| CAD <sup>5</sup> /CABG 72 19.8% | | Other | n cheart disease 135 | 8.5% |
| Hypertension 61 16.8% | | None | 122 | 33.6% |
| Pre-existing Conditions <sup>2</sup> Atrial Fibrillation 53 14.6% Previous MI <sup>6</sup> 45 12.4% Cerebrovascular Disease 36 9.9% Other 234 64.5% 25 22 6.1% | | CAD <sup>5</sup> /CABG | 72 | 19.8% |
| Previous MI <sup>6</sup> 45 12.4% Cerebrovascular Disease 36 9.9% Other 234 64.5% 25 22 6.1% | | Hypertension | 61 | 16.8% |
| Cerebrovascular Disease 36 9.9% Other 234 64.5% 25 22 6.1% | Pre-existing Conditions <sup>2</sup> | Atrial Fibrillation | 53 | 14.6% |
| Other 234 64.5% 25 22 6.1% | The existing conditions | Previous MI <sup>6</sup> | 45 | 12.4% |
| 25 22 6.1% | | Cerebrovascular Disease | 36 | 9.9% |
| | | Other | 234 | 64.5% |
| 27 110 30.3% | | 25 | 22 | 6.1% |
| | | 27 | 110 | 30.3% |
| Valve Size (mm) 29 137 37.7% | Valve Size (mm) | 29 | 137 | 37.7% |
| 31 81 22.3% | | 31 | 81 | 22.3% |
| 33 13 3.6% | | 33 | 13 | 3.6% |

#### Notes:

- 1. n = number of patients in each category; N = total number of study patients
- May be more than one per patient
   CABG = Coronary Artery Bypass Graft
- 4. Permanent or temporary
- CAD = Coronary Artery Disease
   MI = Myocardial Infarction

Table 8: Operative Patient Demographics (Model 6900P)

| | | Study Characteristics (N = 209; 873.18 total pt-yrs.) | |
|---|---|---|---|
| Variable | Category | n | % (n/N) <sup>1</sup> |
| | Calcified | 38 | 18.2% |
| | Congenital | 1 | 0.5% |
| | Degenerative | 105 | 50.2% |
| Etiology <sup>2</sup> | Endocarditis Remote | 10 | 4.8% |
| | Ischemic | 12 | 5.7% |
| | Rheumatic | 64 | 30.6% |
| | Other | 36 | 17.2% |
| | None | 91 | 43.5% |
| | Aortic Valve/Annulus Repair | 3 | 1.4% |
| C | CABG <sup>3</sup> | 58 | 27.8% |
| Concomitant Procedures <sup>2</sup> | Permanent Pacemaker | 1 | 0.5% |
| | Tricuspid Valve/Annulus Repair | 21 | 10.0% |
| | Other | 78 | 37.3% |
| | None | 17 | 8.1% |
| | Arrhythmias | 95 | 45.5% |
| | CAD <sup>4</sup> | 85 | 40.7% |
| | Cardiomyopathy | 13 | 6.2% |
| | Congestive Heart Failure | 66 | 31.6% |
| | Endocarditis | 14 | 6.7% |
| Pre-existing Conditions <sup>2</sup> | Myocardial Infarction | 21 | 10.0% |
| | Peripheral Vascular Disease | 9 | 4.3% |
| | Pulmonary Hypertension | 66 | 31.6% |
| | Rheumatic Fever | 16 | 7.7% |
| | Systemic Hypertension | 49 | 23.4% |
| | TIA <sup>5</sup> /CVA <sup>6</sup> | 24 | 11.5% |
| | Other | 35 | 16.7% |
| | 25 | 28 | 13.4% |
| | 27 | 37 | 17.7% |
| Valve Size (mm) | 29 | 84 | 40.2% |
| | 31 | 43 | 20.6% |
| | 33 | 17 | 8.1% |

#### Notes:

- 1. n = number of patients in each category; N = total number of study patients
- May be more than one per patient
   CABG = Coronary Artery Bypass Graft
   CAD = Coronary Artery Disease
- 5. TIA = Transient Ischemic Attack
- 6. CVA = Cerebral Vascular Accident

Table 9: Effectiveness Outcomes, Functional NYHA (Model 6900)

| | Preoperative<br>Assessment | | Preoperative Postoperative Assessments | | | |
|---|---|---|---|---|---|---|
| | | | 1 to 2 Year | | 5 Year | |
| NYHA Functional Class | n/N <sup>1</sup> | % | n/N | % | n/N | % |
| I | 11/363 | 3.0 | 120/268 | 44.8 | 40/129 | 31.0 |
| II | 73/363 | 20.1 | 90/268 | 33.6 | 25/129 | 19.4 |
| III | 192/363 | 52.9 | 15/268 | 5.6 | 1/129 | 0.8 |
| IV | 84/363 | 23.1 | 0/268 | 0.0 | 0/129 | 0.0 |
| Not Available | 3/363 | 0.8 | 43/268 | 16.0 | 63/129 | 48.8 |

#### Note:

1. n = number of patients in each category; N = total number of study patients.

Table 10: Effectiveness Outcomes, Functional NYHA (Model 6900P)

| | Preoperative<br>Assessment | | | Postoperative | Assessments | |
|---|---|---|---|---|---|---|
| | | | 1 Y | ear | 5 Y | ear |
| NYHA Functional Class | n/N <sup>1</sup> | % | n/N | % | n/N | % |
| l | 6/209 | 2.9 | 86/187 | 46.0 | 30/96 | 31.3 |
| II | 27/209 | 12.9 | 68/187 | 36.4 | 33/96 | 34.4 |
| III | 121/209 | 57.9 | 8/187 | 4.3 | 6/96 | 6.3 |
| IV | 55/209 | 26.3 | 1/187 | 0.5 | 0/96 | 0.0 |
| Not Available | 0/209 | 0.0 | 24/187 | 12.8 | 27/96 | 28.1 |

#### Note:

1. n = number of patients in each category; N = total number of study patients.

Table 11: Effective Outcomes, Hemodynamic Results<sup>1</sup> (Model 6900)

| Hemodynamic<br>Parameter | Results By Valve Size | | | | |
|---|---|---|---|---|---|
| | 25 mm | 27 mm | 29 mm | 31 mm | 33 mm |
| Discharge/Early Post-Im | plant (n = 130, 109 MVR <sup>2</sup> an | d 21 DVR³) | | | |
| Mean gradient <sup>4</sup> | n=3 | n = 23 | n=36 | n = 23 | n=3 |
| • mean ± sd | 5.7 ± 1.2 | 4.2 ± 1.7 | 4.2 ± 1.7 | 3.6 ± 1.0 | 7.5 ± 5.8 |
| • min, max | 5,7 | 2,9 | 1,8 | 2, 5 | 3,14 |
| EOA <sup>5</sup> | n = 1 | n = 17 | n = 22 | n = 25 | n = 5 |
| • mean ± sd | 1.5 | 2.9 ± 0.9 | 3.1 ± 0.9 | 2.5 ± 0.7 | 3.0 ± 1.2 |
| • min, max | 1.5, 1.5 | 1.3, 4.1 | 1.4, 4.2 | 1.5, 3.8 | 1.6, 4.9 |
| Regurgitation <sup>6</sup> | n=3 | n = 28 | n = 51 | n = 40 | n = 8 |
| 0 | 3/3 (100%) | 22/28 (79%) | 36/51 (71%) | 30/40 (75%) | 4/8 (50%) |
| 1+ | 0/3 (0%) | 5/28 (18%) | 13/51 (25%) | 7/40 (18%) | 4/8 (50%) |
| 2+ | 0/3 (0%) | 0/28 (0%) | 1/51 (2%) | 3/40 (7%) | 0/8 (0%) |
| 3+ | 0/3 (0%) | 0/28 (0%) | 1/51 (2%) | 0/40 (0%) | 0/8 (0%) |
| 4+ | 0/3 (0%) | 0/28 (0%) | 0/51 (0%) | 0/40 (0%) | 0/8 (0%) |
| Not available | 0/3 (0%) | 1/28 (3%) | 0/51 (0%) | 0/40 (0%) | 0/8 (0%) |
| 3 to 6 Month Post-Impla | int Interval (n = 49, 42 MVR <sup>2</sup> | and 7 DVR <sup>3</sup> ) | | | |
| Mean gradient <sup>4</sup> | n=5 | n = 19 | n = 15 | n = 5 | n = 2 |
| • mean ± sd | 6.4 ± 1.7 | 5.3 ± 5 | 3.4 ± 1.2 | 4±1.9 | 4±0 |
| • min, max | 5,9 | 2, 25 | 2,6 | 2,7 | 4, 4 |
| E0A <sup>5</sup> | n=5 | n = 18 | n = 13 | n = 5 | n = 2 |
| • mean ± sd | 2.9 ± 0.8 | 2.6 ± 0.7 | 2.8 ± 0.6 | 2.9 ± 0.3 | 2.6 ± 1 |
| • min, max | 1.8, 3.6 | 1.5, 5 | 2, 3.8 | 2.4, 3.3 | 2, 3.3 |
| Regurgitation <sup>6</sup> | n=5 | n = 21 | n = 15 | n=6 | n = 2 |
| 0 | 3/5 (60%) | 17/21 (81%) | 6/15 (40%) | 4/6 (67%) | 1/2 (50%) |
| 1+ | 0/5 (0%) | 4/21 (19%) | 8/15 (53%) | 2/6 (33%) | 0/2 (0%) |
| 2+ | 1/5 (20%) | 0/21 (0%) | 1/15 (7%) | 0/6 (0%) | 1/2 (50%) |
| 3+ | 0/5 (0%) | 0/21 (0%) | 0/15 (0%) | 0/6 (0%) | 0/2 (0%) |
| 4+ | 1/5 (20%) | 0/21 (0%) | 0/15 (0%) | 0/6 (0%) | 0/2 (0%) |
| Not available | 0/5 (0%) | 0/21 (0%) | 0/15 (0%) | 0/6 (0%) | 0/2 (0%) |

Continued on following page.
Table 11: Effective Outcomes, Hemodynamic Results<sup>1</sup> (Model 6900), Continued

| Hemodynamic | | | Results By Valve Size | | |
|---|---|---|---|---|---|
| Parameter | 25 mm | 27 mm | 29 mm | 31 mm | 33 mm |
| 1 to 2 Year Post-Implan | t Interval (n = 131, 114 MVR <sup>2</sup> | and 17 DVR <sup>3</sup> ) | | | |
| Mean gradient <sup>4</sup> | n=3 | n = 40 | n = 47 | n = 27 | n = 4 |
| • mean ± sd | 5.2 ± 0.7 | 4.1 ± 1.6 | 3.5 ± 1.8 | 3.1 ± 1.4 | 2.1 ± 0.5 |
| • min, max | 4.7,6 | 1,7 | 1,10 | 1,7 | 1.5, 2.7 |
| E0A <sup>5</sup> | n = 2 | n=35 | n = 46 | n = 29 | n = 5 |
| • mean ± sd | 1.8 ± 0.4 | 2.3 ± 0.6 | 2.6 ± 0.5 | 2.6 ± 0.7 | 2.5 ± 0.5 |
| • min, max | 1.5, 2.0 | 1.2, 3.5 | 1.1, 3.7 | 1.1, 3.7 | 2.1, 3.2 |
| Regurgitation <sup>6</sup> | n=4 | n = 42 | n = 51 | n = 29 | n = 5 |
| 0 | 2/4 (50%) | 31/42 (74%) | 36/51 (71%) | 17/29 (59%) | 3/5 (60%) |
| 1+ | 1/4 (25%) | 9/42 (21%) | 11/51 (21%) | 8/29 (27%) | 1/5 (20%) |
| 2+ | 1/4 (25%) | 2/42 (5%) | 4/51 (8%) | 2/29 (7%) | 1/5 (20%) |
| 3+ | 0/4 (0%) | 0/42 (0%) | 0/51 (0%) | 2/29 (7%) | 0/5 (0%) |
| 4+ | 0/4 (0%) | 0/42 (0%) | 0/51 (0%) | 0/29 (0%) | 0/5 (0%) |
| Not available | 0/4 (0%) | 0/42 (0%) | 0/51 (0%) | 0/29 (0%) | 0/5 (0%) |
| 5 Year Post-Implant Int | erval ( $n = 11, 9 MVR^2$ and $2 D$ | VR <sup>3</sup> ) | | | |
| Mean gradient <sup>4</sup> | n=0 | n = 6 | n = 5 | n = 0 | n = 0 |
| • mean ± sd | N/A | 8.8 ± 8.1 | 5.1 ± 2.3 | N/A | N/A |
| • min, max | N/A | 4, 25 | 3, 8 | N/A | N/A |
| E0A <sup>5</sup> | n=0 | n = 2 | n = 4 | n = 0 | n = 0 |
| • mean ± sd | N/A | 2.0 ± 1.5 | $2.9 \pm 0.6$ | N/A | N/A |
| • min, max | N/A | 1.0, 3.1 | 2.1, 3.5 | N/A | N/A |
| Regurgitation <sup>6</sup> | n=0 | n = 6 | n = 5 | n = 0 | n = 0 |
| 0 | 0/0 (0%) | 4/6 (66%) | 2/5 (40%) | 0/0 (0%) | 0/0 (0%) |
| 1+ | 0/0 (0%) | 1/6 (17%) | 3/5 (60%) | 0/0 (0%) | 0/0 (0%) |
| 2+ | 0/0 (0%) | 1/6 (17%) | 0/5 (0%) | 0/0 (0%) | 0/0 (0%) |
| 3+ | 0/0 (0%) | 0/6 (0%) | 0/5 (0%) | 0/0 (0%) | 0/0 (0%) |
| 4+ | 0/0 (0%) | 0/6 (0%) | 0/5 (0%) | 0/0 (0%) | 0/0 (0%) |
| Not available | 0/0 (0%) | 0/6 (0%) | 0/5 (0%) | 0/0 (0%) | 0/0 (0%) |

#### Notes:

- 1. Hemodynamic evaluations were performed using transthoracic echocardiography (TTE) and in some cases, transesophageal echocardiography (TEE).
- 2. MVR = mitral valve replacement
- 3. DVR = double valve replacement
- Mean gradient in mmHg
- EOA: Effective Orifice Area, cm<sup>2</sup>
- 6. Regurgitation = none, 0; mild, 1+; moderate, 2+; moderate/severe, 3+; severe, 4+

Table 12: Effectiveness Outcomes, Hemodynamic Results (Model 6900P)<sup>1</sup>

| Hemodynamic | | | Results By Valve Size | | |
|---|---|---|---|---|---|
| Parameter | 25 mm | 27 mm | 29 mm | 31 mm | 33 mm |
| Discharge/Early Post-Impla | nt | | | | |
| Mean gradient <sup>2</sup> | n = 24 | n=35 | n = 83 | n = 42 | n = 16 |
| • mean ± sd | 6.4 ± 1.87 | 4.4 ± 1.52 | 3.4 ± 1.47 | 3.3 ± 1.20 | 4.0 ± 1.38 |
| • min, max | 3,10 | 1.96, 8 | 1.4, 9 | 1,7 | 1.5, 6.91 |
| EOA3 | n=8 | n = 27 | n=77 | n = 41 | n = 16 |
| • mean ± sd | 2.7 ± 0.87 | 2.8 ± 0.58 | 2.9 ± 0.93 | 2.5 ± 0.67 | 2.4 ± 0.52 |
| • min, max | 1.46, 4.4 | 1.5, 3.9 | 1.58, 6 | 1.32, 4.2 | 1.55, 3.31 |
| Regurgitation <sup>4</sup> | n = 27 | n=37 | n = 83 | n = 43 | n = 17 |
| Trivial / None | 19/27 (70%) | 29/37 (78%) | 76/83 (92%) | 39/43 (91%) | 15/17 (88%) |
| 1+ Mild | 6/27 (22%) | 7/37 (19%) | 7/83 (8%) | 4/43 (9%) | 1/17 (6%) |
| 2+ Moderate | 1/27 (4%) | 1/37 (3%) | 0/83 (0%) | 0/43 (0%) | 0/17 (0%) |
| 3+ Moderate/Severe | 0/27 (0%) | 0/37 (0%) | 0/83 (0%) | 0/43 (0%) | 1/17 (6%) |
| 4+ Severe | 0/27 (0%) | 0/37 (0%) | 0/83 (0%) | 0/43 (0%) | 0/17 (0%) |
| Not available | 1/27 (4%) | 0/37 (0%) | 0/83 (0%) | 0/43 (0%) | 0/17 (0%) |
| 3 to 6 Month Post-Implant I | Interval | | | | |
| Mean gradient <sup>2</sup> | n=0 | n = 4 | n=3 | n = 2 | n = 0 |
| • mean ± sd | 0 ± 0 | 4.4 ± 2.25 | 2.3 ± 0.89 | 6.6 ± 2.05 | 0 ± 0 |
| • min, max | 0, 0 | 2.5, 7.5 | 1.3, 3 | 5.1, 8 | 0, 0 |
| EOA <sup>3</sup> | n = 0 | n=3 | n=3 | n = 1 | n = 1 |
| • mean ± sd | 0 ± 0 | 2.4 ± 0.74 | 3.2 ± 0.88 | 2.5 ± 0.00 | 1.2 ± 0.00 |
| • min, max | 0, 0 | 1.6, 3 | 2.3, 4.05 | 2.47, 2.47 | 1.22, 1.22 |
| Regurgitation <sup>4</sup> | n = 0 | n = 5 | n=3 | n = 2 | n=2 |
| Trivial / None | 0 | 3/5 (60%) | 2/3 (67%) | 2/2 (100%) | 2/2 (100%) |
| 1+ Mild | 0 | 1/5 (20%) | 1/3 (33%) | 0/2 (0%) | 0/2 (0%) |
| 2+ Moderate | 0 | 1/5 (20%) | 0/3 (0%) | 0/2 (0%) | 0/2 (0%) |
| 3+ Moderate/Severe | 0 | 0/5 (0%) | 0/3 (0%) | 0/2 (0%) | 0/2 (0%) |
| 4+ Severe | 0 | 0/5 (0%) | 0/3 (0%) | 0/2 (0%) | 0/2 (0%) |
| Not available | 0 | 0/5 (0%) | 0/3 (0%) | 0/2 (0%) | 0/2 (0%) |

Continued on following page.

Table 12: Effectiveness Outcomes, Hemodynamic Results (Model 6900P)<sup>1</sup>, Continued

| Hemodynamic | | | Results By Valve Size | | |
|---|---|---|---|---|---|
| Parameter | 25 mm | 27 mm | 29 mm | 31 mm | 33 mm |
| 1 Year Post-Implant Interval | | | | | |
| Mean gradient <sup>2</sup> | n = 16 | n = 27 | n = 63 | n=34 | n = 15 |
| • mean ± sd | 5.9 ± 2.36 | 4.0 ± 1.45 | 3.0 ± 1.61 | 3.3 ± 1.26 | 3.4 ± 1.25 |
| • min, max | 3, 12 | 2,7 | 1,12 | 1.5, 7 | 1.9, 6.3 |
| E0A3 | n=3 | n = 21 | n = 59 | n=32 | n = 15 |
| • mean ± sd | 2.3 ± 0.16 | 2.4 ± 0.76 | 2.6 ± 0.74 | 2.5 ± 0.67 | 2.3 ± 0.83 |
| • min, max | 2.09, 2.4 | 1.27, 4.76 | 1.5, 5.7 | 1.5, 4 | 1.2, 3.8 |
| Regurgitation <sup>4</sup> | n = 20 | n = 28 | n = 65 | n=34 | n = 16 |
| Trivial / None | 17/20 (85%) | 24/28 (86%) | 53/65 (82%) | 29/34 (85%) | 13/16 (81%) |
| 1+ Mild | 3/20 (15%) | 3/28 (11%) | 6/65 (9%) | 3/34 (9%) | 3/16 (19%) |
| 2+ Moderate | 0/20 (0%) | 0/28 (0%) | 3/65 (5%) | 2/34 (6%) | 0/16 (0%) |
| 3+ Moderate/Severe | 0/20 (0%) | 0/28 (0%) | 1/65 (2%) | 0/34 (0%) | 0/16 (0%) |
| 4+ Severe | 0/20 (0%) | 0/28 (0%) | 0/65 (0%) | 0/34 (0%) | 0/16 (0%) |
| Not available | 0/20 (0%) | 1/28 (4%) | 2/65 (3%) | 0/34 (0%) | 0/16 (0%) |

#### Notes:

- 1. Hemodynamic evaluations were performed using transthoracic echocardiography (TTE) and in some cases, transesophageal echocardiography (TEE).
- Mean gradient in mmHg
   EOA: Effective Orifice Area, cm<sup>2</sup>
- 4. Regurgitation = Trivial/none, 0; mild, 1+; moderate, 2+; moderate/severe, 3+; severe, 4+

## Français

# Bioprothèse mitrale péricardique d'Edwards, modèle 11000M

## Mode d'emploi

ATTENTION : dispositif expérimental. Limité à une utilisation expérimentale en vertu des lois fédérales (États-Unis).

AVERTISSEMENT : dispositif expérimental. Exclusivement à des fins de recherche clinique.

Avertissement : dispositif expérimental. Utilisation limitée à la recherche. Pour une utilisation par des (médecins) chercheurs qualifiés uniquement.

## 1. Description du dispositif et des accessoires

#### 1.1 Description du dispositif

La bioprothèse mitrale péricardique d'Edwards, modèle 11000M, est une bioprothèse trivalve composée d'un péricarde bovin traité installé sur une structure flexible. Elle est disponible dans les tailles suivantes : 25, 27, 29, 31 et 33 mm (tableau 1). Elle est conservée dans un emballage non aqueux et ne nécessite pas de rincage avant l'implantation.

Le fil métallique est fait d'un alliage de chrome-cobalt recouvert d'un matériau tissé en polyester. Une bande laminée en alliage de chrome-cobalt et film en polyester entoure la base de la structure en fil métallique.

Un anneau de suture gaufré en silicone, qui est couvert d'un tissu poreux en polytétrafluoroéthylène (PTFE), est attaché à la structure en fil métallique. L'anneau de suture est crénelé sur sa partie antérieure. Les marqueurs de suture en soie noire de la partie antérieure contribuent à orienter la bioprothèse et à éviter que la voie d'évacuation du ventricule droite ne soit obstruée par un montant.

L'anneau de suture est encerclé par une ligne de guidage de suture en soie noire. L'utilisation de cette ligne pour positionner les sutures à travers l'anneau de suture et dans la région sur la partie externe de l'anneau de suture facilite la pénétration de l'aiguille et donne une compliance variable. Les cellules du gaufrage sont plus larges dans la partie postérieure, là où les calcifications et les irrégularités de l'anneau mitral d'origine sont plus fréquentes (réf. 6).

#### HVT63 25 27 29 31 33 Taille mm mm mm mm mm A. Diamètre de l'endoprothèse 25 27 29 31 31 (fil métallique, mm) B. Diamètre de l'anneau tissulaire 28 29.5 31.5 33.5 33.5 C Diamètre du montant de l'endoprothèse externe 29 31 34 35 35 (embout mm) D. Diamètre de l'anneau de suture 36 38 40 42 externe (en mm) E. Profil effectif antérieur (mm) 7 7.5 ጸ 8.5 8.5 F. Profil effectifpostérieur (mm) 10 10.5 11 11.5 11.5 G. Hauteur profil total (mm) 15 18 Surface de l'orifice (en mm<sup>2</sup>) 474 499 580 653 653

#### 1.2 Description des accessoires

Tableau 1 Dimensions nominales

Les accessoires pouvant être utilisés avec la bioprothèse 11000M sont les suivants :

- Système de support Tricentrix
- Calibreur pour réplique 1173R
- Calibreur pour porteuse 1173B
- Plateau de stérilisation fourni avec le modèle SET1173
- Modèles de poignée 1111, 1117, 1173 et 1126 (pour utilisation unique)

Tous les accessoires sont vendus non stériles, sauf le système de support Tricentrix qui est fixé à la bioprothèse stérile et la poignée 1126 qui est réservée à une utilisation unique.

#### Calibreurs et plateau

Seuls les calibreurs 1173B (figure 1a) et 1173R (figure 1b) peuvent être employés avec la bioprothèse 11000M.

Attention: pour calibrer la bioprothèse 11000M, ne pas utiliser de calibreurs de valves d'autres fabricants ou d'autres prothèses de valves d'Edwards Lifesciences.

N'utiliser que les calibreurs 1173B ou 1173R pour définir la taille à employer pour la bioprothèse 11000M. Les calibreurs 1173B et 1173R permettent de constater immédiatement si la prothèse s'adapte à l'anneau et sont proposés pour chaque taille de bioprothèse 11000M. Le corps des calibreurs 1173B et 1173R indique le diamètre de l'endoprothèse à la base. Grâce à sa partie antérieure crénelée et à ses marqueurs noirs, la lèvre du calibreur 1173R reproduit l'anneau de suture de

Edwards Lifesciences, le logo E stylisé, Edwards, Carpentier-Edwards, Tricentrix, PERIMOUNT, PERIMOUNT Magna, PERIMOUNT Plus, TFX et Magna Mitral Ease sont des marques de commerce d'Edwards Lifesciences Corporation.

la bioprothèse et permet de déterminer les résultats de la suture ou des techniques de préservation de l'appareil sous-valvulaire.

Les calibreurs 1173B et 1173B portent une étiquette indiquant la taille de la bioprothèse. La trousse complète de calibreurs se trouve dans un plateau, modèle SET1173. qui peut être réutilisé et restérilisé.



#### Système de support Tricentrix et poignées

L'ensemble de poignée et support est constitué de deux composants : le système de support Tricentrix (figure 2) monté sur la bioprothèse 11000M, et une poignée (1111, 1117, 1173 ou 1126) fixée au système de support Tricentrix lors de l'opération chirurgicale.



Les poignées suivantes (tableau 2) peuvent être utilisées avec la bioprothèse 11000M.

| 1 | Tableau 2. Poignées accessoires | | | | |
|---|---|---|---|---|---|
| | | | Longue | | |
| | Modèle | Matériau de l'axe | pouces | cm | Réutilisable |
| | 1111 | Acier inoxydable | 7,0 | 17,8 | Oui |
| | 1117 | Nitinol | 9,1 | 23,2 | Oui |
| | 1126 | Acier inoxydable | 11,5 | 29,2 | Non |
| | 1173 | Nitinol | 11,3 | 28,6 | Oui |

Les poignées équipées d'un axe en nitinol sont plus souples que celles en acier inoxydable. Lors de chaque cycle de stérilisation, elles redeviennent droites, ce qui facilite leur fixation au support.

## 2. Mode d'emploi

La bioprothèse mitrale péricardique d'Edwards, modèle 11000M, est destinée aux patients dont il faut remplacer la valve mitrale d'origine ou prothétique.

#### 3. Contre-indications

Ne pas utiliser la bioprothèse si le chirurgien estime que son utilisation est contraire à l'intérêt du patient. La décision finale à ce propos relève du chirurgien qui doit évaluer tous les risques impliqués, y compris l'anatomie et la pathologie observées au moment de l'opération chirurgicale.

## 4. Mises en garde

POUR UTILISATION UNIQUE SEULEMENT. Ce dispositif est conçu, destiné et distribué pour une utilisation unique seulement. Ne pas restériliser ou réutiliser ce dispositif. Aucune donnée n'existe pour corroborer le caractère stérile, la non-pyrogénicité et la fonctionnalité du dispositif après le processus de restérilisation. La bioprothèse et l'emballage deviendront inutilisables en cas d'exposition à des radiations, à la vapeur, à l'oxyde d'éthylène ou à d'autres agents chimiques de stérilisation.

NE PAS CONGELER NI EXPOSER LA BIOPROTHÈSE À UNE CHALEUR EXTRÊME. L'exposition de la bioprothèse à des températures extrêmes rendra le dispositif inutilisable.

## NE PAS UTILISER la bioprothèse :

- si le sachet métallisé, les plateaux scellés ou les lèvres sont ouverts, endommagés ou tachés;
- si la date d'expiration est passée;
- si elle est tombée, endommagée ou mal manipulée de quelle que façon que ce soit. Si une bioprothèse est endommagée lors de l'insertion, ne pas tenter de la réparer.

NE PAS EXPOSER la bioprothèse à des solutions, des produits chimiques, des antibiotiques, etc., à l'exception de solutions salines physiologiques. Le tissu de la valve peut comporter des dommages irréparables non apparents lors d'une inspection visuelle.

NE PAS SAISIR le tissu de la valve de la bioprothèse avec des instruments ni endommager la bioprothèse. Même la plus petite perforation du tissu de la valve peut s'agrandir à terme et compromettre gravement son fonctionnement.

NE PAS CHOISIR UNE TAILLE SUPÉRIEURE. Le choix d'une taille supérieure peut entraîner des dommages à la bioprothèse ou un stress mécanique localisé, susceptible de blesser le cœur ou de causer une panne du tissu de la valve, une distorsion de l'endoprothèse ou une réqurqitation du tissu de la valve.

NE PAS PASSER, à travers la bioprothèse, des cathéters, des sondes électrodes transveineuses ou d'autres instruments chirurgicaux autres qu'un miroir servant à vérifier le positionnement des montants et des sutures. Les autres dispositifs risquent d'endommager le tissu de la valve.

Comme pour tout dispositif médical implanté, il existe un risque de réponse d'immunisation de la part du patient. Certains composants du modèle 11000M sont en alliage contenant du cobalt, du chrome, du nickel, du molybdène, du manganèse, du carbone, du béryllium et du fer. Il faut prendre des précautions avec les patients souffrant d'hypersensibilité à ces matières. Ce dispositif ne contient pas de latex mais peut avoir été fabriqué dans un environnement qui en contient.

#### 5. Évènements indésirables

#### 5.1 Évènements indésirables observés

Comme pour toutes les valves cardiaques prothétiques, des évènements indésirables graves pouvant parfòs aller jusqu'a udécès peuvent survenir. En outre, des évènements indésirables découlant de la réaction du patient au dispositif implanté ou encore d'une modification physique ou chimique de ses composants, plus particulièrement de ceux dont l'origine est biologique, peuvent survenir à des intervalles variables (allant de plusieurs heures à plusieurs jours) et nécessitent une nouvelle opération pour remplacer la prothèse.

La conception de la bioprothèse mitrale péricardique d'Edwards, modèle 11000M, est similaire à celle des bioprothèses péricardiques PERIMOUNT Magna Mitral Ease du modèle 7300TFX de Carpentier-Edwards.

Trois (3) essais cliniques multicentre prospectifs non randomisés ont été effectués hors des États-Unis avec la bioprothèse mitrale péricardique 6900. Sur l'ensemble des patients, trois cent un (301) ont subi un remplacement isolé de la valve mitrale (RVM) tandis que 62 subissaient un double remplacement valvulaire (DRV), la valve aortique étant remplacée par une bioprothèse aortique péricardique PERIMOUNT de Carpentier-Edwards.

Les bioprothèses ont été implantées de 1984 à 1986 dans la première étude, de 1988 à 1994 dans la deuxième et de 1996 à 1997 dans la troisième. Les patients ont été évalués avant l'opération, pendant l'opération, à la sortie, après 1 an et tous les ans par la suite.

Le tableau 3 présente les taux observés d'évènements précoces (≤ 30 jours pour les évènements indésirables en lien avec la valve), le taux linéarisé pour les évènements tardifs (> 30 jours postopératoires) et les taux actuariels d'évènements indésirables 1, 5 et 8 ans après l'opération pour le modèle 6900. Les taux d'évènements indésirables concernaient 363 patients de neuf centres. Le suivi cumulatif était de 1 100 patient-années, avec une moyenne de suivi de 3 années (écart-type = 2,4 années, intervalle = 0 à 8,2 ans). Les données démographiques des patients en période préopératoire et opératoire sont présentées dans les tableaux 5 et 7. Les résultats en matière d'efficacité sont présentées dans les tableaux 9 et 11.

Un (1) essai clinique multicentre prospectif non randomisé a été effectué à l'échelon international auprès de patients ayant reçu la bioprothèse mitrale péricardique PERIMOUNT 6900P de Carpentier-Edwards. Sur l'ensemble des patients, cent soixante-quinze (175) ont subi un remplacement isolé de la valve mitrale (RVM) tandis que trente-quatre (34) subissaient un double remplacement (DRV), la valve aortique étant remplacée par une bioprothèse aortique péricardique PERIMOUNT de Carpentier-Edwards. Dans cette étude, les bioprothèses ont été implantées de 1999 à 2007. Les patients étaient évalués pendant la période péropératoire et à la

sortie, après 1 an et chaque année par la suite. Les évènements indésirables ont été consignés tout au long de la période postopératoire. Le tableau 4 présente les taux observés d'évènements précoces (< 30 jours pour les évènements indésirables en lien avec la valve), le taux linéarisé pour les évènements tardifs (> 30 jours postopératoires) et les taux actuariels d'évènements indésirables 1 et 5 ans après l'opération pour le modèle 6900P. Les taux d'évènements indésirables concernaient deux cent neuf (209) patients de sept centres. Le suivi cumulatif était de 873, 18 patient-années, avec une moyenne de suivi de 4,2 années (écart-type = 2,3 années, intervalle = 0 à 8,2 ans). Les données démographiques des patients en période préopératoire et opératoire sont présentées dans les tableaux 6 et 8. Les résultats en matière d'efficacité sont présentée dans les tableaux 10 et 12.

#### 5.2 Évènements indésirables potentiels

Les évènements indésirables potentiels associés à l'utilisation de biovalves cardiaques prothétiques sont les suivants :

- Angine de poitrine
- Diathèse hémorragique (coagulopathie) en lien avec l'anticoagulothérapie
- Arythmie cardiague
- · Blocage de la valve ostiale coronaire
- Endocardite
- Insuffisance cardiague
- Hémolyse
- Anémie hémolytique
- Hémorragie
- Infection locale et systémique
- · Infarctus du myocarde
- Inadaptation de la prothèse au patient
- · Enclavement de la valve prothétique (coincement)
- · Dysfonction non structurelle de la prothèse
- · Pannus de la prothèse
- Fuite périvalvulaire de la prothèse
- Régurgitation de la prothèse
- · Détérioration de la structure de la prothèse
- Thrombose prothétique
- Accident vasculaire cérébral
- · Thrombo-embolie
- Insuffisance cardiague congestive

Ces complications peuvent avoir les conséquences suivantes :

- Nouvelle opération chirurgicale
- Explantation
- Handicap permanent
- Décès

Voici les autres évènements indésirables en lien avec l'utilisation des bioprothèses mitrales péricardiques PERIMOUNT 6900 de Carpentier-Edwards tirés de la documentation et des rapports issus du système de destion des

plaintes d'Edwards Lifesciences : sténose, régurgitation par une valve insuffisante, perforation du ventricule par les montants de l'endoprothèse, dysfonction de la valve découlant d'une déformation de l'implant et rupture de la structure métallique.

## 6. Études cliniques

Les indicateurs de sécurité mentionnés dans les études prospectives correspondent aux évènements indésirables. Des analyses sanguines ont été utilisées pour confirmer l'absence ou la présence de certains évènements indésirables. Les résultats concernant la sécurité sont détaillés dans le tableau 3 pour le modèle 6900 et dans le tableau 4 pour le modèle 6900P. Les données démographiques préopératoires sont détaillées dans le tableau 5 pour le modèle 6900P. Les données démographiques préopératoires sont détaillées dans le tableau 6 pour le modèle 6900P. Les données démographique pératoires sont détaillées dans le tableau 7 pour le modèle 6900 et dans le tableau 9 pour le modèle 6900P. Les indicateurs d'efficacité correspondent à la classification fonctionnelle de la New York Heart Association (NYHA), résumée dans le tableau 9 pour le modèle 6900 et dans le tableau 10 pour le modèle 6900P, et aux évaluations échocardiographiques résumées dans le tableau 11 pour le modèle 6900 et dans le tableau 12 pour le modèle 6900 et dans

Il n'existe aucune donnée clinique démontrant la résistance accrue à la calcification de la bioprothèse mitrale péricardique d'Edwards, modèle 11000M, par rapport aux autres bioprothèses du marché.

## 7. Individualisation du traitement

Sauf indication contraire, les destinataires de la valve bioprothétique doivent suivre une anticoagulothérapie pendant les premiers stades suivant l'implantation, selon les consignes données à chacun par le médecin. Une anticoagulothérapie ou un traitement antiplaquettaire à long terme doit être envisadé pour les patients montrant des facteurs de risque de thrombo-embolie.

Le jugement final concernant les soins pour un patient donné doit être pris par le fournisseur de santé et le patient à la lumière de l'ensemble de la situation que présente ce dernier (réf. 7). Il est recommandé de poser une bioprothèse en cas de RVA sur des patients de tous âges qui ne prennent pas de warfarine ou pour lesquels il existe une contre-indication importante à la thérapie à base de warfarine. Les préférences du patient sont également à prendre en compte dans une mesure raisonnable lors du choix de l'opération de la valve mitrale et de la valve prothétique. Il est raisonnable d'envisager l'implantation d'une prothèse mécanique pour un RVA de patients de moins de 65 ans pour lesquels l'anticoagulation n'est pas contre-indiquée. Il est également raisonnable d'envisager l'implantation d'une bioprothèse pour un RVA de patients de moins de 65 ans qui ont fait ce choix pour des raisons de mode de vie après avoir été informés dans les détails des risques de l'anticoagulation par rapport à l'éventuelle nécessité d'un deuxième RVA (réf. 7).

#### 7.1 Populations de patients spécifiques

L'innocuité et l'efficacité de la bioprothèse, modèle 11000M, n'ont pas été établies pour les populations suivantes, sur les guelles elles n'ont pas été étudiées :

- patientes enceintes ;
- · mères qui allaitent;
- patients métabolisant le calcium de manière anormale (p. ex., insuffisance rénale, hyperparathyroïdisme);
- patients présentant une insuffisance dégénérative anévrismale de l'aorte (p. ex., nécrose médiale kystique, syndrome de Marfan);
- · enfants, adolescents et jeunes adultes.

Attention: Selon des rapports issus de documentation sur des valves tissulaires (réf. 9, 10, 11, 12 et 13), la fréquence des calcifications de la valve serait supérieure chez les patients de moins de 20 ans. Lorsque cela est possible, il faut

éviter les injections intraveineuses répétées contenant du calcium pendant la période postopératoire. Parallèlement, la consommation excessive de lait ou de produits laitiers doit être évitée chez l'enfant. À cet égard, les recherches effectuées sur les animaux (réf. 14) démontrent qu'un niveau élevé de calcium dans le système peut entraîner une calcification précoce.

## 8. Informations et conseils au patient

Il est conseillé de procéder à un suivi sérieux et continu (au moins par une visite annuelle chez le médecin) afin que les complications liées à la bioprothèse, et plus particulièrement aux problèmes de matériau, puissent faire l'objet d'un diagnostic et d'un traitement adaptés. Les patients porteurs de bioprothèses sont vulnérables à la bactériémie (p. ex., lors de procédures dentaires) et doivent recevoir des conseils concernant l'antibioprophylaxie. Enfin, il faut encourager les patients à porter en permanence leur carte d'identification et à informer les fournisseurs dont ils sollicitent des soins qu'ils possèdent un implant.

#### 9. Présentation

#### 9.1 Conditionnement

La bioprothèse mitrale péricardique d'Edwards, modèle 11000M, est stérile et non pyrogène. Elle est livrée dans un emballage de plateau à double barrière placé dans un sachet métallisé. se trouvant lui-même dans un carton.

Chaque bioprothèse se trouve dans un carton avec un indicateur de température visible à travers une fenêtre sur le panneau latéral. Cet indicateur vise à repérer les produits exposés à des températures extrêmes transitoires. À la réception de la bioprothèse, inspecter immédiatement l'indicateur et consulter l'étiquette du carton pour confirmer l'état « Utiliser ». Si l'état « Utiliser » n'est pas apparent, ne pas se servir de la bioprothèse et contacter le fournisseur local ou le représentant d'Edwards Lifesciences pour organiser une autorisation de retour et un remplacement.

Mise en garde: inspecter soigneusement la bioprothèse avant l'implantation pour trouver des traces d'exposition à des températures extrêmes ou d'autres dégâts.

#### 9.2 Stockage

La bioprothèse mitrale péricardique d'Edwards, modèle 11000M, doit être entreposée à une température comprise entre 10 °C et 25 °C (50 °F et 77 °F), dans son sachet métallisé et son carton de rangement.

#### 10. Directives d'utilisation

#### 10.1 Formation du médecin

Les techniques d'implantation de cette bioprothèse sont semblables à celles du placement d'une bioprothèse mitrale avec endoprothèse. Aucune formation particulière n'est nécessaire pour implanter la bioprothèse mitrale péricardique d'Edwards, modèle 11000M.

#### 10.2 Choix de la taille

Attention: pour calibrer la bioprothèse 11000M, ne pas utiliser de calibreurs de valves d'autres fabricants ou d'autres prothèses de valves d'Edwards Lifesciences.

Attention : vérifier si les calibreurs et les poignées contiennent des traces d'usure comme des ternissures, des fissurations ou des craquelures.
Remplacer le calibreur ou la poignée en cas de détériorations.

Mise en garde : les fragments des poignées et des calibreurs ne sont pas radio-opaques et ne peuvent pas être détectés par un imageur externe.

Vérifier que les accessoires ont été stérilisés conformément aux recommandations fournies avec les articles réutilisables.

Les marques noires sur la lèvre reproduisent les marqueurs noirs de l'anneau de suture. Elles délimitent la partie antérieure de l'anneau de suture de la bioprothèse, qui doit être positionnée en face de la partie de l'anneau d'origine située entre les commissures de manière à enjamber la région de la voie d'évacuation du ventricule gauche. Sur le calibreur pour la réplique 1173R, la hauteur et l'emplacement des montants de l'endoprothèse sont marqués de manière à faciliter l'alignement et le bon positionnement.

Les calibreurs sont équipés de poignées déjà fixées dont la longueur est augmentée pour un meilleur accès en cas d'exposition difficile, pour les patients ayant une cage thoracique profonde et pour permettre une procédure moins invasive. La manière dont l'arrière de la poignée est fixée au calibreur permet d'avoir une vue dégagée du ventricule à travers le corps afin de mieux évaluer les structures sous-valvulaires. Les calibreurs 1173B et 1173R portent une étiquette indiquant la taille de la bioprothèse.

| Étape | Procédure |
|---|---|
| 1 | Choix de la taille à l'aide du calibreur pour porteuse<br>1173B :<br>Pour choisir la taille à l'aide du calibreur pour porteuse 1173B,<br>passer son corps à travers l'anneau mitral. Vérifier qu'il repose<br>directement sur la partie plane de l'anneau. |
| 2 | Choix de la taille à l'aide du calibreur pour réplique<br>1173R :<br>Pour choisir la taille à l'aide du calibreur pour réplique 1173R,<br>passer son corps à travers l'anneau mitral de manière à ce que<br>l'embout du calibreur, qui reproduit l'anneau de suture de la<br>bioprothèse, repose sur la partie supérieure de l'anneau mitral.<br>HVT61 |

Certaines techniques, comme l'utilisation de petites compresses, l'enroulement de la valve ou la préservation de l'appareil mitral sous-valvulaire peuvent également réduire la taille de l'anneau mitral et permettre le choix d'une bioprothèse plus petite (réf. 8). Lors de l'utilisation de ces techniques, il est conseillé de réviser la taille de l'anneau pour éviter de choisir une bioprothèse trop grande. Le rendement constant des bioprothèse mitrales péricardiques d'Edwards, modèle 11000M, évite de devoir choisir une taille supérieure pour obtenir le rendement hémodynamique recherché chez la plupart des patients (tableaux 11 et 12).

Il peut arriver que la membrure, qui est élastique, soit étirée par le système de support Tricentrix au cours de l'implantation. Elle se rétractera alors autour du montant lorsque le support sera retiré, coinçant ainsi les valves et génant leur fonctionnement. Les calibreurs 1173B et 1173B sont faits d'un matériau transparent qui permet de voir l'appareil sous-valvulaire au cours du choix de la taille. Veiller à ce qu'aucune membrane ne gêne le passage des montants.

Attention : faire preuve d'une attention toute particulière lors du recours à des techniques de préservation de l'appareil sous-valvulaire, afin d'éviter que la membrane ne se coince dans un montant.

Mise en garde: éviter de choisir une bioprothèse trop grande. Le choix d'une taille supérieure peut entraîner des dommages à la bioprothèse ou un stress mécanique localisé, susceptible de blesser le cœur ou de causer une panne du tissu de la valve, une distorsion de l'endoprothèse ou une réquigitation du tissu de la valve.

#### 10.3 Instructions de manipulation et de préparation

Il est conseillé de suivre une formation sur le tas avant de manipuler et de préparer la bioprothèse mitrale péricardique d'Edwards, modèle 11000M.

| Étape | Procédure |
|---|---|
| 1 | Attention : ne pas ouvrir pas l'emballage de la<br>bioprothèse mitrale péricardique d'Edwards, modèle<br>11000M, avant d'avoir l'assurance que l'implantation<br>aura lieu. |
| | Mise en garde : Ne pas ouvrir le sachet métallisé dans<br>une zone stérile. Ce sachet ne sert qu'à protéger la<br>bioprothèse. Seul l'emballage le plus à l'intérieur peut<br>pénétrer dans la zone stérile. |
| | Une fois que la bonne taille de bioprothèse a été choisie, retirer<br>le sachet métallisé du carton dans la zone non stérile. Avant<br>d'ouvrir, examiner l'emballage pour vérifier s'il y a des<br>dommages et des scellés cassés ou manquants. |
| 2 | Près de la zone stérile, tenir la base du plateau extérieur et retirer son couvercle. |
| 3 | Le plateau intérieur et son contenu sont stériles. Transférer le<br>plateau interne sur la zone stérile. Il faut manipuler le contenu du<br>plateau intérieur en recourant à une technique chirurgicale<br>stérile afin d'éviter la contamination. |
| | HVT26 |

| Étape | Procédure | | Étape | Procédure |
|---|---|---|---|---|
| 4 | d'avoir l'assurance que l'implantation a ura lieu et que<br>le chirurgien est prêt à mettre la valve en place. | | | Attention : il faut éviter d'enchevêtrer l'étiquette avec<br>le numéro de série dans la poignée lors de la fixation.<br>Attention : l'ensemble poignée-support est indispensable |
| | Attention : la bioprothèse n'est pas fixée sur le plateau<br>intérieur. Il faut faire attention en ouvrant le couvercle<br>et en tirant sur le couvercle en plastique. | L | | pour l'implantation et ne doit pas être retiré jusqu'à ce<br>que la bioprothèse soit suturée sur l'anneau mitral. |
| | Avant d'ouvrir, examiner le plateau intérieur et le couvercle<br>pour vérifier s'il y a des dommages, des tâches et des scellés<br>cassés ou manquants. Tenir la base du plateau intérieur et<br>retirer son couvercle. | | 7 | Une fois la poignée fixée, retirer l'ensemble du plateau (cà-d,<br>le manchon de plastique, le clip, le système de support Tricentrix<br>et la bioprothèse). Le manchon de plastique n'est pas solidement<br>fixé au clip. Il se peut qu'il reste sur le plateau. Le déploiement<br>n'en sera pas compromis. |
| 5 | Pour atteindre la bioprothèse, retirer le couverde en plastique en tirant sur les deux languettes. Jeter le couverde en plastique. HAVTSA HAVTS4 | | | Attraper le manchon de plastique ou le clip pour poursuivre la rotation jusqu'à ressentir une résistance, jusqu'à ce que le montant blanc du support soit en position déverrouillée. CP1089-23 Ou CP1089-6 |
| 6 | Fixer la poignée au système de support Tricentrix alors que la bioprothèse repose toujours sur le plateau. Pour cela, insérer la poignée dans le support et la tourner vers la droite jusqu'à sentir une résistance. HVT52 | | | CP1089-8 CP1089-9 Verrouillé Déverrouillé |

Attention : ne pas saisir la bioprothèse avec les mains ou des instruments chirurgicaux.

| Étape | Procédure | Étape | Procédure |
|---|---|---|---|
| 8 | Pousser la poignée jusqu'à ce que le montant blanc du support coulisse face aux valves et s'enclenche en position complètement déployée. Un déclic peut se faire entendre lorsque la position de déploiement est atteinte. (P1089-24 | 11 | Retirer le clip en le faisant glisser hors du support, vers le côté. CP1089-26 |
| 9 | Attention : si la poignée n'est pas suffisamment poussée<br>lors du déploiement du système de support Tricentrix, il<br>se peut que le système échoue à réduire les risques de | | Jeter le manchon et le clip. |
| | coincement de la suture. Toujours vérifier que le déploiement est effectif. Il ne devrait plus exister aucun espace entre l'adaptateur bleu et le support gris. L'ensemble poignée-montant ne devrait plus pouvoir coulisser. Le montant blanc du support devrait dépasser à travers les valves, tandis que les trois commissures devraient être légèrement inclinées vers le centre de la bioprothèse. Le montant blanc du support déployé va plisser les valves de manière temporaire. Lorsque le support sera retiré après l'implantation, elles reprendront leur position normale. HVTS6 | 12 | Une étiquette avec le numéro de série est fixée à l'anneau de suture de chaque bioprothèse par une suture. Ce numéro de série doit être comparé avec le numéro se trouvant sur l'emballage de la bioprothèse et sur la carte de données d'implantation de la bioprothèse. L'étiquette ne doit pas être détachée de la bioprothèse jusqu'à ce que l'implantation soit sûre. Attention: si les numéros de série sont différents, la bioprothèse doit être renvoyée sans avoir été utilisée. Attention: il faut faire attention en coupant ou déchirant le tissu de l'anneau de suture lorsque l'étiquette du numéro de série est retirée. Attention: pour éviter d'endommager le tissu de l'anneau de suture, ne pas tirer sur la suture à travers l'anneau. |
| | | 13 | IL EST INUTILE DE RINCER la bioprothèse mitrale péricardique<br>d'Edwards, modèle 11000M, avant l'implantation.<br>Attention : si la bioprothèse est rincée avant<br>l'implantation, elle doit être ensuite conservée hydratée<br>à l'aide d'une irrigation saline physiologique stérile sur<br>les deux côtés du tissu de la valve pendant toute la durée |
| 10 | Après le déploiement, retirer le manchon (s'il est fixé) en<br>tenant la poignée et en la tirant hors du clip.<br>(P1089-25 | | de la procédure chirurgicale. Il est recommandé de la<br>rincer toutes les une à deux minutes.<br>Attention : éviter que le tissu de la valve entre en<br>contact avec des serviettes, des linges ou d'autres<br>sources de particules susceptibles de s'y transférer. |
| | 7 | | |

## 10.4 Implantation du dispositif

#### Étape Procédure Étape Procédure 2 Orientation adéquate de la bioprothèse : Le chirurgien doit être familier avec les recommandations Attention : le fil métallique de la bioprothèse, modèle concernant la mesure et le positionnement supra-annulaire 11000M, est symétrique, et les trois supports des (voir la section 10.2 Choix de la taille.) commissures (montants) sont équidistants. L'anneau de suture est cependant concu en fonction d'une orientation À cause de la complexité et de la variété du remplacement donnée de la bioprothèse. La partie crénelée de l'anneau chirurgical de la valve cardiague, le choix de la technique de suture, entre les deux protubérances en silicone, doit chirurgicale, correctement modifiée selon les mises en garde être placée face à la partie intercommissurale antérieure décrites précédemment, est à la discrétion du chirurgien de l'anneau et eniamber la région de la voie d'évacuation individuel. En général, les étapes suivantes doivent être suivies : du ventricule gauche. 1. Retirer par chirurgie les valves malades ou endommagées Les marqueurs de suture en contraste de l'anneau de suture ainsi que toutes les structures associées au besoin. indiquent la bonne orientation et la distance type entre les commissures. Cette distance peut cependant varier d'un patient 2. Retirer par chirurgie le calcium de l'anneau afin d'assurer un à l'autre. Sur le côté gauche, deux sutures noires rapprochées bon positionnement de l'anneau de suture de la bioprothèse indiquent où placer le premier point et correspondent à la pour éviter d'endommager le tissu délicat de la valve. commissure antérieure 3. Choisir la bonne taille. Mesurer l'anneau exclusivement à l'aide du calibreur mitral 1173B ou 1173R (figures 1a et 1b). Le côté droit comporte une seule suture noire qui indique l'emplacement approximatif de la commissure postérieure. 4. Bien positionner la prothèse. Lorsque ces guides d'orientation sont utilisés, le troisième montant se positionne naturellement vers le milieu de 5. Nouer les sutures une fois le support en place pour éviter l'emplacement de la valve postérieure. qu'elles ne forment une boucle ou que la membrane ne se coince. Attention : il convient de bien faire attention à ne pas placer un montant en face de la voie d'évacuation du 6. Examiner les valves de la bioprothèse pour repérer les ventricule gauche, car il pourrait compromettre le déformations ou les fuites pouvant être survenues lors de rendement hémodynamique sur le long terme. l'étane précédente 3 Positionnement de la suture : Attention: lors d'un choix d'une bioprothèse, il faut prendre en compte la taille, l'âge et l'état physique par L'anneau de suture est encerclé par une ligne de guidage de rapport à la taille de la bioprothèse, afin de minimiser suture en soie noire. Lors du positionnement des sutures à le risque d'hémodynamique sous-optimale. Toutefois, travers l'anneau de suture, la force de glissement est réduite le choix final revient au médecin après l'évaluation des lorsque les sutures sont placées directement à travers l'anneau risques et des avantages pour le patient. de suture et dans la région, de la ligne de guidage à la partie externe de l'anneau de suture. Attention : il faut éliminer adéquatement les calcifications de l'anneau du patient avant Il faut maintenir une tension sur les sutures pendant que la l'implantation pour éviter que le tissu délicat de la valve bioprothèse est enfoncée dans l'anneau, afin de réduire les bioprothétique ne s'endommage à leur contact. Insérer risques de formation de boucles susceptibles de coincer une le calibreur dans l'anneau mitral. Le corps devrait valve. Une fois les montants d'endoprothèse complètement touiours s'v adapter dans peine. rétractés après la mise en place du système de support

Attention: n'utiliser que des calibreurs 1173B ou 1173R

pour choisir la taille de la bioprothèse. L'emploi d'autres calibreurs peut conduire à un choix non adapté (voir 1.2 Description des accessoires). Comme pour les autres bioprothèses mitrales, l'implantation de la bioprothèse mitrale péricardique d'Edwards, modèle 11000M, s'effectue généralement par la technique de suture discontinue matelassée. Cette technique est recommandée pour choisir la taille de l'anneau après le placement des sutures, ces dernières pouvant réduire la taille de la bioprothèse pouvant être implantée.

Tricentrix, il sera plus facile de guider les sutures vers la position

adaptée derrière les montants et sur l'anneau de suture.

#### Étape Procédure

Retirer la poignée avant de nouer les sutures. La poignée et l'adaptateur bleu doivent être retirés en même temps. Maintenir la position de la bioprotitése dans l'anneau en plaçant délicatement le forceps ou les mains recouvertes de gants sur le support et en coupant le fil vert de l'adaptateur bleu. Retirer l'adaptateur bleu et la poignée en une seule opération.





Attention: éviter d'enrouler ou de coincer une suture autour des cages ouvertes, des montants libres ou des supports de commissures de la bioprothèse, sous peine de compromettre le bon fonctionnement de la valve. Pour réduire les risques d'enroulement des sutures, il est essentiel de laisser le support déployé en place iusau'à ce que tous les nœuds soient faits.

Cependant, si le support gêne la vision du chirurgien, il faut nouer toutes les sutures proches des trois montants du cadre avant de couper les trois fils de fixation du support vert pour enlever le support.

Attention: si les fils de fixation du support déployé sont coupés avant que les sutures adjacentes ne soient nouées, le support n'empêchera plus l'enroulement des sutures autour des montants de la structure.

Il faut bien prendre soin d'éviter de nouer les sutures en haut des coins des tiges grises du support. Avant de nouer chaque suture, examiner les valves tout en tenant les deux brins sous tension. La déformation ou le déplacement des valves pendant cette étape indique que la suture est enroulée autour d'un montant. Il ne faut pas relâcher la tension sur les sutures avant ou après le retrait du support, sous peine de favoriser la formation de boucles et de coincer les sutures. Il est conseiller de passer un miroir chirurgical à travers les valves après le retrait du support afin d'examiner chaque montant ainsi que le nostitionnement des sutures.

Attention: lors de sutures séparées, il est important de les couper près des nœuds et de veiller à ce que le bout exposé n'entre pas en contact avec le tissu de la valve (réf. 8).

#### Étape Procédure

Voici comment retirer le système de support Tricentrix en une seule opération à la fin des sutures :

CP1089-14



- À l'aide d'un scalpel ou de ciseaux placés uniquement dans le canal de coupe, couper chacune des trois (3) sutures vertes exposées. Ne jamais tenter de couper une suture sous un support partiellement détaché, car un fragment pourrait tomber dans le ventricule. Éviter de couper ou d'endommager l'endoprothèse ou le tissu de la valve en même temps que les sutures.
- Après avoir coupé les trois (3) sutures du support, retirer le système de support Tricentrix de la bioprotthèse en une seule opération, en même temps que vous nouez les sutures, en utilisant des gants ou des forceps protégés.
- 3. Après l'implantation, retirer et jeter la baquette.

## 10.5 Nettoyage et stérilisation des accessoires

Les accessoires de la bioprothèse mitrale péricardique d'Édwards, modèle 11000M, sont emballés à part. La poignée du modèle 1126 est stérile et est destinée à un usage unique. Les poignées des modèles 1111, 1117 et 1173 et les calibreurs 11738 et 11738 ne sont pas stériles et doivent être nettoyés et stérilisés avant l'utilisation. Les poignées, les calibreurs, la base et le couvercle du plateau doivent être nettoyés et stérilisés à nouveau avant chaque utilisation. Consulter le mode d'emploi fourni avec les accessoires réutilisables pour connaître les consignes de nettoyage et de stérilisation.

## 10.6 Retour de la bioprothèse

Edwards Lifesciences souhaite obtenir des échantillons cliniques recouverts de la bioprothèse mitrale péricardique d'Edwards, modèle 11000M, à des fins d'analyse. Pour retourner des bioprothèses recouvertes, contacter votre représentant.

- Emballage non ouvert avec la barrière stérile intacte: si le sachet métallisé ou les plateaux n'ont pas été ouverts, retourner la bioprothèse dans son emballage d'origine.
- Emballage ouvert, mais avec la bioprothèse non implantée: si le plateau est ouvert, la bioprothèse n'est plus stérile. Si la bioprothèse n'est pas implantée, elle doit être placée dans un fixateur histologique adapté comme du méthanediol à 10 % ou du glutaraldéhyde à 2 %, puis retournée à l'entreprise. La réfrigération n'est pas nécessaire dans ces circonstances.
- Bioprothèse explantée: la bioprothèse explantée doit être placée dans un fixateur histologique adapté comme du méthanediol à 10 % ou du glutaraldéhyde à 2 %, puis retournée à l'entreprise. La réfrigération n'est pas nécessaire dans ces circonstances.

## Sécurité dans l'environnement de résonance magnétique (RM)



#### Condition RM

Les tests non cliniques ont montré que la bioprothèse mitrale péricardique d'Edwards, modèle 11000M, est conforme à la condition RM. Un patient possédant la bioprothèse, modèle 11000M, peut subir un balayage sans danger immédiatement après l'implantation, dans les conditions suivantes :

- Champ magnétique statique de 3 teslas ou moins
- Champ gradient spatial maximum de 720 gauss/cm
- Taux d'absorption spécifique maximal signalé par le système RM pour tout le corps de 3 W/kg pour un balayage de 15 minutes.

Pour les tests non cliniques, la bioprothèse mitrale péricardique d'Edwards, modèle 11000M, a produit une augmentation de température inférieure ou égale à 0,5 °C à un taux d'absorption spécifique (TAS) moyen maximum reporté par le système RM de 3 W/kg pendant un balayage RM de 15 minutes dans un système RM de 3 teslas (Excite, logiciel G3.0-052B, General Electric Healthcare).

Il est possible que la qualité de l'image RM soit compromise si la zone d'intérêt correspond à l'emplacement de la bioprothèse modèle 11000M ou en est relativement proche. Il est recommandé d'optimiser les paramètres d'imagerie RM.

## 12. Informations du patient

#### 12.1 Carte d'identification de la recherche

Une carte d'identification de la recherche est remise à chaque sujet implanté avec la bioprothèse mitrale péricardique d'Edwards, modèle 11000M.

#### 12.2 Documents d'information du patient

Il est possible d'obtenir des documents d'information du patient d'Edwards ou de l'un de ses spécialistes des ventes cliniques.

#### 13. Références

- Marchand MA., et al. Fifteen-year Experience with the Mitral Carpentier-Edwards PERIMOUNT Pericardial Bioprosthesis. Ann Thorac Surg. 2001; 71:S236-9.
- Liao K., et al. Bovine Pericardium versus Porcine Aortic Valve: Comparison of Tissue Biological Properties As Prosthetic Valves; Artificial Organs. 1992:16(4):361-5.
- Vesely I., et al. Comparison of the Compressive Buckling of Porcine Aortic Valve Cusps and Bovine Pericardium. J. Heart Valve Dis. January 1998; 7(1):34-9.
- Carpentier A. From Valvular Xenograft to Valvular Bioprosthesis (1965-1977). Med. Instrum. 1977; 11(2):98-101.
- Carpentier A., et al. Continuing Improvements in Valvular Bioprostheses. J. Thorac. Cardiovasc. Surg. 1982; 83(1):27-42.
- Arounlangsy P., et al. Histopathogenesis of early stage mitral annular calcification. J. Med Dent Sci. 2004; 51(1):35-44.
- Bonow RO., et al. ACC/AHA Guidelines for the Management of Patients With Valvular Heart Disease: A Report of the American College of Cardiology/ American Heart Association Task Force on Practice Guidelines (Committee on Management of Patients with Valvular Heart Disease). J. Am Coll Cardiol. 2006; 48:e1-148.

- Aagaard J., et al. Mitral valve replacement with total preservation of native valves and subvalvular apparatus. J. Heart Valve Dis. May 1997; 6(3):274-8; discussion 279-80.
- Jamieson, W.R.E., et al. Carpentier-Edwards Standard Porcine Bioprosthesis: Primary Tissue Failure (Structural Valve Deterioration) by Age Groups. Ann Thorac Surg 1988, 46:155-162.
- Odell, J.A. Calcification of Porcine Bioprostheses in Children. In Cohn, L. and V. Gallucci (eds): Cardiac Bioprostheses. Yorke Medical Books. New York, 1982, pp 231-237.
- Reul, G.J., et al. Valve Failure with the lonescu-Shiley Bovine Pericardial Bioprosthesis: Analysis of 2680 Patients. J. Vasc Surg 1985, 2(1):192-204.
- Sanders, S.P., et al. Use of Hancock Porcine Xenografts in Children and Adolescents. Am J. Cardiol 1980, 46(3):429-438.
- Silver, M.M., et al. Calcification in Porcine Xenograft Valves in Children. Am J. Cardiol 1980, 45:685-689.
- Carpentier, A., et al. Continuing Improvements in Valvular Bioprostheses. J. Thorac Cardiovasc Surg 1982, 83(1):27-42.

Les prix peuvent être modifiés sans préavis. Ce produit est fabriqué et distribué selon au moins une brevets américains suivants : n°S de brevets américains 5,928,281; 5,931,969; 5,961,549; 6,102,94; 6,245,105; 6,413,275; 6,416,547; 6,561,970; 6,585,766; 6,837,902; 6,945,997; 6,966,925; RE 40570; 7,214,344; 7,658,763; 7,682,391; 7,972,376; 8,007,992; 8,357,387; et 8,632,608; ainsi que les brevets étrangers correspondants. De plus, des brevets supplémentaires sont en attente.

Se référer à la légende des symboles à la fin du document.

Tableau 3 : Taux observés d'évènements indésirables pour les RVM et les DRV (modèle 6900)

Tous les patients étudiés : N = 363 Suivi cumulatif : 1 100 patient-années

| | Évènemen | ts précoces | Évènements tardifs <sup>1</sup> | | Absence d'évènements (%) [IC de 95 %] <sup>2</sup> | | |
|---|---|---|---|---|---|---|---|
| Complication | n <sup>3</sup> | % | n | %/pt-an | 1 an (n = 287) | 5 ans (n = 141) | 8 ans (n = 18) |
| Mortalité (tous) | 34 | 9,4 | 50 | 4,7 | 85,5 [81,8,89,2] | 75,4 [70,3, 80,6] | 65,4 [57,6, 73,2] |
| Évènements en lien avec la valve | | | | | | | |
| Mortalité (en lien avec la valve) | 0 | 0 | 16 | 1,5 | 97,7 [96,0, 99,4] | 95,3 [92,8, 97,8] | 91,9 [87,5, 96,4] |
| Explantations | 0 | 0 | 8 | 0,7 | 98,7 [98,0, 99,3] | 96,7 [95,3, 98,0] | 95,6 [93,9, 97,3] |
| Nouvelles opérations chirurgicales | 2 | 0,6 | 12 | 1,1 | 97,1 [96,2, 98,1] | 95,1 [93,6, 96,6] | 93,0 [90,9, 95,1] |
| Hémorragie en lien avec<br>l'anticoagulothérapie | 2 | 0,6 | 9 | 0,8 | 97,1 [95,2,99,0] | 97,1 [95,2, 99,0] | 94,1 [88,2, 100] |
| Endocardite | 1 | 0,3 | 3 | 0,3 | 99,0 [97,9, 100] | 98,7 [97,4, 98,9] | 98,7 [97,4, 98,9] |
| Hémolyse | 0 | 0,0 | 1 | 0,1 | 99,7 [99,0, 100] | 99,7 [99,0, 100] | 99,7 [99,0, 100] |
| Dysfonction non structurelle | 0 | 0,0 | 3 | 0,3 | 100 [100, 100] | 99,3 [98,0, 100] | 98,3 [95,9, 100] |
| Fuite périvalvulaire (tous) | 1 | 0,3 | 5 | 0,5 | 98,4 [97,0, 99,8] | 98,4 [97,0, 99,8] | 97,3 [94,9, 99,8] |
| Détérioration de la structure de la valve | 0 | 0,0 | 5 | 0,5 | 100,0 [100, 100] | 97,6 [95,2, 100] | 92,8 [85,3, 100] |
| Thrombo-embolie | 5 | 1,4 | 8 | 0,7 | 97,5 [95,8, 99,2] | 96,1 [93,8, 98,5] | 96,1 [93,8, 98,5] |
| Thrombose | 0 | 0,0 | 0 | 0,0 | 100,0 [100, 100] | 100,0 [100, 100] | 100,0 [100, 100] |

#### Remarques:

- 1. Les taux d'évènements tardifs sont calculés sous forme de taux linéarisés (%/pt-an) sur la base de 1 072,5 patient-années tardifs (> 30 jours après l'opération).
- Les taux d'absence d'évènements ont été calculés avec la méthode Kaplan-Meier. La formule de Greenwood a été utilisée pour calculer les erreurs-types de ces estimations.
- n = nombre d'évènements.

Tableau 4: Taux observés d'évènements indésirables (modèle 6900P)

Tous les patients étudiés : N = 209 Suivi cumulatif : 873.18 total pt-an

| | Évènemen | ts précoces | Évènen | nents tardifs1 | Absence d'évèneme | nts (%) [IC de 95 %] <sup>2</sup> |
|---|---|---|---|---|---|---|
| Complication | n <sup>3</sup> | % | n | %/pt-an | 1 an | 5 ans |
| Mortalité (tous) | 3 | 1,4 | 45 | 5,3 | 93,2 [88,8, 95,9] | 74,4 [66,9,80,5] |
| Évènements en lien avec la valve | | | | | | |
| Mortalité (en lien avec la valve) | 1 | 0,5 | 12 | 1,4 | 98,5 [95,5, 99,5] | 92,0 [86,2,95,5] |
| Explantations | 1 | 0,5 | 8 | 0,9 | 97,5 [94,0, 98,9] | 96,5 [92,2,98,5] |
| Nouvelles opérations chirurgicales | 0 | 0,0 | 0 | 0,0 | 100,0 [100, 100] | 100,0 [100, 100] |
| Saignements | 5 | 2,4 | 13 | 1,5 | 96,1 [92,3, 98,0] | 91,9 [86,5,95,2] |
| Endocardite | 1 | 0,5 | 3 | 0,4 | 99,5 [96,6, 99,9] | 97,1 [92,1,98,9] |
| Dysfonction non structurelle | 0 | 0,0 | 1 | 0,1 | 99,5 [96,4, 99,9] | 99,5 [96,4,99,9] |
| Fuite périvalvulaire (tous) | 1 | 0,5 | 2 | 0,2 | 99,5 [96,7, 99,9] | 98,4 [95,2,99,5] |
| Détérioration de la structure de la valve | 0 | 0,0 | 2 | 0,2 | 100,0 [100, 100] | 99,0 [93,2,99,9] |
| Thrombo-embolie | 4 | 1,9 | 12 | 1,4 | 97,0 [93,5, 98,7] | 91,3 [85,8,94,7] |
| Thrombose | 0 | 0,0 | 0 | 0,0 | 100,0 [100, 100] | 100,0 [100, 100] |

#### Remarques:

- 1. Les taux d'évènements tardifs sont calculés sous forme de taux linéarisés (%/pt-an) sur la base de 856,24 patient-années tardifs (> 30 jours après l'opération).
- Les taux d'absence d'évènements ont été calculés avec la méthode Kaplan-Meier. La formule de Greenwood a été utilisée pour calculer les erreurs-types de ces
  estimations.
- n = nombre d'évènements.

Tableau 5 : Données démographiques préopératoires (modèle 6900)

| | | Caractéristiques de l'étude (N = 363; 1 100 total pt-an) | |
|---|---|---|---|
| Variable | Catégorie | Catégorie n % (r | |
| Âge lors de l'implantation (N = 363) | Moyenne ± écart-type | 66,1 ± 10,7 | |
| Sexe | Fém./masc. | 212/151 | 58,4%/41,6% |
| | Aucune | 30 | 8,3% |
| Diamantinus/faialania | Sténose | 91 | 25,1% |
| Diagnostique/étiologie | Régurgitation | 184 | 50,7% |
| | Maladies mixtes | 58 | 16,0% |

## Remarque:

1. n = nombre de patients pour chaque catégorie; <math>N = total de patients de l'étude.

Tableau 6 : Données démographiques préopératoires (modèle 6900P)

| | | Caractéristiques de l'étude (N = 209; 873,18 total pt-an) | |
|---|---|---|---|
| Variable | Catégorie | n | % (n/N) <sup>1</sup> |
| Âge lors de l'implantation (N = 209) | Moyenne ± écart-type | 71,4 ± 9,4 | |
| Sexe | Fém./masc. | 138/71 | 66,0%/34,0% |
| | Maladies mixtes | 48 | 23,0% |
| Diagnostique/étiologie | Régurgitation | 121 | 57,9% |
| | Sténose | 32 | 15,3% |
| | Dysfonction de la valve | 8 | 3,8% |

## Remarque:

1. n =nombre de patients pour chaque catégorie; N =total de patients de l'étude.

Tableau 7 : Données démographiques des patients en période opératoire (modèle 6900)

| | | Caractéristiqu<br>(N = 363; 1 10 | |
|---|---|---|---|
| Variable | Catégorie | n | % (n/N) <sup>1</sup> |
| | Rhumatisme cardiaque | 135 | 37,2% |
| | Calcification | 82 | 22,6% |
| | Dégénération | 50 | 13,8% |
| 6 | Endocardite | 39 | 10,7% |
| Étiologie <sup>2</sup> | Bioprothèse défectueuse | 15 | 4,1% |
| | Cardiopathie ischémique | 14 | 3,9% |
| | Anomalies congénitales | 8 | 2,2% |
| | Autre | 44 | 12,1% |
| | Aucune | 200 | 55,1% |
| | PA <sup>3</sup> | 78 | 21,5% |
| | Réparation tricuspidienne | 61 | 16,8% |
| D. (1 | Pompe à ballonnet intra aortique | 17 | 4,7% |
| Procédures concomitantes <sup>2</sup> | Stimulateur cardiaque <sup>4</sup> | 6 | 1,7% |
| | Réparation/remplacement aortique | 5 | 1,4% |
| | Réparation d'un anévrisme | 4 | 1,1% |
| | Autre | 31 | 8,5% |
| | Aucune | 122 | 33,6% |
| | C <sup>5</sup> /PA | 72 | 19,8% |
| | Hypertension | 61 | 16,8% |
| Affections préexistantes <sup>2</sup> | Fibrillation auriculaire | 53 | 14,6% |
| | IM antérieur <sup>6</sup> | 45 | 12,4% |
| | Maladie cérébrovasculaire | 36 | 9,9% |
| | Autre | 234 | 64,5% |
| | 25 | 22 | 6,1% |
| | 27 | 110 | 30,3% |
| Taille de la valve (mm) | 29 | 137 | 37,7% |
| | 31 | 81 | 22,3% |
| | 33 | 13 | 3,6% |

#### Remarques:

- 1. n = nombre de patients pour chaque catégorie; N = total des patients de l'étude
- Possibilité de plus d'un par patient
   PA = Pontage aortocoronarien
- 4. Permanent ou temporaire
- 5. C = Coronaropathie
  6. IM = Infarctus du myocarde

Tableau 8 : Données démographiques des patients en période opératoire (modèle 6900P)

| | | Caractéristique<br>(N = 209; 873,1 | |
|---|---|---|---|
| Variable | Catégorie | n | % (n/N) <sup>1</sup> |
| | Calcification | 38 | 18,2% |
| | Congénital | 1 | 0,5% |
| | Dégénératif | 105 | 50,2% |
| Étiologie <sup>2</sup> | Endocardite récente | 10 | 4,8% |
| | Ischémique | 12 | 5,7% |
| | Rhumatismal | 64 | 30,6% |
| | Autre | 36 | 17,2% |
| | Aucune | 91 | 43,5% |
| | Réparation valve/anneau aortique | 3 | 1,4% |
| | PA <sup>3</sup> | 58 | 27,8% |
| Procédures concomitantes <sup>2</sup> | Stimulateur cardiaque permanent | 1 | 0,5% |
| | Réparation de la valve/anneau tricuspide | 21 | 10,0% |
| | Autre | 78 | 37,3% |
| | Aucune | 17 | 8,1% |
| | Arythmie | 95 | 45,5% |
| | C <sub>6</sub> | 85 | 40,7% |
| | Myocardiopathie | 13 | 6,2% |
| | Insuffisance cardiaque congestive | 66 | 31,6% |
| | Endocardite | 14 | 6,7% |
| uffections préexistantes <sup>2</sup> | Infarctus du myocarde | 21 | 10,0% |
| | Maladie vasculaire périphérique | 9 | 4,3% |
| | Hypertension artérielle pulmonaire | 66 | 31,6% |
| | Fièvre rhumatismale | 16 | 7,7% |
| | Hypertension généralisée | 49 | 23,4% |
| | AIT <sup>4</sup> /AVC <sup>5</sup> | 24 | 11,5% |
| | Autre | 35 | 16,7% |
| | 25 | 28 | 13,4% |
| | 27 | 37 | 17,7% |
| aille de la valve (mm) | 29 | 84 | 40,2% |
| | 31 | 43 | 20,6% |
| | 33 | 17 | 8,1% |

#### Remarques:

- 1. n = nombre de patients pour chaque catégorie; N = total des patients de l'étude
- Possibilité de plus d'un par patient
   PA = Pontage aortocoronarien
- 4. AIT = accident ischémique transitoire
- 5. AVC = accident vasculaire cérébral
- 6. C = Coronaropathie

Tableau 9 : Résultats en matière d'efficacité, classification fonctionnelle NYHA (modèle 6900)

| | Évaluation | | Évaluations postopératoires | | | |
|---|---|---|---|---|---|---|
| Classification fonctionnelle | préopé | ratoire | 1 à 2 | 2 ans | 5 ans | |
| de la NYHA | n/N <sup>1</sup> | % | n/N | % | n/N | % |
| I | 11/363 | 3,0 | 120/268 | 44,8 | 40/129 | 31,0 |
| II | 73/363 | 20,1 | 90/268 | 33,6 | 25/129 | 19,4 |
| III | 192/363 | 52,9 | 15/268 | 5,6 | 1/129 | 0,8 |
| IV | 84/363 | 23,1 | 0/268 | 0,0 | 0/129 | 0,0 |
| Non disponible | 3/363 | 0,8 | 43/268 | 16,0 | 63/129 | 48,8 |

#### Remarque:

1. n = nombre de patients pour chaque catégorie; <math>N = total de patients de l'étude.

Tableau 10 : Résultats en matière d'efficacité, classification fonctionnelle NYHA (modèle 6900P)

| | Évaluation | | Évaluations postopératoires | | | |
|---|---|---|---|---|---|---|
| Classification fonctionnelle | préopé | ratoire | 1 | an | 5 a | ins |
| de la NYHA | n/N <sup>1</sup> | % | n/N | % | n/N | % |
| 1 | 6/209 | 2,9 | 86/187 | 46,0 | 30/96 | 31,3 |
| II | 27/209 | 12,9 | 68/187 | 36,4 | 33/96 | 34,4 |
| Ш | 121/209 | 57,9 | 8/187 | 4,3 | 6/96 | 6,3 |
| IV | 55/209 | 26,3 | 1/187 | 0,5 | 0/96 | 0,0 |
| Non disponible | 0/209 | 0,0 | 24/187 | 12,8 | 27/96 | 28,1 |

## Remarque:

1. n = nombre de patients pour chaque catégorie; N = total de patients de l'étude.

Tableau 11 : Résultats en matière d'efficacité, résultats hémodynamiques 1 (modèle 6900)

| Paramètre | Résultats par taille de valve | | | | |
|---|---|---|---|---|---|
| hémodynamique | 25 mm | 27 mm | 29 mm | 31 mm | 33 mm |
| Sortie/précoce post-implanta | tion (n = 130, 109 RVM | <sup>2</sup> et 21 DRV <sup>3</sup> ) | | | |
| Gradient moyen <sup>4</sup> | n=3 | n = 23 | n=36 | n = 23 | n=3 |
| • moyenne ± écart-type | 5,7 ± 1,2 | 4,2 ± 1,7 | 4,2 ± 1,7 | 3,6 ± 1,0 | 7,5 ± 5,8 |
| • min., max. | 5,7 | 2,9 | 1, 8 | 2,5 | 3,14 |
| SEO <sup>5</sup> | n = 1 | n = 17 | n = 22 | n = 25 | n = 5 |
| • moyenne ± écart-type | 1,5 | 2,9 ± 0,9 | 3,1 ± 0,9 | 2,5 ± 0,7 | 3,0 ± 1,2 |
| • min., max. | 1,5, 1,5 | 1,3, 4,1 | 1,4,4,2 | 1,5, 3,8 | 1,6, 4,9 |
| Régurgitation <sup>6</sup> | n=3 | n = 28 | n = 51 | n = 40 | n = 8 |
| 0 | 3/3 (100%) | 22/28 (79%) | 36/51 (71%) | 30/40 (75%) | 4/8 (50%) |
| 1+ | 0/3 (0%) | 5/28 (18%) | 13/51 (25%) | 7/40 (18%) | 4/8 (50%) |
| 2+ | 0/3 (0%) | 0/28 (0%) | 1/51 (2%) | 3/40 (7%) | 0/8 (0%) |
| 3+ | 0/3 (0%) | 0/28 (0%) | 1/51 (2%) | 0/40 (0%) | 0/8 (0%) |
| 4+ | 0/3 (0%) | 0/28 (0%) | 0/51 (0%) | 0/40 (0%) | 0/8 (0%) |
| Non disponible | 0/3 (0%) | 1/28 (3%) | 0/51 (0%) | 0/40 (0%) | 0/8 (0%) |
| Intervalle de 3 à 6 mois post-i | implantation (n = 49, 42 | 2 RVM <sup>2</sup> et 7 DRV <sup>3</sup> ) | | | |
| Gradient moyen <sup>4</sup> | n = 5 | n = 19 | n = 15 | n = 5 | n = 2 |
| • moyenne ± écart-type | 6,4 ± 1,7 | 5,3 ± 5 | 3,4 ± 1,2 | 4±1,9 | 4 ± 0 |
| • min., max. | 5, 9 | 2,25 | 2, 6 | 2,7 | 4, 4 |
| SEO <sub>2</sub> | n = 5 | n = 18 | n = 13 | n = 5 | n = 2 |
| • moyenne ± écart-type | 2,9 ± 0,8 | $2,6 \pm 0,7$ | 2,8 ± 0,6 | 2,9 ± 0,3 | 2,6 ± 1 |
| • min., max. | 1,8, 3,6 | 1,5,5 | 2, 3,8 | 2,4, 3,3 | 2, 3,3 |
| Régurgitation <sup>6</sup> | n = 5 | n = 21 | n = 15 | n=6 | n = 2 |
| 0 | 3/5 (60%) | 17/21 (81%) | 6/15 (40%) | 4/6 (67%) | 1/2 (50%) |
| 1+ | 0/5 (0%) | 4/21 (19%) | 8/15 (53%) | 2/6 (33%) | 0/2 (0%) |
| 2+ | 1/5 (20%) | 0/21 (0%) | 1/15 (7%) | 0/6 (0%) | 1/2 (50%) |
| 3+ | 0/5 (0%) | 0/21 (0%) | 0/15 (0%) | 0/6 (0%) | 0/2 (0%) |
| 4+ | 1/5 (20%) | 0/21 (0%) | 0/15 (0%) | 0/6 (0%) | 0/2 (0%) |
| Non disponible | 0/5 (0%) | 0/21 (0%) | 0/15 (0%) | 0/6 (0%) | 0/2 (0%) |

Suite sur la page suivante.

Tableau 11 : Résultats en matière d'efficacité, résultats hémodynamiques (modèle 6900), suite

| Paramètre | | | Résultats par taille de valve | e | |
|---|---|---|---|---|---|
| hémodynamique | 25 mm | 27 mm | 29 mm | 31 mm | 33 mm |
| Intervalle de 1 à 2 ans après i | mplantation (n = 131, 1 | 14 RVM <sup>2</sup> et 17 DRV <sup>3</sup> ) | | | |
| Gradient moyen <sup>4</sup> | n=3 | n = 40 | n = 47 | n = 27 | n = 4 |
| • moyenne ± écart-type | 5,2 ± 0,7 | 4,1 ± 1,6 | 3,5 ± 1,8 | 3,1 ± 1,4 | 2,1 ± 0,5 |
| • min., max. | 4,7,6 | 1,7 | 1,10 | 1,7 | 1,5, 2,7 |
| SEO <sub>2</sub> | n=2 | n=35 | n = 46 | n = 29 | n = 5 |
| • moyenne ± écart-type | 1,8 ± 0,4 | 2,3 ± 0,6 | 2,6 ± 0,5 | 2,6 ± 0,7 | 2,5 ± 0,5 |
| • min., max. | 1,5, 2,0 | 1,2, 3,5 | 1,1,3,7 | 1,1,3,7 | 2,1,3,2 |
| Régurgitation <sup>6</sup> | n = 4 | n = 42 | n = 51 | n = 29 | n = 5 |
| 0 | 2/4 (50%) | 31/42 (74%) | 36/51 (71%) | 17/29 (59%) | 3/5 (60%) |
| 1+ | 1/4 (25%) | 9/42 (21%) | 11/51 (21%) | 8/29 (27%) | 1/5 (20%) |
| 2+ | 1/4 (25%) | 2/42 (5%) | 4/51 (8%) | 2/29 (7%) | 1/5 (20%) |
| 3+ | 0/4 (0%) | 0/42 (0%) | 0/51 (0%) | 2/29 (7%) | 0/5 (0%) |
| 4+ | 0/4 (0%) | 0/42 (0%) | 0/51 (0%) | 0/29 (0%) | 0/5 (0%) |
| Non disponible | 0/4 (0%) | 0/42 (0%) | 0/51 (0%) | 0/29 (0%) | 0/5 (0%) |
| Intervalle de 5 ans après imp | lantation (n = 11,9 RVA | M <sup>2</sup> et 2 DRV <sup>3</sup> ) | | | |
| Gradient moyen <sup>4</sup> | n=0 | n = 6 | n = 5 | n = 0 | n = 0 |
| • moyenne ± écart-type | S.O. | 8,8 ± 8,1 | 5,1 ± 2,3 | S.O. | S.O. |
| • min., max. | S.O. | 4, 25 | 3, 8 | S.O. | S.O. |
| SEO <sub>2</sub> | n = 0 | n = 2 | n = 4 | n = 0 | n = 0 |
| • moyenne ± écart-type | S.O. | 2,0 ± 1,5 | 2,9 ± 0,6 | S.O. | S.O. |
| • min., max. | S.O. | 1,0,3,1 | 2,1, 3,5 | S.O. | S.O. |
| Régurgitation <sup>6</sup> | n=0 | n=6 | n = 5 | n = 0 | n = 0 |
| 0 | 0/0 (0%) | 4/6 (66%) | 2/5 (40%) | 0/0 (0%) | 0/0 (0%) |
| 1+ | 0/0 (0%) | 1/6 (17%) | 3/5 (60%) | 0/0 (0%) | 0/0 (0%) |
| 2+ | 0/0 (0%) | 1/6 (17%) | 0/5 (0%) | 0/0 (0%) | 0/0 (0%) |
| 3+ | 0/0 (0%) | 0/6 (0%) | 0/5 (0%) | 0/0 (0%) | 0/0 (0%) |
| 4+ | 0/0 (0%) | 0/6 (0%) | 0/5 (0%) | 0/0 (0%) | 0/0 (0%) |
| Non disponible | 0/0 (0%) | 0/6 (0%) | 0/5 (0%) | 0/0 (0%) | 0/0 (0%) |

- 1. Les évaluations hémodynamiques ont été effectuées par échocardiographie transthoracique et, dans certains cas, par échocardiographie transoesophagienne.
- RVM = remplacement de la valve mitrale
   DRV = double remplacement de la valve
- 4. Gradient moyen en mm Hg
- 5. SEO: surface effective d'orifice, cm<sup>2</sup>
- 6. Régurgitation = aucune, 0; bénigne, 1+; modérée, 2+; modérée à grave, 3+; grave, 4+

Tableau 12 : Résultats en matière d'efficacité, résultats hémodynamiques (modèle 6900P)<sup>1</sup>

| Paramètre | | | Résultats par taille de valv | e | |
|---|---|---|---|---|---|
| hémodynamique | 25 mm | 27 mm | 29 mm | 31 mm | 33 mm |
| Sortie/précoce post-implanta | ation | | | | |
| Gradient moyen <sup>2</sup> | n = 24 | n=35 | n = 83 | n = 42 | n = 16 |
| • moyenne ± écart-type | 6,4 ± 1,87 | 4,4 ± 1,52 | 3,4 ± 1,47 | 3,3 ± 1,20 | 4,0 ± 1,38 |
| • min., max. | 3,10 | 1,96, 8 | 1,4,9 | 1,7 | 1,5,6,91 |
| 2E03 | n = 8 | n = 27 | n=77 | n = 41 | n = 16 |
| • moyenne ± écart-type | 2,7 ± 0,87 | 2,8 ± 0,58 | 2,9 ± 0,93 | 2,5 ± 0,67 | 2,4 ± 0,52 |
| • min., max. | 1,46, 4,4 | 1,5, 3,9 | 1,58, 6 | 1,32, 4,2 | 1,55, 3,31 |
| Régurgitation <sup>4</sup> | n = 27 | n=37 | n = 83 | n = 43 | n = 17 |
| Anodine/aucune | 19/27 (70%) | 29/37 (78%) | 76/83 (92%) | 39/43 (91%) | 15/17 (88%) |
| 1+ Bénigne | 6/27 (22%) | 7/37 (19%) | 7/83 (8%) | 4/43 (9%) | 1/17 (6%) |
| 2+ Modérée | 1/27 (4%) | 1/37 (3%) | 0/83 (0%) | 0/43 (0%) | 0/17 (0%) |
| 3+ Modérée à grave | 0/27 (0%) | 0/37 (0%) | 0/83 (0%) | 0/43 (0%) | 1/17 (6%) |
| 4+ Grave | 0/27 (0%) | 0/37 (0%) | 0/83 (0%) | 0/43 (0%) | 0/17 (0%) |
| Non disponible | 1/27 (4%) | 0/37 (0%) | 0/83 (0%) | 0/43 (0%) | 0/17 (0%) |
| Intervalle de 3 à 6 mois post- | implantation | | | | |
| Gradient moyen <sup>2</sup> | n = 0 | n = 4 | n=3 | n = 2 | n = 0 |
| • moyenne ± écart-type | 0 ± 0 | 4,4 ± 2,25 | 2,3 ± 0,89 | 6,6 ± 2,05 | 0 ± 0 |
| • min., max. | 0, 0 | 2,5,7,5 | 1,3, 3 | 5,1,8 | 0, 0 |
| SEO3 | n = 0 | n=3 | n=3 | n = 1 | n = 1 |
| • moyenne ± écart-type | 0 ± 0 | 2,4 ± 0,74 | 3,2 ± 0,88 | 2,5 ± 0,00 | 1,2 ± 0,00 |
| • min., max. | 0, 0 | 1,6,3 | 2,3,4,05 | 2,47, 2,47 | 1,22, 1,22 |
| Régurgitation <sup>4</sup> | n = 0 | n = 5 | n=3 | n = 2 | n = 2 |
| Anodine/aucune | 0 | 3/5 (60%) | 2/3 (67%) | 2/2 (100%) | 2/2 (100%) |
| 1+ Bénigne | 0 | 1/5 (20%) | 1/3 (33%) | 0/2 (0%) | 0/2 (0%) |
| 2+ Modérée | 0 | 1/5 (20%) | 0/3 (0%) | 0/2 (0%) | 0/2 (0%) |
| 3+ Modérée à grave | 0 | 0/5 (0%) | 0/3 (0%) | 0/2 (0%) | 0/2 (0%) |
| 4+ Grave | 0 | 0/5 (0%) | 0/3 (0%) | 0/2 (0%) | 0/2 (0%) |
| Non disponible | 0 | 0/5 (0%) | 0/3 (0%) | 0/2 (0%) | 0/2 (0%) |

Suite sur la page suivante.

Tableau 12 : Résultats en matière d'efficacité, résultats hémodynamiques (modèle 6900P)<sup>1</sup>, suite

| Paramètre | | Résultats par taille de valve | | | |
|---|---|---|---|---|---|
| hémodynamique | 25 mm | 27 mm | 29 mm | 31 mm | 33 mm |
| Intervalle de 1 an après imp | lantation | | | | |
| Gradient moyen <sup>2</sup> | n = 16 | n = 27 | n = 63 | n=34 | n = 15 |
| • moyenne ± écart-type | 5,9 ± 2,36 | 4,0 ± 1,45 | 3,0 ± 1,61 | 3,3 ± 1,26 | 3,4 ± 1,25 |
| • min., max. | 3,12 | 2,7 | 1,12 | 1,5,7 | 1,9,6,3 |
| 2E03 | n=3 | n = 21 | n = 59 | n=32 | n = 15 |
| • moyenne ± écart-type | 2,3 ± 0,16 | 2,4 ± 0,76 | 2,6 ± 0,74 | 2,5 ± 0,67 | 2,3 ± 0,83 |
| • min., max. | 2,09, 2,4 | 1,27, 4,76 | 1,5, 5,7 | 1,5, 4 | 1,2,3,8 |
| Régurgitation <sup>4</sup> | n = 20 | n = 28 | n = 65 | n=34 | n = 16 |
| Anodine/aucune | 17/20 (85%) | 24/28 (86%) | 53/65 (82%) | 29/34 (85%) | 13/16 (81%) |
| 1+ Bénigne | 3/20 (15%) | 3/28 (11%) | 6/65 (9%) | 3/34 (9%) | 3/16 (19%) |
| 2+ Modérée | 0/20 (0%) | 0/28 (0%) | 3/65 (5%) | 2/34 (6%) | 0/16 (0%) |
| 3+ Modérée à grave | 0/20 (0%) | 0/28 (0%) | 1/65 (2%) | 0/34 (0%) | 0/16 (0%) |
| 4+ Grave | 0/20 (0%) | 0/28 (0%) | 0/65 (0%) | 0/34 (0%) | 0/16 (0%) |
| Non disponible | 0/20 (0%) | 1/28 (4%) | 2/65 (3%) | 0/34 (0%) | 0/16 (0%) |

## Remarques:

- 1. Les évaluations hémodynamiques ont été effectuées par échocardiographie transthoracique et, dans certains cas, par échocardiographie transoesophagienne.
- Gradient moyen en mm Hg
   SEO: surface effective d'orifice, cm<sup>2</sup>
- 4. Régurgitation = anodine/aucune 0; bénigne, 1+; modérée, 2+; modérée à grave, 3+; grave, 4+

## Polski

## Osierdziowa bioproteza mitralna Edwards model 11000M

## Instrukcja użytkowania

PRZESTROGA: Urządzenie badawcze. Prawo federalne (Stanów Zjednoczonych Ameryki) ogranicza użytkowanie tego urządzenia do celów badawczych.

PRZESTROGA: Urządzenie badawcze. Wyłącznie do badań klinicznych.

Przestroga: Urządzenie badawcze. Przeznaczone wyłącznie do celów badawczych. Do stosowania wyłącznie przez wykwalifikowanych badaczy (lekarzy).

#### Opis urządzenia i akcesoriów

#### 1.1 Opis urządzenia

Osierdziowa bioproteza mitralna Edwards model 11000M jest trójpłatkową bioprotezą wykonaną z odpowiednio przygotowanego wołowego osierdzia, umocowaną na elastycznej ramie. Jest dostępna w rozmiarach 25, 27, 29, 31 i 33 mm (Tabela 1). Bioproteza jest przechowywana w opakowaniu niewodnym i nie wymaga przemywania przed wszczepieniem.

Prowadnica druciana jest wykonana ze stopu kobaltowo-chromowego i jest pokryta tkaniną poliestrową. Stop kobaltowo-chromowy/warstwa laminatu poliestrowego otacza podstawe ramy prowadnicy drucianei.

Silikonowy pierścień do wszywania o strukturze waflowej, pokryty porowatą tkaniną politetrafluoroetylenową (PTFE), jest przymocowany do ramy prowadnicy drucianej. Pierścień do wszywania jest obrębiony wzdłuż przedniej części. Szwy znacznikowe z czarnego jedwabiu na przedniej części ułatwiają ułożenie bioprotezy i pomagają zapobiec zablokowaniu drogi odpływu z lewej komory przez rozpórkę.

Linia prowadząca szew z czarnego jedwabiu otacza pierścień do wszywania. Umieszczanie szwów przechodzących przez pierścień do wszywania i w regionie od linii prowadzącej szew do zewnętrznej części pierścienia do wszywania ułatwia penetrację igły i zapewnia zmienną zgodność. W strukturze waflowej komórki są szersze wzdłuż części tylnej, gdzie w naturalnym pierścieniu mitralnym częstsze są zwapnienia i nieregularności (poz. 6).

| | - 0 | | | | HVT63 |
|---|---|---|---|---|---|
| Rozmiar | 25<br>mm | 27<br>mm | 29<br>mm | 31<br>mm | 33<br>mm |
| A. Średnica stentu (prowadnica druciana, mm) | 25 | 27 | 29 | 31 | 31 |
| B. Średnica pierścienia tkanki (mm) | 28 | 29,5 | 31,5 | 33,5 | 33,5 |
| C. Zewnętrzna średnica wspornika<br>stentu (końcówka, mm) | 29 | 31 | 34 | 35 | 35 |
| D. Zewnętrzna średnica pierścienia<br>do wszywania (mm) | 36 | 38 | 40 | 42 | 44 |
| E. Efektywny profil – część<br>przednia (mm) | 7 | 7,5 | 8 | 8,5 | 8,5 |
| E. Efektywny profil — część tylna<br>(mm) | 10 | 10,5 | 11 | 11,5 | 11,5 |
| G. Całkowita wysokość profilu (mm) | 15 | 16 | 17 | 18 | 18 |
| Powierzchnia geometryczna<br>otworu (mm²) | 424 | 499 | 580 | 653 | 653 |

#### 1.2 Opis akcesoriów

Do bioprotezy 11000M dostępne są następujące akcesoria:

- · system uchwytu Tricentrix
- kalibrator replikuiacy 1173R

Tabela 1: Wymiary nominalne

- kalibrator cylindra 1173B
- taca do wviaławiania dostarczana z modelem SET1173
- modele rekojeści 1111, 1117, 1173 i 1126 (do jednorazowego użytku)

Wszelkie akcesoria są dostarczane jako niejałowe, z wyjątkiem systemu uchwytu Tricentrix, dostarczanego w postaci jałowej i dołączonego do jałowej bioprotezy, oraz rękojeści 1126, dostarczanej w postaci jałowej i przeznaczonej do iednokrotnego użvcia.

#### Kalibratory i taca

Z bioprotezą 11000M można stosować wyłącznie modele kalibratorów 1173B (Rysunek 1a) lub 1173R (Rysunek 1b).

Przestroga: Do określania rozmiaru bioprotezy 11000M nie należy używać kalibratorów zastawkowych innych producentów ani kalibratorów przeznaczonych do innych protez zastawkowych firmy Edwards Lifesciences.

Do ustalenia odpowiedniego rozmiaru bioprotezy 11000M należy używać wyłącznie kalibratorów model 1173B i 1173R. Kalibratory 1173B i 1173R umożliwiają bezpośrednią obserwację dopasowania w pierścieniu włóknistym. Są dostarczane dla każdego z dostępnych rozmiarów bioprotezy 11000M. Cylindry kalibratorów model 1173B i 1173R wskazują zewnętrzną średnicę stentu przy

Edwards Lifesciences, logo stylizowanej litery E, Edwards, Carpentier-Edwards, Tricentrix, PERIMOUNT, PERIMOUNT Magna, PERIMOUNT Plus, TFX i Magna Mitral Ease to znaki towarowe firmy Edwards Lifesciences Corporation.

podstawie. Krawędź kalibratorów replikujących 1173R powiela kształt pierścienia do wszywania bioprotezy z jego przednią, obrębioną częścią oraz czarnymi onacznikami. Ma to na celu lepsze ustalenie wyników stosowania specyficznych technik wszywania lub technik zabezpieczenia aparatu podzastawkowego.

Kalibratory 1173B i 1173R są oznaczone rozmiarem bioprotezy. Kompletny zestaw kalibratorów jest umieszczony na tacy model SET1173, którą można ponownie wykorzystywać i sterylizować.



## System uchwytu Tricentrix i rękojeści

Zespół uchwyt/rękojeść składa się z dwóch części: systemu uchwytu Tricentrix (Rysunek 2), który jest mocowany do bioprotezy 11000M, i rękojeści (1111, 1117, 11173 lub 1126), która jest dołączana do systemu uchwytu Tricentrix podczas zabiegu.





Poniższe rękojeści (Tabela 2) mogą być stosowane z bioprotezą 11000M:

| Tabela 2. R | Tabela 2. Rękojeści akcesoriów | | | |
|---|---|---|---|---|
| | | Całkowit | a długość | Do<br>wielokrotnego |
| Model | Materiał korpusu | cale | cm | użytku |
| 1111 | Stal nierdzewna | 7,0 | 17,8 | Tak |
| 1117 | Nitinol | 9,1 | 23,2 | Tak |
| 1126 | Stal nierdzewna | 11,5 | 29,2 | Nie |
| 1173 | Nitinol | 11,3 | 28,6 | Tak |

Rękojeści o trzonie nitinolowym są elastyczniejsze od uchwytów ze stali nierdzewnej. Po każdym cyklu wyjaławiania powracają do oryginalnego, prostego kształtu, co pozwala na łatwiejsze przymocowanie uchwytu.

## 2. Wskazania do stosowania

Osierdziowa bioproteza mitralna Edwards model 11000M jest przeznaczona dla pacjentów wymagających wymiany naturalnej lub protetycznej zastawki mitralnej.

#### 3. Przeciwwskazania

Nie należy stosować produktu, jeżeli chirurg sądzi, że jego użycie jest sprzeczne z dobrem pacjenta. To on powinien podjąć decyzję dotyczącą zastosowania tej bioprotezy lub zrezygnowania z jej użycia, ponieważ może ocenić różne czynniki ryzyka związane z jej wszczepieniem, w tym również budowę anatomiczną pacjenta oraz zmiany patologiczne widoczne podczas operacji.

#### 4. Ostrzeżenia

WYŁĄCZNIE DO JEDNORAZOWEGO UŻYTKU. Opisywane urządzenie jest zaprojektowane i rozprowadzane wyłącznie z zamiarem jednorazowego użytku i takie jest jego przeznaczenie. Urządzenia nie wolno sterylizować ani stosować ponownie. Nie istnieją żadne dane potwierdzające jałowość, niepirogenność i sprawność produktu po ponownej sterylizacji. Wystawienie bioprotezy lub pojemnika na działanie promieniowania, pary, tlenku etylenu lub innych chemicznych środków sterylizujących spowoduję, że bioproteza będzie niezdatna do użytku.

NIE WOLNO ZAMRAŻAĆ BIOPROTEZY ANI PODDAWAĆ DZIAŁANIU SKRAJNIE WYSOKIEJ TEMPERATURY. Narażenie bioprotezy na skrajne temperatury uczyni urządzenie niezdatnym do użycia.

Bioprotezy NIE NALEŻY UŻYWAĆ:

- jeśli torebka foliowa, zapieczętowane tace lub pokrywy są otwarte, uszkodzone lub zabrudzone
- · jeśli minął termin ważności lub
- jeśli została upuszczona, zniszczona lub postępowano z nią w niewłaściwy sposób. Jeśli podczas wszczepiania bioproteza ulegnie zniszczeniu, nie należy podeimować próby iei naprawy.

NIE NALEŻY NARAŻAĆ bioprotezy na działanie jakichkolwiek roztworów, środków chemicznych, antybiotyków itp., z wyjątkiem jałowego roztworu soli fizjologicznej. Może nastąpić nienaprawialne uszkodzenie tkanki płatków, które może nie być widoczne gołym okiem.

NIE WOLNO CHWYTAĆ tkanki płatków bioprotezy narzędziami ani w żaden sposób uszkadzać bioprotezy. Nawet najmniejsza perforacja ktanki płatków może z czasem ulec powiększeniu, powodując znaczne upośledzenie czynności zastawki. NIE NALEŻY STOSOWAĆ ZBYT DUŻEGO ROZMIARU. Stosowanie zbyt dużego rozmiaru może spowodować uszkodzenie bioprotezy lub miejscowe naprężenia mechaniczne, których efektem może być uszkodzenie serca, zniszczenie tkanki płatków, zniekształcenie stentu i przepływ fali zwrotnej przez zastawke.

NIE PRZEPROWADZAĆ PRZEZ BIOPROTEZĘ CEWNIKÓW, wprowadzanych do żył elektrod stymulujących ani żadnych narzędzi chirurgicznych, z wyjątkiem lusterka chirurgicznego używanego do sprawdzania umieszczenia rozpórek i szwów. Pozostałe narzędzia chirurgiczne moga spowodować uszkodzenie tkanki płatków.

Podobnie jak w przypadku każdego implantowanego przyrządu medycznego, istnieje ryzyko odpowiedzi immunologicznej u pacjenta. Do składników modelu 11000M należy stop metalu, który zawiera kobalt, chrom, nikiel, molibden, mangan, węgiel, beryl oraz żelazo. Należy zachować ostrożność u pacjentów z nadwrażliwościami na te materiały. Urządzenie zostało wytworzone bez lateksu, ale mogło być produkowane w środowisku zawierajacym lateks.

## 5. Zdarzenia niepożądane

#### 5.1 Zaobserwowane zdarzenia niepożądane

Podobnie jak w przypadku wszystkich sztucznych zastawek serca, stosowanie zastawek tkankowych może wiązać się z poważnymi działaniami niepożądanymi, niekiedy prowadzącymi do zgonu. Ponadto po upływie różnych okresów czasu (godzin lub dni) mogą występować zdarzenia niepożądane wynikające z indywidualnej reakcji pacjenta na wszczepione urządzenie lub fizycznych i chemicznych zmian jego komponentów, zwłaszcza pochodzenia biologicznego; moga one powodować konieczność ponownej operacji i wymiany protezy.

Osierdziowa bioproteza mitralna Edwards model 11000M jest podobna w konstrukcji do bioprotez osierdziowych Carpentier-Edwards PERIMOUNT Magna Mitral Ease model 7300TFX.

Przeprowadzono trzy (3) wieloośrodkowe, nierandomizowane, prospektywne badania kliniczne, poza terenem Stanów Zjednoczonych, u pacjentów z zaimplantowaną bioprotezą osierdziową zastawki mitralnej model 6900. Trzystu jeden (301) pacjentów poddanych zostało izolowanej wymianie zastawki mitralnej (MVR), a 62 wymianie dwóch zastawek (DVR), przy czym zastawka wortalna była wymieniana na bioprotezę osierdziową PERIMOUNT firmy Carpentier-Edwards model aortalny.

W pierwszym badaniu bioprotezy wszczepiano w latach od 1984 do 1986, w drugim badaniu bioprotezy wszczepiano w latach od 1989 do 1994, w trzecim badaniu bioprotezy wszczepiano w latach od 1996 do 1997. Stan pacjentów oceniano przedoperacyjnie, śródoperacyjnie, przy wypisywaniu ze szpitala, po 1 roku i następnie corocznie. Przez cały okres pooperacyjny notowano występowanie zdarzeń niepożądanych.

Tabela 3 przedstawia częstość obserwowanych zdarzeń wczesnych dla modelu 6900 (< 30 dni w przypadku zdarzeń niepożądanych związanych z zastawką), liniowo przedstawia częstość zdarzeń późnych (> 30 dni po zabiegu) oraz aktuarialną częstość zdarzeń niepożądanych po 1 roku, 5 latach i 8 latach po zabiegu. Częstość występowania zdarzeń niepożądanych pochodzą od 363 pacjentów w dziewięciu ośrodkach. Zbiorczy czas obserwacji wyniósł 1100 pacjentolat ze średnim czasem obserwacji wynoszącym 3,0 roku (SD = 2,4 roku, zakres = 0 do 8,2 lat). Przedoperacyjne i pochodzące z okresu operacji dane demograficzne pacjentów zostały przedstawione w tabelach 5 i 7. Wyniki dotyczące skuteczności operacji zostały przedstawione w tabelach 9 i 11.

Przeprowadzono jedno (1) wieloośrodkowe, nierandomizowane, prospektywne, międzynarodowe badanie kliniczne u pacjentów z zaimplantowaną bioprotezą osierdziową zastawki mitralnej Carpentier-Edwards PERIMOUNT Plus model 6900P. U stu siedemdziesięciu pięciu (175) pacjentów przeprowadzono zabieg izolowanej wymiany zastawki mitralnej (MVR), a u 34 pacjentów zabieg wymiany

dwóch zastawek (DVR) z wymianą zastawki aortalnej na bioprotezę osierdziową zastawki aortalnej Carpentier-Edwards PERIMOUNT. W tym badaniu implantacje przeprowadzano w latach 1999-2007. Stan pacjentów oceniano przedoperacyjnie, śródoperacyjnie/przy wypisywaniu ze szpitala, po 1 roku, a następnie orocznie. Przez cały okres pooperacyjny notowano występowanie zdarzeń niepożądanych. Tabela 4 przedstawia częstość obserwowanych zdarzeń wczesnych dla modelu 6000P (s 30 dni w przypadku zdarzeń niepożądanych związanych z zastawką), liniowo przedstawia częstość zdarzeń późnych (> 30 dni po zabiegu) oraz aktuarialną częstość zdarzeń niepożądanych po 1 roku i 5 latach po zabiegu. Częstości zdarzeń niepożądanych podano w oparciu o dane dotyczące dwustu dziewięciu (209) pacjentów z siedmiu ośrodków. Łączny okres obserwacji wyniósł 873,18 pacjentolat ze średnim okresem obserwacji 4,2 roku (SD = 2,3 roku, zakres = 0 do 8,2 lat). Przedoperacyjne i pochodzące z okresu operacji dane demograficzne pacjentów zostały przedstawione w tabelach 6 i 8. Wyniki dotyczące skuteczności operacji zostały przedstawione w tabelach 10 i 12.

#### 5.2 Możliwe zdarzenia niepożadane

Zdarzenia niepożądane potencjalnie związane z zastosowaniem bioprotez zastawek serca to:

- Dławica piersiowa
- Skazy krwotoczne związane z leczeniem przeciwzakrzepowym (koagulopatia)
- Zaburzenia rytmu serca
- Zablokowanie uiścia wieńcowego
- · Zapalenie wsierdzia
- Niewydolność serca
- Niedokrwistość hemolityczna
- Hemoliza
- Krwotok
- · Miejscowe i/lub uogólnione zakażenie
- Zawał mięśnia sercowego
- Niedopasowanie protezy do pacjenta (PPM)
- · Usidlenie płatka zastawki (wklinowanie)
- · Niestrukturalna dysfunkcja protezy
- Wytworzenie łuszczki
- Przeciek okołozastawkowy
- Niedomykalność protezy
- Strukturalne uszkodzenie protezy
- · Zakrzepica protezy
- Udar mózgu
- · Zaburzenia zakrzepowo-zatorowe
- Przemijające niedokrwienie mózgu (TIA)

Wymienione powikłania mogą prowadzić do:

- · Powtórnego zabiegu operacyjnego
- Usunięcia zastawki
- Trwałej niepełnosprawności
- Zgonu

Inne zdarzenia niepożądane, związane z zastosowaniem osierdziowej bioprotezy zastawki mitralnej Carpentier-Edwards PERIMOUNT model 6900, zebrane w literaturze oraz pochodzące z doniesień otrzymanych z systemu obsługi reklamacji firmy Edwards Lifesciences obejmują: stenozę, niedomykalność niewydolnej zastawki, perforację komory wspornikami stentów, niesprawność zastawki z powodu odkształcenia implantu, pęknięcie ramy prowadnicy drucianej.

#### 6. Badania kliniczne

Punktami końcowymi bezpieczeństwa uchwyconymi w badaniach prospektywnych były zdarzenia niepożądane; stosowano analizy krwi w celu potwierdzenia nieobecności lub obecności określonych zdarzeń niepożądanych. Wyniki bezpieczeństwa dla modelu 6900 zaprezentowano w tabeli 3, a dla modelu 6900 w tabeli 4. Przedoperacyjne dane demograficzne pacjentów dla modelu 6900 zostały przedstawione w tabeli 5, a dla modelu 6900P w tabeli 6. Operacyjne dane demograficzne pacjentów, którym wszczepiono model 6900, podano w tabeli 7, a model 6900P — w tabeli 8. Punktami końcowymi skuteczności były klasyfikacja funkcjonalna Nowojorskiego Towarzystwa Kardiologicznego (NYHA) i badania echokardiograficzne. Podsumowanie wyników klasyfikacji zawarto w tabeli 9 dla modelu 6900 i tabeli 10 dla modelu 6900 tabeli 12 dla modelu 6900 tabeli 12 dla modelu 6900 tabeli 12 dla modelu 6900 tabeli 12 dla modelu 6900.

Brak danych klinicznych wskazujących na zwiększoną odporność osierdziowej bioprotezy mitralnej Edwards model 11000M na zwapnienie, w porównaniu do innych dostępnych na rynku bioprotez.

## 7. Indywidualizacja leczenia

Biorcy bioprotez zastawek serca powinni kontynuować leczenie przeciwzakrzepowe (z wyjątkiem przypadków, w których jest ono przeciwwskazane) w pierwszym okresie po wszczepieniu — w każdym przypadku według oceny lekarza. Długoterminowe leczenie przeciwzakrzepowe i/lub przeciwpłytkowe należy rozważyć u pacjentów z czynnikami ryzyka zaburzeń zakrzepowo-zatorowych.

Ostateczną decyzję w sprawie opieki nad konkretnym pacjentem powinien podjąć personel medyczny oraz pacjent, w świetle wszystkich okoliczności dotyczących tego pacjenta (poz. 7). Bioproteza jest zalecana do MVR u pacjentów w każdym wieku, którzy nie będą przyjmować warfaryny lub mają poważne przeciwwskazania medyczne do leczenia warfaryną. Preferencje pacjenta to racjonalne kryterium przy wyborze operacji wymiany zastawki mitralnej oraz wyborze protezy mitralnej. Mechaniczna proteza jest rozsądnym wyborem do MVR u pacjentów poniżej 65 roku życia, którzy nie mają przeciwwskazania do leczenia przeciwzakrzepowego. Bioproteza jest rozsądnym wyborem do MVR u pacjentów poniżej 65 roku życia, którzy wybrali wymianę zastawki ze względów związanych ze stylem życia po szczegółowym omówieniu ryzyka leczenia przeciwzakrzepowego względem prawdopodobieństwa konieczności przeprowadzenia kolejnego zabiegu MVR (poz. 7).

#### 7.1 Szczególne grupy pacjentów

Nie potwierdzono bezpieczeństwa ani skuteczności stosowania modelu bioprotez 11000M w następujących szczególnych populacjach, ponieważ nie przebadano ich w takich grupach:

- kobiety ciężarne;
- matki karmiące;
- pacjenci z nieprawidłowym metabolizmem wapnia (np. z przewlekłą niewydolnościa nerek lub nadczynnościa przytarczyc):
- pacjenci ze schorzeniami zwyrodnieniowymi aorty powodującymi powstawanie tętniaków (np. martwica torbielowata błony środkowej, zespół Marfana);
- dzieci, młodzież lub młode osoby dorosłe.

Przestroga: Na podstawie doniesień w piśmiennictwie na temat zastawek tkankowych (poz. 9, 10, 11, 12 i 13) wydaje się występować zwiększony odsetek zwapnienia listków u pacjentów w wieku poniżej 20 lat. Jeśli jest to możliwe, należy unikać powtarzanych dożylnych wstrzyknięć preparatów zawierających wapń w okresie pooperacyjnym, a u dzieci także nadmiernego spożycia mleka oraz nabiału. Wyniki badań prowadzonych na zwierzętach (poz. 14) wskazują, że wysoki poziom wapnia w organizmie może prowadzić do wczesnego powstawania zwapnień.

## 8. Informacja dla pacjenta

Po operacji zaleca się uważną i stałą obserwację lekarską (przynajmniej jedna wizyta rocznie), aby umożliwić rozpoznanie i właściwe leczenie powikłań związanych z bioprotezą, szczególnie wynikających z uszkodzenia materiału. Pacjentom z bioprotezą, którzy są w grupie podwyższonego ryzyka bakteriemii (np. mają być poddani zabiegom stomatologicznym), warto doradzić profilaktyczną terapię antybiotykową. Pacjentom należy doradzać, aby zawsze nosili przy sobie Kartę danych wszczepu oraz informowali pracowników służby zdrowia o posiadanym implancie przy zasięganiu porady lekarskiej.

#### Sposób dostarczania

#### 9.1 Opakowanie

Osierdziowa bioproteza mitralna Edwards model 11000M jest dostarczana w postaci jałowej i niepirogennej w opakowaniu tacowym z podwójną ochroną. Opakowanie tacowe z podwójną ochroną mieści się w torebce foliowej, która znaiduie się w kartonie.

Każda bioproteza umieszczona jest w kartonie ze wskaźnikiem temperatury widocznym przez okienko na panelu bocznym. Wskaźnik temperatury przeznaczony jest do umożliwienia identyfikacji produktów narażonych na przejściowe skrajne warunki temperaturowe. W chwili otrzymania bioprotezy należy niezwłocznie sprawdzić wskaźnik i zapoznać się z etykietą kartonu, aby potwierdzić stan "Do wykorzystania". Jeśli stan "Do wykorzystania" nie jest oczywisty, nie należy używać bioprotezy i skontaktować się z lokalnym dostawcą lub przedstawicielem firmy Edwards Lifesciences w celu dokonania ustaleń dotyczących potwierdzenia zwrotu i wymiany.

Ostrzeżenie: Dokładnie sprawdzić bioprotezę przed implantacją pod kątem dowodów ekspozycji na skrajne temperatury lub innych uszkodzeń.

## 9.2 Przechowywanie

Osierdziową bioprotezę mitralną Edwards model 11000M należy przechowywać w temperaturze 10°C do 25°C (50-77°F), w torebce foliowei i kartonie, na półce.

## 10. Wskazówki dotyczące użycia

## 10.1 Szkolenia lekarzy

Techniki wszczepiania niniejszej bioprotezy są zbliżone do technik stosowanych przy wszczepianiu innych stentowych bioprotez zastawki mitralnej. Specjalne przeszkolenie lekarzy nie jest konieczne do wykonywania implantacji osierdziowei bioprotezy mitralnei Edwards model 11000M.

#### 10.2 Kalibrowanie

Przestroga: Do określania rozmiaru bioprotezy 11000M nie należy używać kalibratorów zastawkowych innych producentów ani kalibratorów przeznaczonych do innych protez zastawkowych firmy Edwards Lifesciences.

Przestroga: Sprawdzić kalibratory i rękojeści pod kątem zużycia, takiego jak stępienie, pękanie lub spękanie włoskowate. W razie zauważenia jakichkolwiek objawów zużycia kalibrator lub rękojeść należy wymienić.

Ostrzeżenie: Fragmenty rękojeści i kalibratorów nie są radiologicznie nieprzezroczyste i nie można ich lokalizować za pomocą zewnętrznego urządzenia obrazującego.

Sprawdzić, czy akcesoria zostały wyjałowione zgodnie z zalecanymi instrukcjami dostarczonymi z akcesoriami wielorazowymi.

Czarne znaczniki na krawędzi odpowiadają czarnym szwom znacznikowym na pierścieniu do wszywania. Wyznaczają one przednią część pierścienia do wszywania bioprotezy, która powinna zostać umieszczona naprzeciw przednie międzyspoidłowej części naturalnego pierścienia, aby objąć obszar odpływu z lewej komory. Wysokość i lokalizacja wsporników stentów jest oznaczona na kalibratorze 1173R, aby pomóc w optymalnym wyrównaniu i osadzeniu.

Kalibratory są dostarczane z wstępnie przymocowanymi rękojeściami, które wydłużają rękojeść dla lepszego dostępu w przypadku trudnych warunków, głębokiej klatki piersiowej lub dostępu minimalnie inwazyjnego. Przyłączenie do kalibratora rękojeści tylnej zapewnia nieograniczany wgląd przez cylinder do komory celem oceny struktur podzastawkowych. Kalibratory 1173B i 1173R są oznaczone rozmiarem bioprotezy.

## Krok Postępowanie

Ustalanie wymiarów za pomocą kalibratora cylindra 1173B:

Aby ustalić wymiary za pomocą kalibratora cylindra 1173B, należy przełożyć część cylindryczną kalibratora przez pierścień zastawki mitralnej. Upewnić się, że część cylindryczna jest położona bezpośrednio w płaszczyźnie pierścienia zastawki mitralnej.



Ustalanie wymiarów za pomocą kalibratora 1173R: Aby ustalić wymiary za pomocą kalibratora 1173R, należy przeprowadzić część cylindryczną kalibratora przez pierścień zastawki mitralnej w taki sposób, aby końcówka kalibratora (symulująca część pierścienia do wszywania bioprotezy) spoczywała na górnej krawedzi pierścienia.



Inne techniki, jak zastosowanie podkladek, fałdowanie (reefing) płatków lub zachowywanie mitralnego aparatu podzastawkowego mogą dodatkowo zmniejszać rozmiar pierścienia zastawki mitralnej, a tym samym rozmiar bioprotezy do wszczepienia (poz. 8). Przy stosowaniu tych technik zaleca się ponownie określić rozmiar pierścienia dla uniknięcia wszczepienia zbyt dużej bioprotezy. Spójna wydolność osierdziowych bioprotez mitralnych Edwards model 11000M czyni wszczepianie zbyt dużego rozmiaru protezy niepotrzebnym do osiągnięcia pożądanej wydolności hemodynamicznej u wiekszości pacientów (tabela 11 i 12).

Ze względu na elastyczne właściwości struna może zostać wydłużona przez system uchwytu Tricentrix podczas implantacji, jednak skurczy się po usunięciu uchwytu, chwytając płatki i zaburzając funkcję zastawki. Kalibratory 1173B i 1173B są wykonane z przezroczystego materiału, aby aparat podzastawkowy był widoczny podczas dobierania rozmiaru. Należy upewnić się, że żadna ze strun nie znaidzie się na drodze rozpórek.

Przestroga: Przy stosowaniu technik zachowania aparatu podzastawkowego należy zachować szczególną ostrożność, aby nie doszło do uchwycenia strun ścięgnistych w rozpórce.

Ostrzeżenie: Unikać stosowania zbyt dużego rozmiaru bioprotezy. Stosowanie zbyt dużego rozmiaru może spowodować uszkodzenie bioprotezy lub miejscowe naprężenia mechaniczne, których skutkiem może być uszkodzenie serca, zniszczenie tkanki płatków, zniekształcenie stentu i przepływ fali zwrotnej.

## 10.3 Instrukcje dotyczące manipulacji i przygotowania

Zaleca się przeprowadzenie szkolenia w miejscu pracy przed rozpoczęciem manipulacji i przygotowania osierdziowej bioprotezy mitralnej Edwards, model 11000M.

| Krok | Postępowanie |
|---|---|
| 1 | Przestroga: Nie otwierać opakowania osierdziowej<br>bioprotezy mitralnej Edwards model 11000M przed<br>upewnieniem się, że dojdzie do implantacji. |
| | Ostrzeżenie: Nie otwierać torebki foliowej w polu<br>jałowym. Torebka foliowa stanowi jedynie osłonę<br>zabezpieczającą. Jedynie najbardziej wewnętrzne<br>opakowanie tacowe można wprowadzać do pola<br>jałowego. |
| | Po wyborze odpowiedniego rozmiaru bioprotezy należy, poza<br>polem jałowym, wyjąć z kartonu torebkę foliową. Przed<br>otwarciem należy sprawdzić, czy opakowanie nie jest<br>uszkodzone i czy nie brakuje pieczęci lub czy nie są one<br>uszkodzone. |
| 2 | Należy przytrzymać podstawę tacy zewnętrznej w pobliżu pola jałowego i oderwać pokrywe tacy zewnętrznej. |

## Krok Postepowanie 3 Taca wewnętrzna i jej zawartość sa jałowe. Należy przełożyć tace wewnetrzna do pola jałowego. Przy postępowaniu z wewnetrzną tacą należy stosować jałowe techniki chirurgiczne w celu unikniecia skażenia. Przestroga: Nie otwierać wewnętrznego opakowania przed upewnieniem się, że dojdzie do implantacji, a

także dopóki chirurg nie przygotuje się do umieszczenia zastawki.

> Przestroga: Bioproteza nie jest przymocowana do tacy wewnętrznej. Należy ostrożnie odrywać pokrywe i usuwać plastikowa osłonę.

Przed otwarciem należy sprawdzić, czy taca wewnętrzna i pokrywa nie sa uszkodzone, poplamione i czy nie brakuje pieczeci lub czy nie są one uszkodzone. Należy przytrzymać podstawę tacy wewnętrznej i oderwać pokrywę tacy wewnętrznej.

5 Aby uzyskać dostęp do bioprotezy, należy usunąć plastikową osłonę przez pociągnięcie za obie zakładki. Wyrzucić plastikową osłonę.





#### Krok Postepowanie

Przymocować rekojeść do systemu uchwytu Tricentrix, gdy bioproteza znajduje się jeszcze na tacy. W celu połaczenia należy włożyć rekojeść do uchwytu i obracać zgodnie z ruchem wskazówek zegara do momentu napotkania wyraźnego oporu.



Przestroga: Bioprotezy nie należy chwytać rękoma ani za pomoca narzedzi chirurgicznych.

Przestroga: Należy zwrócić uwagę, by w trakcie mocowania nie dopuścić do zaplątania etykiety z numerem servinym wokół rekojeści.

Przestroga: Zespół rękojeść/uchwyt jest potrzebny w trakcie implantacji i nie należy go usuwać do momentu przyszycia bioprotezy do pierścienia.

7 Po zamocowaniu rękojeści wyjąć cały zespół (tj. plastikowy rękaw, zaczep, system uchwytu Tricentrix i bioproteze) z tacy. Rękaw plastikowy jest luźno nałożony na zacisk i może pozostać na tacy. Nie wpłynie to na stosowanie produktu.

HVT53



# Krok Postonowanie Krok Postępowanie Uchwyciwszy plastikowy rękaw lub zacisk, kontynuować rotację w celú przezwyciężenia oporu do momentu, gdy biały słupek uchwytu znajdzie się w pozycji odblokowanej. CP1089-23 Lub CP1089-6 CP1089-8 CP1089-9 Zablokowany **Odblokowany** Należy nacisnąć z wymaganą siłą uchwyt, tak aby biały słupek uchwytu wsunął się między płatki i zabłokował się w ostatecznej pozycji otwartej. Osiągnięcie ostatecznej pozycji jest sygnalizowane odgłosem kliknięcia. 8 CP1089-24

| Krok | Postępowanie |
|---|---|
| 9 | Przestroga: Jeżeli podczas otwierania systemu uchwytu<br>Tricentrix nie popchnięto rękojeści z odpowiednią siłą,<br>układ namiotowy nie będzie zabezpieczony i nie będzie<br>w stanie zminimalizować możliwości uchwycenia szwów. |
| | Zawsze należy sprawdzać właściwe rozstawienie. Pomiędzy<br>niebieskim adapterem i szarym uchwytem nie powinno być<br>wolnego miejsca. Zespół uchwyt-słupek nie powinien być w<br>stanie się dalej przesuwać. |
| | Biały słupek uchwytu powinien wystawać przez płatki, podczas<br>gdy trzy spoidla powinny być lekko odchylone w stronę<br>centralnej częśd bioprotezy. Płatki będą chwilowo zmarszczone<br>przez opuszczony biały słupek uchwytu. Po wyjęciu uchwytu po<br>wszczepieniu płatki powrócą do normalnej pozycji. HVT56 |
| 10 | Po opuszczeniu wyjąć rękaw (jeżeli jest przyłączony) przez<br>przytrzymanie rękojeści i wyciągnięcie rękawa z zacisku.<br>(P1089-25 |
| 11 | Zdjąć zacisk przez zsunięcie go z uchwytu w kierunku bocznym.<br>CP1089-26 |
| | CF1000-20 |
| | Należy wyrzucić rękaw i zacisk. |

| Krok | Destanavania |
|---|---|
| Krok | Postępowanie |
| 12 | Do każdego pierścienia do wszywania bioprotezy dołączona jest etykieta z numerem seryjnym. Należy sprawdzić, czy numer seryjny jest zgodny z numerem na opakowaniu bioprotezy i kartą danych implantacji bioprotezy. Etykiety nie należy odrywać od bioprotezy przed upewnieniem się, że dojdzie do wszczepienia. |
| | Przestroga: W przypadku zauważenia jakiejkolwiek<br>różnicy w numerze seryjnym należy zwrócić nieużywaną<br>bioprotezę. |
| | Przestroga: Należy zwrócić szczególną uwagę na to, aby<br>podczas usuwania etykiety z numerem seryjnym<br>uniknąć nacięcia lub rozerwania tkaniny pierścienia do<br>wszywania. |
| | Przestroga: By uniknąć uszkodzenia tkaniny pierścienia<br>do wszywania, nie należy przeciągać supła szwu z<br>etykietą z numerem seryjnym przez pierścień do<br>wszywania. |
| 13 | Osierdziowa bioproteza mitralna Edwards model 11000M <b>NIE WYMAGA PŁUKANIA</b> przed implantacją. |
| | Przestroga: Jeśli bioproteza zostanie wypłukana przed implantacją, należy ją utrzymywać w stanie nawodnienia jałowym roztworem soli fizjologicznej po obu stronach tkanki płatka przez pozostały czas trwania zabiegu chirurgicznego. Zaleca się przepłukiwanie co jedną lub dwie minuty. |
| | Przestroga: Należy unikać kontaktu tkanki płatka z<br>ręcznikami, płótnem i innymi źródłami materii pylastej,<br>która może zostać przeniesiona na tkankę płatka. |

| Krok | Postępowanie |
|---|---|
| 1 | Chirurg powinien znać zalecenia dotyczące doboru rozmiarów oraz umiejscowienia protezy ponad pierścieniem (Patrz 10.2 Kalibrowanie). |
| | Ze względu na złożoność i rodzaje operacji wymiany zastawki<br>serca wybór techniki chirurgicznej, odpowiednio<br>zmodyfikowanej zgodnie z wcześniej opisanymi<br>Ostrzeżeniami, zależy od decyzji chirurga. Zasadniczo należy<br>wykonać następujące kroki: |
| | Chirurgicznie usunąć zmienione chorobowo lub uszkodzone<br>płatki zastawki i wszystkie związane z nią struktury<br>konieczne do usunięcia. |
| | Chirurgicznie usunąć wapń z pierścienia w celu<br>zapewnienia odpowiedniego umieszczenia pierścienia do<br>wszywania bioprotezy i niedopuszczenia do uszkodzenia<br>delikatnej tkanki płatka. |
| | Odpowiednio dobrać rozmiar. Zmierzyć pierścień,<br>posługując się wyłącznie modelami kalibratorów<br>mitralnych 1173B i 1173R (Rysunki 1a–1b). |
| | 4. Prawidłowo osadzić protezę. |
| | Założyć szwy z umieszczonym na miejscu uchwytem w celu<br>zminimalizowania możliwości zapętlenia szwów lub<br>uchwycenia strun ściegnistych. |

#### Krok Postepowanie

Upewnić sie, że nie nastapiło uszkodzenie płatków bioprotezy podczas zakładania szwów i że nie występuje przeciek.

Przestroga: Podczas doboru wymiarów bioprotezy dla danego pacienta należy wziać pod uwage jego wymiary anatomiczne, wiek i kondycie fizyczna, aby zmnieiszyć do minimum możliwość uzvskania suboptymalnego wyniku hemodynamicznego. Jednak ostatecznego doboru bioprotezy w poszczególnych przypadkach powinien dokonać lekarz po starannym rozważeniu wszystkich zagrożeń i korzyści dla określonego pacienta.

Przestroga: Przed implantacja protezy należy w dostatecznym stopniu usunać złogi wapnia z pierścienia włóknistego u pacienta, aby uniknać uszkodzenia delikatnych płatków bioprotezy w wyniku ich kontaktu ze złogami wapnia. Należy wprowadzić kalibrator do pierścienia zastawki mitralnei. Cylinder kalibratora powinien zawsze mieścić sie swobodnie w pierścieniu.

Przestroga: Do wyboru rozmiaru bioprotezy stosować wyłacznie kalibratory 1173B lub 1173R: inne kalibratory mogą prowadzić do wyboru niewłaściwej zastawki (patrz 1.2 Opis akcesoriów). Podobnie do innych bioprotez mitralnych, osierdziowa bioproteze mitralna Edwards model 11000M wszczepia się zazwyczaj za pomocą zakładkowych szwów materacowych. Zaleca się dokonanie pomiaru pierścienia po założeniu szwów. ponieważ mogą one zmniejszyć rozmiar bioprotezy przeznaczonej do wszczepienia.

2 Prawidłowe zorientowanie bioprotezy:

> Przestroga: Rama prowadnicy drucianej bioprotezy model 11000M jest symetryczna, a trzy podpórki spoidła (rozpórki) sa rozmieszczone w równych odstepach. Jednak pierścień do wszywania został tak zaprojektowany, aby można go było użyć w określonym położeniu bioprotezy. Obrebiona cześć pierścienia do wszywania, znajdująca się pomiędzy dwoma silikonowymi wybrzuszeniami, powinna być umieszczona naprzeciw przedniej miedzyspojdłowej cześci pierścienia, obeimujac droge odpływu z lewej komory.

Kontrastujące szwy znacznikowe na pierścieniu do wszywania są przeznaczone do ułatwienia właściwego ułożenia i wskazują typowa odległość miedzyspoidłowa. Jednak odległość ta może różnić się u poszczególnych pacientów. Po lewei stronie, dwa sasiadujące ze soba czarne szwy wskazują miejsce, w którym powinien być wykonany pierwszy szew i odzwierciedlaja spoidło przednie. Po prawei stronie pojedynczy czarny szew wskazuje przybliżona lokalizacje spojdła tylnego. Dzieki wykorzystaniu powyższych pomocy w ułożeniu trzeci element powinien w sposób naturalny wypaść w miejscu (lub w pobliżu) tvlnego płatka.

Przestroga: Należy zwrócić szczególna uwage, aby nie umieścić rozpórki na wprost drogi odpływu z lewei komory, ponieważ mogłoby to upośledzić długookresowa wydolność hemodynamiczną.

#### Krok Postepowanie

## 3 Założenie szwu:

Czarna linia prowadząca szew obiega pierścień do wszywania. Przy zakładaniu szwów na pierścieniu do wszywania można zredukować siły przesuwające pierścień przez rozmieszczanie szwów na wprost przez pierścień i w obszarze od linii prowadzącej szwy do zewnętrznej części pierścienia do wszywania.

Należy utrzymywać szwy naprężone podczas obniżania bioprotezy do pierścienia; minimalizuje to możiwoutworzenia się zapętleń szwu, które mogłyby uchwycić płatek. Wraz z w pełni wsuniętymi wspornikami stentu, gdy system uchwytu Tricentrix znajduje się na miejscu, pomaga to we wprowadzeniu szwów do ich właściwych pozycji poza rozpórkami oraz na pierścieniu do wszywania.

Przed zawiązaniem szwów należy usunąć rękojeść. Rękojeść i niebieski adapter muszą zostać usunięte razem jako zespół. Utrzymać rozmieszczenie bioprotezy w obrębie pierścienia przez delikatne chwycenie uchwytu kleszczykami lub dłonią w rękawiczce i przecięcie zielonej nitki na niebieskim adapterze. Zestaw niebieskiego adaptera i rękojeści należy wyjąć w całości jako zespół.

CP1089-27



4 Przestroga: Należy unikać zapętlenia lub uwięzienia szwu wokół otwartych elementów szkieletu, wolnych rozpórek lub wsporników spoideł bioprotezy, co mogłoby zakłócać prawidłowe działanie zastawki. Dla zminimalizowania ryzyka zapętlenia szwów należy koniecznie pozostawić uchwyt w sercu do momentu zakończenia szycia.

Jeżeli jednak pozostawienie uchwytu na miejscu ogranicza pole widzenia chirurga, wszystkie szwy przylegające do każdej z trzech rozpórek szkieletu muszą zostać związane przed przecięciem trzech zielonych nici utrzymujących uchwyt (w celu jego usuniecia).

Przestroga: Jeżeli szwy utrzymujące umieszczony uchwyt zostaną przecięte przed związaniem tych przylegających szwów, uchwyt nie będzie już minimalizować możliwości zapetlenia szwów wokół rozpórek szkieletu.

#### Krok Postepowanie

Należy w szczególności uważać, aby nie zawiązać szwów na szczytach rogów szarych odnóg uchwytu. Przed zawiązaniem każdego ze szwów trzeba sprawdzić płatki, utrzymując oba końce nici w stanie naprężenia. Odkształcenie lub ruch płatków podczas tej czynności może świadczyć o zapętleniu szwu wokół rozpórki. W żadnym momencie przed usunięciem uchwytu lub po jego usunięciu nie wolno zmniejszyć naprężenia nići, gdyż mogłoby to spowodować powstanie pętli na szwach i ewentualnie uwięzienie. Zaleca się umieszczenie lusterka chirurgicznego za płatkami po usunięciu uchwytu, aby sprawdzić każda rozpórke i właściwe umieszczenie szwów.

Przestroga: Podczas zakładania szwów przerywanych istotne jest, aby uciąć nici blisko punktów wiązania i upewnić się, aby odsłonięte końcówki nici nie stykały się z tkanka płatków (poz. 8).

System uchwytu Tricentrix usuwa się jako jedną część po zakończeniu zakładania szwów w następujący sposób:

CP1089-14



- Należy przeciąć każdy z trzech (3) widocznych zielonych szwów, używając skalpela lub nożyczek wprowadzonych wyłącznie do kanału cięcia. Nigdy nie wolno podejmować prób przecięcia szwów pod częściowo oddzielonym uchwytem, ponieważ część szwów mocujących może wpaść do komory serca. Należy unikać przecięcia oraz uszkodzenia stentu lub tkanki płatków podczas przecinania szwów.
- Po prawidłowym przecięciu wszystkich trzech (3) szwów mocujących należy usunąć z bioprotezy (jako jedną część) system uchwyth ricentrix wraz ze szwami mocującymi, używając jałowych rękawic lub zabezpieczonych kleszczyków.
- 3. Po implantacji wyjąć i wyrzucić uchwyt.

## 10.5 Czyszczenie i sterylizacja akcesoriów

Akcesoria do osierdziowej bioprotezy mitralnej Edwards, model 11000M, są pakowane oddzielnie. Rękojeść model 1126 dostarczana jest w stanie jałowym i jest przeznaczona wyłącznie do jednorazowego użytku. Rękojeści model 1111, 1117 i 1173 oraz kalibratory model 1173B i 1173B są dostarczane w stanie niejałowym i przed użyciem trzeba je umyć i wyjałowić. Należy wyczyścić i ponownie wysterylizować rękojeśći, kalibratory, podstawę i pokrywę tacy przed każdym użyciem. Instrukcje dotyczące mycia i wyjaławiania zawarte są w instrukcji stosowania dostarczanej z akcesoriami wielorazowymii.

#### 10.6 Zwrot bioprotez

Firma Edwards Lifesciences jest zainteresowania otrzymaniem odzyskanych klinicznych egzemplarzy osierdziowej bioprotezy mitralnej model 11000M do analizy. W celu zwrotu odzyskanych bioprotez należy skontaktować się z lokalnym przedstawicielem firmy.

- Nieotwarte opakowanie z nienaruszoną barierą jałową: Jeśli torebka foliowa ani tace nie zostały otwarte, bioprotezę należy zwrócić w oryginalnym opakowaniu.
- Otwarte opakowanie, lecz bioproteza nie została wszczepiona: Jeśli taca została otwarta, bioproteza nie jest już jalowa. Jeśli bioproteza nie zostanie wszczepiona, należy ją umieścićw odpowiednim utrwalaczu histologicznym, takim jak 10% formalina lub 2% aldehyd glutarowy, i zwrócić do firmy. W takich okolicznościach schłodzenie nie jest konieczne.
- Eksplantowana bioproteza: Usunięte bioprotezy należy umieszczać w odpowiednim utrwalaczu histologicznym, takim jak 10% formalina czy 2% aldehyd glutarowy, a następnie zwrócić do firmy. W takich okolicznościach schłodzenie nie jest konieczne.

## Zasady bezpieczeństwa w środowisku rezonansu magnetycznego (MR)



#### Warunki w badaniu MR

Badania pozakliniczne wykazały, że osierdziowa bioproteza mitralna Edwards model 11000M może być stosowana w środowisku MR. Pacjent z bioprotezą zastawki mitralnej 11000M może być bezpiecznie skanowany bezpośrednio po umieszczeniu implantu przy zachowaniu następujących warunków:

- Statyczne pole magnetyczne o indukcji nieprzekraczającej 3 tesli.
- Maksymalny gradient przestrzenny pola wynoszący 720 gausów/cm.
- Maksymalny raportowany w systemie MR, uśredniony dla całego ciała współczynnik absorpcji promieniowania (SAR) wynosi 3 W/kg na 15 minut skanowania.

W badaniach pozaklinicznych osierdziowa bioproteza mitralna Edwards model 11000M wywołała wzrost temperatury o nie więcej niż o 0,5°C przy maksymalnym raportowanym w systemie MR, uśrednionym dla całego ciała współczynniku absorpcji promieniowania (SAR) wynoszącym 3 W/kg na 15 minut skanowania MR w systemie o indukcji 3 T (Excite, Software G3.0-052B, General Electric Healthcare).

Jakość obrazu MR może być nieprawidłowa, jeżeli obszar badania mieści się w tym samym obszarze lub blisko bioprotezy mitralnej 11000M. Zalecana jest optymalizacja parametrów obrazowania MR.

## 12. Informacje dla pacjentów

#### 12.1 Karta identyfikacyjna badania

Karta identyfikacyjna badania jest przekazywana każdemu pacjentowi ze wszczepioną osierdziową protezą mitralną Edwards model 11000M.

#### 12.2 Materiały informacyjne dla pacjenta

Materiały informacyjne dla pacjenta można uzyskać w firmie Edwards lub u przedstawiciela klinicznego firmy Edwards.

#### 13. Piśmiennictwo

- Marchand MA., et al. Fifteen-year Experience with the Mitral Carpentier-Edwards PERIMOUNT Pericardial Bioprosthesis. Ann Thorac Surg. 2001: 71:5236-9.
- Liao K., et al. Bovine Pericardium versus Porcine Aortic Valve: Comparison of Tissue Biological Properties As Prosthetic Valves; Artificial Organs. 1992:16(4):361-5.
- Vesely I., et al. Comparison of the Compressive Buckling of Porcine Aortic Valve Cusps and Bovine Pericardium. J. Heart Valve Dis. January 1998; 7(1):34-9.
- Carpentier A. From Valvular Xenograft to Valvular Bioprosthesis (1965-1977). Med. Instrum. 1977; 11(2):98-101.
- Carpentier A., et al. Continuing Improvements in Valvular Bioprostheses. J. Thorac. Cardiovasc. Surg. 1982; 83(1):27-42.
- Arounlangsy P., et al. Histopathogenesis of early stage mitral annular calcification. J. Med Dent Sci. 2004; 51(1):35-44.
- Bonow RO., et al. ACC/AHA Guidelines for the Management of Patients With Valvular Heart Disease: A Report of the American College of Cardiology/ American Heart Association Task Force on Practice Guidelines (Committee on Management of Patients with Valvular Heart Disease). J. Am Coll Cardiol. 2006; 48:e1-148.
- Aagaard J., et al. Mitral valve replacement with total preservation of native valves and subvalvular apparatus. J. Heart Valve Dis. May 1997; 6(3):274-8; discussion 279-80.
- Jamieson, W.R.E., et al. Carpentier-Edwards Standard Porcine Bioprosthesis: Primary Tissue Failure (Structural Valve Deterioration) by Age Groups. Ann Thorac Surg 1988, 46:155-162.
- Odell, J.A. Calcification of Porcine Bioprostheses in Children. In Cohn, L. and V. Gallucci (eds): Cardiac Bioprostheses. Yorke Medical Books. New York, 1982, pp 231-237.
- Reul, G.J., et al. Valve Failure with the lonescu-Shiley Bovine Pericardial Bioprosthesis: Analysis of 2680 Patients. J. Vasc Surg 1985, 2(1):192-204.
- Sanders, S.P., et al. Use of Hancock Porcine Xenografts in Children and Adolescents. Am J. Cardiol 1980, 46(3):429-438.
- Silver, M.M., et al. Calcification in Porcine Xenograft Valves in Children. Am J. Cardiol 1980, 45:685-689.
- Carpentier, A., et al. Continuing Improvements in Valvular Bioprostheses. J. Thorac Cardiovasc Surg 1982, 83(1):27-42.

Ceny mogą ulec zmianie bez powiadomienia. Niniejszy produkt jest wytwarzany i sprzedawany zgodnie z co najmien jednym sposód następujących patentów amerykańskich: nr patentu w USA 5,928,281; 5,931,969; 5,961,549; 6,102,944; 6,245,105; 6,413,275; 6,416,547; 6,561,970; 6,585,766; 6,837,902; 6,945,997; 6,966,925; RE 40570°, 7,214,344; 7,658,763; 7,682,391; 7,972,376; 8,007,992; 8,357,387 oraz 8,632,608; i odpowiadających im patentów zarejestrowanych za granica. Ponadto trwa uzyskiwanie innych patentów.

Należy zapoznać się z objaśnieniami symboli, umieszczonymi na końcu niniejszego dokumentu.

Tabela 3: Zaobserwowane częstotliwości zdarzeń niepożądanych – MVR i DVR (Model 6900)

Wszyscy pacjenci poddani analizie: N = 363

Skumulowana liczba obserwacji: 1100 pacjentolat

| | Zdarzenia wczesne | | Zdarzenia późne <sup>1</sup> | | Bez zdarzeń niepożądanych (%) [95% CI] <sup>2</sup> | | |
|---|---|---|---|---|---|---|---|
| Powikłanie | n <sup>3</sup> | % | n | %/pacjentorok | 1 rok (n = 287) | 5 lat (n = 141) | 8 lat (n = 18) |
| Śmiertelność (całkowita) | 34 | 9,4 | 50 | 4,7 | 85,5 [81,8; 89,2] | 75,4 [70,3; 80,6] | 65,4 [57,6; 73,2] |
| Zdarzenia związane z zastawką | | | | | | | |
| Śmiertelność (związana z zastawką) | 0 | 0 | 16 | 1,5 | 97,7 [96,0; 99,4] | 95,3 [92,8;97,8] | 91,9 [87,5; 96,4] |
| Eksplantacje | 0 | 0 | 8 | 0,7 | 98,7 [98,0; 99,3] | 96,7 [95,3;98,0] | 95,6 [93,9; 97,3] |
| Powtórne operacje | 2 | 0,6 | 12 | 1,1 | 97,1 [96,2;98,1] | 95,1 [93,6; 96,6] | 93,0 [90,9; 95,1] |
| Krwotok związany z antykoagulacją | 2 | 0,6 | 9 | 0,8 | 97,1 [95,2;99,0] | 97,1 [95,2;99,0] | 94,1 [88,2; 100] |
| Zapalenie wsierdzia | 1 | 0,3 | 3 | 0,3 | 99,0 [97,9; 100] | 98,7 [97,4;98,9] | 98,7 [97,4; 98,9] |
| Hemoliza | 0 | 0,0 | 1 | 0,1 | 99,7 [99,0; 100] | 99,7 [99,0; 100] | 99,7 [99,0; 100] |
| Dysfunkcja pozastrukturalna | 0 | 0,0 | 3 | 0,3 | 100 [100; 100] | 99,3 [98,0; 100] | 98,3 [95,9; 100] |
| Przeciek okołozastawkowy<br>(wszystkie) | 1 | 0,3 | 5 | 0,5 | 98,4 [97,0; 99,8] | 98,4 [97,0; 99,8] | 97,3 [94,9; 99,8] |
| Strukturalne pogorszenie stanu<br>zastawki | 0 | 0,0 | 5 | 0,5 | 100,0 [100; 100] | 97,6 [95,2; 100] | 92,8 [85,3; 100] |
| Zaburzenia zakrzepowo-zatorowe | 5 | 1,4 | 8 | 0,7 | 97,5 [95,8;99,2] | 96,1 [93,8;98,5] | 96,1 [93,8; 98,5] |
| Zakrzepica | 0 | 0,0 | 0 | 0,0 | 100,0 [100; 100] | 100,0 [100; 100] | 100,0 [100; 100] |

#### Uwagi:

- 1. Częstości zdarzeń późnych zostały obliczone jako częstości przedstawione liniowo (%/pacjentorok) w oparciu o 1072,5 późnych pacjentolat (> 30 dni po zabiegu).
- Przebieg bez zdarzeń niepożądańych został obliczony przy użyciu metody Kaplana-Meiera. Do obliczenia standardowego blędu tych zmiennych zastosowany został wzór Greenwooda.
- n = liczba zdarzeń.

#### Tabela 4: Zaobserwowane częstotliwości zdarzeń niepożądanych (Model 6900P)

Wszyscy pacjenci poddani analizie: N = 209

Skumulowana liczba obserwacji: 873,18 pacjentolat ogółem

| Zdarzenia wczesne Zdarzenia późne¹ Bez zdarzeń niepożądanych (%) [95% CI]² | | | | danuch (OC) FOEOC (FII) | | |
|---|---|---|---|---|---|---|
| D 11 : | | | | | | , |
| Powikłanie | n <sup>3</sup> | % | n | %/pacjentorok | 1 rok | 5 lat |
| Śmiertelność (całkowita) | 3 | 1,4 | 45 | 5,3 | 93,2 [88,8; 95,9] | 74,4 [66,9; 80,5] |
| Zdarzenia związane z zastawką | | | | | | |
| Śmiertelność (związana z zastawką) | 1 | 0,5 | 12 | 1,4 | 98,5 [95,5;99,5] | 92,0 [86,2; 95,5] |
| Eksplantacje | 1 | 0,5 | 8 | 0,9 | 97,5 [94,0;98,9] | 96,5 [92,2; 98,5] |
| Powtórne operacje | 0 | 0,0 | 0 | 0,0 | 100,0 [100; 100] | 100,0 [100; 100] |
| Zdarzenia związane z krwawieniem | 5 | 2,4 | 13 | 1,5 | 96,1 [92,3; 98,0] | 91,9 [86,5; 95,2] |
| Zapalenie wsierdzia | 1 | 0,5 | 3 | 0,4 | 99,5 [96,6;99,9] | 97,1 [92,1; 98,9] |
| Dysfunkcja pozastrukturalna | 0 | 0,0 | 1 | 0,1 | 99,5 [96,4;99,9] | 99,5 [96,4; 99,9] |
| Przeciek okołozastawkowy<br>(wszystkie) | 1 | 0,5 | 2 | 0,2 | 99,5 [96,7; 99,9] | 98,4 [95,2; 99,5] |
| Strukturalne pogorszenie stanu<br>zastawki | 0 | 0,0 | 2 | 0,2 | 100,0 [100;100] | 99,0 [93,2; 99,9] |
| Zaburzenia zakrzepowo-zatorowe | 4 | 1,9 | 12 | 1,4 | 97,0 [93,5;98,7] | 91,3 [85,8; 94,7] |
| Zakrzepica | 0 | 0,0 | 0 | 0,0 | 100,0 [100; 100] | 100,0 [100; 100] |

## Uwagi:

- Czestości zdarzeń późnych zostały obliczone jako czestości przedstawione liniowo (%/pacjentorok) w oparciu o 856,24 późnych pacjentolat (> 30 dni po zabiegu).
- Przebieg bez zdarzeń niepożądanych został obliczony przy użyciu metody Kaplana-Meiera. Do obliczenia standardowego blędu tych zmiennych zastosowany został wzór Greenwooda.
- n = liczba zdarzeń.

Tabela 5: Przedoperacyjne dane demograficzne pacjentów (Model 6900)

| | | Charakterystyka badania (N = 363; łącznie 1100 pacjentolat) | |
|---|---|---|---|
| Parametr | Kategoria | n | % (n/N) <sup>1</sup> |
| Wiek w momencie wszczepienia (N = 363) | Średnia ± SD | 66,1 ± 10,7 | |
| Płeć | Kobieta/mężczyzna | 212/151 | 58,4%/41,6% |
| | Brak | 30 | 8,3% |
| Poznoznanio/stielogia | Stenoza | 91 | 25,1% |
| Rozpoznanie/etiologia | Niedomykalność | 184 | 50,7% |
| | Wada złożona | 58 | 16,0% |

#### Uwaga:

1. n = liczba pacjentów w każdej kategorii; N = liczba pacjentów w badaniu ogółem.

## Tabela 6: Przedoperacyjne dane demograficzne pacjentów (Model 6900P)

| | | | Charakterystyka badania (N = 209; łącznie 873,18 pacjentolat) |
|---|---|---|---|
| Parametr | Kategoria | n | % (n/N) <sup>1</sup> |
| Wiek w momencie wszczepienia (N = 209) | Średnia ± SD | 71,4 ± 9,4 | |
| Płeć | Kobieta/mężczyzna | 138/71 | 66,0%/34,0% |
| | Wada złożona | 48 | 23,0% |
| D | Niedomykalność | 121 | 57,9% |
| Rozpoznanie/etiologia | Stenoza | 32 | 15,3% |
| | Dysfunkcja zastawki | 8 | 3,8% |

## Uwaga:

1. n = liczba pacjentów w każdej kategorii; N = liczba pacjentów w badaniu ogółem.

Tabela 7: Operacyjne dane demograficzne pacjentów (Model 6900)

| | | Charakterystyka badania<br>(N = 363; łącznie 1100 pacjentolat) | |
|---|---|---|---|
| Parametr | Kategoria | n | % (n/N) <sup>1</sup> |
| | Choroba reumatyczna serca | 135 | 37,2% |
| | Zwapnienie | 82 | 22,6% |
| | Degeneracja | 50 | 13,8% |
| For Love 2 | Zapalenie wsierdzia | 39 | 10,7% |
| Etiologia <sup>2</sup> | Uszkodzenie bioprotezy | 15 | 4,1% |
| | Choroba niedokrwienna serca | 14 | 3,9% |
| | Nieprawidłowości wrodzone | 8 | 2,2% |
| | Inna | 44 | 12,1% |
| | Brak | 200 | 55,1% |
| | CABG <sup>3</sup> | 78 | 21,5% |
| | Zabieg naprawczy zastawki trójdzielnej | 61 | 16,8% |
| D 1 | Kontrapulsacja wewnątrzaortalna | 17 | 4,7% |
| Procedury towarzyszące <sup>2</sup> | Rozrusznik <sup>4</sup> | 6 | 1,7% |
| | Zabieg naprawczy aorty/wymiana | 5 | 1,4% |
| | Zabieg naprawczy tętniaka | 4 | 1,1% |
| | Inna | 31 | 8,5% |
| | Brak | 122 | 33,6% |
| | CAD <sup>5</sup> /CABG | 72 | 19,8% |
| | Nadciśnienie | 61 | 16,8% |
| Występujące wcześniej schorzenia <sup>2</sup> | Migotanie przedsionków | 53 | 14,6% |
| | Przebyty MI <sup>6</sup> | 45 | 12,4% |
| | Choroba naczyń mózgowych | 36 | 9,9% |
| | Inna | 234 | 64,5% |
| | 25 | 22 | 6,1% |
| | 27 | 110 | 30,3% |
| Rozmiar zastawki (mm) | 29 | 137 | 37,7% |
| | 31 | 81 | 22,3% |
| | 33 | 13 | 3,6% |

#### Uwagi:

- 1. n = liczba pacjentów w każdej kategorii; N = liczba pacjentów w badaniu ogółem
- Może być więcej niż jeden na pacjenta
   CABG = Coronary Artery Bypass Graft (Pomostowanie aortalno-wieńcowe)
- 4. Utrwalone lub napadowe
- CAD = Coronary Artery Disease (Choroba wieńcowa)
   MI = Myocardial Infarction (Zawał serca)

Tabela 8: Operacyjne dane demograficzne pacjentów (Model 6900P)

| | | Charakterystyka badania<br>(N = 209; łącznie 873,18 pacjentolat) | |
|---|---|---|---|
| Parametr | Kategoria | n | % (n/N) <sup>1</sup> |
| | Zwapnienie | 38 | 18,2% |
| | Wada wrodzona | 1 | 0,5% |
| | Zmiany zwyrodnieniowe | 105 | 50,2% |
| Etiologia <sup>2</sup> | Odległe następstwa zapalenia wsierdzia | 10 | 4,8% |
| | Niedokrwienne | 12 | 5,7% |
| | Reumatyczne | 64 | 30,6% |
| | Inna | 36 | 17,2% |
| | Brak | 91 | 43,5% |
| | Korekta zastawki/pierścienia włóknistego | 3 | 1,4% |
| | CABG <sup>3</sup> | 58 | 27,8% |
| Procedury towarzyszące <sup>2</sup> | Stały stymulator serca | 1 | 0,5% |
| | Korekta zastawki trójdzielnej/pierścienia<br>włóknistego | 21 | 10,0% |
| | Inna | 78 | 37,3% |
| | Brak | 17 | 8,1% |
| | Arytmie | 95 | 45,5% |
| | CAD <sup>4</sup> | 85 | 40,7% |
| | Kardiomiopatia | 13 | 6,2% |
| | Zastoinowa niewydolność serca | 66 | 31,6% |
| | Zapalenie wsierdzia | 14 | 6,7% |
| Występujące wcześniej schorzenia <sup>2</sup> | Zawał mięśnia sercowego | 21 | 10,0% |
| | Choroba naczyń obwodowych | 9 | 4,3% |
| | Nadciśnienie płucne | 66 | 31,6% |
| | Gorączka reumatyczna | 16 | 7,7% |
| | Nadciśnienie uogólnione | 49 | 23,4% |
| | TIA5/CVA6 | 24 | 11,5% |
| | Inna | 35 | 16,7% |
| | 25 | 28 | 13,4% |
| | 27 | 37 | 17,7% |
| Rozmiar zastawki (mm) | 29 | 84 | 40,2% |
| | 31 | 43 | 20,6% |
| | 33 | 17 | 8,1% |

## Uwagi:

- 1. n= liczba pacjentów w każdej kategorii; N= liczba pacjentów w badaniu ogółem 2. Może być więcej niż jeden na pacjenta
- CABG = Coronary Artery Bypass Graft (Pomostowanie aortalno-wieńcowe)
   CAD = Coronary Artery Disease (Choroba wieńcowa)
- 5. TIA = przejściowy atak niedokrwienny
- 6. CVA = udar mózgu
Tabela 9: Skuteczność według kryterium klasyfikacji NYHA (Model 6900)

| | Ocena<br>przedoperacyjna | | Oceny pooperacyjne | | | |
|---|---|---|---|---|---|---|
| | | | 1 do | 1 do 2 lat | | lat |
| Klasa funkcjonalna NYHA | n/N <sup>1</sup> | % | n/N | % | n/N | % |
| 1 | 11/363 | 3,0 | 120/268 | 44,8 | 40/129 | 31,0 |
| II | 73/363 | 20,1 | 90/268 | 33,6 | 25/129 | 19,4 |
| III | 192/363 | 52,9 | 15/268 | 5,6 | 1/129 | 0,8 |
| IV | 84/363 | 23,1 | 0/268 | 0,0 | 0/129 | 0,0 |
| Niedostępne | 3/363 | 0,8 | 43/268 | 16,0 | 63/129 | 48,8 |

#### Uwaga:

1. n = liczba pacjentów w każdej kategorii; N = liczba pacjentów w badaniu ogółem.

Tabela 10: Skuteczność według kryterium klasyfikacji NYHA (Model 6900P)

| | Ocena<br>przedoperacyjna | | Oceny pooperacyjne | | | |
|---|---|---|---|---|---|---|
| | | | 11 | rok | 5 lat | |
| Klasa funkcjonalna NYHA | n/N <sup>1</sup> | % | n/N | % | n/N | % |
| I | 6/209 | 2,9 | 86/187 | 46,0 | 30/96 | 31,3 |
| II | 27/209 | 12,9 | 68/187 | 36,4 | 33/96 | 34,4 |
| III | 121/209 | 57,9 | 8/187 | 4,3 | 6/96 | 6,3 |
| IV | 55/209 | 26,3 | 1/187 | 0,5 | 0/96 | 0,0 |
| Niedostępne | 0/209 | 0,0 | 24/187 | 12,8 | 27/96 | 28,1 |

#### Uwaga:

1. n = liczba pacjentów w każdej kategorii; N = liczba pacjentów w badaniu ogółem.

Tabela 11: Skuteczność, wyniki badań hemodynamicznych<sup>1</sup> (Model 6900)

| Parametr | | Wyniki w zależności od rozmiaru zastawki | | | |
|---|---|---|---|---|---|
| hemodynamiczny | 25 mm | 27 mm | 29 mm | 31 mm | 33 mm |
| Przy wypisie/krótko po in | nplantacji (n = 130 <i>,</i> 109 MV | R <sup>2</sup> i 21 DVR <sup>3</sup> ) | | | |
| Średni gradient <sup>4</sup> | n=3 | n = 23 | n=36 | n = 23 | n=3 |
| •Średnia ± SD | 5,7 ± 1,2 | 4,2 ± 1,7 | 4,2 ± 1,7 | 3,6 ± 1,0 | 7,5 ± 5,8 |
| • min., maks. | 5,7 | 2,9 | 1,8 | 2,5 | 3,14 |
| E0A <sup>5</sup> | n=1 | n = 17 | n = 22 | n = 25 | n = 5 |
| •Średnia ± SD | 1,5 | 2,9 ± 0,9 | 3,1 ± 0,9 | 2,5 ± 0,7 | 3,0 ± 1,2 |
| • min., maks. | 1,5; 1,5 | 1,3;4,1 | 1,4;4,2 | 1,5;3,8 | 1,6;4,9 |
| Fala zwrotna <sup>6</sup> | n=3 | n = 28 | n=51 | n = 40 | n = 8 |
| 0 | 3/3 (100%) | 22/28 (79%) | 36/51 (71%) | 30/40 (75%) | 4/8 (50%) |
| 1+ | 0/3 (0%) | 5/28 (18%) | 13/51 (25%) | 7/40 (18%) | 4/8 (50%) |
| 2+ | 0/3 (0%) | 0/28 (0%) | 1/51 (2%) | 3/40 (7%) | 0/8 (0%) |
| 3+ | 0/3 (0%) | 0/28 (0%) | 1/51 (2%) | 0/40 (0%) | 0/8 (0%) |
| 4+ | 0/3 (0%) | 0/28 (0%) | 0/51 (0%) | 0/40 (0%) | 0/8 (0%) |
| Niedostępne | 0/3 (0%) | 1/28 (3%) | 0/51 (0%) | 0/40 (0%) | 0/8 (0%) |
| 3–6 miesięcy po implanta | acji (n = 49, 42 MVR² i 7 DVF | R <sup>3</sup> ) | | | |
| Średni gradient <sup>4</sup> | n=5 | n = 19 | n = 15 | n=5 | n = 2 |
| • Średnia ± SD | 6,4 ± 1,7 | 5,3 ± 5 | 3,4 ± 1,2 | 4±1,9 | 4 ± 0 |
| • min., maks. | 5,9 | 2,25 | 2,6 | 2,7 | 4, 4 |
| E0A <sup>5</sup> | n=5 | n = 18 | n = 13 | n = 5 | n = 2 |
| • Średnia ± SD | 2,9 ± 0,8 | 2,6 ± 0,7 | 2,8 ± 0,6 | 2,9 ± 0,3 | 2,6 ± 1 |
| • min., maks. | 1,8;3,6 | 1,5;5 | 2;3,8 | 2,4;3,3 | 2;3,3 |
| Fala zwrotna <sup>6</sup> | n=5 | n = 21 | n = 15 | n=6 | n = 2 |
| 0 | 3/5 (60%) | 17/21 (81%) | 6/15 (40%) | 4/6 (67%) | 1/2 (50%) |
| 1+ | 0/5 (0%) | 4/21 (19%) | 8/15 (53%) | 2/6 (33%) | 0/2 (0%) |
| 2+ | 1/5 (20%) | 0/21 (0%) | 1/15 (7%) | 0/6 (0%) | 1/2 (50%) |
| 3+ | 0/5 (0%) | 0/21 (0%) | 0/15 (0%) | 0/6 (0%) | 0/2 (0%) |
| 4+ | 1/5 (20%) | 0/21 (0%) | 0/15 (0%) | 0/6 (0%) | 0/2 (0%) |
| Niedostępne | 0/5 (0%) | 0/21 (0%) | 0/15 (0%) | 0/6 (0%) | 0/2 (0%) |

Ciąg dalszy na następnej stronie.

Tabela 11: Skuteczność, wyniki badań hemodynamicznych<sup>1</sup> (Model 6900), ciąg dalszy

| Parametr | | Wyniki w zależności od rozmiaru zastawki | | | |
|---|---|---|---|---|---|
| hemodynamiczny | 25 mm | 27 mm | 29 mm | 31 mm | 33 mm |
| 1-2 lat po implantacji (n | = 131, 114 MVR <sup>2</sup> i 17 DVR <sup>3</sup> ) | | | | |
| Średni gradient <sup>4</sup> | n=3 | n = 40 | n = 47 | n = 27 | n = 4 |
| •Średnia ± SD | 5,2 ± 0,7 | 4,1 ± 1,6 | 3,5 ± 1,8 | 3,1 ± 1,4 | 2,1 ± 0,5 |
| • min., maks. | 4,7;6 | 1,7 | 1,10 | 1,7 | 1,5; 2,7 |
| E0A <sup>5</sup> | n=2 | n=35 | n = 46 | n = 29 | n = 5 |
| •Średnia ± SD | 1,8 ± 0,4 | 2,3 ± 0,6 | 2,6 ± 0,5 | 2,6 ± 0,7 | 2,5 ± 0,5 |
| • min., maks. | 1,5; 2,0 | 1,2;3,5 | 1,1;3,7 | 1,1;3,7 | 2,1;3,2 |
| Fala zwrotna <sup>6</sup> | n=4 | n = 42 | n = 51 | n = 29 | n = 5 |
| 0 | 2/4 (50%) | 31/42 (74%) | 36/51 (71%) | 17/29 (59%) | 3/5 (60%) |
| 1+ | 1/4 (25%) | 9/42 (21%) | 11/51 (21%) | 8/29 (27%) | 1/5 (20%) |
| 2+ | 1/4 (25%) | 2/42 (5%) | 4/51 (8%) | 2/29 (7%) | 1/5 (20%) |
| 3+ | 0/4 (0%) | 0/42 (0%) | 0/51 (0%) | 2/29 (7%) | 0/5 (0%) |
| 4+ | 0/4 (0%) | 0/42 (0%) | 0/51 (0%) | 0/29 (0%) | 0/5 (0%) |
| Niedostępne | 0/4 (0%) | 0/42 (0%) | 0/51 (0%) | 0/29 (0%) | 0/5 (0%) |
| 5 lat po implantacji (n = | 11, 9 MVR <sup>2</sup> i 2 DVR <sup>3</sup> ) | | | | |
| Średni gradient <sup>4</sup> | n = 0 | n = 6 | n = 5 | n = 0 | n = 0 |
| •Średnia ± SD | nie dotyczy | 8,8 ± 8,1 | 5,1 ± 2,3 | nie dotyczy | nie dotyczy |
| • min., maks. | nie dotyczy | 4, 25 | 3, 8 | nie dotyczy | nie dotyczy |
| E0A <sup>5</sup> | n = 0 | n = 2 | n = 4 | n = 0 | n = 0 |
| •Średnia ± SD | nie dotyczy | 2,0 ± 1,5 | 2,9 ± 0,6 | nie dotyczy | nie dotyczy |
| • min., maks. | nie dotyczy | 1,0;3,1 | 2,1;3,5 | nie dotyczy | nie dotyczy |
| Fala zwrotna <sup>6</sup> | n = 0 | n = 6 | n = 5 | n = 0 | n = 0 |
| 0 | 0/0 (0%) | 4/6 (66%) | 2/5 (40%) | 0/0 (0%) | 0/0 (0%) |
| 1+ | 0/0 (0%) | 1/6 (17%) | 3/5 (60%) | 0/0 (0%) | 0/0 (0%) |
| 2+ | 0/0 (0%) | 1/6 (17%) | 0/5 (0%) | 0/0 (0%) | 0/0 (0%) |
| 3+ | 0/0 (0%) | 0/6 (0%) | 0/5 (0%) | 0/0 (0%) | 0/0 (0%) |
| 4+ | 0/0 (0%) | 0/6 (0%) | 0/5 (0%) | 0/0 (0%) | 0/0 (0%) |
| Niedostępne | 0/0 (0%) | 0/6 (0%) | 0/5 (0%) | 0/0 (0%) | 0/0 (0%) |

#### Uwani

- Oceny hemodynamiczne wykonane były z zastosowaniem przezklatkowego badania echokardiograficznego (TTE) oraz w niektórych przypadkach przezprzełykowego badania echokardiograficznego (TEE).
- MVR = wymiana zastawki mitralnej
- 3. DVR = wymiana dwóch zastawek
- 4. Średni gradient wyrażony w mmHg
- EOA: Efektywne pole ujścia, cm<sup>2</sup>
- 6. Fala zwrotna = brak, 0; łagodna, 1+; umiarkowana, 2+; umiarkowana/ciężka, 3+; ciężka, 4+

Tabela 12: Skuteczność, wyniki badań hemodynamicznych (Model 6900P)<sup>1</sup>

| Parametr | Wyniki w zależności od rozmiaru zastawki | | | | |
|---|---|---|---|---|---|
| hemodynamiczny | 25 mm 27 mm | | 29 mm | 31 mm | 33 mm |
| Przy wypisie/krótko po impla | ntacji | | | | |
| Średni gradient <sup>2</sup> | n = 24 | n=35 | n = 83 | n = 42 | n = 16 |
| • Średnia ± SD | 6,4 ± 1,87 | 4,4 ± 1,52 | 3,4 ± 1,47 | 3,3 ± 1,20 | 4,0 ± 1,38 |
| • min., maks. | 3,10 | 1,96; 8 | 1,4;9 | 1,7 | 1,5; 6,91 |
| EOA3 | n = 8 | n = 27 | n=77 | n = 41 | n = 16 |
| •Średnia ± SD | 2,7 ± 0,87 | 2,8 ± 0,58 | 2,9 ± 0,93 | 2,5 ± 0,67 | 2,4 ± 0,52 |
| • min., maks. | 1,46; 4,4 | 1,5;3,9 | 1,58; 6 | 1,32; 4,2 | 1,55;3,31 |
| Fala zwrotna <sup>4</sup> | n = 27 | n=37 | n = 83 | n = 43 | n = 17 |
| Nieznaczna/brak | 19/27 (70%) | 29/37 (78%) | 76/83 (92%) | 39/43 (91%) | 15/17 (88%) |
| 1+ łagodna | 6/27 (22%) | 7/37 (19%) | 7/83 (8%) | 4/43 (9%) | 1/17 (6%) |
| 2+ umiarkowana | 1/27 (4%) | 1/37 (3%) | 0/83 (0%) | 0/43 (0%) | 0/17 (0%) |
| 3+ umiarkowana/ciężka | 0/27 (0%) | 0/37 (0%) | 0/83 (0%) | 0/43 (0%) | 1/17 (6%) |
| 4+ ciężka | 0/27 (0%) | 0/37 (0%) | 0/83 (0%) | 0/43 (0%) | 0/17 (0%) |
| Niedostępne | 1/27 (4%) | 0/37 (0%) | 0/83 (0%) | 0/43 (0%) | 0/17 (0%) |
| 3–6 miesięcy po implantacji | | | | | |
| Średni gradient <sup>2</sup> | n = 0 | n = 4 | n=3 | n = 2 | n = 0 |
| •Średnia ± SD | 0 ± 0 | 4,4 ± 2,25 | 2,3 ± 0,89 | 6,6 ± 2,05 | 0 ± 0 |
| • min., maks. | 0, 0 | 2,5;7,5 | 1,3;3 | 5,1;8 | 0, 0 |
| E0A <sup>3</sup> | n = 0 | n=3 | n=3 | n = 1 | n = 1 |
| •Średnia ± SD | 0 ± 0 | 2,4 ± 0,74 | 3,2 ± 0,88 | 2,5 ± 0,00 | 1,2 ± 0,00 |
| • min., maks. | 0, 0 | 1,6;3 | 2,3; 4,05 | 2,47; 2,47 | 1,22; 1,22 |
| Fala zwrotna <sup>4</sup> | n = 0 | n = 5 | n=3 | n = 2 | n = 2 |
| Nieznaczna/brak | 0 | 3/5 (60%) | 2/3 (67%) | 2/2 (100%) | 2/2 (100%) |
| 1+łagodna | 0 | 1/5 (20%) | 1/3 (33%) | 0/2 (0%) | 0/2 (0%) |
| 2+ umiarkowana | 0 | 1/5 (20%) | 0/3 (0%) | 0/2 (0%) | 0/2 (0%) |
| 3+ umiarkowana/ciężka | 0 | 0/5 (0%) | 0/3 (0%) | 0/2 (0%) | 0/2 (0%) |
| 4+ ciężka | 0 | 0/5 (0%) | 0/3 (0%) | 0/2 (0%) | 0/2 (0%) |
| Niedostępne | 0 | 0/5 (0%) | 0/3 (0%) | 0/2 (0%) | 0/2 (0%) |

Ciąg dalszy na następnej stronie.

Tabela 12: Skuteczność, wyniki badań hemodynamicznych (Model 6900P)<sup>1</sup>, ciąg dalszy

| | ı | | | | |
|---|---|---|---|---|---|
| Parametr | | Wyniki | w zależności od rozmiaru z | astawki | |
| hemodynamiczny | 25 mm | 27 mm | 27 mm 29 mm | | 33 mm |
| 1 rok po implantacji | | | | | |
| Średni gradient <sup>2</sup> | n = 16 | n = 27 | n = 63 | n=34 | n = 15 |
| • Średnia ± SD | 5,9 ± 2,36 | 4,0 ± 1,45 | 3,0 ± 1,61 | 3,3 ± 1,26 | 3,4 ± 1,25 |
| • min., maks. | 3, 12 | 2,7 | 1, 12 | 1,5;7 | 1,9;6,3 |
| E0A3 | n=3 | n = 21 | n = 59 | n=32 | n = 15 |
| • Średnia ± SD | 2,3 ± 0,16 | 2,4 ± 0,76 | 2,6 ± 0,74 | 2,5 ± 0,67 | 2,3 ± 0,83 |
| • min., maks. | 2,09; 2,4 | 1,27;4,76 | 1,5;5,7 | 1,5;4 | 1,2;3,8 |
| Fala zwrotna <sup>4</sup> | n = 20 | n = 28 | n = 65 | n=34 | n = 16 |
| Nieznaczna/brak | 17/20 (85%) | 24/28 (86%) | 53/65 (82%) | 29/34 (85%) | 13/16 (81%) |
| 1+ łagodna | 3/20 (15%) | 3/28 (11%) | 6/65 (9%) | 3/34 (9%) | 3/16 (19%) |
| 2+ umiarkowana | 0/20 (0%) | 0/28 (0%) | 3/65 (5%) | 2/34 (6%) | 0/16 (0%) |
| 3+ umiarkowana/ciężka | 0/20 (0%) | 0/28 (0%) | 1/65 (2%) | 0/34 (0%) | 0/16 (0%) |
| 4+ ciężka | 0/20 (0%) | 0/28 (0%) | 0/65 (0%) | 0/34 (0%) | 0/16 (0%) |
| Niedostępne | 0/20 (0%) | 1/28 (4%) | 2/65 (3%) | 0/34 (0%) | 0/16 (0%) |

#### Uwagi:

- 1. Oceny hemodynamiczne wykonane były z zastosowaniem przezklatkowego badania echokardiograficznego (TTE) oraz w niektórych przypadkach przezprzełykowego badania echokardiograficznego (TEE).

  Średni gradient wyrażony w mmHg

  EOA: Efektywne pole ujścia, cm²

- 4. Fala zwrotna = Nieznaczna/brak, 0; łagodna, 1+; umiarkowana, 2+; umiarkowana/ciężka, 3+; ciężka, 4+

This page intentionally left blank. ■ Cette page est intentionnellement laissée blanche. ■ Niniejsza strona pozostaje pusta.

## Symbol Legend • Légende des symboles • Legenda Symboli

| | English | Français | Polski | Γ | | English | Français | Polski |
|---|---|---|---|---|---|---|---|---|
| REF | Catalogue<br>Number | Numéro de<br>référence | Numer<br>Katalogowy | | STER <b>I</b> LE EO | Ethylene<br>Oxide<br>Sterilized | Stérilisé<br>à l'oxyde<br>d'éthylène | Wysterylizowano<br>Przy Użyciu<br>Tlenku Etylenu |
| <u>^</u> | Caution | Attention | Przestroga | | | Do not use | Ne pas utiliser | Nie używać, |
| Ţ <u>i</u> | Consult<br>instructions<br>for use | Consulter<br>le mode<br>d'emploi | Zapoznać się<br>z instrukcją<br>użycia | 11 | 8 | if package<br>is opened or<br>damaged. | si l'emballage<br>est ouvert ou<br>endommagé. | jeśli opakowanie<br>jest otwarte<br>lub uszkodzone. |
| 2 | Single Use | À usage<br>unique | Do<br>jednorazowego<br>użytku | | EC REP | European<br>Authorized<br>Representative | Mandataire<br>européen | Autoryzowany<br>przedstawiciel<br>w Europie |
| # | Quantity | Quantité | llość | | | Contents<br>sterile and | Contenu stérile et<br>apyrogène si le | Zawartość<br>sterylna i |
| $\square$ | Use By | Utiliser avant | Zużyć Do | | STERILE 388 | nonpyrogenic<br>if package is<br>unopened or | conditionnement<br>n'est ni ouvert ni<br>endommagé. | niepirogenna, o ile<br>opakowanie nie<br>zostało otwarte |
| SN | Serial<br>Number | Numéro<br>de série | Numer<br>Serii | | | undamaged. | | ani uszkodzone. |
| | Manufacturer | Fabricant | Producent | | <b>₽</b> 25 °C | Do not freeze -<br>Store between | Ne pas<br>congeler- | Nie zamrażać -<br>Przechowywać w |
| SZ | Size | Taille | Rozmiar | | 10-7 | 10 °C and 25 °C | Conserver entre<br>10°C et 25°C | temperaturze od<br>10 °C do 25 °C |

Note: Not all symbols may be included in the labeling of this product. • Remarque: il est possible que certains symboles n'apparaissent pas sur les étiquettes de ce produit. • Uwaga: Nie wszystkie symbole muszą być użyte na etykietach niniejszego produktu.

GLX3SL5x7.1



EC REP

Edwards Lifesciences Services GmbH Edisonstr. 6

85716 Unterschleissheim Germany

Manufacturer \*\*\* Edwards Lifesciences LLC One Edwards Way Irvine, CA 92614-5688 USA Made in USA

Telephone 949.250.2500 FAX

800.424.3278 949.250.2525

3/14 199663003 A ©Copyright 2014, Edwards Lifesciences LLC All rights reserved.

> DATA MATRIX BARCODE FPO

# Vendor: Do Not Print this page. For Internal Edwards Lifesciences Use Only.

| | Title: IFU, 11000N | Title: IFU, 11000M, IDE, E, F, P | | | |
|---|---|---|---|---|---|
| | Part Number: 19966 | 53003 Rev.: A | | Page <b>61</b> of <b>61</b> | ECR: 118879 |
| Edwards<br>Irvine, CA 92614 | Graphic Artist: Glen | n Getler | | | Date: 3/6/14 |
| First<br>Proofer: Lenor | e Dunn | Date: 3/7/14 | Second<br>Proofer | | Date: |
| Full Proofed Against Redline Docuproof X | | | | Full X Proofed Against Redline X Docuproof | |
| First n/a Date: n/a | | | Second Proofer: Theresa Menchaca Date: 3/7/14 | | |
| Pages: n/a | | | | Pages: 1 - 19, 49 - 61 | |
| First n/a | | Date: <b>n/a</b> | Second | | Date: 3/7/14 |
| Proofer: n/a Date: n/a | | | | Proofer: Lee VIDDER Date: 3///14 | |
| Pages: <b>n/a</b> | | | Pages: 20 - 48 | | |

#### NOTE

- 1. ALL ART PRINTS 100% BLACK UNLESS OTHERWISE NOTED.
- 2. PROOF IS 100% OF ACTUAL PRINTED SIZE.

<u>INK</u> Black **EDWARDS LIFESCIENCES LLC**CLINICAL INVESTIGATIONAL PLAN

## ATTACHMENT C - INFORMED CONSENT FORM TEMPLATE

REVISION J: 03 MARCH 2021

#### SAMPLE INFORMED CONSENT – Model 11000A

## **Subject Information**

## CLINICAL TRIAL # 2012-02 (AORTIC CONSENT FORM, CONTINUED FOLLOW-UP)

Prospe**C**tive, n**O**n-rando**M**ized, **M**ultic**EN**ter **C**linical evaluation of the **E**dwards Pericardial Aortic & Mitral Bioprostheses (Models 11000A and 11000M) with a new tissue treatment platform (COMMENCE TRIAL)

You are invited to take part in a clinical research trial. This information sheet tells you why the research is being done and what it would involve for you if you chose to take part. Please read the following information carefully and feel free to discuss this with your family or your doctor. If you are unclear about anything or would like more information, please contact, <Name> on <Tel. number>. Give yourself time to decide whether or not you wish to take part. Your participation in this research trial is voluntary. If you decide to participate, we will ask you to sign this document in order to state your agreement. This trial is given a favorable opinion by the Institutional Review Board and by the US Food and Drug Administration (FDA). It will be conducted according to the regulations governing clinical research. A description of this clinical trial will be available on http://www.ClinicalTrials.gov, as required by U.S. Law. This Web site will not include information that can identify you. At most, the Web site will include a summary of the results. You can search this Web site at any time.

#### Introduction

The heart contains four (4) valves, which allow the blood to flow in the correct direction. When a valve does not work properly, the heart has to work harder in order to pump the required amount of blood to the body. This may cause symptoms that depend on the valve that is damaged and the amount of the damage. If the damage is serious, surgery to remove and replace the damaged valve with a new valve is recommended.

## What is the purpose of this trial?

The objective of this trial is to confirm that modifications to tissue processing, valve sterilization, and packaging of the FDA-approved (P860057/S042) Carpentier-Edwards PERIMOUNT Magna Ease Pericardial Bioprosthesis, Model 3300TFX (designated as the Edwards Pericardial Aortic Bioprosthesis, Model 11000A) do not raise any new questions of safety and effectiveness in subjects who require replacement of their native or prosthetic aortic valve. The only differences between the Model 3300TFX and the Model 11000A are modifications in tissue processing, valve sterilization, and packaging. Data collected in this clinical investigation was submitted to the FDA, and the Model 11000A valve is now approved to sell in the United States. In order to obtain sufficient long-term data on the valve, up to 250 Subjects at up to 10 hospitals that consent to extended follow-up will continue to be followed in this trial for up to 10 years (an additional 5 years from original study design).

## Why am I asked to participate to this research trial?

You are being asked to continue to participate in this trial because continued follow up beyond the original 5 year duration is a request by the FDA so that Edwards may obtain long term

performance data on the valve that you received. This new aortic valve was developed to treat subjects having aortic valve disease like you.

## Trial design

Up to 700 aortic valve replacement subjects and up to 175 mitral valve replacement subjects in up to 40 hospitals located throughout the United States, Canada, Europe and Asia Pacific will be enrolled in this trial. Your participation in this trial will not change your planned surgical treatment as all enrolled subjects will receive the Model 11000A valve, unless contraindicated by the trial doctor. The entire length of the trial is expected to last up to 10.5 years. Your participation will last for 10 years. You will be asked to return to the hospital where the surgery was done and be checked by the trial doctor or his/her colleagues. You will be assessed at discharge, 1 month, at 3 months, 12 months, and annually thereafter for 10 years from the time of implant of the Model 11000A valve into your heart. Please note the 1 month visit will be conducted by phone.

## Description of the Edwards Pericardial Aortic Bioprosthesis, Model 11000A

The Edwards Pericardial Aortic Bioprosthesis, Model 11000A is an FDA-approved device. The Model 11000A valve is an FDA-approved Carpentier-Edwards PERIMOUNT Magna Ease 3300TFX valve, with modifications in tissue processing, valve sterilization, and packaging.

The Magna Ease valve consists of three tissue leaflets made of bovine (cow) pericardium (heart tissue). These leaflets have been treated with a new Edwards tissue process, built on the FDA-approved Edwards ThermaFix process to stabilize and preserve tissue. This process also allows the Model 11000A to be stored in non-liquid packaging and to not require rinsing prior to implant.

## How was the valve under investigation tested?

The valve was tested, on animals and in bench-top laboratory testing, in conformity with the U.S. Regulations. The valve also has been implanted in 133 patients in Europe. Preliminary results of these tests to date have shown that the valve is suitable for implant in humans.

The technique used for implanting the valve is the same as your doctor uses with other biological heart valves. Each of the trial doctors involved in this clinical trial is properly trained on how to implant the Model 11000A valve.

The Model 11000A valve is being tested in ongoing clinical trials inside and outside the United States.

## What will happen to me if I take part?

If you agree to participate in this trial, you will be treated like any other subject having a similar operation and you also will have some more tests (described below) to collect more information about the valve and the surgery.

The decision about participating in this trial is entirely yours. Please make sure that all your questions are addressed before you make a decision. If you consent to participate, we will ask you to sign and date this informed consent form. A copy of this form will be given to you.

The trial doctor will then ask you questions and will run tests and procedures to see if you qualify for trial participation. These tests and procedures include:

- Your blood pressure, heart rate, height, and weight will be measured (physical exam)
- Your medical history and your current medications will be reviewed
- Your blood will be collected for laboratory testing. The blood draw will consist of a needle being stuck into a vein in your arm (or other area where a vein can be accessed). Approximately two tablespoons (30 mL) of blood will be drawn at this visit for routine tests including a complete blood count, plasma free hemoglobin, or haptoglobin or serum LDH, coagulation profile, and serum creatinine to test for kidney function. Any remaining blood sample will be discarded according to hospital regulations.
- An electrocardiogram (a test using a machine that records the electrical activity of your heart. The recording is done by putting self adhesive discs on your chest)
- An echocardiogram (a test using a machine that creates sound waves creating pictures of inside your heart. A small probe is put on the outside of your chest)
- The severity of your health will be graded using a standard scale by the New York Heart Association (NYHA) based on your ability to do physical activities
- You will complete a questionnaire to assess your quality of life
- If you are a woman of child-bearing age (and are not sterile) a small amount of blood or urine will be obtained to check for pregnancy

If the results of the tests and examinations do not meet the trial requirements and your doctor assesses that you are not qualified to participate in the trial, you will be excluded from the trial and the trial doctor will discuss with you an alternative treatment for your disease. No further commitments related to this trial will be requested from you.

If, as a result of the above mentioned tests and examinations, your doctor assesses that you are qualified to participate in the trial, you will be scheduled for surgery. Upon your approval, your personal physician will be informed of your participation in the clinical trial.

Similar to other aortic valve replacement operations, this surgical procedure is performed under general anesthesia. The cardiac surgeon reaches the heart by making a cut in the chest and opening the sternum [breast bone]. The beating of the heart is stopped and the blood circulation will continue using a "heart-lung" machine.

If during surgery your trial doctor finds a reason not to implant the Model 11000A valve, you will receive an FDA-approved aortic valve. You will not have any further commitments related to this trial.

If your trial doctor determines that there are no contraindications, you will receive the Model 11000A valve and you will be considered enrolled in the trial.

During your surgery after the Model 11000A valve is implanted, a small tube used as a probe for a transesophageal echocardiogram (TEE) will be entered through your mouth and advanced down to the area of the heart. The doctor will use this echocardiogram to take pictures of your heart. This is part of every surgery to replace a heart valve.

If the Model 11000A valve is replaced with another FDA-approved aortic valve at any time after enrollment, you will be followed for 30 days or until any symptoms or side effects you may

experience have resolved. Your investigational valve may be removed or explanted and sent to the Sponsor or an independent lab for further analysis.

After your surgery and before you go home, you will have some more tests and examinations as described below:

- Your blood pressure, heart rate and weight will be measured (physical exam)
- Your current medications will be recorded
- Blood tests (including a complete blood count, plasma free hemoglobin or haptoglobin or serum LDH and coagulation profile)
- An electrocardiogram (once right after your procedure, and once before you go home)
- An echocardiogram will be obtained to see that the newly implanted Model 11000A valve sits well in its position and that it works well
- You will be asked if you have experienced any unusual symptoms or side effects since the procedure any finding will be recorded in order to control your health status

At 1 month after your surgery, you will be called and asked to provide information about your health status:

- Your current medications will be recorded
- Your health condition will be graded based on your ability to perform physical activities (NYHA class)
- You will be asked if you have experienced any unusual symptoms or side effects since your last assessment
- An appointment will be scheduled for you to return to the trial center approximately at 3 months from your procedure date

During your 3 month and subsequent annual follow-up visits, you will be asked to provide information about your health status and you will undergo the following procedures:

- Your blood pressure, heart rate and weight will be measured (physical exam)
- Your current medications will be recorded
- Blood tests (including a complete blood count, plasma free hemoglobin or haptoglobin or serum LDH, and coagulation profile)
- An electrocardiogram
- An echocardiogram
- Your health condition will be graded based on your ability to perform physical activities (NYHA class)
- You will complete a questionnaire that will help your doctor to assess your quality of life (only at 12 month follow-up)
- You will be asked if you have experienced any unusual symptoms or side effects since your last assessment

## Participant responsibilities

If you decide to participate in this research trial, you will have to follow the instructions given by your trial doctor and his colleagues and return to the hospital for all the follow-up visits until the tenth follow up year. Completing all trial visits is important to make sure that the trial results are complete and accurate. If you wish to stop participating in the trial or if you find you have not followed instructions listed above, it is important that you notify the trial doctor or research staff.

Your participation in this research trial is **entirely voluntary** and it is your right to refuse to participate or withdraw at any time without penalty or loss of benefits to which you are otherwise entitled. You are free to withdraw from the trial at any time without giving any reason, even if you have confirmed in writing that you want to take part. Your decision to withdraw will not have any adverse effect whatsoever on your further treatment in our hospital.

Giving false, incomplete, or misleading information about your medical history, including past and present use of medications, could have a very serious effect on your health. It is very important that you give a true and complete medical history.

## What are the possible benefits of taking part?

There are no guaranteed benefits from participation in this clinical investigation.

Potential benefits resulting from this clinical trial include:

- improvement of aortic valve function
- acute relief of symptoms related to aortic stenosis
- improvement in morbidity and mortality compared to similar/conventional devices

In addition, information gained from the conduct of this trial may be of benefit to other people with the same medical condition in the future. The long-term results of using the investigational valve are not known at the present time.

Alternative treatments include palliative medical therapy, aortic balloon valvuloplasty (opening the narrowed aortic valve with a balloon catheter) and surgical replacement of the aortic valve with another brand of prosthesis.

## What are the possible risks/inconveniences of taking part?

You must understand that the treatment of choice for your condition is a heart valve replacement and that alternative valves are available.

As with all prosthetic heart valves, there is a possibility that serious complications, sometimes leading to death, could develop that were not anticipated. In addition, complications and inconveniences due to individual subject reaction to an implanted device, or to physical or chemical changes in the components, particularly those of biological origin may occur, necessitating reoperation and replacement of the prosthetic device. These risks will be explained to you by your trial doctor. Unforeseeable risks may also occur. Should any side effects occur, they will be fully assessed and you will be monitored closely.

You may experience events and/or outcomes that may include, but are not necessarily limited to, the following:

## Known/potential risks associated with the use of stented bioprosthetic heart valves include but are not limited to:

- Angina (chest pain or other pain from the heart)
- Bleeding diatheses/coagulopathy related to anticoagulant therapy (increased susceptibility to bleeding)
- Cardiac arrhythmias (change in or blockage of the heartbeat rhythm)
- Cardiac failure
- Coronary ostial blockage (blockage of opening of coronary artery)
- Endocarditis (infection of the valve)
- Hemolysis/Hemolytic anemia (breaking open of red blood cells with release of hemoglobin)
- Hemorrhage (bleeding)
- Immunological response
- Leaflet entrapment (impingement)
- Myocardial infarction (heart attack)
- Nonstructural valve dysfunction
- Malfunctions of valve due to distortion at implant, fracture of wireform, physical and or chemical deterioration of valve components

- Paravalvular/Perivalvular leak (blood leaking around the valve when it is closed)
- Patient prosthetic mismatch (PPM)
   (inappropriate sizing)
- Regurgitation/insufficiency (blood leaking through the valve when it is closed)
- Stenosis (narrowing of the valve)
- Thromboembolism/stroke
   (blood clot breaking off from the
   valve and causing blockage in the
   circulation downstream)
- Tissue deterioration including infection, calcification, thickening, perforation, degeneration, suture abrasion, instrument trauma, and or leaflet detachment
- Transient ischemic attack (TIA) (mini-stroke)
- Valve pannus (excessive tissues growth around the valve)
- Valve thrombosis (blood clot attachment to the valve)

## <u>Potential risks associated with aortic valve replacement surgery include but are not limited to</u>:

- Allergic reaction
- Annular dissection (tear in the tissue around valve opening)
- Aortic/arterial dissection (tear in the artery)
- Bleeding, anticoagulant related (related to blood thinners)
- Bleeding, procedural/postprocedural (during or after surgery)

- Cardiac arrest (heart stops beating)
- Cardiogenic shock (not enough blood being pumped by the heart)
- Disseminated intravascular coagulation (DIC) (the blood clots too much)
- Esophageal rupture (tear or hole in the tube that connects the mouth to the stomach)

- Heart failure
- Hematoma (localized collection of blood)
- Heparin induced thrombocytopenia (HITs) (low platelet count in blood due to medication)
- Hypertension/Hypotension (blood pressure that is too low or too high)
- Hypoxemia (lack of oxygen)
- Infection, local or wound
- Infection, systemic (body-wide, called septicemia)
- Myocardial Infarction (heart attack)
- Multi-system organ failure (MOF) (example liver and or kidneys stop working)
- Pericardial effusion (fluid around the heart)
- Pericardial tamponade (a large amount of fluid around the heart

- such that is interferes with its normal performance)
- Pleural effusion (fluid around the lungs)
- Pulmonary edema (fluid in the lungs)
- Pneumonia (infection of the lungs)
- Renal dysfunction (kidney function worsening)
- Respiratory failure (lung failure where the level of oxygen in the blood becomes dangerously low)
- Thromboembolism (blood clot)
  - Venous, peripheral or central (blood clot in vein)
  - Arterial, peripheral or central (blood clot in artery)
  - Pulmonary, thrombus (blood clot in lung)

These complications may manifest clinically as symptoms including but not limited to abnormal heart murmur, exercise intolerance, shortness of breath, anemia, and/or fever.

It is possible that these complications could lead to:

- Reoperation
- Explant (removal of the valve)
- Permanent disability
- Death

Risks associated with the Model 11000A are anticipated to be the same as listed above for other aortic bioprosthetic valves and valve replacement surgery.

You may require anti-coagulant therapy (a substance that prevents clotting of the blood) as a result of having your aortic valve replaced with the Model 11000A valve. You may require long-term anti-platelet therapy (aspirin, unless there is a reason you should not take it) even if long-term anti-coagulant therapy is not required.

Post procedural anti-coagulant and anti-platelet medications include the risk of causing severe bleeding and heavy blood loss. Because of this risk, anyone taking these drugs must take care to avoid injuries. Any falls, blows to the body or head, or other injuries should be reported to a physician, as internal bleeding may occur without any obvious symptoms. Post procedural anti-coagulation and associated risks are no different with the investigational valve than with valves already approved by the FDA.

## Risks from taking a blood sample

You will have routine blood samples taken from a vein in your arm by a needle stick. Risks associated with drawing blood from your arm include slight discomfort and/or bruising. Infection, bleeding, clotting, or fainting also are possible, although unlikely. The number of times that you will have a blood sample drawn for this trial is maximal 8 times over approximately 5 years. At maximum, two tablespoons (30 mL) of blood will be taken at a single visit.

## Risks from an electrocardiogram

In rare circumstances, a rash or irritation at the location of the electrocardiogram electrode placement can occur due to the adhesive. If this should occur, it will be assessed and treated using clinical standards of care with appropriate medication(s) and/or compresses.

## Risks from an echocardiogram

A lubricant (gel) is used on the skin to improve picture quality and this may feel cold. There are no known risks associated with receiving a transthoracic echocardiogram.

## Risks from an transesophageal echocardiography (TEE)

The few risks of TEE involve passing the probe from your mouth down into your throat and esophagus. You may have a sore throat for a day or two. In very rare cases, TEE causes the esophagus to bleed.

## If I decide against participating in the clinical trial what other options do I have?

If you decide not to participate in this trial, you can discuss with your doctor which options of heart valve replacement best suit your requirements. There are a number of brands of bioprosthetic valves available. Alternatives available to you may include continuation of your current heart medications and treatments without having surgery to replace your aortic valve. It is important that you discuss these other options with your doctor. This does not in any way affect your further clinical care.

## What if something goes wrong?

Your doctor and Edwards Lifesciences LLC will take all appropriate efforts to prevent any injury or illness which may occur as a result of your participation in this trial. If you suffer any injury or illness as a direct result of participating in this trial, you will receive medical care and treatment at this hospital. Call your trial doctor immediately. Signing this consent does not affect any legal rights you have.

### Will my taking part in this trial be kept confidential?

The records of this trial will be kept confidential. This section explains how your medical records might be used and disclosed if you agree to participate in this trial.

All physicians involved in the trial follow a strict clinical protocol. You have the right to determine who has access to your health records. Records collected in this trial includes your medical history, the results of physical exams, lab tests and other diagnostic procedures as described

above in this consent form, as well as basic demographic information and data related to your trial treatment.

By signing this form:

- You allow the research staff and/or the trial doctor to use your medical records for the trial and to disclose your health information to the Sponsor, Edwards Lifesciences LLC, or to the sponsor's representatives, in order to review the results of the trial and to monitor the safety of participants.
- You allow the trial doctor and/or sponsor to publish the results of the trial or discuss the
  results at conferences. If this is done, no information will be included that would reveal
  your identity.

The information sent by the trial doctor and/or research staff to the Sponsor will not include your name, address, or other identifiers. Instead, the trial doctor will assign a coded number to the records that are provided to the Sponsor. However, your entire medical record may be reviewed at the trial doctor's office and/or hospital by the Sponsor and/or Sponsor representatives, by regulatory/government agencies including the Food and Drug Administration (FDA) and the independent Institutional Review Board (IRB - a committee formally selected to approve, review and monitor research involving human subjects), and/or other regulatory agencies in other countries. The purpose of these reviews is to assure the safety and well-being of trial participants and the quality of the clinical trial.

The trial doctor and/or research staff will make every effort to protect the privacy of your information. However, absolute confidentiality cannot be guaranteed because of the need to disclose information as described above.

This authorization does not have an expiration date. If you do not cancel this authorization then it will remain in effect indefinitely.

You can cancel this authorization at any time by giving a written notice to the trial doctor. If you cancel this authorization, then you no longer will be able to participate in the trial, and the information that was collected prior to canceling the authorization may still be used and disclosed to the above-mentioned parties. You will receive a signed copy of this consent for your records.

All data collected within the scope of the trial may be forwarded to other persons or institutions not authorized for direct data inspection in an anonymized form only.

## Participation and Withdrawal

You have the right to choose not to be in this trial or to stop being a part of this trial at any time without any consequences. This means that there will be no penalty or loss of medical benefits to which you are entitled.

If you choose to stop being a part of this trial, you must first notify the trial doctor immediately so that a plan can be provided for your continued medical care. At the time you stop taking part in the trial, you will be asked to return for a final safety evaluation that will include gathering information about your current medical condition and conducting any required procedures. For your own safety, you should go through the trial exit procedures any time you leave the trial and make arrangements for your continued medical care.

It is possible that your participation in this trial may be stopped at any time without asking you. This might happen if you do not follow the instructions given by the trial doctor or if the trial Sample Informed Consent

Page 9

doctor believes it is in your best interest. The trial also may be stopped for administrative, medical, or other reasons as determined by the trial doctor, the Sponsor, or regulatory authorities. Any significant new findings developed during the course of this research that might affect your willingness to participate in the trial will be provided to you and the trial doctor.

While participating in this trial, you should not take part in any other clinical trial. This is to protect you from possible injury that may arise.

## Who is organizing and funding the research?

This trial/research is organized by Edwards Lifesciences LLC, the Sponsor and the company that makes the Model 11000A valve. The clinical research staff will not be paid to include you in this trial but the hospital will be reimbursed for the costs incurred in conducting this research.

## **Costs and Compensation**

You will be billed for all charges normally associated with heart valve replacement (including trial-related visits) — only those required procedures outside of the routine standard of care will be paid for by the sponsor. There will be no financial compensation for your participation in this clinical trial.

You will be reimbursed for the travel expenses you have in order to return to the hospital for the follow-up visits required during the trial. You will still be responsible for the cost of your usual ongoing medical care, including procedures and/or non-trial drugs that are not required by this clinical research trial. If you have any questions, please ask the trial doctor, or a member of the research staff.

You understand that all forms of medical diagnosis and treatment, whether routine or trial-related, involve some risk of injury. In spite of all precautions, you might develop medical complications from participating in this research trial. You understand that the Sponsor or the hospital cannot assume liability for injury caused by the use of this particular valve or any other valve. In the event physical injury occurs as a result of participating in this research trial, the necessary facilities, emergency treatment and professional medical services will be available to you, just as they are to anyone. In the event of an unexpected injury directly related to the investigational device or the procedures described in the Clinical Research Protocol, the Sponsor will reimburse the hospital for the cost of treatment for any such injury, under the following conditions:

- The costs of treatment are not paid for by your medical or hospital insurance or coverage; and
- The injury is not due to negligence of the Investigator or the hospital;
- The Investigator and the hospital have followed the Clinical Protocol requirements; and
- You have followed the instructions of the Investigator

You further understand that you do not waive any liability rights for personal injury by signing this form.

### Contact details for further information

| If you require any further information before or during the trial, or if you have any questions afte you have read this Subject Information Sheet/ Informed Consent, please contact the trial docto responsible for you: |
|---|
| Trial Doctor: Phone: |
| Further information |
| You consent to participate in a research trial and your data will be used in the statistical analysi |
| of that clinical trial. It is understood that your personal identifiable data continues to be subjec |
| to data protection and shall not be disclosed to any third parties. Participation in this clinical |
| trial is voluntary, and you can discontinue participation at any time without giving reasons, and |
| without penalty. The Principal Investigator or the Sponsor also may decide on your premature |
| discontinuation in this trial. |
| Signature of subject or his/her legal representative |
| I have received written information about the clinical trial or the information was read out to me and I had sufficient time to read this through and think about it. I also was orally informed in detail by (name of clinical investigator) about the nature significance and scope of the clinical trial; in particular about the objectives, conduct, benefit risk, and insurance coverage including the associated obligations. All my questions were answered in an understandable way. I do not have any further questions right now. I know that I can ask questions at any time, including during and after the clinical trial. |
| • I declare my voluntary consent to the clinical trial. I am aware that I can refuse to participate or withdraw my consent at any time without incurring any penalties or disadvantages. |
| <ul> <li>I agree that my medical data may be recorded in the context of this clinical trial. I agree that the medical data may be forwarded in anonymous form to authorized specialists for data processing and scientific evaluation and to the competent authorities for review.</li> </ul> |
| <ul> <li>At the same time, I agree that my health data may be recorded in the context of this clinical<br/>trial and representatives of the Sponsor or the regulatory agencies may inspect my data for<br/>review purposes.</li> </ul> |
| <ul> <li>Finally, I agree to scientific publication of the research results in compliance with provision<br/>of data protection legislation.</li> </ul> |
| I agree / I do not agree that my primary care physician may be informed about my participation in this trial. |

| Print name of trial participant | Date | Time <sup>1</sup> |
|---|---|---|
| Signature of trial participant | | |
| Print name of legal representative (if required) | Date | Time |
| Signature of legal representative (if required) | | |
| Signature of Person Obtaining Consent I have explained the clinical trial to the su his/her questions. I have the impression this document and gives his/her consent t given a copy of the signed consent form. | that he/she under | stands the information contained in |
| Name of Person Obtaining Consent (printed) | Date | Time |
| Signature of Person Obtaining<br>Consent | Clinic | |

<sup>&</sup>lt;sup>1</sup> Required only if consent is taken on the same day as the trial procedure

#### SAMPLE INFORMED CONSENT- Model 11000M

## **Subject Information**

## CLINICAL TRIAL # 2012-02 (MITRAL CONSENT FORM, CONTINUED FOLLOW-UP)

Prospe**C**tive, n**O**n-rando**M**ized, **M**ultic**EN**ter **C**linical evaluation of the **E**dwards Pericardial Aortic & Mitral Bioprostheses (Models 11000A & 11000M) with a new tissue treatment platform (COMMENCE TRIAL)

You are invited to take part in a clinical research trial. This information sheet tells you why the research is being done and what it would involve for you if you chose to take part. Please read the following information carefully and feel free to discuss this with your family or your doctor. If you are unclear about anything or would like more information, please contact, <Name> on <Tel. number>. Give yourself time to decide whether or not you wish to take part. Your participation in this research trial is voluntary. If you decide to participate, we will ask you to sign this document in order to state your agreement. This trial is given a favorable opinion by the Institutional Review Board and by the US Food and Drug Administration (FDA). It will be conducted according to the regulations governing clinical research. A description of this clinical trial will be available on http://www.ClinicalTrials.gov, as required by U.S. Law. This Web site will not include information that can identify you. At most, the Web site will include a summary of the results. You can search this Web site at any time.

## Introduction

The heart contains four (4) valves, which allow the blood to flow in the correct direction. When a valve does not work properly, the heart has to work harder in order to pump the required amount of blood to the body. This may cause symptoms that depend on the valve that is damaged and the amount of the damage. If the damage is serious, surgery to remove and replace the damaged valve with a new valve is recommended.

## What is the purpose of this trial?

The objective of this trial is to confirm that modifications to tissue processing, valve sterilization, and packaging of the FDA-approved (P860057/S068) Carpentier-Edwards PERIMOUNT Magna Mitral Ease Pericardial Bioprosthesis, Model 7300TFX, which will be designated as the Edwards Pericardial Mitral Bioprosthesis Model 11000M, do not raise any new questions of safety and effectiveness in subjects who require replacement of their native or prosthetic mitral valve. The only differences between the Model 7300TFX and the Model 11000M are modifications in tissue processing, valve sterilization, and packaging. Data collected in this clinical investigation was submitted to the FDA, and the Model 11000M valve is now approved to sell in the United States. In order to obtain sufficient long-term data on the valve, up to 25 Subjects at select hospitals that consent to extended follow-up will continue to be followed in this trial for up to 10 years (an additional 5 years from original study design).

## Why am I asked to participate to this research trial?

You are being asked to continue to participate in this trial as requested by the FDA so that Edwards may obtain long term safety and performance data on the valve that you received. This new mitral valve was developed to treat subjects having mitral valve disease like you.

### Trial design

Up to 700 aortic valve replacement subjects and up to 175 mitral valve replacement subjects in up to 40 hospitals located throughout the United States, Canada, Europe and Asia Pacific will be enrolled in this trial. Your participation in this trial will not change your planned surgical treatment as all enrolled subjects will receive the Model 11000M valve, unless contraindicated by the trial doctor. The entire length of the trial is expected to last up to 10.5 years. Your participation will last for 10 years. You will be asked to return to the hospital where the surgery was done and be checked by the trial doctor or his/her colleagues. You will be assessed at discharge, 1 month, 3 months, 12 months, and annually thereafter for 10 years from the time of implant of the Model 11000M valve into your heart. Please note the 1 month visit will be conducted by phone.

### Description of the Edwards Pericardial Mitral Bioprosthesis, Model 11000M

The Edwards Pericardial Mitral Bioprosthesis, Model 11000M is an FDA-approved device. The Model 11000M valve is an FDA-approved Carpentier-Edwards PERIMOUNT Magna Mitral Ease 7300TFX valve, with modifications in tissue processing, valve sterilization, and packaging.

The Magna Mitral Ease valve consists of three tissue leaflets made of bovine (cow) pericardium (heart tissue). These leaflets have been treated with a new Edwards tissue process, built on the FDA-approved Edwards ThermaFix process to stabilize and preserve tissue. This process also allows the Model 11000M to be stored in non-liquid packaging and to not require rinsing prior to implant.

## How was the valve under investigation tested?

The valve was tested on animals and in bench-top laboratory testing, in conformity with the U.S. Regulations. The results of these tests to date have shown that the valve is suitable for implant in humans.

The technique used for implanting the valve is the same as your doctor uses with other biological heart valves. Each of the trial doctors involved in this clinical trial is properly trained on how to implant the Model 11000M valve.

The Model 11000M valve is being tested in ongoing clinical trials.

## What will happen to me if I take part?

If you agree to participate in this trial, you will be treated like any other subject having a similar operation and you also will have some more tests (described below) to collect more information about the valve and the surgery.

The decision about participating in this trial is entirely yours. Please make sure that all your questions are addressed before you make a decision. If you consent to participate, we will ask you to sign and date this informed consent form. A copy of this form will be given to you.

The trial doctor will then ask you questions and will run tests and procedures to see if you qualify for trial participation. These tests and procedures include:

- Your blood pressure, heart rate, height, and weight will be measured (physical exam)
- Your medical history and your current medications will be reviewed
- Your blood will be collected for laboratory testing. The blood draw will consist of a needle being stuck into a vein in your arm (or other area where a vein can be accessed). Approximately two tablespoons (30 mL) of blood will be drawn at this visit for routine tests including a complete blood count, plasma free hemoglobin or haptoglobin or serum LDH coagulation profile, and serum creatinine to test for kidney function. Any remaining blood sample will be discarded according to hospital regulations.
- An electrocardiogram (a test using a machine that records the electrical activity of your heart. The recording is done by putting self-adhesive discs on your chest)
- An echocardiogram (a test using a machine that creates sound waves creating pictures of inside your heart. A small probe is put on the outside of your chest)
- The severity of your health will be graded using a standard scale by the New York Heart Association (NYHA) based on your ability to do physical activities
- You will complete a questionnaire to assess your quality of life
- If you are a woman of child-bearing age (and are not sterile) a small amount of blood or urine will be obtained to check for pregnancy

If the results of the tests and examinations do not meet the trial requirements and your doctor assesses that you are not qualified to participate in the trial, you will be excluded from the trial and the trial doctor will discuss with you an alternative treatment for your disease. No further commitments related to this trial will be requested from you.

If, as a result of the above mentioned tests and examinations, your doctor assesses that you are qualified to participate in the trial, you will be scheduled for surgery. Upon your approval, your personal physician will be informed of your participation in the clinical trial.

Similar to other mitral valve replacement operations, this surgical procedure is performed under general anesthesia. The beating of the heart is stopped and the blood circulation will continue using a "heart-lung" machine.

If during surgery your trial doctor finds a reason not to implant the Model 11000M valve, you will receive an FDA-approved mitral valve. You will not have any further commitments related to this trial.

If your trial doctor determines that there are no contraindications, you will receive the Model 11000M valve and you will be considered enrolled in the trial.

During your surgery after the Model 11000M valve is implanted, a small tube used as a probe for a transesophageal echocardiogram (TEE) will be entered through your mouth and advanced down to the area of the heart. The doctor will use this echocardiogram to take pictures of your heart. This is part of every surgery to replace a heart valve.

If the Model 11000M valve is replaced with another FDA-approved mitral valve at any time after enrollment, you will be followed for 30 days or until any symptoms or side effects that you may experience have resolved. Your investigational valve may be removed or explanted and sent to the Sponsor or an independent lab for further analysis.

After your surgery and before you go home, you will have some more tests and examinations as described below:

- Your blood pressure, heart rate and weight will be measured (physical exam)
- Your current medications will be recorded
- Blood tests (including a complete blood count, plasma free hemoglobin or haptoglobin or serum LDH and coagulation profile)
- An electrocardiogram (once right after your procedure, and once before you go home)
- An echocardiogram will be obtained to see that the newly implanted Model 11000M valve sits well in its position and that it works well
- You will be asked if you have experienced any unusual symptoms or side effects since the procedure – any finding will be recorded in order to control your health status

At 1 month after your surgery, you will be called and asked to provide information about your health status:

- Your current medications will be recorded
- Your health condition will be graded based on your ability to perform physical activities (NYHA class)
- You will be asked if you have experienced any unusual symptoms or side effects since your last assessment
- An appointment will be scheduled for you to return to the trial center approximately at 3 months from your procedure date

During your 3 month and subsequent annual follow-up visits, you will be asked to provide information about your health status and you will undergo the following procedures:

- Your blood pressure, heart rate and weight will be measured (physical exam)
- Your current medications will be recorded
- Blood tests (including a complete blood count, plasma free hemoglobin or haptoglobin or serum LDH, and coagulation profile)
- An electrocardiogram
- An echocardiogram
- Your health condition will be graded based on your ability to perform physical activities (NYHA class)
- You will complete a questionnaire that will help your doctor to assess your quality of life (only at 12 month follow-up)
- You will be asked if you have experienced any unusual symptoms or side effects since your last assessment

## Participant responsibilities

If you decide to participate in this research trial, you will have to follow the instructions given by your trial doctor and his colleagues and return to the hospital for all the follow-up visits until the tenth follow up year. Completing all trial visits is important to make sure that the trial results are complete and accurate. If you wish to stop participating in the trial or if you find you have not followed instructions listed above, it is important that you notify the trial doctor or research staff.

Your participation in this research trial is **entirely voluntary** and it is your right to refuse to participate or withdraw at any time without penalty or loss of benefits to which you are otherwise entitled. You are free to withdraw from the trial at any time without giving any reason, even if you have confirmed in writing that you want to take part. Your decision to withdraw will not have any adverse effect whatsoever on your further treatment in our hospital.

Giving false, incomplete, or misleading information about your medical history, including past and present use of medications, could have a very serious effect on your health. It is very important that you give a true and complete medical history.

## What are the possible benefits of taking part?

There are no guaranteed benefits from participation in this clinical investigation.

Potential benefits resulting from this clinical trial include:

- improvement of mitral valve function
- acute relief of symptoms related to mitral stenosis
- improvement in morbidity and mortality compared to similar/conventional devices

In addition, information gained from the conduct of this trial may be of benefit to other people with the same medical condition in the future. The long-term results of using the investigational valve are not known at the present time.

Alternative treatments include palliative medical therapy, mitral balloon valvuloplasty (opening the narrowed mitral valve with a balloon catheter) and surgical replacement of the mitral valve with another brand of prosthesis.

### What are the possible risks/inconveniences of taking part?

You must understand that the treatment of choice for your condition is a heart valve replacement and that alternative valves are available.

As with all prosthetic heart valves, there is a possibility that serious complications, sometimes leading to death, could develop that were not anticipated. In addition, complications and inconveniences due to individual subject reaction to an implanted device, or to physical or chemical changes in the components, particularly those of biological origin may occur, necessitating reoperation and replacement of the prosthetic device. These risks will be explained to you by your trial doctor. Unforeseeable risks may also occur. Should any side effects occur, they will be fully assessed and you will be monitored closely.

You may experience events and/or outcomes that may include, but are not necessarily limited to, the following:

## Known/potential risks associated with the use of stented bioprosthetic heart valves include but are not limited to:

- Angina (chest pain or other pain from the heart)
- Bleeding diatheses/coagulopathy related to anticoagulant therapy (increased susceptibility to bleeding)
- Cardiac arrhythmias (change in or blockage of the heartbeat rhythm)
- Cardiac failure
- Coronary ostial blockage (blockage of opening of coronary artery)
- Endocarditis (infection of the valve)
- Hemolysis/Hemolytic anemia (breaking open of red blood cells with release of hemoglobin)
- Hemorrhage (bleeding)
- Immunological response
- Leaflet entrapment (impingement)
- Myocardial infarction (heart attack)
- Nonstructural valve dysfunction
- Malfunctions of valve due to distortion at implant, fracture of wireform, physical and or chemical deterioration of valve components

- Paravalvular/Perivalvular leak (blood leaking around the valve when it is closed)
- Patient prosthetic mismatch (PPM)
   (inappropriate sizing)
- Regurgitation/insufficiency (blood leaking through the valve when it is closed)
- Stenosis (narrowing of the valve)
- Thromboembolism/stroke (blood clot breaking off from the valve and causing blockage in the circulation downstream)
- Tissue deterioration including infection, calcification, thickening, perforation, degeneration, suture abrasion, instrument trauma, and or leaflet detachment
- Transient ischemic attack (TIA) (mini-stroke)
- Valve pannus (excessive tissues growth around the valve)
- Valve thrombosis (blood clot attachment to the valve)

## <u>Potential risks associated with mitral valve replacement surgery include but are not limited to</u>:

- Allergic reaction
- Annular dissection (tear in the tissue around valve opening)
- Aortic/arterial dissection (tear in the artery)
- Bleeding, anticoagulant related (related to blood thinners)
- Bleeding, procedural/postprocedural (during or after surgery)
- Cardiac arrest (heart stops beating)

- Cardiogenic shock (not enough blood being pumped by the heart)
- Disseminated intravascular coagulation (DIC) (the blood clots too much)
- Esophageal rupture (tear or hole in the tube that connects the mouth to the stomach)
- Heart failure
- Hematoma (localized collection of blood)
- Heparin induced thrombocytopenia (HITs) (low platelet count in blood due to medication)
- Hypertension/Hypotension (blood pressure that is too low or too high)
- Hypoxemia (lack of oxygen)
- Infection, local or wound
- Infection, systemic (body-wide, called septicemia)
- Myocardial Infarction (heart attack)
- Multi-system organ failure (MOF) (example liver and or kidneys stop working)

- Pericardial effusion (fluid around the heart)
- Pericardial tamponade (a large amount of fluid around the heart such that is interferes with its normal performance)
- Pleural effusion (fluid around the lungs)
- Pulmonary edema (fluid in the lungs)
- Pneumonia (infection of the lungs)
- Renal dysfunction (kidney function worsening)
- Respiratory failure (lung failure where the level of oxygen in the blood becomes dangerously low)
- Thromboembolism (blood clot)
  - Venous, peripheral or central (blood clot in vein)
  - Arterial, peripheral or central (blood clot in artery)
  - Pulmonary, thrombus (blood clot in lung)

These complications may manifest clinically as symptoms including but not limited to abnormal heart murmur, exercise intolerance, shortness of breath, anemia, and/or fever.

It is possible that these complications could lead to:

- Reoperation
- Explant (removal of the valve)
- Permanent disability
- Death

Risks associated with the Model 11000M are anticipated to be the same as listed above for other mitral bioprosthetic valves and valve replacement surgery.

You may require anti-coagulant therapy (a substance that prevents clotting of the blood) as a result of having your mitral valve replaced with the Model 11000M valve. You may require long-term anti-platelet therapy (aspirin, unless there is a reason you should not take it) even if long-term anti-coagulant therapy is not required.

Post procedural anti-coagulant and anti-platelet medications include the risk of causing severe bleeding and heavy blood loss. Because of this risk, anyone taking these drugs must take care to avoid injuries. Any falls, blows to the body or head, or other injuries should be reported to a Sample Informed Consent

Page 7

physician, as internal bleeding may occur without any obvious symptoms. Post procedural anticoagulation and associated risks are no different with the investigational valve than with valves already approved by the FDA.

## Risks from taking a blood sample

You will have routine blood samples taken from a vein in your arm by a needle stick. Risks associated with drawing blood from your arm include slight discomfort and/or bruising. Infection, bleeding, clotting, or fainting also are possible, although unlikely. The number of times that you will have a blood sample drawn for this trial is maximal 8 times over approximately 5 years. At maximum, two tablespoons (30 mL) of blood will be taken at a single visit.

## Risks from an electrocardiogram

In rare circumstances, a rash or irritation at the location of the electrocardiogram electrode placement can occur due to the adhesive. If this should occur, it will be assessed and treated using clinical standards of care with appropriate medication(s) and/or compresses.

## Risks from an echocardiogram

A lubricant (gel) is used on the skin to improve picture quality and this may feel cold. There are no known risks associated with receiving a transthoracic echocardiogram.

## Risks from an transesophageal echocardiography (TEE)

The few risks of TEE involve passing the probe from your mouth down into your throat and esophagus. You may have a sore throat for a day or two. In very rare cases, TEE causes the esophagus to bleed.

## If I decide against participating in the clinical trial what other options do I have?

If you decide not to participate in this trial, you can discuss with your doctor which options of heart valve replacement best suit your requirements. There are a number of brands of bioprosthetic valves available. Alternatives available to you may include continuation of your current heart medications and treatments without having surgery to replace your mitral valve. It is important that you discuss these other options with your doctor. This does not in any way affect your further clinical care.

## What if something goes wrong?

Your doctor and Edwards Lifesciences LLC will take all appropriate efforts to prevent any injury or illness which may occur as a result of your participation in this trial. If you suffer any injury or illness as a direct result of participating in this trial, you will receive medical care and treatment at this hospital. Call your trial doctor immediately. Signing this consent does not affect any legal rights you have.

## Will my taking part in this trial be kept confidential?

The records of this trial will be kept confidential. This section explains how your medical records might be used and disclosed if you agree to participate in this trial.

All physicians involved in the trial follow a strict clinical protocol. You have the right to determine who has access to your health records. Records collected in this trial includes your medical

history, the results of physical exams, lab tests and other diagnostic procedures as described above in this consent form, as well as basic demographic information and data related to your trial treatment.

## By signing this form:

- You allow the research staff and/or the trial doctor to use your medical records for the trial and to disclose your health information to the Sponsor, Edwards Lifesciences LLC, or to the sponsor's representatives, in order to review the results of the trial and to monitor the safety of participants.
- You allow the trial doctor and/or sponsor to publish the results of the trial or discuss the
  results at conferences. If this is done, no information will be included that would reveal
  your identity.

The information sent by the trial doctor and/or research staff to the Sponsor will not include your name, address, or other identifiers. Instead, the trial doctor will assign a coded number to the records that are provided to the Sponsor. However, your entire medical record may be reviewed at the trial doctor's office and/or hospital by the Sponsor and/or Sponsor representatives, by regulatory/government agencies including the Food and Drug Administration (FDA) and the independent Institutional Review Board (IRB - a committee formally selected to approve, review and monitor research involving human subjects), and/or other regulatory agencies in other countries. The purpose of these reviews is to assure the safety and well-being of trial participants and the quality of the clinical trial.

The trial doctor and/or research staff will make every effort to protect the privacy of your information. However, absolute confidentiality cannot be guaranteed because of the need to disclose information as described above.

This authorization does not have an expiration date. If you do not cancel this authorization then it will remain in effect indefinitely.

You can cancel this authorization at any time by giving a written notice to the trial doctor. If you cancel this authorization, then you no longer will be able to participate in the trial, and the information that was collected prior to canceling the authorization may still be used and disclosed to the above-mentioned parties. You will receive a signed copy of this consent for your records.

All data collected within the scope of the trial may be forwarded to other persons or institutions not authorized for direct data inspection in an anonymized form only.

## **Participation and Withdrawal**

You have the right to choose not to be in this trial or to stop being a part of this trial at any time without any consequences. This means that there will be no penalty or loss of medical benefits to which you are entitled.

If you choose to stop being a part of this trial, you must first notify the trial doctor immediately so that a plan can be provided for your continued medical care. At the time you stop taking part in the trial, you will be asked to return for a final safety evaluation that will include gathering information about your current medical condition and conducting any required procedures. For your own safety, you should go through the trial exit procedures any time you leave the trial and make arrangements for your continued medical care.

It is possible that your participation in this trial may be stopped at any time without asking you. This might happen if you do not follow the instructions given by the trial doctor or if the trial doctor believes it is in your best interest. The trial also may be stopped for administrative, medical, or other reasons as determined by the trial doctor, the Sponsor, or regulatory authorities. Any significant new findings developed during the course of this research that might affect your willingness to participate in the trial will be provided to you and the trial doctor.

While participating in this trial, you should not take part in any other clinical trial. This is to protect you from possible injury that may arise.

## Who is organizing and funding the research?

This trial/research is organized by Edwards Lifesciences LLC, the Sponsor and the company that makes the Model 11000M valve. The clinical research staff will not be paid to include you in this trial but the hospital will be reimbursed for the costs incurred in conducting this research.

## **Costs and Compensation**

You will be billed for all charges normally associated with heart valve replacement (including trial-related visits) — only those required procedures outside of the routine standard of care will be paid for by the sponsor. There will be no financial compensation for your participation in this clinical trial.

You will be reimbursed for the travel expenses you have in order to return to the hospital for the follow-up visits required during the trial. You will still be responsible for the cost of your usual ongoing medical care, including procedures and/or non-trial drugs that are not required by this clinical research trial. If you have any questions, please ask the trial doctor, or a member of the research staff.

You understand that all forms of medical diagnosis and treatment, whether routine or trial-related, involve some risk of injury. In spite of all precautions, you might develop medical complications from participating in this research trial. You understand that the Sponsor or the hospital cannot assume liability for injury caused by the use of this particular valve or any other valve. In the event physical injury occurs as a result of participating in this research trial, the necessary facilities, emergency treatment and professional medical services will be available to you, just as they are to anyone. In the event of an unexpected injury directly related to the investigational device or the procedures described in the Clinical Research Protocol, the Sponsor will reimburse the hospital for the cost of treatment for any such injury, under the following conditions:

- The costs of treatment are not paid for by your medical or hospital insurance or coverage; and
- The injury is not due to negligence of the Investigator or the hospital;
- The Investigator and the hospital have followed the Clinical Protocol requirements; and
- You have followed the instructions of the Investigator

You further understand that you do not waive any liability rights for personal injury by signing this form.

## **Contact details for further information**

| yo | you require any further information before or during the trial, or if you have any questions after u have read this Subject Information Sheet/ Informed Consent, please contact the trial doctor sponsible for you: |
|---|---|
| Tri | ial Doctor: Phone: |
| Fu | rther information |
| Yo | ou consent to participate in a research trial and your data will be used in the statistical analysis |
| of | that clinical trial. It is understood that your personal identifiable data continues to be subject |
| to | data protection and shall not be disclosed to any third parties. Participation in this clinical |
| tri | al is voluntary, and you can discontinue participation at any time without giving reasons, and |
| wi | thout penalty. The Principal Investigator or the Sponsor also may decide on your premature |
| dis | scontinuation in this trial. |
| I h<br>an<br>de | ave received written information about the clinical trial or the information was read out to me d I had sufficient time to read this through and think about it. I also was orally informed in trial by (name of clinical investigator) about the nature, gnificance and scope of the clinical trial; in particular about the objectives, conduct, benefit, |
| ris<br>an | k, and insurance coverage including the associated obligations. All my questions were swered in an understandable way. I do not have any further questions right now. I know that an ask questions at any time, including during and after the clinical trial. |
| • | I declare my voluntary consent to the clinical trial. I am aware that I can refuse to participate or withdraw my consent at any time without incurring any penalties or disadvantages. |
| • | I agree that my medical data may be recorded in the context of this clinical trial. I agree that the medical data may be forwarded in anonymous form to authorized specialists for data processing and scientific evaluation and to the competent authorities for review. |
| • | At the same time, I agree that my health data may be recorded in the context of this clinical trial and representatives of the Sponsor or the regulatory agencies may inspect my data for review purposes. |
| • | Finally, I agree to scientific publication of the research results in compliance with provisions of data protection legislation. |
| <br>pa | I agree / I do not agree that my primary care physician may be informed about my rticipation in this trial. |

| Print name of trial participant | Date | Time <sup>1</sup> |
|---|---|---|
| Signature of trial participant | | |
| Print name of legal representative (if required) | Date | Time |
| Signature of legal representative | | |
| (if required) | | |
| Signature of Person Obtaining Consent | | |
| I have explained the clinical trial to the sublisher questions. I have the impression this document and gives hisher consent to given a copy of the signed consent form. | that he/she unders | stands the information contained in |
| Name of Person Obtaining Consent (printed) | Date | Time |
| Signature of Person Obtaining<br>Consent | Clinic | |

<sup>&</sup>lt;sup>1</sup> Required only if consent is taken on the same day as the trial procedure Sample Informed Consent

EDWARDS LIFESCIENCES LLC
CLINICAL INVESTIGATIONAL PLAN


**ATTACHMENTS** 

## **ATTACHMENT D – CASE REPORT FORMS**

REVISION J: 03 MARCH 2021



# TRIAL NUMBER 2012-02 COMMENCE™ TRIAL - REV H

STUDY SCREENING

| Subject Study ID | | y ID | 201202 - Site# |
|---|---|---|---|
| Inc | lusio | n Crit | eria DATE OF SCREENING DE MAN MAN MAN DE L'ANDRE DE L'A |
| YES | NO | NAP | |
| | | | 1. SUBJECT IS 18 YEARS OR OLDER |
| | | | SUBJECT HAS PROVIDED WRITTEN INFORMED CONSENT PRIOR TO TRIAL PROCEDURES 2. |
| | | | IF YES, DATE OF CONSENT: |
| | | | SAME IRB OR THE SAME HEALTHCARE SYSTEM 4. SUBJECT IS DIAGNOSED WITH AORTIC OR MITRAL VALVE DISEASE REQUIRING VALVE REPLACEMENT BASED ON PRE- OPERATIVE EVALUATION |
| | | | 5. SUBJECT IS SCHEDULED TO UNDERGO PLANNED AORTIC OR MITRAL VALVE REPLACEMENT WITH OR WITHOUT CONCOMITANT BYPASS SURGERY |
| | | | SUBJECT IS SCHEDULED TO UNDERGO PLANNED AORTIC VALVE REPLACEMENT WITH OR WITHOUT RESECTION AND REPLACEMENT OF THE ASCENDING AORTA FROM THE SINOTUBULAR JUNCTION AND WITHOUT THE NEED FOR CIRCULATORY ARREST FOR HEMI ARCH OR ARCH REPLACEMENT |
| IF AN | Y RES | PONS | E BELOW IS "YES" THE SUBJECT IS NOT ELIGIBLE FOR THE STUDY |
| EXCLUSION CRITERIA | | | |
| EXCESSION CRITERIA | | | |
| YES | NO | | |
| | | 1. | SUBJECT REQUIRES EMERGENCY SURGERY |
| | | 2. | SUBJECT REQUIRES PLANNED MULTIPLE VALVE REPLACEMENT/REPAIR (WITH THE EXCEPTION OF MITRAL VALVE REPLACEMENT WITH TRICUSPID VALVE REPAIR) |
| | | 3. | SUBJECT HAS PRIOR VALVE SURGERY, WHICH INCLUDED IMPLANT OF A BIOPROSTHETIC VALVE, MECHANICAL VALVE, OR ANNULOPLASTY RING THAT WILL REMAIN IN SITU |
| | | 4. | SUBJECT REQUIRES A SURGICAL PROCEDURE OUTSIDE OF THE CARDIAC AREA (E.G. VASCULAR BYPASS) |
| | | 5. | SUBJECT REQUIRES SURGICAL REPLACEMENT OF THE AORTIC ROOT |
| | | 6. | subject has active endocarditis/myocarditis or endocarditis/myocarditis within $3$ months prior to the scheduled avr surgery |
| | | 7. | SUBJECT HAS RENAL INSUFFICIENCY AS DETERMINED BY CREATININE (S-CR) $\geq 2.5$ Mg/DL OR END-STAGE RENAL DISEASE REQUIRING CHRONIC DIALYSIS AT SCREENING VISIT |
| | | 8. | SUBJECT HAS AN MRI OR CT-SCAN CONFIRMED STROKE, CEREBROVASCULAR ACCIDENT (CVA), OR TRANSIENT ISCHEMIC ATTACK (TIA) WITHIN 6 MONTHS (180 DAYS) OF THE VALVE SURGERY |
| | | 9. | SUBJECT HAS ACUTE MYOCARDIAL INFARCTION (MI) WITHIN 30 DAYS PRIOR TO THE SCHEDULED AORTIC OR MITRAL VALVE REPLACEMENT SURGERY |
| | | 10. | SUBJECT HAS PRESENCE OF NON-CARDIAC DISEASE LIMITING LIFE EXPECTANCY TO LESS THAN 12 MONTHS |
| | | 11. | SUBJECT IS DIAGNOSED WITH HYPERTROPHIC OBSTRUCTIVE CARDIOMYOPATHY (HOCM) |
| | | 12. | SUBJECT IS DIAGNOSED WITH ABNORMAL CALCIUM METABOLISM AND HYPERPARATHYROIDISM |
| | | 13. | SUBJECT EXHIBITS A LEFT VENTRICULAR EJECTION FRACTION $\leq 20\%$ AS VALIDATED BY DIAGNOSTIC PROCEDURE PRIOR TO PLANNED VALVE SURGERY |


# TRIAL NUMBER 2012-02 COMMENCE™ TRIAL - REV H

STUDY SCREENING

| S | ubjed | ct Stud | ly ID | 201202 | | | | - | | | | Site# |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | | | 14. | SUBJECT WITH E | СНОС | ARDIO | GRAPI | HIC EVI | DENCE | OF A | N INTR | A-CARDIAC MASS, THROMBUS, OR VEGETATION |
| | | | 15. | SUPPORT, OR ME | ECHAN | NICAL \ | /ENTIL | ATION | WITHIN | <b>130</b> D | AYS PE | REQUIRING INOTROPIC SUPPORT, MECHANICAL CIRCULATORY<br>RIOR TO THE PROCEDURE |
| | | | 16. | | PENIA | | | | | | | NEMIA (HGB < 10.0 GM/L OR 6 MMOL/L), OR OMPANIED BY HISTORY OF BLEEDING DIATHESIS OR |
| | | | 17. | SUBJECT HAS A | PRIOR | ORGA | N TRA | NSPLA | NT OR | IS CUF | RRENTI | LY AN ORGAN TRANSPLANT CANDIDATE |
| | | | 18. | CURRENT OR RE | CENT | PARTI | CIPATI | ON (WI | тнім 6 | WEE | (S PRIC | OR TO SURGERY) IN ANOTHER DRUG OR DEVICE TRIAL |
| | | | 19. | SUBJECT WAS PI | REVIO | USLYI | MPLAN | ITED W | ITH TR | IAL DE | VICE ( | MODEL 11000A OR MODEL 11000M) |
| | | | 20. | SUBJECT IS PREC<br>PREGNANT DURI | | | | | | | | POTENTIAL ONLY), LACTATING, OR PLANNING TO BECOME<br>AL |
| | | | 21. | SUBJECT IS CUR | RENTL | Y INC | ARCER | ATED ( | OR UNA | ABLE T | O GIVE | VOLUNTARY INFORMED CONSENT |
| | | | 22. | SUBJECT HAS A | DOCUI | MENTE | D HIST | TORY O | F SUB | STANC | E (DRI | JG OR ALCOHOL) ABUSE WITHIN THE LAST 5 YEARS |
| | | | 23. | SUBJECT REQUIR | RES C | ONCO | MITANT | LEFT | VENTR | ICULA | R ASSI | ST DEVICE (LVAD) PLACEMENT |
| | | | BASED ON ANSWERS ABOVE, IS THIS SUBJECT ELIGIBLE FOR INTRA-OPERATIVE EVALUATION? IF YES, HAS A SURGERY DATE FOR THIS SUBJECT BEEN SCHEDULED? | | | | | | | | | |
| | | | | DATE: | | | | | | | | |
| | | | | DID THE SUBJECT PROCEDURE? | T'S EL | IGIBILI | TY FOI | R THE S | STUDY | CHAN | GE PRI | OR TO ENTERING THE OPERATING ROOM FOR THE STUDY |
| | | | | IF YES, WHY DID ADVERSE EV | | STATUS | CHAN | IGE PR | IOR TO | ENTE | RING T | HE OR? |
| | | | | SUBJECT WIT | | | NSENT | | | | | |
| II | NTRA | -OPE | RATIV | E EXCLUSIO | | | RIA | | | | | |
| | ES | NO | | | | | | | | | | |
| | | | | SUBJECT WAS HI | | | CALLY | UNSTA | BLE D | JRING | THE P | ROCEDURE REQUIRING THE PROCEDURE TO BE ABORTED PRIOR |
| | | | | SURGEON DETER<br>VALVE IMPLANT I | | | | | | E IMPL | ANTED | AFTER INTRA-OPERATIVE EVALUATION AND PRIOR TO TRIAL |
| | | | | IF YES, WHY WAS | UIRE | S A SIZ | E NOT | | | | E TRIA | L VALVE |
| | | | | IF YES, WE | | | | TIOLO | GY? | DEG | ENER | ATIVE SCHEMIC MIXED DISEASE RHEUMATIC |
| | | | | OTHER REAS | ON | | | | | ОТН | IER | |
| | | | | WAS THE SUBJEC | CT EN | ROLLE | D IN TH | HE STU | DY? | | | |
| | | | | | | | | | | | _ | |
| elet. | IATUR | | | | | | | | | • | | PATE NAME NAME NAME NAME NAME NAME NAME NAM |
| SIGN | IATURE | = | | | | | | | | | | D D M M M Y Y Y Y |

| Sub | ject Stud | y ID <b>2012</b> ( | 02 | - | | Site# | | |
|---|---|---|---|---|---|---|---|---|
| VISIT | DATE: | / | | | | | | |
| 1. Pri | mary m | | tact with subjec | | | | | |
| | | ☐ HOSPITAL/ | CLINIC VISIT | | | | | |
| | | ☐ PHONE IN | NTERVIEW | | | | | |
| | | ☐ IN-PATIEN | NT ADMISSION | | | | | |
| PHYS | SICAL A | SSESSMENT | ·<br>/ VITAL SIGNS: | 1 | | | | |
| | WEIGH | T: | | | | lbs | | |
| | HEART | RATE: | | bpm | | | | |
| | SYSTO | LIC BLOOD PF | RESSURE | mmHg | | | | |
| | DIASTO | DLIC BLOOD P | RESSURE | mmHg | | | | |
| CURR | ENT NYI | HA CLASSIFIC | CATION | | | | | |
| | | CLASS I | | | | NOT DONE | | |
| | | CLASS II | | | | NOT APPLICABLE A | T DISCHARGE | |
| | | CLASS III | | | | | | |
| | | CLASS IV | | | | | | |
| CANA | DIAN CA | ARDIOVASCUI | LAR SOCIETY (CO | S) ANGINA C | LASS | | | |
| | ☐ CLAS | S 0 | ☐ CLASS I | ☐ CLAS | S II | ☐ CLASS III | | CLASS IV |
| | ☐ UNKN | IOWN | NOT APPLICAE | BLE AT DISCHA | RGE | | | |
| CURF | RENT MI | EDICATIONS | | | | | | |
| YES | | EDICATION LIS | T WAS COLLECTED | ) | | | | |
| _ | | | | | | | | |
| ECHC | CARDI | OGRAPHY | | | | | | |
| YES | | CHOCARDIOGR | AM WAS COMPLET | ED | | | | |
| DATE | OF EXAI | M: | | _ (DD/MMM/Y | YYY) | | | |

| Sub | ject S | Study ID | 201202 | | | - | | | | Site# | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| ELEC | TRO | CARDIO | OGRAM (EC | G): | | | | | | | | | | <u> </u> |
| YES | NO | · | (20 | <b>-</b> | | | | | | | | | | |
| | | ECG W | AS COMPLETE | D | | | | | | | | | | |
| DATE | OF E\ | / A N A . | | | | | | N 4N 4 /N | ^^^ | <b>N</b> | | | | |
| | | | / CONDUCTI | | | | • | IVIIVI/ 1 | 1111 | ) | | | | |
| YES | NO | | 7 00110011 | ON DI | OTOIL | )AI10 | LO | | | | | | | |
| | | | ED WITH PERI | ЛANEN | T PACE | EMAKI | ER (IF | YES | . SPE | CIFY TYPE) | | | | |
| _ | _ | | CONTINUOUS | | | | ( | | , | , | | | | |
| | ☐ INTERMITTENT (Rate responsive/ On demand) ☐ IMPLANTED WITH IMPLANTABLE CARDIOVERTER DEFIBRILLATOR (ICD/AICD) | | | | | | | | | | | | | |
| | | IMPLAN | TED WITH IMP | LANTAI | BLE CA | RDIO' | VERT | ER D | EFIBI | RILLATOR (ICD/AICD) | | | | |
| | | SINUS R | HYTHM | | | | | | | | | | | |
| | | SINUS T | ACHYCARDIA | | | | | | | | | | | |
| | | ATRIAL | FIBRILLATION | SUPR | AVENT | RICUL | AR T | ACHY | ′CAR | DIA (INDICATE EPISODAL | - PAT | TERN | ) | |
| | | | PAROXYSMAL | (SELF- | TERMI | NATIN | IG) | | | | | | | |
| | | | PERSISTENT ( | NON-S | ELF TE | RMINA | ATING | 6) | | | | | | |
| | | ATRIAL F | LUTTER | | | | | | | | | | | |
| | | TACHYO | ARDIA-BRADY | 'CARDI | IA SYNI | DROM | ΙE | | | | | | | |
| | | VENTRI | CULAR TACHY | CARDI | A (IF YE | ES, INI | DICAT | E EP | ISOD | OAL PATTERN) | | | | |
| | | | | D/PRE | MATUF | RE VEI | NTRIC | CULAI | R CO | MPLEXES (PVC) | | | | |
| | _ | _ | SUSTAINED | | | | | | | | | | | |
| | | | | | | | SPECI | FY) | | | | | | |
| Ш | Ш | | CK (IF YES, IND | DICATE | | • | <b></b> . | | | | | | | |
| | | _ | 1 <sup>ST</sup> | l | UNI | KNOW | /N | | | | | | | |
| | | _ | 2 <sup>ND</sup><br>3 <sup>RD</sup> | | | | | | | | | | | |
| П | | _ | | ^k/ INIT | BAVEN | ITRICI | IΙΙΔR | CON | חור. | TION DELAY (IF YES, IND | I∩∆TE | RRΔ | NCH) | |
| | ш | | LEFT - COMPL | | TVAVEI | 11110 | OLAIN | 0011 | | RIGHT - COMPLETE | IOATE | DIVA | | |
| | | | LEFT- INCOMP | | | | | | | RIGHT- INCOMPLETE | | | | |
| | | | CONDUCTION | | JBANCF | E, SPF | ECIFY | : | J | 2 | | | | |
| _ | _ | | | | | | • | | | | | | | |

| Subject Study ID | 201202 | | | - | | | | | S | Site# | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| BLOOD DATA | | | | | | | | | | | | | | | | |
| YES NO BLOOD | LABS WERE I | DRAWI | N AT THI | S VIS | SIT | | | | | | | | | | | |
| QUALITY OF LIFE S | URVEY | | | | | | | | | | | | | | | |
| YES NO | RVEY COMPL | _ETED <sup>'</sup> | ? | | | | | | | | | | | | | |
| OID ANY ADVERSE | EVENTS OC | CCUR | SINCE - | THE | LAST | FOL | LOW | -UP ASS | SESSM | ENT? | | | YES | 8 | | ] NO |
| F YES, COMPLETE ADV | ERSE EVENT F | ORM | | | | | | | | | | | | | | |
| Categories include: | | | | | | | | | | | | | | | | |
| Blood and lymphatic (inclu | ding ALL bleedi | ng comp | olications) | | | | | | | | | | | | | |
| Cardiovascular –Arrhythm | ia | | | | | | | | | | | | | | | |
| Cardiovascular - Regurgita | ation | | | | | | | | | | | | | | | |
| Cardiovascular - Stenosis | | | | | | | | | | | | | | | | |
| Cardiovascular - Embolic I | Event/Valve Thro | ombosis | 3 | | | | | | | | | | | | | |
| Cardiovascular - Misc | | | | | | | | | | | | | | | | |
| Device Dysfunction | | | | | | | | | | | | | | | | |
| Gastrointestinal/Hepatic | | | | | | | | | | | | | | | | |
| Genitourinary/Renal | | | | | | | | | | | | | | | | |
| Pulmonary/Respiratory | | | | | | | | | | | | | | | | |
| Peripheral Vascular | | | | | | | | | | | | | | | | |
| Psychiatric | | | | | | | | | | | | | | | | |
| Muscular Skeletal/Dermato | ologic | | | | | | | | | | | | | | | |
| Nonspecific or Unknown B | ody System | | | | | | | | | | | | | | | |
| | | | | | | | DATE | SIGNED | | | | | | | | |
| SIGNATURE | | | | | | | | _ | D [ | _ | M | M | | Y | Y | Y |

SIGNATURE

| Subject Study ID | 201202 | | - | | | Site# | | | |
|---|---|---|---|---|---|---|---|---|---|
| VISIT DATE: D D | ./ | - <sup>/</sup> | - <sub>Y</sub> - <sub>Y</sub> | | | | | | |
| DATE OF BIRTH | / _ M | M M | / <sub>Y</sub> <del>Y</del> | | R YEAR | | AND AGE | <del>Y</del> <del>Y</del> <del>-</del> | Y |
| GENDER MALE | : FEMALE | | | | | | | | |
| _<br>□ PERI | (IF FEMALE) PERFORMED POST-MEN OTHER FORMED POSITIVE | IOPAUSAL | EGATIVE | | | | | | |
| RACE/ ETHNICITY | | | | | | | | | |
| ETHNICITY HISPANI NOT HIS RACE AMEF ASIA | CAN AMERICA<br>VE HAWAIIAN | TINO<br>OR ALASK<br>AN OR BLA | CK | SLANDER | | | | | |
| SUBJECT HEIGHT: | | | c | m 🗌 in | | | | | |
| CURRENT LEFT VEN | ITRICULAR E. | JECTION F | RACTION ( | LVEF) | % | | | | |
| □NO | E WITHIN THE N | NORMAL RAI | NGE? | ιт? | | | | | |
| | | | | | DATE _ | / | M M | / | |
| SIGNATURE | | | | | D | D M | M M | / <u>Y</u> <u>Y</u> | Y Y |

| Subject Study ID | | <b>201202</b> - Si | te# | | |
|---|---|---|---|---|---|
| Blood D | raw Date: | $\frac{1}{10^{\circ}}$ $\frac{1}$ | | | |
| Blood Para | ameters | Is this value | a within | Was the r | esult clinically |
| DONE | NOT<br>DONE | Values normal r<br>Yes | | signit | ficant? No |
| | | WHITE BLOOD CELLS (WBC): 10 <sup>3</sup> / μL | | | |
| | | RED BLOOD CELLS (RBC): ☐ 10 <sup>6</sup> /µL ☐ 10 <sup>12</sup> /L | | | |
| | | HEMOGLOBIN : | | | |
| | | HEMATOCRIT: % | | | |
| | | PLATELET COUNT : 10 <sup>3</sup> / µL | | | |
| | | COAGULATION PROFILE: INR PTT PT | | | |
| | | PLASMA FREE HEMOGLOBIN : mg/dL mmol/L g/dL OR | | | |
| | | ☐ 10 <sup>6</sup> /uL HAPTOGLOBIN: ☐ mg/dL ☐ OR | | | |
| | | SERUM LDH: IU/L | | | |
| | | DATE SIGNED | | | |
| | | | D MMM YYYY | | |

SIGNATURE

| Subje | ct Study II | 201202 | 201202 - Site# | | | | | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | | TION COLLECT | | | | | | | | | | | | IMM/ | |
| YES | NO | | | | | | | | | | | | | | |
| | | ACE OR ARB INHIE | BITOF | RS | | | | | | | | | | | |
| | | ANTICOAGULANTS | | | | | | | | | | | | | |
| | | ANTICOAGULANTS | ] W. | | | | | | DERIV <i>i</i> | | | | | | |
| | | ANTIPLATELETS | AS<br>TIC | SPIRIN<br>CLOPI<br>OPID | N – EC<br>IDINE<br>OGRE | OTRII<br>TIC<br>ELPI | LID<br>LAVIX | ENTR | OPHEI | | | | | | |
| | | CALCIUM BLOCKE<br>DIURETIC<br>LIPID LOWERING | :R | | | | | | | | | | | | |
| | | NITRATES<br>STEROIDS | | | | | | | | | | | | | |
| SIGNATU | IRE | | | | | | | | DATE | D | D | M | M | M | Y |

| | | | _ |
|------------------|--------|---|-------|
| Subject Study ID | 201202 | ı | Site# |
| | L | | |

| CARDIOVASCUL | AR ME | DICAL | HISTORY |
|--------------|-------|-------|---------|

| CARDI | OVAS | CULAR MEDICAL HISTORY |
|---|---|---|
| YES | NO | |
| П | | CORONARY ARTERY DISEASE – (INDICATE WHICH NATIVE CORONARY VESSEL HAS ≥ 50% |
| _ | _ | NARROWING) LEFT ANTERIOR DESCENDING (LAD) CORONARY ARTERY |
| | | ☐ CIRCUMFLEX CORONARY ARTERY |
| | | ☐ RIGHT CORONARY ARTERY |
| | | ☐ LEFT MAIN CORONARY ARTERY |
| | | CAROTID ARTERY DISEASE – (INDICATE THE SEVERITY OF DISEASE) |
| | Ш | CAROTID OCCLUSION (>79% DIAMETER OCCLUSION) |
| | | ☐ ≥ 50% STENOSIS BUT NO OCCLUSION |
| | | ☐ < 50% STENOSIS |
| | П | PERIPHERAL ARTERY /VASCULAR DISEASE (INDICATE WHICH SYMPTOMS THE SUBJECT HAS EXPERIENCED) |
| <u>—</u> | | ☐ CLAUDICATION |
| | | ☐ AORTIC ANEURYSM |
| | | PULMONARY HYPERTENSION |
| | ш | WHAT IS THE SEVERITY OF THE CONDITION? |
| | | ☐ MILD (PULMONARY ARTERY SYSTOLIC PRESSURE <31mmHg) |
| | | ☐ MODERATE (PULMONARY ARTERY SYSTOLIC PRESSURE 31-55mmHg) |
| | | ☐ SEVERE (PULMONARY ARTERY SYSTOLIC PRESSURE IS >55mHg) |
| | | SYSTEMIC HYPERTENSION |
| _ | _ | ☐ HAS A DOCUMENTED HISTORY OF HYPERTENSION DIAGNOSED AND TREATED WITH MEDICATION, DIET, AND/OR EXERCISE |
| | | HAS PRIOR DOCUMENTATION OF BLOOD PRESSURE >140 MMHg SYSTOLIC OR 90 MMHg DIASTOLIC FOR PATIENTS WITHOUT |
| | | DIABETES OR CHRONIC KIDNEY DISEASE; OR PRIOR DOCUMENTATION OF BLOOD PRESSURE >130 MMHG SYSTOLIC OR 80 MMHG DIASTOLIC ON AT LEAST 2 OCCASIONS FOR PATIENTS WITH DIABETES OR CHRONIC KIDNEY DISEASE |
| | | ☐ IS CURRENTLY ON PHARMACOLOGIC THERAPY TO CONTROL HYPERTENSION |
| | | CARDIOMYOPATHY |
| | Ш | PRIMARY/INTRINSIC (HYPERTROPHIC, DILATED, ETC) |
| | | ☐ SECONDARY/EXTRINSIC (ISCHEMIC, DIABETIC, ETC) |
| | П | CONGESTIVE HEART FAILURE |
| | Ш | AORTIC STENOSIS |
| | | IF YES: ☐ MILD |
| | | ☐ MODERATE |
| | | □ SEVERE |
| | | UNKNOWN |
| Ш | Ш | AORTIC INSUFFICIENCY |

| Subje | ct Study ID | 201202 | | | | - | | | | | | Site# | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | | [<br>[<br>[<br>MITRAL STENOS | +2<br>+3<br>+4<br><b>IS</b><br>YES: | TRAC<br>MILD<br>MOD<br>SEVE | ERAT | Ē | | | | | | | |
| | | [ | SE | ODER<br>EVERE | ≣ | | | | | | | | |
| | | MITRAL INSUFFI<br>[<br>[<br>[ | +1<br>+2<br>+3<br>+4 | TRAC<br>MILD<br>MOD<br>SEVE | E<br>ERAT | Έ | | | | | | | |
| | | [ | ] МО | ILD<br>ODER<br>EVERE | | | | | | | | | |
| | | PULMONARY INS<br>[<br>[<br>[<br>[ | +1<br>+2<br>+3<br>+4<br>- | NKNC<br>TRAC<br>MILD<br>MOD<br>SEVE | Y<br>E<br>ERAT | | | | | | | | |
| | | | ] МО | ILD<br>ODER<br>EVERE | | | | | | | | | |
| | | TRICUSPID INSU<br>[<br>[<br>[<br>[ | U FFICIE | NKNC<br>ENCY<br>TRAC<br>MILD<br>MOD | OWN<br>E<br>ERAT | | _ | | | | | | |
| | ☐ MY€ | | ] STE | EMI<br>N STE | _<br>MI _ | D D | / M | M<br>- M | /<br>/ | <u>Y</u> <u>Y</u> | F LAST ( | Y | CE) |

| Subject | t Study ID | 201202 | | | | - | | | | | | Si | te# | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | | | ☐ UN | | | | | | | ′ HO\ | | Y Y<br>Y MONTH<br>AGO | is ago | DID TI | HE LAS | ST MI ( | OCCUR? |
| | | IF | UNKN | NOWN | l, DID | THE E | VENT | occ | UR >5 | YEA | RS AGO | O? YES | S NO | | | | |
| | Ш | | CT EV SI SI T/ A T/ VI | ER HAINUS INUS INUS INUS INUS INUS INUS INUS | AD TH TACHY BRADY CARD FIBRI IS FLUT CARD ICULA CARD | E FOL<br>YCARI<br>YCARI<br>IA- BRI<br>ILLATI<br>PAF<br>THIS<br>TER<br>IA-BR.<br>IR TAC<br>NON<br>SUS | LOWII DIA DIA AADYO ON/SI ROXYS RSISTE A PEF ADYCA CHYCA NSUST | ARDI<br>BMAL<br>ENT<br>RMANI<br>ARDIA<br>FAINE<br>ED | A SYNVENTE | C RH | HYTHMS ME LAR TA HITION? | | NO □ | | XES | | |
| SUSTAINED OTHER CARDIAC ARRHYTHMIA PLEASE SPECIFY: HAS THE SUBJECT EVER SHOWN SIGNS OF THE FOLLOWING CONDUCTION DISTURBANCES? AV BLOCK INDICATE THE LAST RECORDED DEGREE OF AV BLOCK 1st 2nd 2nd 3rd UNKNOWN BUNDLE BRANCH BLOCK/ INTRAVENTRICULAR BLOCKS INDICATE BRANCH LEFT-COMPLETE LEFT-INCOMPLETE RIGHT-COMPLETE RIGHT-INCOMPLETE RIGHT-COMPLETE RIGHT-INCOMPLETE LEFT ANTERIOR FASCULAR BLOCK LEFT POSTERIOR FASICULAR BLOCK NONSPECIFIC INTRAVENTRICULAR CONDUCTION DEFECTS OTHER CONDUCTION DISTURBANCE | | | | | | | | | | | | | | | | | |
| | _ | TRANSIENT ISO<br>IS THE DATE W<br>DA | | THE L | AST K | NOW | N TIA | occı | IRRED | KNO | OWN? | MM/YYY | Y) | | | | |

IF DATE IS UNKNOWN, APPROXIMATELY HOW MANY MONTHS AGO DID THE LAST MI OCCUR?

| Subjec | t Stud | ly ID | 20120 | 2 | | | - | | | | | | Site# | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | | | | | | | | | | | MON | NTHS AG | 9O | | | | | |
| | | | | IF UNI | KNOV | VN, DID | THE E | VENT | occi | JR >5 ` | YEAR | S AGO? | YES NO | ) <u> </u> | | | | |
| | | c | EREBROVA | ASCUL | LAR A | CCIDE | NT (CV | A/STR | OKE; | DID N | OT RE | COVER | WITHIN 24 HO | OURS) | | | | |
| | | ( | (IF YES, IND | ICATE | TYPE | E OF E | /ENTS | AND D | ATE ( | OF LAS | ST OC | CURRE | NCE) | | | | | |
| | | | | | DATE | OF LA | ST KN | OWN C | CVA | | | | | | | | | |
| | | | | | | | <u>D</u> | /_<br>D I | <u>—</u> — | | / <del>_</del> | <u></u> | - <del>- Y</del> | | | | | |
| | | | | IF DA | ATE IS | UNKN | OWN, | APPRO | XIMA | TELY | HOW | MANY <b>W</b> | EEKS AGO D | D THE | LAST | TIA O | CCUR? | |
| | | | | | | | | | | | WE | EKS AGO | ) | | | | | |
| | | | | IF UN | NKNO' | WN, DII | ) THE | EVENT | occ | UR >5 | YEAR | RS AGO? | YES N | 0 🗆 | | | | |
| | | | | OES T<br>YSFUI | | | | SEVER<br>'ES 🗌 | | _ | ENT O | F MOBIL | ITY AS A RES | ULT O | F A NE | UROL | OGICAL | |
| | | EN | NDOCARDIT | 'IS | | | | | | | | | | | | | | |
| | | | | | CUF | RENTLY | BEING | G TREA | ATED | | | | | | | | | |
| | | | | | | | | | | 3 MON | ITHS ( | NOT CU | RRENTLY BEI | NG TR | EATE | ) | | |
| | | | | | TRE | EATED : | > 3 MO | NTHS . | AGO | | | | | | | | | |
| | | MYO | CARDITIS | | | | | | | | | | | | | | | |
| | | | | | CUF | RENTLY | BEING | G TREA | ATED | | | | | | | | | |
| | | | | | | | | | | 3 MON | ITHS ( | NOT CU | RRENTLY BEI | NG TR | EATE | D) | | |
| | | | | | | ATED : | | | | | | | | | | | | |
| 닏 | | | RLIPIDEMIA | | IYPEF | RCHOLI | ESTER | OLEMI | IA | | | | | | | | | |
| | Ш | RHEU | IMATIC FEV | ER | | | | | | | | | | | | | | |
| PRIOR | CARD | OIOVA | CULAR S | URG | ICAL | . INTE | RVE | NTION | IS | | | | | | | | | |
| | | | dovascular a | | | | IE SUE | SJECT | PREV | IOUSL | -Y HAI | D? (Any | vascular interv | ention i | ncludir | ng CAE | BG, PTCA, Sten | t, |
| | | _ | 1 | | | | | | | | | | | | | | | |
| | | | 2 | | | | | | | | | | | | | | | |
| | | | 3 | | | | | | | | | | | | | | | |
| | | | ≥ 4 | | | | | | | | | | | | | | | |
| | | | HEART SUR<br>and PFO rep<br>0 | | | | | | REVIO | USLY | HAD? | (Valve re | eplacements/ r | epairs/ | valvulo | plastie | s/ | |
| | | | 1 | | | | | | | | | | | | | | | |
| | | | 2 | | | | | | | | | | | | | | | |
| | | | 3 | | | | | | | | | | | | | | | |
| | | | ≥ 4 | | | | | | | | | | | | | | | |
| HAS THE | SUBJE | ECT RE | QUIRED AN | IPUTA | TION | OF A L | IMB D | JE TO | ARTE | RIAL I | DISEA | SE? YE | S NO | | | | | |

| Subjec | ct Study ID | 201202 | | | | - | | | | | | Site# | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| HAS THE | SUBJECT | BEEN IMPLANTE | D WITI | H A PI | ERMA | NENT | PACI | EMAK | ER OF | F A | N IMPLAN | TABLE CARI | DIOVE | RTER | EFRIB | RILLATOR? |
| Yes | No | | | | | | | | | | | | | | | |
| | | AICD / PACEM | VKED | IMDI A | ΔNIT | | | | | | | | | | | |
| Ш | | SPECIFY THE | | | | IT THE | = SLIB | IECT | ндс. | | | | | | | |
| | | OI LOII I IIIL | | | | | | | | SIVE | E/ON DEMA | AND) PACEM | AKER | | | |
| | | | | | | US P | ACEM | AKER | | | | | | | | |
| | | | | ICD/A | AICD | | | | | | | | | | | |
| | | IF YES, | INDICA | ATE D | ATE ( | OF IMI | PLANT | | /_ | M | | / <sub>Y</sub> <sub>Y</sub> , | <u>Y</u> Y | - | | |
| | | IF DATE IS UNKN<br>MPLANTED? | OWN, | APPF | ROXIM | IATEL | Y HO\ | IAM V | NY MC | TNC | THS AGO W | VAS THE SU | BJECT | | | |
| | · | | | | | | | | | | MONTHS | S AGO | | | | |
| | | | IF UN | IKNOV | NN, D | ID TH | E EVE | NT O | CCUR | >5 | YEARS AC | GO? YES [ | □ NO | | | |
| WERE S | URGICAL | INTERVENTION | IS PE | RFO | RME | O ON | ANY | OF T | HE FO | OL | LOWING | CARDIOVA | SCUL | AR CO | MPON | IENTS? |
| | | CAROTID ART | ERIES | 3 | | | | | | | | | | | | |
| | П | WHAT TYPES | | END/<br>END/<br>OTHE | ARTE<br>OVAS | RECT<br>CULA | OMY<br>R ANG | SIOPL | ASTY | ΑN | AROTIDS? ND STENTIN ROTIDS: | | | | | |
| | | THORACIC AC | | • | | | | | | | | | | | | |
| | | LIMB ARTERIE | | | | | | | | | | | | | | |
| | | CORONARY A | RTER | IES | | | | | | | | | | | | |
| | | WHAT TYPE O | F INTE | RVEN | NTION | IS HA | VE BE | EN PE | ERFOR | RM | ED? | | | | | |
| | | CABG | YES [ | ] NO | | | | | | | | | | | | |
| | | PTCA (BALLOC | □<br>□<br>DN ANG | UNKI<br>GIOPL | AFTS<br>NOWI<br>ASTY | N<br>/)/ PEF | | RAFT: | s<br>Js co | | | | (PTCI) | | S□ N<br>S□ N | _ |
| | | WAS A STERM | | 0120 | . 011 | , | J | _ | | , ,, | | ,,,,,,,,,,,,,,,,,,,,,,,,,,,,,,,,,,,,,,, | | | о | |
| | | OTHER INTERV | /ENTIC | NO NC | I THE | COR | ONAR | Y AR1 | TERIES | S: | YES N | 0 🗆 | | | | |
| | | AORTIC VALVE | | | | | | | | | | | | | | |
| | | | □ ∨<br>□ ∨<br>□ c | | REPL | ACEN | | | | | | | | | | |

| Subjec | t Study IE | 201202 | | - | | | | | Site# | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | | MITRAL VALVE | | | | | | | | | | | |
| | | | VALVU VALVE | OPLASTY<br>LOPLAST\<br>REPLACE<br>.REPAIR:_ | MENT | | | | | | | | |
| | | PULMONARY VAL | .VE | | | | | | | | | | |
| | | | ] VALVU | LOPLASTY | , | | | | | | | | |
| | | | VALVE | REPLACE | MENT | | | | | | | | |
| | | | ] OTHER | REPAIR:_ | | | | | | | | | |
| | | TRICUSPID VALVE | E | | | | | | | | | | |
| | | | VALVU | OPLASTY<br>LOPLASTY<br>REPLACE<br>REPAIR:_ | | | | | | | | | |
| | | OTHER CARDIOVA | ASCULAR | COMPON | ENT, SF | PECIF | Y (LO | CATION ANI | D TYPE OF F | ROCE | DURE I | PERFOR | RMED): |

| Subjec | ct Study ID | 201202 | | | | - | | | | | Site# | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| NON-C | ARDIOVAS | CULAR RISK | ( FAC | TOF | RS | | | | | | | | | | | |
| DOES T | HE SUBJEC | T CURRENTL | Y HAV | /E OF | R HA | S TH | E SUI | BJEC | T EVE | ER HAD TH | E FOLLOWING | G DISE | ASES | <b>5</b> ? | | |
| | | BLEEDING DIA | THESI | S | | | | | | | | | | | | |
| | | ☐ ACUTE ANE ☐ BLEEDING D ☐ COAGULOP ☐ LEUKOPENI ☐ THROMBOC ☐ OTHER TYP | OIATHE<br>ATHIES<br>A (WBO<br>YTOPE | ESIS<br>S<br>C <3.5<br>ENIA ( | 5 x 10 <sup>,</sup><br>(PLAT | ^3/ uL<br>ELET | .) | NT < 5 | 60 x 10 | ^3 /uL) | | | | | | _ |
| | | CALCIUM META | ABOLI | C DIS | ORDE | ERS | | | | | | | | | | |
| | | CANCER, SPEC | CIFY: _ | | | | | | | | | | | | | |
| | | HAS THE SUBJ<br>STUDY PROCE | | | | | | E SUE | BJECT | RECEIVE CH | HEMOTHERAPY | WITHI | N 30 E | YAS P | RIOR TO | ) THE |
| | | CHRONIC OBS | TRUCT | TIVE P | PULM | ONAF | RY DIS | EASE | (COP | D)/ CHRONIC | C LUNG DISEAS | E | | | | |
| | | PLEASE INDICA GO-75% 50-59% <sow availa="" chronic="" in="" not="" of="" other="" oxygen="" st="" th="" tre<="" treath="" what=""><th>BLE<br/>IENT D<br/>HALEI<br/>I'EROII<br/>R VENT</th><th>DID TH<br/>D OR D<br/>D THE</th><th><b>IE SU</b><br/>ORAL<br/>ERAP'<br/>ON</th><th>I<b>BJEC</b><br/>BRC</th><th>CT REC</th><th>DILA<sup>-</sup></th><th>TOR T</th><th></th><th>TION?</th><th></th><th></th><th></th><th></th><th>_</th></sow> | BLE<br>IENT D<br>HALEI<br>I'EROII<br>R VENT | DID TH<br>D OR D<br>D THE | <b>IE SU</b><br>ORAL<br>ERAP'<br>ON | I <b>BJEC</b><br>BRC | CT REC | DILA <sup>-</sup> | TOR T | | TION? | | | | | _ |
| | Ш | DIABETES | | <b></b> | | | | | | | | | | | | |
| | | | | | | | | | | NT THE PAT | IENT IS RECEIN | /ING) | | | | |
| | | OBESITY (BMI | ≥ 30) | | | | | | | | | | | | | |
| | | LIVER DISEASE | <b>.</b> | | | | | | | | | | | | | |
| | | MUSCULOSKE | LETAL | . DYSI | FUNC | TION | | | | | | | | | | |
| | | DOES THE SUE | JECT | HAVE | SEV | ERE I | MPAIF | RMEN | T OF N | MOBILITY DU | E TO THIS CON | DITION | N? YE | s □ ı | NO 🗆 | |
| | | RENAL FAILUR | E/INS | SUFFI | CIEN | CY | | | | | | | | | | |
| | | DATE SUBJEC | T WAS | DIAG | SNOS | ED: | | | | | | | | | | |
| | | | | | - | D D | _/ <u></u> | | / | <u>Y</u> <u>Y</u> <u>Y</u> | - <u>Y</u> | | | | | |
| | | IF UNKNOWN, | APPR | OXIM | ATEL | Y HO | IAM W | NY MC | ONTHS | AGO WAS 1 | HE SUBJECT D | IAGNO | SED? | | | |
| | | IF UNKNOWN | WAS T | THE S | SUBJE | CT D | IAGNO | OSED | > 5 YF | ARS AGO? | YES□ NO□ | | | | | |

| Subject Study ID | 201202 | | - | | | | S | ite# | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | YES NO | SUBJEC | T CURREN | ITLY RE | CEIVING D | IALYSIS | | | | | | | | |
| | OTHER DISEASE<br>CHEMOTHERAPY | | | | | | PY INHA | LED OR | SYST | EMIC S | TERO | ID TH | IERAP | Y OR |
| | SMOKER, CU | JRRENT | | | | | | | | | | | | |
| | IF NO, WHE | EN DID SU | BJECT QUI | T: | | | | | | | | | | |
| | | □ Q | UIT > 1 MO | NTH AG | Ю | | | | | | | | | |
| | | ☐ Q | UIT ≤ 1 MO | NTH AG | SO | | | | | | | | | |
| | ALCOHOL/DF | RUG ABUS | SE . | | | | | | | | | | | |
| | | | | | DATE | | | | | | | | | |
| SIGNATURE | | | | | | D | D | M | M | M | Υ | Υ | Υ | Υ |

| S | ubject Study ID | 201202 | | - | | | Sit | e# | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|
| qu<br>mi | ualityMetric's SF<br>estions to meas<br>nutes to comple<br>vers the same | sure functional<br>ete. The SF-12 | health and<br>2v2 is a prac | well-beii<br>ctical, re | ng from<br>liable, a | n the subj<br>and valid | ect's point<br>measure o | of view.<br>f physica | It takes or<br>I and mer | nly 2-3 | |
| Da | ite of Assessme | nt: | D M M - | M / — | <u>Y</u> <u>Y</u> | <u>Y</u> | | | | | |
| 1. | In general, w | ould you say | your health | is: | | | | | | | |
| | Excellent1 | Very good | _ | ood<br>3 | | Fair<br>□₄ | | Poor <sub>5</sub> | | | |
| 2. | The following you in these a | questions are a | | - | might d | o during | a typical da | y. Does y | your healt | h now li | <u>mit</u> |
| | Madauska | ::A: | | | mited a<br>ot | Yes, lin | | No, not<br>nited at all | I | | |
| a. | Moderate active table, pushing or playing golf. | <u>vities,</u> sucn as<br>a vacuum clear | • | | <b>1</b> 1 | | 2 | $\square_3$ | | | |
| b. | Climbing severa | <u>al</u> flights of stairs | S. | | <b>]</b> 1 | | 2 | $\square_3$ | | | |
| 3. | . J <u> </u> | st 4 weeks, how<br>daily activities <u>a</u> | | | _ | = | of the follo | wing prot | olems with | n your w | ork or |
| | | | All of the | e Mos | | Some of the time | A little of the time | None o | | | |
| | a. Accomplish would like. | <u>ied less</u> than y | ou<br> | | <b>]</b> 2 | $\square_3$ | <b></b> 4 | $\square_5$ | | | |
| | | ed in the <u>kind</u><br>er activities. | of $\square_1$ | | $\mathbf{l}_2$ | <b></b> 3 | <b></b> 4 | <b></b> 5 | | | |
| 4. | During the pas | st 4 weeks, how | much of the | e time ha | ave you | ı had any | of the follo | wing prob | olems with | ı your w | ork or |

other regular daily activities as a result of any emotional problems (such as feeling depressed or anxious)?

<sup>&</sup>lt;sup>1</sup>SF-12v2<sup>™</sup> Health Survey<sup>®</sup> 1994, 2002 by QualityMetric incorporated and Medical Outcomes Trust. SF-12<sup>®</sup> a registered trademark of Medical Outcomes Trust. (SF12v2 Standard, US version 2.0).

| S | ubject Study ID | 201202 | - | | | Site | # | | |
|---|---|---|---|---|---|---|---|---|---|
| | | | All of the time | Most of the time | Some of the time | A little of the time | None of the time | | |
| | a. <u>Accomplish</u> would like. | hed less than you | | $\square_2$ | <b></b> 3 | <b></b> 4 | $\square_5$ | | |
| | b. Did work carefully th | or activities <u>less</u><br>an usual? | | $\square_2$ | $\square_3$ | $\square_4$ | <b></b> 5 | | |
| 5. | | ast 4 weeks, how<br>nome and housew | | <u>pain</u> inter | fere with y | our norma | l work (inc | luding b | oth work |
| | Not at all ☐1 | A little bit | Modera<br>□₃ | • | Quite a bit | Ext | remely<br>□₅ | | |
| 6. | weeks. For e | ions are about ho<br>ach question, ple<br>much of the time | ase give o | ne answe | er that come | | • | _ | |
| | J | | All of the time | Most of the time | Some of the time | A little of the time | None of the time | | |
| | a. Have you f | elt calm and | | $\square_2$ | $\square_3$ | $\square_4$ | $\square_5$ | | |
| | b. Did you ha | ve a lot of energy? | | | $\square_3$ | $\square_4$ | $\square_5$ | | |
| | c. Have you f | elt downhearted | | $\square_2$ | <b></b> 3 | $\square_4$ | $\square_5$ | | |
| 7. | | <u>ast 4 weeks,</u> how<br>th your social act | | | | | | ional pro | <u>oblems</u> |
| | All of the | Most of the | Some of | the | A little of the | Non | e of the | | |
| | time<br>1 | time<br> | time | | time<br> | | ime<br>D <sub>5</sub> | | |
| | | | | | DATE SIGNED | | | | |
| SIG | NATURE | | | | | D D | M M I | M Y | YYY |

| | | CO | MM | IENC | E <sup>TM</sup> 1 | RIAI | _ | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Subject Study ID 201 | 202 | | | - | | | | | Site# | | | | |
| | ECHO SITI | ETRAC | CKIN | NG/E | VAL | JATI | ON | | | | Page | e 1 o | of 4 |
| ECHO SITE TRACKING FORM | | | | | | | | | | | | | |
| Date ECHO exam | | | | / | | | | / | | (DD/ | МММ | /YYYY | <b>')</b> |
| Name of the echocardiographer | | | • | | | • | • | | | 1 | | | |
| Echocardiograph equipment use | d (check one | e): | | | | | | | | | | | |
| GE Vivid | | | | | | | | | | | | | |
| Other GE, specify | | | | | | | | | | | | | |
| Philips IE33 | | | | | | | | | | | | | |
| Other Philips, specify: | | | | | | | | | | | | | |
| Siemens | | | | | | | | | | | | | |
| Other model, specify: | | | | | | | | | | | | | |
| Please provide the following ph | ysical assess | ment p | arar | neter | s: | | | | | | | | |
| Subject weight | | □ | kg | [ | ] lb | | | | | | | | |
| Heart rate | | bpr | m | | | | | | | | | | |
| Blood pressure | | / | | r | nmHg | | | | | | | | |
| Cardiac rhythm (check one): | Paced | Indeterr | minato | e | | | | | | | | | |
| Miscellaneous | | | | | | | | | | | | | |
| Is subject enrolled in aortic or m | itral arm of t | rial? | | | | | | | | | | | |
| Did the echocardiographer asses | ss the study v | /alve? | | | | | | | | | | | |
| Date echocardiographs shipped/<br>the Core Lab | uploaded to | | | / | | | | / | | (DD/ | МММ | /YYYY | ') |
| Shipping | | | | _ | | | | • | | | | | |
| Shipping method (check one): | | | | | | | | | | | | | |
| Images uploaded | | | | | | | | | | | | | |
| Study 2012-02 | | | | | | | | | | | | | 1 |

| | | | | C | OMMENC | E™ TRI | AL | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | Subject S | Study ID | 201202 | | - | | | | | Sit | :e# | | | |
| | • | | ECHO : | SITE TRA | CKING/E | VALUA <sup>.</sup> | TION | | | | | Pa | ge 2 ( | of 4 |
| | Shipping track | | vider, specify:<br>r: | | | | | | | | | | | |
| SIGNATI | URE | | | | | DATE | D | D | M | M M | \ | Y | Y | Y |

Study 2012-02

| | | | | СОММЕ | NCE | E™ TR | RIA | L | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Subje | ect Study ID | 201202 | 2 | - | • | | | | | | Site# | | | | |
| | | ECH | O SITE T | RACKING | i/E\ | VALUA | ΑTI | ON | | | | | Page | e 3 o | f۷ |
| ECHO SI | TE EVALUATIO | N FORM | | | | | | | | | | | | | |
| Please inc | dicate the result | s of the LVO | T assessm | ent: | | | | | | | | | | | |
| Peak veloc | city | | | m/sec | | [ | | Not eva | luable | | | | | | |
| Peak gradi | ent | _ | | —<br>mmHg | | [ | | Not eva | luable | | | | | | |
| Mean grad | dient | _ | | —<br>mmHg | | [ | | Not eva | luable | | | | | | |
| VTI | | _ | | cm | | [ | | Not eva | luable | | | | | | |
| | dicate the result<br>only indicate resultity | | | | | | | comple<br>Not eva | | on for tria | al arm p | ositic | n): | | |
| Peak gradi | ent | _ | | mmHg | | [ | | Not eva | luable | | | | | | |
| Mean grad | dient | _ | | mmHg | | [ | | Not eva | luable | | | | | | |
| VTI | | _ | | cm | | [ | | Not eva | luable | | | | | | |
| Annulus si | ze | _ | | cm | | [ | | Not eva | luable | | | | | | |
| Valve area | l | _ | | cm <sup>2</sup> | | [ | | Not eva | luable | | | | | | |
| Please inc | dicate the AR se | verity: | | | | | | | | | | | | | |
| | 0 None | | | | | | | | | | | | | | |
| | +1 Trivial/Trac | e | | | | | | | | | | | | | |
| | +2 Mild | | | | | | | | | | | | | | |
| | +3 Moderate | | | | | | | | | | | | | | |
| | +4 Severe | | | | | | | | | | | | | | |
| | Indeterminate | | | | | | | | | | | | | | |
| Please inc | dicate the MR se | everity: | | | | | | | | | | | | | |
| | 0 None | | | | | | | | | | | | | | |
| | +1 Trivial/Trac | e | | | | | | | | | | | | | |
| | +2 Mild | | | | | | | | | | | | | | |
| | +3 Moderate | | | | | | | | | | | | | | |
| | +4 Severe | | | | | | | | | | | | | | |
| | Indeterminate | | | | | | | | | | | | | | |
| LVEF | | | | % | | [ | | Not eva | luable | | | | | | |
| LVEF range | e (max, min) | | _ | | % | [ | | Not eva | luable | | | | | | |

| Study 2012-02 |
|---------------|

| Sul | oject Study ID | 201202 | | | - | | | | | | | Site | # | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | | ЕСНО | SITE TR | RACKIN | IG/E | VALU | JATIC | )N | | | | | | Pa | age |
| What m | nethod was used f | for LVEF? | | | | | | | | | | | | | |
| | Single plane | | | | | | | | | | | | | | |
| | Biplane | | | | | | | | | | | | | | |
| | Quinones | | | | | | | | | | | | | | |
| | Visual | | | | | | | | | | | | | | |
| Please i | ndicate the sever | ity of paravalvu | lar leak ( | PVL) of | the s | tudy v | alve: | | | | | | | | |
| | 0 None | | | | | - | | | | | | | | | |
| | +1 Trivial/Trac | ce | | | | | | | | | | | | | |
| | +2 Mild | | | | | | | | | | | | | | |
| | +3 Moderate | | | | | | | | | | | | | | |
| | +4 Severe | | | | | | | | | | | | | | |
| | Indeterminate | è | | | | | | | | | | | | | |
| | Not applicable | e at baseline | | | | | | | | | | | | | |
| What w | as the assessmer | nt of RV function | 1? | | | | | | | | | | | | |
| | Normal | | | | | | | | | | | | | | |
| | Mildly reduce | d | | | | | | | | | | | | | |
| | Moderately re | educed | | | | | | | | | | | | | |
| | Severely redu | ced | | | | | | | | | | | | | |
| | Indeterminate | 2 | | | | | | | | | | | | | |
| | | | | | | DATE | . [ | | | | | | | | |
| JRE | | | | | | J/ (11 | | | ) | M | M | M | Y | Y | Y |

Study 2012-02

COMMENCE™ TRIAL

| Subje | ct Study | ID 201202 - Site# |
|---|---|---|
| DATE O | | PITAL ADMISSION: D D / M M M M / Y Y Y Y Y Y Y Y Y Y Y Y |
| IMPLAN | ITING S | URGEON: |
| PREOP | ERATIV | E CONDITION |
| YES | NO | |
| | | DID A MYOCARDIAL INFARCTION (MI) OCCUR WITHIN 21 DAYS PRIOR TO SURGERY? INDICATE THE TIME INTERVAL WHEN THE LAST MI OCCURRED: □ <6 HOURS □ 6-24 HOURS □ 1-7 DAYS □ 8-21 DAYS |
| | | WITHIN 2 WEEKS PRIOR TO THE SURGICAL PROCEDURE: WAS THE SUBJECT IN CONGESTIVE HEART FAILURE? |
| | | WITHIN 2 WEEKS PRIOR TO THE SURGICAL PROCEDURE: DID THE SUBJECT EXPERIENCE AN ARRHYTHMIA? WAS THE OBSERVED ARRHYTHMIA CONSIDERED ATRIAL FIBRILLATION OR ATRIAL FLUTTER? YES NO |
| | | WAS THE SUBJECT EXPERIENCING CARDIAC/CHEST PAIN AT ADMISSION? WHAT IS THE LIKELY CAUSE OF THESE SYMPTOMS? STABLE ANGINA UNSTABLE ANGINA UNLIKELY DUE TO ISCHEMIA NON-STEMI STEMI |
| | | DID THE SUBJECT RECEIVE IV INOTROPIC AGENTS WITHIN 48 HOURS PRECEDING SURGERY OR ADMINISTRATION OF THIS MEDICATION DOCUMENTED AS CONTRAINDICATED? |
| DID THE<br>ANESTH | | T EXPERIENCE OR REQUIRE ANY OF THE FOLLOWING AFTER ADMISSION BUT PRIOR TO GOING UNDER |
| | | VENTRICULAR FIBRILLATION |
| | | VENTRICULAR TACHYCARDIA |
| | | CARDIOGENIC SHOCK |
| | | ABORTED SUDDEN DEATH |
| | | ACUTE RENAL FAILURE (ANURIA OR OLIGURIA <10 ML/HR) |
| | | CARDIOPULMONARY RESUSCITATION < 1 HOUR PRIOR TO SURGERY |
| | | VENTILATION PRIOR TO ARRIVAL IN THE ANESTHETIC ROOM |
| | | INOTROPIC SUPPORT OR IABP |
| | | ANOTHER CARDIAC INTERVENTION <6 HOURS PRIOR TO SCHEDULED SURGERY |

WHAT IS THE URGENCY OF THE SURGERY BEING PERFORMED? (CHECK ONE)


| Subje | ect Study ID | 201202 | | | | - | | | | | Site# |
|---|---|---|---|---|---|---|---|---|---|---|---|
| | ELECTIVE | | | | | | | | | | |
| | URGENT | | | | | | | | | | |
| | SALVAGE | | | | | | | | | | |
| | EMERGENCY | ( | | | | | | | | | |
| PLEAS | E CONFIRM | THE DIAGNOS | SIS FO | OR TH | IE CL | JRRE | NT R | EPLA | CEME | ENT (CHECK ( | ONE) |
| | STENOSIS | | | | | | | | | | |
| | STENOSIS V | VITH INSUFFICI | ENCY | | | | | | | | |
| | PURE INSUF | FICIENCY | | | | | | | | | |
| | PROSTHETIC | VALVE DYSFU | INCTIO | NC | | | | | | | |
| | OTHER DIAG | NOSIS, SPECIF | Y: | | | | | | | | |
| SURG | ICAL APPRO | OACH (CHEC | K ON | E) | | | | | | | |
| | FULL S | STERNOTOMY | | | | | | | | | |
| | MINI U | PPER STERNO | TOMY | | | | | | | | |
| | RIGHT | THORACOTOM | ΙΥ | | | | | | | | |
| | OTHER | R MIS, SPECIFY | : | | | | | | | | |
| SURG | SICAL APPI | ROACH AN | D AN | NNU | LUS | PRE | PAF | RATIO | NC | | |
| WERE | THE FOLLO | OWING CON | COM | ITAN | IT PF | ROCE | DUR | ES P | ERFO | ORMED? | |
| YES | NO | | | | | | | | | | |
| | | RONARY ART | ERY | BYPA | ASS ( | GRAF | TNG | (CAB | 3 = Di | istal | |
| | | W MANY GRAF | | | | | | | | | |

| Subjec | t Study | ID 201202 - Site# |
|---|---|---|
| YES | NO | |
| | | PERMANENT PACEMAKER IMPLANT |
| | | WAS CARDIAC RESYNCHRONIZATION TECHNIQUE (CRT) USED? YES NO |
| | | WAS THIS PROCEDURE PLANNED? □ YES □ NO |
| | | IF NO, WHY WERE TEMOPRARY PACER LINES NOT EMPLOYED? |
| | | AUTOMATED IMPLANTED CARDIOVERTER (AICD) IMPLANT |
| | | WAS CARDIAC RESYNCHRONIZATION TECHNIQUE (CRT) USED? YES NO |
| | | ATRIAL ABLATION |
| | | WHAT TYPE OF ABLATION PROCEDURE WAS DONE? PRIMARY EPICARDIAL PRIMARILY INTRACARDIAC |
| | | AORTIC ANEURYSM/ DISSECTION REPAIR |
| | | ATRIAL SEPTAL DEFECT (ASD) REPAIR |
| | | WHAT WAS THE TYPE OF DEFECT REPAIRED? PATENT FORAMEN OVALE |
| | | ☐ SECUNDUM ASD |
| | | ☐ SINUS VENOSUS ASD ☐ MULTIPLE DEFECTS |
| | | ROOT SINUS ENLARGEMENT |
| | | AORTIC ANNULAR ENLARGMENT |
| | | WHAT METHOD WAS USED? NICKS MANOUGUIAN KONNO |
| | | TRICUSPID VALVE REPAIR (WITH MITRAL VALVE REPLACEMENT) |
| | | OTHER PROCEDURE, PLEASE SPECIFY: |

| Subje | ct Study | ID | 201202 | | | | - | | | | Site# | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| YES | NO | | | | | | | | | | | | |
| | | WEF | RE ANY UNF | LANN | ED P | ROC | EDUR | RES P | ERFO | RMEI | D DURING THIS OPERATI | ON? | |
| | | WHY | WAS THIS P | ROCED | URE | NECE | SSAR | Υ? | | | | | |
| | | | UNSUSPE | CTED | SUBJ | ECT D | ISEAS | SE OR | ANAT | YMC | | | |
| | | | SURGICA | L COM | PLICA | TION | | | | | | | |
| | | | S AN INTRA<br>OCEDURE? | AORTI | СВА | LLO | ON PU | JMP ( | IABP) | USE | D IN RELATION TO THIS S | SURG | ICAL |
| | | WHE | N WAS THE I | ABP IN | SERT | ED? | | | | | | | |
| | | | PREOPER | RATIVE | LY | | | | | | | | |
| | | | INTRAOP | ERATIV | 'ELY | | | | | | | | |
| | | | POSTOPE | RATIV | ELY | | | | | | | | |
| | | WAS | ANNULAR D | EBRID | EMEN | T PEF | RFORM | MED? | | | | | |
| | | DEG | REE: | | | | | | | | | | |
| | | | ] ROUTINI | Ē | | | | | | | | | |
| | | | EXTENS | IVE – N | OT RI | EQUIF | RING A | NNUL | AR RE | PAIR | | | |
| | | | EXTENS | IVE – R | EQUI | RING | ANNU | LAR R | EPAIR | /RECC | ONSTRUCTION | | |
| | | LOC | ATION: | | | | | | | | | | |
| | | | FULL AN | NULAR | CIRC | UMFE | ERENC | CE | | | | | |
| | | | ] PARITAL | ANNU | LAR C | IRCU | MFER | ENCE | (>= 50 | %) | | | |
| | | | PARTIAL | ANNU | LAR C | IRCU | MFER | ENCE | (<50% | ) | | | |
| | | CAL | CIFICATION F | REMOV | AL: | | | | | | | | |
| | | | ] COMPLE | TE | | | | | | | | | |
| | | | ] INCOMP | LETE ( | >= 50 | %) | | | | | | | |
| | | | ] INCOMP | LETE ( | <50% | ) | | | | | | | |
| WHAT: | STUDY V | /ALVI | E MODEL W | AS EM | IPLO' | YED? | (CHE | ECK C | NE) | | | | |
| | 11000A | | | | | | | | | | | | |
| | 11000M | | | | | | | | | | | | |
| HOW M | IANY AT | TEMF | TS WERE N | IADE 1 | TO IM | IPLAI | NT TH | IE VA | LVE? | (CHE | CK ONE) | | |
| | 2 | | | | | | | | | | | | |
| | 1 | | | | | | | | | | | | |

| Subject Study ID | 201202 | | | | - | | | | Site# | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| WHY WAS | A SECOND AT | ГЕМРТ | TO IN | MPLAI | ит тн | E STU | JDY VA | LVE | NOT PERFORMED? | | | |
| | FIRST ATTEMP | PT SUC | CCESS | SFUL | | | | | | | | |
| | A STUDY VALV | /E OF <sup>-</sup> | THE C | ORRE | ECT S | IZE IS | NOT A | VAILA | ABLE AT THE SITE | | | |
| | NONE OF THE | SIZES | S AVAI | LABLE | E FOR | THE | STUDY | / VAL\ | /E ARE SUITABLE FOR THE | SUBJE | CT | |
| | SURGEON CHO | | от то | O ATTI | EMPT | TO IN | 1PLAN | T THE | STUDY VAVLE AGAIN DUE | TO A M | IEDICA | <b>AL</b> |
| | OTHER REASO | ON: SP | ECIFY | /:<br> | | | | | | | | |
| WAS THE HEART R | ESTARTED W | тн ті | HE S | TUDY | VAL | VE IN | IPLAN | ITED1 | ? | | | |
| □ NO | | | | | | | | | | | | |
| WAS A CO | MMERCIAL VAI | LVE SU | JCCE | SSFUI | LLY IN | /IPLAI | NTED? | | | | | |
| | NO (PLEASE F | ILL OL | JT A S | STUDY | EXIT | FOR | M) | | | | | |
| | YES | | | | | | | | | | | |
| | PLEASE PROV | /IDE TI | HE FO | LLOV | VING I | NFOF | RMATIC | N AB | OUT THE COMMERCIAL VAI | VE: | | |
| | MANUFACTUR | RER AN | ID MO | DEL: | | | | | | | | |
| | VALVE SIZE (M | ИМ): | | | | | | | | | | |
| | SERIAL NUMB | ER: | | | | | | | | | | |
| YES | | | | | | | | | | | | |
| WAS A PO | ST-IMPLANT TE | RANSE | SOPF | IAGE/ | AL EC | HOCA | ARDIO | GRAM | PERFORMED? | | | |
| | NO | | | | | | | | | | | |
| | YES | | | | | | | | | | | |
| | TIME ECHOCA | RDIO | GRAM | STAF | RTED: | | | | : (2 | 4 HR F | FORMA | AT) |
| | WHAT TYPE O | | | RDIOG | RAM | WAS | DONE | ? | | | | |
| | WAS ANY OBS | SERVE | | GURG | ITATO | ON CL | INICAL | LY AC | CCEPTABLE? | | | |
| WAS SERI | JM GLYCEROL | ANALY | YSIS F | REQUI | RED I | FOR T | HIS SU | JBJEC | T? | | | |


| Subject Study ID | 201 | 202 | | | | - | | | | Site# |
|---|---|---|---|---|---|---|---|---|---|---|
| WAS A PO | | RATIVE<br>YES | ELEC | TROC | CARDI | OGR <i>A</i> | AM PE | RFORI | MED U | UPON ARRIVAL TO THE ICU? |
| YES NO | | | | | | | | | | |
| | WAS T | HERE A | BLEE | DING | -RELA | ATED | REOP | ERATI | ON WI | /ITHIN THE FIRST 24 HOURS AFTER SURGERY? |
| | | NY ADVE | | | | | | | | Υ? |
| SURGICAL PROC | EDUR | E TIMII | NG | | | | T | | | |
| SKIN INCISION: | | | | : | | | | (2 | 24 HR | R FORMAT) |
| START ECC (PUMP): | | | | : | | | | (2 | 24 HR | R FORMAT) |
| START CROSS CLAMP | <b>P</b> : | | | - : | | | | (2 | 24 HR | R FORMAT) |
| START SIZING: | | | | : | | | | (2 | 24 HR | R FORMAT) |
| REMOVAL CROSS CLA | AMP: | | | : | | | | (2 | 24 HR | R FORMAT) |
| END ECC (PUMP): | | | | : | | | | (2 | 24 HR | R FORMAT) |
| SKIN CLOSURE: | | | | : | | | | (2 | 24 HR | R FORMAT) |
| COMMENTS: | | | | | | | | | | |
| SIGNATURE | | | | | | | | D | ATE S | SIGNED N M M M Y Y Y Y |


| Subje | ect Study | / ID | 2012 | 02 | | | | - | | | | | | | Site | # | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| AORT | IC VAL | /E ET | riolog | Y | | | | | | | | | | | | | | | | | | | |
| YES | NO | | | | | | | | | | | | | | | | | | | | | | |
| | | DEGI | ENERATI\ | VΕ | | | | | | | | | | | | | | | | | | | |
| | | DYS | TROPHIC | CALC | IFICA | TION | | | | | | | | | | | | | | | | | |
| | | CON | GENITAL | | | | | | | | | | | | | | | | | | | | |
| | | RHE | UMATIC | | | | | | | | | | | | | | | | | | | | |
| | | REM | OTE END | OCAR | DITIS | | | | | | | | | | | | | | | | | | |
| | | OTH | ER ETIOL | OGY, | SPEC | IFY: | | | | | | | | | | | | | | | | | |
| COND | ITION C | F TH | IE AORT | TIC V | 'ALV | E AN | ID SI | JRRC | DUNE | DING | ANA | TOM | Y | | | | | | | | | - | |
| YES | NO | | | | | | | | | | | | | | | | | | | | | | |
| | | WAS | CALCIFIC | CATIO | N OB | SERVI | ED? | | | | | | | | | | | | | | | | |
| | | YE | S N | 0 | | | | | | | | | | | | | | | | | | | |
| | | | | | ANN | JLUS | | | | | | | | | | | | | | | | | |
| | | | | | LEAF | LETS | | | | | | | | | | | | | | | | | |
| | | | | | AOR <sup>3</sup> | TIC W | ALL | | | | | | | | | | | | | | | | |
| | | | | | COR | ONAR | Y ART | ERIE | 3 | | | | | | | | | | | | | | |
| | | | | | LEAF | LET F | USIOI | N | | | | | | | | | | | | | | | |
| | | | | | LEAF | LET P | PERFC | RATIO | NC | | | | | | | | | | | | | | |
| | | | | | MYX | TAMC | OUS ( | LEAFL | ET) | | | | | | | | | | | | | | |
| | | | | | VEGI | ETATI | ON | | | | | | | | | | | | | | | | |
| | | | | | CON | GENIT | AL VA | LVE [ | DEFEC | CT | | | | | | | | | | | | | |
| | | | | | | ] BI | CUSPI | D AOF | RTIC \ | /ALVE | | | | | | | | | | | | | |
| | | | | | | ] UN | NICUS | PID A | ORTIC | VALV | E | | | | | | | | | | | | |
| | | | | | OTH | ER DIS | SEASE | CON | DITIO | N, SPE | CIFY: | | | | | | | | | | | - | |
| COMM | MENTS: | | | | | | | | | | | | | | | | | | | | | | |
| 0011111 | | | | | | | | | | | | | | | | | | | | | | | |
| | | | | | | | | | | | DAT | E SIGN | NED | | | | | | | | | | |
| SIGNATU | RE | | | | | | | | | | | | L | D | D | M | М | М | · _ , | Υ | Υ | Υ | Υ |

| Subjec | ct Study | / ID | 201202 | | | | - | | | | Site# |
|---|---|---|---|---|---|---|---|---|---|---|---|
| MITRAI | L VAL\ | /E ET | IOLOGY | | | | | | | | |
| YES | NO | | | | | | | | | | |
| | | DEGE | NERATIVE | | | | | | | | |
| | | DYST | ROPHIC CAL | CIFICA | TION | | | | | | |
| | | FUNC | TIONAL DISE | ASE | | | | | | | |
| | | CONG | SENITAL | | | | | | | | |
| | | RHEU | IMATIC | | | | | | | | |
| | | REMO | TE ENDOCA | RDITIS | | | | | | | |
| | | ISCHE | EMIC HEART I | DISEAS | SE | | | | | | |
| | | MITRA | AL VALVE PRO | DLAPS | E | | | | | | |
| | | | ANTERIOF | 2 | | | | | | | |
| | | | _ | | | | | | | | |
| | | OTHE | | | IEV. | | | | | | |
| | | | R ETIOLOGY | | | _ | 100 | | | | |
| | | )F TH | E MITRAL ' | /ALV | E AN | ID SU | JRRC | JUNI | DING | ANA | ГОМҮ |
| YES | NO | \A/A C / | CAL CIEICATIO | | SED\/E | -D2 | | | | | |
| | Ш | | CALCIFICATIO | IN OB | SERVE | יט? | | | | | |
| | | YES | S NO | ANNU | 11 1 1 1 2 | | | | | | |
| | | Ш | | _ | | NTERI | OR | | | | |
| | | | | | | DSTE | | | | | |
| | | | | | ] ВІ | LATE | RAL | | | | |
| | | | | LEAF | LETS | | | | | | |
| | | | | | | NTERI | | | | | |
| | | | | | | OSTEF<br>LEAFL | | | | | |
| | | | | _ | RDAE | | | | | | |
| | | | | | LLARY | | | | | | |
| | | | | DILA <sup>-</sup> | TED A | NNUL | US | | | | |
| | | | | | LET F | | | | | | |
| | | | | LEAF | LET P | ERFC | RATIO | ON | | | |
| | | | | MYX | OMAT | OUS ( | LEAFL | LET) | | | |
| | | | | | OELAS | | | | , | | |
| | | | | VEGE | ETATIO | NC | | | | | |
| | | | | CON | GENIT | AL MI | TRAL | VALV | E DEF | ECT | |

| Subject Study ID | 201202 | | | - | | | | | | Site# | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| YE | s no | | | | | | | | | | | | | | | | |
| | | CHORDA | AE DYSFU | JNCT | ION | | | | | | | | | | | | |
| | | | ELONGA | TED | | | | | | | | | | | | | |
| | | | TETHER | ED | | | | | | | | | | | | | |
| | | | RUPTUR | RED | | | | | | | | | | | | | |
| | | OTHER I | DISEASE | CON | DITIO | N, SPE | CIFY:_ | | | | | | | | | - | |
| MITRAL VALVE RI | EPLACEMEN | NT TECH | HNIQUE | <b>E</b> | | | | | | | | | | | | | |
| | | | Α | NTER | IOR L | EAFLE | ΞT | | | | | | | | | | |
| | | | | | | | | RESERVA | | | | | | | | | |
| | | | | | | | | SERVATIO | N | | | | | | | | |
| | | | | | | | | EMOVAL | | | | | | | | | |
| | | | PC | | | LEAFL | | DEOED\/A | TION | | | | | | | | |
| | | | | | | | | RESERVA<br>SERVATIO | | | | | | | | | |
| | | | | | | | | EMOVAL | 'IN | | | | | | | | |
| | | | ΔΝ | | | HORDS | | LIVIOVAL | | | | | | | | | |
| | | | Air | | | RESEF | | | | | | | | | | | |
| | | | | | | EMOVI | | | | | | | | | | | |
| | | | PC | | | CHORE | | | | | | | | | | | |
| | | | | | □Р | RESEF | RVED | | | | | | | | | | |
| | | | | | □R | EMOVI | ED | | | | | | | | | | |
| COMMENTS: | | | | | | | | | | | | | | | | | |
| | | | | | | | | - 0.0 | | | | | | | | | |
| | | | | | | | DAT | E SIGNED | | | | | | | | | |
| SIGNATURE | | | | | | | | | D | D | M | M | M | Υ | Υ | Υ | Υ |

| | | | C | ОММЕ | NCE | ™ TRI | AL – | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Sı | ıbject Study ID | 201202 | | | - | | | | | Site# | | | |
| , | | | DEVICE | PERF | ORM | ANCE | | | | | Page | 1 o | f <b>2</b> |
| Wha | t study valve impla | nt attempt was | being pe | rforme | d? | | <u> </u> | L <sup>st</sup> att | empt | 2 <sup>nd</sup> attempt | | | |
| Pleas | e provide the follo | wing information | on about | the stu | dy val | ve: | | | | | | | |
| Valve | e size: | | | | | | | | | | | | |
| | 19mm | m 🗌 23mm | | 25mm | | 27mm | n [ | | 29mm [ | 31mm | 33mm | | |
| Seria | l Number: | | | | | | | | | | | | _ |
| Wha | t type of sizer was i | used? | | | | | | | | | | | |
| | Model 1133 [AC | ORTIC] | | | | | | | | | | | |
| | Model 1173 [M | IITRAL] | | | | | | | | | | | |
| | Universal sizer | | | | | | | | | | | | |
| | Other sizer, spe | cify: | | | | | | | | | | | |
| What | was the barrel size o | f the valve sizer? | 1 | | mm | | | | | | | | _ |
| What | suture technique wa | s used to secure | the valve | (check o | ne)? | | | | | | | | |
| | Single simple interr | upted without p | edgets | | | | | | | | | | |
| | Horizontal interrup | ted mattress wit | hout pled | gets (intr | a-ann | ular) | | | | | | | |
| | Horizontal interrup | ted without pled | gets (supr | a-annula | ar) | | | | | | | | |
| | Horizontal interrup | ted with pledget | s (intra-an | nular) | | | | | | | | | |
| | Horizontal interrup | ted with pledget | s (supra-a | nnular) | | | | | | | | | |
| | Continuous running | g sutures without | pledgets | strip | | | | | | | | | |
| | Continuous running | g sutures with ple | edgets/stri | р | | | | | | | | | |
| | Interrupted figure | of eight without p | oledgets | | | | | | | | | | |
| | Other technique, sp | pecify: | | | | | | | | | | | |
| | Not attempted | | | | | | | | | | | | _ |
| How | was the valve position | ned? 🔲 S | upra-annula | ar [ | ] In | tra-annu | ar | | Not attempte | d | | | |
| Did th | ne study valve perfori | m as intended? | | lo [ | ☐ Ye | es | | | | | | | |
| | Please indicate | the types of valve | e failures o | bserved | d (sele | ct all tha | it apply | /): | | | | | |
| | Study 2012-02 | | | | | | | | | | | | |

| | | | СО | ММЕ | NCE | ™ TF | RIAL | - | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Subject Study II | 201202 | | | | - | | | | | | Site | # | | | |
| | | DEV | ICE I | PERF | ORM | IANC | Έ | | | | | | Pag | ge 2 c | of 2 |
| | Device function, un | able to | place | sutur | es thre | ough t | he sev | wing rir | ng | | | | | | |
| | Device function, un | able to | posit | ion or | the a | ortic a | nnulu | S | | | | | | | |
| | Device function, bio | prosth | nesis a | nd ho | lder se | parate | e durii | ng prod | edure | | | | | | |
| | Device function, otl | ner, spe | ecify: | | | | | | | | | | | | |
| | Device use, sizing to | echniqu | ue | | | | | | | | | | | | |
| | Device use, sterility | compr | romise | ed | | | | | | | | | | | |
| | Device use, used ex | pired p | orodu | ct | | | | | | | | | | | |
| | Device use, compor | nent da | amage | d by c | perato | or | | | | | | | | | |
| | Device use, improp | er post | ionin | 3 | | | | | | | | | | | |
| | Device use, other, s | pecify: | | | | | | | | | | | | | |
| DEVICE TECHNICA | L SUCCESS | | | | | | | | | | | | | | |
| Was the heart resta | rted with the valve | e in pla | ace at | fter th | nis imp | olant a | attem | pt? | | No | ☐ Yes | | | | |
| Did the subject leave | e the operating ro | om wi | th th | e stuc | dy valv | e in p | lace | for thi | s attem | pt? | ☐ No | ) | Ye: | 5 | |
| If No, Why | did the implant atte | mpt fai | 1? | | | | | | | | | | | | |
| | Valve failure (Please | e indica | ate th | e valve | e failur | e type | on th | is form | n) | | | | | | |
| | Subject died | | | | | | | | | | | | | | |
| | Other reason, speci | fy: | | | | | | | | | | | | | |
| Please provide the | time at which eac | n step | in th | e stu | dy dev | ice p | roced | lure o | ccurred | in HH | :MM:SS f | orma | t: | | |
| Start of study procedure | (first stitch placed) | | | | | : | | $ bracket{:}$ | | | Not attem | | | | |
| First stitch placed on valv | ve ring | | | | | : | | | | | Not attem<br>Not availab | | | | |
| Complete the study procurative) | edure (last stitch tied c | lown on | the | | | : | | ]:[ | | | Not attem | | | | |
| Comments: | | | | | | | | | | | | | | | |
| | | | | | | DAT | | | | | | | | | |
| SIGNATURE | | | | | | 0.0. | | | ) D | M | ММ | Y | ′ Y | Υ | Υ |
| Study 2012-02 | 2 | | | | | | | | | | | | | | 7 |

| Subject Study ID <b>201202</b> - | Site | # | | | |
|---|---|---|---|---|---|
| VISIT TYPE: ☐ DISCHARGE ☐ 10 DAY FOLLOW UP (ECH | O REQUIRED) | | | | |
| DATE OF DISCHARGE: $\_D / \_M / \_M / \_M / \_Y / \_Y / \_Y / \_Y$ | | | | | |
| DISCHARGED TO: | | | | | |
| HOME | | | | | |
| ANOTHER HOSPITAL | | | | | |
| EXTENDED CARE | | | | | |
| POST OPERATIVE HOSPITALIZATION INFORMATION | | | | | |
| DURATION OF TIME IN INTENSIVE CARE UNIT | D/ | YS AN | 1D | HOUR | ≀S |
| DURATION FO TIME IN INTERMEDIATE CARE / HIGH DEPENDENCY | Y UNIT DA | YS AN | D | HOUR | .S |
| DURATION OF TIME IN GENERAL WARD | D | YS AN | ND | HOUR | ≀S |
| ******COMPLETE ASSESSI | MENT FORM******* | • | | | |
| SIGNATURE | D D | M | M M | YYY | Y |

| Sı | ubject Study ID 20120 | 02 | | | - | | | | | | Sit | e# | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | | REC | CORI | D ON | ILY ( | ONE | ADV | ERS | E EV | ENT I | PER | FORI | VI | | | | | | |
| 1. | EVENT ONSET DATE | | | | | | | | | | | | | | | | | | |
| | | D D | M | M | M | Υ | Υ | Υ | Υ | l | | | | | | | | | |
| 2. | SITE AWARENESS DATE | | | | | | | | | | | | | | | | | | |
| | 1 | D D | M | M | M | Υ | Υ | Υ | Υ | | | | | | | | | | |
| 3. | TIMING OF EVENT ONSET | | | | [ | ] INT | RA-OF | ERATI | VΕ | □ P( | OST-OF | PERATI | VΕ | | | | | | |
| 4. | IS THIS A NEW OR WORSEN | IING ADV | ERSE | EVEN | T? [ | <br>NE' | W | | | _<br>_ w | ORSEN | IING | | | | | | | |
| 5.<br>(S | EVENT NAME<br>SEE ADVERSE EVENT LISTING*) | | | | | | | | | | | | | | | | | | |
| 6. | EVENT SUMMARY | | | | | | | | | | | | | | | | | | |
| 7. | METHOD OF DETECTION (C | HECK ALL T | HAT AF | PLY) | | LAB FI | NDING | - E | ЕСНО | | ANGIO | GRAM | | ] MRI | | ]EC | G | | |
| | | ПА | UTOPS | SY | | OBSER | NOITAV | 1 🔲 E | EXAM | | REOPE | | | | | ( | (DD/ <b>I</b> . | /MM/Y | YYY) |
| | OBSERVATION (Date of reoperation:(DD/MMM/YYYY) | | | | | | | | , | | | | | | | | | | |
| | | | | | - | | | | | | | | | | | | - | | |
| | DATE OF TEST/ EXAM: | | | | | _ | | | | | | | | | | | | | |
| 8. | CAUSALITY: IS THIS EVENT | RELATE | D TO | ANY O | F THE | FOLL | OWIN | IG? | | | | DID AN | | | | LIC | MEDI | CATIC | ON |
| | SURGICAL PROCEDURE | YE | ES | | ] NO | | | UNDE | TERMI | NED | | | | YE | s [ | N | 0 | | |
| | | | | | | | | | | | | ANTI | COAG | ULAN | Γ MED | ICA | TION | I | |
| | STUDY VALVE | YE | ES | | _ NO | | | UNDE | TERMI | NED | | ASPII | RIN | | | | | | |
| | STUDY VALVE PROCEDURE | YE | ES | L | NO | | | UNDE | TERMI | NED | 1 - | , | | | TELET | | | | |
| | USER ERROR | YE | ES | | NO | | | UNDE | TERMI | NED | MED | ICATIO | | | ОМВО | | BOLI | <u></u> | |
| | DEFICIENCY IN INSTRUCTIONS | S YE | ES | | ] NO | | | UNDE | TERMI | NED | | THIS | | CATIO | N PRE | SCI | RIBE | D DUI | Е ТО |
| | UNDERLYING CONDITION | YE | ΞS | | NO | | | UNDE | TERMI | NED | | [ | YE | S | | | NO | ) | |
| | IF YES, WHAT WAS THE UND | ERLYING ( | CONDI | TION: | | | | | | | | NON- | | | | 3OLI | IC ME | DICA | TION |
| | | | | _ | _ | | | | | | | /ES | | | NO | | | | |
| 10. | SERIOUS ADVERSE EVENT | _ | | | _ NO | | | | | | | IF | YES, | SPEC | IFY: | _ | | | |
| | | ED IN DEA | | | | | | | | | | | | | | | | | |
| | <u> </u> | D IN LIFE- | | | | | R INJU | JRY | | | | | | | | | | | |
| | RESULTE | D IN PERI | MANEN | IT IMPA | AIRMEI | NT | | | | | | | | | | | | | |

| Subject Study ID 201202 - | Site | ‡ | | | |
|---|---|---|---|---|---|
| RESULTED IN HOPSITALIZATION OR PROLONGING OF CURRED RESULTED IN SURGICAL INTERVENTION TO PREVENT PERMAPE RESULTED IN FETAL DISTRESS OR DEATH, CONGENITAL ABNORMANTICIPATED DEVICE RELATED ADVERSE DEVICE YES NO BEFFECT? | ANENT IMPAIRMENT<br>IORMALITY OR BIRTI | TO BODY S | | | |
| 11. ACTION TAKEN/TREATMENT (MULTIPLE RESPONSES POSSIBLE) CARDIOVERSION TRANSFUSION IF YES, NUMBER OF PRBC UNITS TRANSFUSED MEDICATION GIVEN, SPECIFY PACEMAKER/ICD IMPLANT (NOT PLANNED PRIOR TO AVR - PROVIDE DA | | | (DD/MMM/Y | YYY) | |
| PROLONGED HOSPITALIZATION RE-HOSPITALIZATION REQUIRED ADMISSION DATE: | RVENTION ON STUD | | COMPLETE EX | | EPORT) |
| 12. OUTCOME ONGOING UNRESOLVED AT STUDY EXIT UNKNOWN AT STUDY EXIT CHRONIC CONDITION RESOLVED WITH OUT SEQUELAE RESOLVED WITH SEQUELAE DEATH (PRIMARY CAUSE) DEATH (NOT PRIMARY CAUSE) | DATE: D D D D D D D D D D D D D D D D D D | M M | | | Y Y |
| DATE SIGNED SIGNATURE | D D M | M | M Y | Y | YY |

| | | | - |
|------------------|--------|---|-------|
| Subject Study ID | 201202 | - | Site# |

\*AE Categories include:

Blood and lymphatic (including ALL bleeding complications)

Cardiovascular - Arrhythmia

Cardiovascular - Regurgitation

Cardiovascular - Stenosis

Cardiovascular - Embolic Event/Valve Thrombosis

Cardiovascular - Misc

**Device Dysfunction** 

Gastrointestinal/Hepatic

Genitourinary/Renal

Pulmonary/Respiratory

Peripheral Vascular

Psychiatric

Muscular Skeletal/Dermatologic

Nonspecific or Unknown Body System

Select ONE Adverse event from listing in applicable category
| Subject Study | / ID | 2012 | 02 | | | | - | | | | | | Site | # | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| DATE OF REC | PER | ATION/ | REM | OVA | L/ E | XPL | ANT | | | | D D | M M | / | | Y Y | / <u>Y</u> | | | |
| SURGERY OC | CUR | RED AT | INV | ESTI | GAT | ION | AL C | ENT | ER: | | ] YE | S | | NO | | | | | |
| TYPE OF PRO | CED | URE PE | RFO | RME | D: | | | | | | | | | | | | | | |
| EVDI ANT DDO | 0055 | | | E IN V<br>MANUF<br>ER, SP | FACT | UREF | and | MODE | L: | | | | | | ZE (M | M): | | | |
| EXPLANT PRO | | | | _ | NAP | | | | <b>500</b> | | VDI 411 | | | • | | | | | |
| | | AT WAS T<br>FULL STE<br>MINI UPF<br>AT TYPE ( | ERNOT | TOMY<br>TERNO | ОТОМ | ΙΥ | | RIGI<br>NOT | HT TH | ORAC<br>LABLE | OTOMY | PROC | EDURE | · | | | | | |
| | WHA | AT WAS R | EMOV | ED? | | NOT | AVAI | LABLE | Ī | | | | | | | | | | |
| | | BIOPROS<br>BIOPROS | | | | | } | | | | | | | | | | | | |
| | WAS | S A ROOT | ABSC | ESS F | PRES | ENT A | AT RE | OPER | ATIO | N? | □NO | | □YES | 8 | | | | | |
| | | E OF STU<br>S A REPLA | | | | | | | ]3 🔲 | 4 □5 | □N/A | ( | (5 is the e | easies | t/best | ) | | | |
| | □N | IO 🗆YI | ES N | /ANUF | FACT | UREF | and | MODE | L: | | | | | \$ | SIZE (I | MM): | | | |
| DEVICE GRO<br>ANSWER EACH<br>YES NO | | | TION | l (API | PEAF | RANC | E O | - VAL | VE P | RIOR | TO OR | IMME | DIATEL | _Y FC | )LLO | WING | EXPL | ANT) | |
| | | THROM | //BUS | | | | | | | | | | | | | | | | |
| | | VEGET | ATION | 1 | | | | | | | | | | | | | | | |
| | | SUTUR | E INT | ERFEF | RENC | E | | | | | | | | | | | | | |
| | | CALCIF | FICATI | ON | | | | | | | | | | | | | | | |
| | | FIBROS | SIS | | | | | | | | | | | | | | | | |
| | | DEHIS | CENCE | Ξ | | | | | | | | | | | | | | | |
| | | OTHER | R, SPE | CIFY: | | | | | | | | | | | | | | | |
| DID EXCISIO | _ | | | | | | | | | | TRUCT | | | | 5? □ | NOT A | VAILA | BLE | |
| WAS EXPLAN | TED S | STUDY V | ALVE | RET | URN | ED? | □ NC | ) 🗆 | YES, | RGA#: | : | | | | | | | | |
| | | | | | | | | | | DAT | E SIGNE | D | | | | | | | |
| SIGNATURE | | | | | | | | | | | | | ) D | M | 1 M | l M | Y | / Y | YY |

| Subj | ect Stu | ıdy ID | 201202 | | | - | | | | | Site# | <i>‡</i> [ | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | REASO | | OY EXIT EXIT (SELECT | - | OI PEO | IIDEN | FOLL | OW LIPS | | D | / | M | M | _ / | Y | Y | Υ | Y |
| | 2.<br>3.<br>4. | SUBJE<br>REQUIF<br>STUDY<br>SUBJE | CT DID NOT RE<br>RED FOLLOW-U<br>VALVE EXPLA<br>CT MET AN EX | CEIVE STU<br>JP PERIOD<br>NTED AND<br>CLUSION C | DY VAL'<br>SUBJEC<br>RITERIO | VE DU | RING '<br>MPLET<br>'ER ST | THE IND<br>TED THE<br>TUDY EN | EX PROCE<br>PROTOCO<br>ROLLMEN | OL RE | QUIRED | | | | | OCOL | | |
| | <b>5</b> . | a. | CT VOLUNTAR POST STUDY | | | | | | | ESTIGA | ATOR | | | | | | | |
| | | b. | POST DISCH | | | | - | RAWAI · | | | | | | | | | | |
| | | | | | | | | | | | | | | | | _ | | |
| | 6. | SUBJE | CT LOST TO FO | DLLOW-UP | (SUBJI | ECT M | ISSED | 2 SEQU | ENTIAL FO | OLLOW | V-UP VI | SITS) | | | | | | |
| | 7. | DEATH | | | | | | | | | | | | | | | | |
| | | А | DATE OF | DEATH | 1 | 1 | | (DD/ | MMM/YYY | Y) | | | | | | | | |
| | | В | | _ | | | | | | | PROCE | DURE' | ? □\ | /ES Γ | 1 NO | | | |
| | | С | . DID THE S | | E PRIOR | TO DI | SCHAF | | | | | | _ | | | | | |
| | | D | . CAUSE OF | DEATH: | | | | | | | | | | | | _ | | |
| | | | DATE REF | PORTED TO | SPONS | OR: | | | | (DI | D/MMM/ | YYYY | <b>'</b> ) | | | | | |
| | | ASE PRO<br>CEDURE | VIDE THE FOLI | LOWING IN | FORMAT | ION AI | BOUT | THE SUI | BJECT'S H | OSPIT | ALIZAT | ION A | FTER | THE S | TUDY | ′ VALVE | Ξ | |
| | DUR | ATION A | ND TIME IN THI | E INTENSIV | E CARE | UNIT ( | (ICU) | | D/ | AYS AI | ND | | _HOU | RS | | | | |
| | DUR | ATION A | ND TIME IN THI | E INTERME | DIATE C | ARE/ H | HIGH D | EPEND | ENCY UNIT | Γ | | | | | | | | |
| | | | | | | | | | D | DAYS A | AND | | _HOU | JRS | | | | |
| | DUR | ATION A | ND TIME IN THI | E GENERAL | . WARD | | | | | DAYS / | AND | | HO | URS | | | | |
| | | | DATE OF A | UTOPSY:_ | | | | | (DD/MMM/ | YYYY) | <u> </u> | NOT A | PPLIC | ABLE | | | | |
| | | | WAS A S | STUDY VAL | VE REMO | OVED / | AT AU | TOPSY? | ☐ YES ☐<br>(IF YES, F | | UT REC | P_EX | P FOF | RM) | | | | |
| | 8. | OTHER I | REASON, SPEC | CIFY: | | | | | | | | | | | | _ | | |
| | | | | | | | | DAT | E SIGNED | | | | | | | | | |

SIGNATURE

| Subje | et Study ID 201202 - | Site# |
|---|---|---|
| 1. | <b>DATE OF DEVIATION:</b> $\frac{1}{D} \frac{1}{D} \frac{1}{M} \frac{1}{M} \frac{1}{M} \frac{1}{M}$ | <u></u> |
| 2. | PLEASE SELECT PROTOCOL DEVIATION CODE (PI | ROTOCOL DEVIATION CODE LIST) |
| | EVENT CODE: | |
| | IF MISSED VISIT, SPECIFY: | |
| | 1 <sup>st</sup> ATTEMPTED CONTACT | (DD/MMM/YYYY), TIME (HH:MM) |
| | 2 <sup>nd</sup> ATTEMPTED CONTACT | (DD/MMM/YYYY), TIME (HH:MM) |
| | 3 <sup>rd</sup> ATTEMPTED CONTACT | (DD/MMM/YYYY), TIME (HH:MM) |
| | CAN YOU CONFIRM THROUGH ANY SOURC | CES THAT THE SUBJECT IS ALIVE? |
| | IF OTHER DEVIATION, SPECIFY: | |
| 3. | REASON: | |
| | ☐ NOT ORDERED BY PHYSICIAN | |
| | OVERSIGHT | |
| | ☐ PATIENT NOT AVAILABLE | |
| | ☐ PATIENT TOO SICK TO HAVE TEST | |
| | ☐ OTHER, SPECIFY: | |
| 4. | CORRECTIVE ACTION: | |
| | ☐ STUDY STAFF RE-TRAINED | |
| | OTHER, SPECIFY: | |
| | | DATE SIGNED |
| SIGNATU | RE | D D M M M Y Y Y |

| EDW | ARDS | | | L NUMBI | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|
| Sub | ject Study ID | 201202 | | - | | | | Site | # | |
| | | ECH | IO CORE LA | B EVAL | JATIOI | ١ | | | | |
| ЕСНО С | ORE LAB TRACI | KING FORM | | | | | | | | |
| Date ECI | HO received by c | ore lab | | / | | | / | | | (DD/MMM/YYYY) |
| Date of r | eadability assess | sment | | / | | | ]/ | | | (DD/MMM/YYYY) |
| Please in | dicated whether | r or not the imag | ges were read | lable (che | ck one): | | | | | |
| | Readable | | | | | | | | | |
| | Partially readab | ole | | | | | | | | |
| | Not readable | | | | | | | | | |
| | | sent to the site to | resend the ima | ages? | | | | | | |
| | No Date of r | Yes esend request: | | / | | | ]/[ | | | (DD/MMM/YYYY) |
| | Was the readab | oility issue resolve | d? | | | | | | | |

(DD/MMM/YYYY)

Was the ECHO assessed by the core lab?

Yes

Date readability issue resolved:

☐ No

☐ No ☐ Yes

#### 2

| EDWARDS | | TRIAL NUMBER 2012-02 COMMENCE <sup>TM</sup> TRIAL | |
|---|---|---|---|
| Subject Study ID | 201202 | - | Site# |
| | FCHO CORF LAB EVALUATION | | |

#### **ECHO CORE LAB EVALUATION**

| Physical | l Assess | ment | |
|---|---|---|---|
| Subject v | veight | | ☐ kg ☐ lb |
| Body Sur | face Are | (BSA) | m <sup>2</sup> Not evaluable |
| Heart rat | e | | bpm |
| Blood pre | essure | · | / mmHg |
| Does the | e ECHO | indicate the sub | ject has the following cardiac rhythm/conducting system disturbances? |
| No | Yes | Indeterminate | |
| | | | Normal sinus rhythm |
| | | | Atrial fibrillation |
| | | | Atrial flutter |
| | | | Ventricular tachycardia |
| | | | Ventricular fibrillation |
| | | | AV Block |
| | | | Please indicate the degree: 1st 2nd 3 <sup>rd</sup> Unknown |
| | | | Bundle branch block |
| | | | Please specify the location: Left Right Not evaluable |
| | | | Paced rhythm Please specify the location: Atrial Ventricular Atrioventricular |
| Valve A | ssessme | ent: Stenosis | |
| Please in | dicate th | ne level of aortic st | enosis (check one): |
| | None | | |
| | Study | 2012-02 | |

| | WARDS | | | | TRIAL | | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Su | bject | Study ID | 201202 | | | - | | | | Site# | | | | |
| | | | ECI | но со | RE LAE | EVA | LUAT | ION | | | P | age : | 3 of 1 | 10 |
| | М | ild | | | | | | | | | | | | |
| | М | oderate | | | | | | | | | | | | |
| | Se | vere | | | | | | | | | | | | |
| | No | ot evaluable | | | | | | | | | | | | |
| s there | mitra | l stenosis? | | | | | | | | | | | | |
| ☐ Yes | | ] No | | | | | | | | | | | | |
| f Yes, | | | | | | | | | | | | | | |
| | М | ild | | | | | | | | | | | | |
| | М | oderate | | | | | | | | | | | | |
| | Se | vere | | | | | | | | | | | | |
| | No | ot evaluable | | | | | | | | | | | | |
| tiology | of mi | tral stenosis: | | | | | | | | | | | | |
| | Ca | lcific | | | | | | | | | | | | |
| | Rh | eumatic | | | | | | | | | | | | |
| | Ot | her: Specify | | | | | | | <br> | _ | | | | |
| | In | determinate | | | | | | | | | | | | |
| .V Stru | ıcture | /Regional Fu | ınction | | | | | | | | | | | |
| Please i | ndicat | e if any of the | following abnorr | nalities v | vere obs | erved: | | | | | | | | |
| No | Yes | | | | | | | | | | | | | |
| | | LV aneurysm | | | | | | | | | | | | |
| | | Please speci | ify the location: | | | | | | | | | | | |
| | | Wall motion | abnormality | | | | | | | | | | | |
| | | Please spec | ify: | | | | | | | | | | | |

Study 2012-02

Cavity dilation

| EDWARDS | | | | | BER 2012- | | |
|---|---|---|---|---|---|---|---|
| Subject Study ID | 201202 | | - | • | | | Site# |
| | ECI | HO CORE | LAB E | VAL | LUATION | | |
| Apical and/o | r left atrial throm | nbi | | | | | |
| Please speci | fy: | | | | | | |
| Other abnorn | mality | | | | | | |
| Global LV Structure/Fu | ınction | | | | | | |
| What method of calculation | was used for LV | function as | sessment | t (che | eck one)? | | |
| Biplane | | | | | | | |
| Single | | | | | | | |
| Quinones | | | | | | | |
| Visual | | | | | | | |
| LVEDV | | | ml | | | Not evaluable | |
| LVESV | | | ml | | | Not evaluable | |
| LVEF | | | % | | | Not evaluable | |
| LV Dimension | | | _ | | | | |
| Septal thickness (end-diasto | lic) | | cm | | | Not evaluable | |
| Posterior wall thickness (end | d-diastolic) | | cm | | | Not evaluable | |
| LV end-diastolic dimension | | | cm | | | Not evaluable | |
| LV end-systolic dimension | | | cm | | | Not evaluable | |
| LV mass | | | g | | | Not evaluable | |
| LV mass index (BSA Correcte | ed LV Mass) | | g/m² | | | Not evaluable | |
| Left Atrium (LA) | | | mm | | | Not evaluable | |
| Aortic Dimensions | | | | | | | |
| LVOT diameter | | | cm | | | Not evaluable | |
| Aortic annulus | | | cm | | | Not evaluable | |
| Aortic root diameter | | | cm | | | Not evaluable | |

Study 2012-02

| EDWARDS | | TRIAL | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|
| Subject Study ID | 201202 | | - | | | | Site# | | |
| | ЕСНО | CORE LA | B EVA | LUAT | ION | | _ | Page | 5 of 1 |
| STJ diameter | | cr | n | | | Not evalua | ble | | |
| Valve Assessment: M<br>Please fill out this section | | position | | | | | | | |
| $V_{peak}$ | | | | m/se | С | | Not evaluable | | |
| TVI | | | | cm | | | Not evaluable | | |
| Peak gradient (by continuo | us wave) | | | mmH | g | | Not evaluable | | |
| Mean gradient (by continuo | ous wave) | | | mmH | g | | Not evaluable | | |
| TVI (LVOT) | | | | cm | | | Not evaluable | | |
| Maximum V(LVOT) | | | | m/se | С | | Not evaluable | | |
| Mean V(LVOT) | | | | m/se | С | | Not evaluable | | |
| Stroke volume<br>[LVOT derived for aortic pos<br>valve for mitral position] | sition; across mitral | | | ml | | | Not evaluable | | |
| Transvalvular flow | | | | mL/s | | | Not evaluable | | |
| Cardiac output (LVOT deriv | ed) | | | L/mir | 1 | | Not evaluable | | |
| Cardiac index | | | | L/mir | ı/m² | | Not evaluable | | |
| EOA (continuity equation) | | | | cm <sup>2</sup> | | | Not evaluable | | |
| EOA index | | | | -<br>cm²/r | m² | | Not evaluable | | |
| Performance index | | | | cm²/c | :m² | | ] Not evaluable | | |
| Valve Assessment: Re<br>Please fill out this section | | position | | _ | | | | | |
| Please identify all the me | ethods of calculatio | n used: | | | | | | | |
| No Yes | | | | | | | | | |

| 140 | 103 | |
|-----|-----|--------------------------|
| | | Color doppler |
| | | Regurgitant fraction |
| | | Proximal convergent flow |

Study 2012-02

| EDWARD | S | | | NUMBER | 2012-02 M TRIAL | | |
|---|---|---|---|---|---|---|---|
| | ct Study ID | 201202 | | - | | | Site# |
| _ | ' | ECH | IO CORE LAI | B EVALUA | TION | | |
| | ] Continuous | s wave Doppler (p | oressure half-tin | ne, only appli | cable to aortic | regurgitation) | |
| | ] Aortic/pulr | monary flow reve | rsal | | | | |
| Please indi | cate the parava | alvular leak seve | erity: | | | | |
| | 0 None | | | | | | |
| | +1 Trivial/Trace | e | | | | | |
| | +2 Mild | | | | | | |
| | +3 Moderate | | | | | | |
| | +4 Severe | | | | | | |
| | Not evaluable | | | | | | |
| | Not applicable | | | | | | |
| If the parav | valvular leak se | everity is +2, +3, | or +4, please | indicate the | following: | | |
| Num | ber of jets: | 1 | 3 🗆 | 4 🔲 | Other, specify: | | |
| Pleas | se indicate the lo | ocation of the jets | s: | | | | |
| Pleas | se indicate the ir | mage view of the | jets: 🔲 PI | _AX 🔲 | PSAX | A5C A3C | |
| Please indi | cate the transv | valvular leak sev | erity: | | | | |
| | 0 None | | | | | | |
| | +1 Trivial/Trace | e | | | | | |
| | +2 Mild | | | | | | |
| | +3 Moderate | | | | | | |
| | +4 Severe | | | | | | |
| | Not evaluable | | | | | | |

Study 2012-02

Please indicate the total regurgitation severity:

0 None

+1 Trivial/Trace

| 11 | TRIAL NUMBER 2012-02 | | | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|
| EDWAR | DS | | | С | OM | MEN | ICE <sup>T</sup> | M TF | RIAL | | |
| Subject Study ID 201202 - Site# | | | | | | | | | | | |
| | ECHO CORE LAB EVALUATION | | | | | | | | | | |
| П | +2 Mild | | | | | | | | | | |
| | +3 Moderate | | | | | | | | | | |
| | +4 Severe | | | | | | | | | | |
| | Not evaluable | | | | | | | | | | |
| Primary me | chanism of mitra | al valve regurgita | ition ( | Note: | Only a | applica | ble if s | ubjec | t is in t | the mitral arm at baseline visit) | |
| | Type I – Norm | al Leaflet Motior | า | | | | | | | | |
| | Type II – Leafle | et Prolapse | | | | | | | | | |
| | Type IIIa – Restricted leaflet opening | | | | | | | | | | |
| | Type IIIb – Restricted leaflet closure | | | | | | | | | | |
| | Not evaluable | | | | | | | | | | |
| | Not applicable | | | | | | | | | | |
| Valve Mo | orphology | | | | | | | | | | |
| Please ind | icate the degre | e of calcification | n: | | | | | | | | |
| | Not evaluable | | | | | | | | | | |
| | None | | | | | | | | | | |
| | Mild | | | | | | | | | | |
| | Moderate | | | | | | | | | | |
| | Heavy | | | | | | | | | | |
| Please ind | icate the degre | e of annular ca | lcific | ation | (only | appli | cable 1 | to mi | tral ar | m): | |
| | Not applicable | • | | | | | | | | | |
| | Not evaluable | | | | | | | | | | |
| | None | | | | | | | | | | |
| | Mild | | | | | | | | | | |
| | Moderate | | | | | | | | | | |
| | | | | | | | | | | | 7 |
| | Study 2012-02 | | | | | | | | | | 1 |

| | TRIAL NUMBER 2012-02 COMMENCE™ TRIAL | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|
| Subje | ct Study ID | 201202 | | | - | | | Site# | <u> </u> |
| | ECHO CORE LAB EVALUATION | | | | | | | | |
| | _ | | | | | | | | |
| | Heavy | | | | | | | | |
| Please ind | icate whether t | the following m | orpholog | gies we | re obs | erved | l: | | |
| No Yes | ; | | | | | | | | |
| | Cusp perfora | tion | | | | | | | |
| | Pannus form | ation | | | | | | | |
| | Thrombus | | | | | | | | |
| | Vegetation | | | | | | | | |
| | Ring abscess | | | | | | | | |
| | Pseudoaneur | rysm | | | | | | | |
| Non-Trial | Arm Valve A | ssessment | | | | | | | |
| Please ind | icate the level | of tricuspid valv | e regurg | itation | | | | | |
| | 0 None | | | | | | | | |
| | +1 Trivial/Trac | ce | | | | | | | |
| | +2 Mild | | | | | | | | |
| | +3 Moderate | | | | | | | | |
| | +4 Severe | | | | | | | | |
| | Not evaluable | | | | | | | | |
| | | of mitral valve I | | | m] | | | | |
| | 0 None | | | | | | | | |
| | +1 Trivial/Trac | ce | | | | | | | |
| | +2 Mild | | | | | | | | |
| | +3 Moderate | | | | | | | | |
| | Study 2012-02 | | | | | | | | 7 |

| EDWARDS | TRIAL NUMBER 2012-02 COMMENCE <sup>TM</sup> TRIAL | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|
| Subject | Study ID | 201202 | | | | - | Site# | | |
| _ | ECHO CORE LAB EVALUATION | | | | | | | | |
| | +4 Severe | | | | | | | | |
| | Not evaluable | | | | | | | | |
| | Not applicable | | | | | | | | |
| Please indicate the level of aortic valve regurgitation [Note: Select 'Not applicable' if subject is in the Aortic Trial arm] | | | | | | | | | |
| | 0 None | e ii subject is iii | the A | ortic i | ilai ail | 11] | | | |
| _ | +1 Trivial/Trac | e | | | | | | | |
| | +2 Mild | | | | | | | | |
| | +3 Moderate | | | | | | | | |
| _ | +4 Severe | | | | | | | | |
| | Not evaluable | | | | | | | | |
| | Not applicable | | | | | | | | |
| Pericardial | effusion | | | | | | | | |
| Please indica | ite the level o | of pericardial e | ffusio | n: | | | | | |
| | None | | | | | | | | |
| <u> </u> | Small | | | | | | | | |
| | Moderate | | | | | | | | |
| | Large | | | | | | | | |
| | Tamponade | | | | | | | | |
| | Not evaluable | | | | | | | | |
| | Other, specify: | : | | | | | | | |
| RV Function | n | | | | | | | | |
| Please indica | ite the overa | ll assessment c | of the | right | ventr | icle | | | |
| | | | | | | | | <br> | <br>_ |
| Stu | dy 2012-02 | | | | | | | | |

| Ŕ | | | | | BER 2012<br>CE <sup>TM</sup> TF | | |
|---|---|---|---|---|---|---|---|
| EDWARE | OS . | | | | | \'\\ <b>_</b> | |
| Subjec | ct Study ID | 201202 | | - | | | Site# |
| | | EC | HO CORE L | AB EVA | LUATION | J | |
| | Normal | | | | | | |
| | Abnormal | | | | | | |
| ECHO Qua | ality | | | | | | |
| Please indi | cate the overa | ll quality of the | e ECHOs | | | | |
| | Good | | | | | | |
| | Fair | | | | | | |
| | Poor | | | | | | |
| | Inadequate | | | | | | |
| COMMEN | ITS: | | | | | | |

**EDWARDS LIFESCIENCES LLC**CLINICAL INVESTIGATIONAL PLAN

### ATTACHMENT E - CORE LABORATORY PROCEDURE MANUAL

REVISION J: 03 MARCH 2021

# Core Laboratory Procedure Manual (For Model 11000A)

ProspeCtive, nOn-randoMized, MulticENter Clinical Evaluation of the Edwards Pericardial Aortic & Mitral Bioprostheses (Models 11000A & 11000M) with a New Tissue Treatment Platform

(COMMENCE TRIAL)

# **Clinical Protocol Number 2012-02**

Revision E

# Table of Contents

# **Contents**

| 1. | Introduction and General Objectives | 3 |
|----|-----------------------------------------------------------|------|
| | Echo Timeline | |
| 3. | Examination Protocol – Cardiac Echo-Doppler | 4 |
| 4. | Site Echocardiographer Checklist | . 12 |
| 5. | Core Lab Echo Tracking Form | . 14 |
| 6. | Site Data Collection/ Entry into EDC (Echo Tracking Form) | . 14 |
| 7. | Shipping & Contact Information | . 16 |

#### 1. Introduction and General Objectives

Echocardiographic measures of aortic valve function, mitral valve function and left ventricular size and function are used as markers of success in this trial. The echocardiogram will be performed at specified time points. The majority of the echocardiograms will be transthoracic echocardiograms and this document focuses on this technique. The details of the image planes and the measurement conventions are described below.

#### 2. Echo Timeline

Each subject enrolled in the trial will have a completed echo at all of the following time points:

| Follow-up Visit | Visit Window |
|---|---|
| Screening | Day -60 to Day 0 |
| Operative (TEE) | Within 1 hr from cross clamp removal |
| Discharge | Prior to POD +10, or prior to Discharge, whichever is earlier |
| POD 105 | -15/+10 days |
| POD 390 | -25/+45 days |
| POD 730 | -25/+45 days |
| POD 1095 | -25/+45 days |
| POD 1460 | -25/+45 days |
| POD 1825 | -25/+45 days |
| POD 2190 (6 yr)* | -55/+75 days |
| POD 2555 (7 yr)* | -55/+75 days |
| POD 2920 (8 yr)* | -55/+75 days |
| POD 3285 (9 yr)* | -55/+75 days |
| POD 3650 (10yr)* | -55/+75 days |

<sup>\*</sup> Only required for subjects who have consented to continued follow-up with the Model 11000A valve at the top 3 enrolling sites.

All echocardiograms should be full transthoracic echocardiograms (TTE) except at the operative interval, where a full transesophageal echocardiogram (TEE) should be performed. A TEE may also be accepted for the baseline/screening echocardiogram.

If applicable, always label the echo (or CD) with Subject ID, Visit Interval, and Exam Date and attach the Echo (Site) worksheet with vitals/ heart rhythm information. Please check to see that the demographic information on the images matches the data sheet.

#### 3. Examination Protocol – Cardiac Echo-Doppler

#### **OBJECTIVES:**

- The primary objective of the initial echo-Doppler examination is to establish baseline cardiac anatomy and function with an emphasis on the aortic valve, aortic root and left ventricular size and function
- The primary goals of the follow-up post-implantation studies are to reassess the aortic valve prosthesis (structure and function) and to determine the impact of the implantation on the parameters evaluated.
- Complete Echo-Doppler examinations are required at the time points specified in the table above.
- Two-dimensional ultrasound imaging systems with pulsed, continuous wave and color Doppler capability, and permanent recording capabilities are required.
- The only accepted storage format is DICOM standard digital.
- You should have transducers with both fundamental and harmonic capability with frequency ranges that are suitable for most adult subjects (approximately 2 to 7 mHz).

#### EXAMINATION PREPARATION, POSITIONING, AND GENERAL PROCEDURES:

- A qualified physician or sonographer must perform all ultrasound exams. If possible, participating sites should attempt to utilize the same person as well as the same machine for image acquisition throughout the trial.
- Prior to starting the study, the physician/sonographer should provide the subject with an overview of the study (duration, general procedure etc).
- Subjects will typically be studied while they are in the left lateral decubitus position although occasionally the best images will be obtained with the subject supine.
- EKG leads will be applied and the EKG control setting of the machine optimized to ensure a high quality EKG with adequate amplitude QRS complex for reliable digital capture (lead II equivalent preferred).
- All views will be acquired with 2 captures OF EACH VIEW as follows:
  - o Sinus rhythm (up to 90 bpm): 3 beat capture
  - o Sinus rhythm (more than 90 bpm): 5 beat capture
  - o Frequent atrial or ventricular ectopy: 3 second capture
  - o Atrial fibrillation or flutter, paced rhythm: 5 second capture
- It is essential that the view be optimized and stabilized before recording. Images are typically acquired during quiet respiration. Breath-holding during recording is not required unless necessary to ensure a stable high quality image.
- The spatial resolution of the images should be optimized using the highest frequencies capable of providing adequate penetration. For each view, the gain, compression and focus should be optimized so that the best echocardiographic image of the endocardial borders is obtained.
- Use echo contrast if available for images with suboptimal endocardial definition

- The sweep speed for all spectral Doppler and M-mode recordings should be 100 mm/sec. NOTE: at least 3 consecutive sinus beats and at least 5 consecutive "irregular rhythm" beats must be captured, so adjust the number of captures accordingly.
- As defined in the ASE Guidelines for the Quantification of Native Valve Regurgitation, Nyquist settings for color Doppler assessment of the cardiac valves should be 50-60 cm/sec.
- We encourage you to perform measurements as needed for clinical feedback to treating physicians. If you do perform on-line measurements, please do not obscure the flow profiles of subsequent beats. We suggest storing BOTH measured and unmeasured Doppler spectra and images.
- Once the data storage/file save operation is complete, transmit the data to the Core Lab, utilizing the instruction documentation provided in the AG Mednet Desktop Agent.
  - De-identify the images through the AG Mednet while uploading data. Enter the subject information as specified on the Echo Tracking Form. Importantly, the height and weight will have to be entered at every follow-up interval. Please measure and note the blood pressure on the subject ID screen or as an annotation on one or more images.

#### **EXAMINATION SEQUENCE:**

#### 1. Parasternal Long Axis of LV, LVOT and AV

- 2D (Image A below)
- Color Doppler of MR
- Color Doppler of LVOT and aortic valve (AV) for aortic insufficiency
- Magnified views of LVOT and aortic valve to identify the true LVOT dimension, AV annulus and stent diameter (Image B below)
- · High parasternal view to see ascending aorta
- Off-axis views to search for aortic paravalvular leak
- Obtain an RV inflow view
- · Color flow Doppler of triscuspid valve
- Pulse wave Doppler of inflow 1-2cm below the valve
- · Continuous wave Doppler of TV
- Obtain RV outflow to include bifurcation if possible
- Color flow Doppler of PA
- Pulse wave Doppler of the pulmonary valve 1-2 cm below the valve in the outflow tract
- · Continuous wave Doppler of PA



#### II. Parasternal Short axis at LV level

- 2D should be obtained at 3 levels: apex, mid-papillary muscle and base
- Color Doppler of MR from the basal view is also requested

#### III. Parasternal Short axis at aortic valve level

- 2D
- Color Doppler of aortic valve including sewing ring of prosthesis to search for paravalvular leak
- Color Doppler of TR is optional in this view



#### IV. Apical 4 chamber

- 2D optimizing LV endocardial borders: Need to see all aspects of the lateral wall, septum, and apex
- Show a loop with decreased depth such that LV occupies most of the imaging sector ensuring all walls are visualized
- Color Doppler of MR showing entire left atrium (to allow jet dimension/LA measurement)
- If there is more than mild MR, provide components for PISA calculation
  - o CW of MR jet
  - o Zoomed PISA display (baseline shift down to optimize hemispherical PISA shell)
  - The aliasing velocity of color scale should be shifted down or towards MR jet to around 40cm/sec

o If possible, provide split screen (color suppress) images (i.e. one side with color, one without)

• Color Doppler of TR with CW



#### V. Apical 5 chamber view

- Pulse wave Doppler of LVOT (to avoid the region of flow acceleration sample volume should be positioned at valve level and then moved apically until valve noise or "clicks" are no longer detected and then recorded for the baseline study)
- For post-implantation studies, it is imperative that the sample volume be placed proximal to the valve frame AND at a second position within the valve frame but proximal to the valve cusps. Studies in which there are no clips with the sample volume proximal to the valve frame will be considered INADEQUATE.
- Note: record a full screen 2D image showing the pulse wave sample position (either as moving
  image or still frame) as well as the Pulse Wave Spectral Doppler for each position. It is very
  difficult to establish the sample volume position from the small image that is available when
  image and spectral display are provided simultaneously.
- Color Doppler of LVOT and aortic valve for AI (use off axis views to ensure that all AI jets are demonstrated)
- Continuous wave and pulse wave Doppler through the aortic valve
- Continuous wave Doppler through the aortic valve
- Pulse Wave Doppler the left ventricular outflow tract

#### VI. Apical 2 chamber

- 2D optimizing LV endocardial borders: Need to see all aspects of the anterior wall, inferior wall, and apex
- Show a loop with decreased depth such that LV occupies most of the imaging sector ensuring all walls are visualized
- Color Doppler of MR



\* Image A shows the traditional 2 chamber while image B shows the 2 chamber with decreased depth

#### VII. Apical long axis view (also known as 3 chamber view)

- Color Doppler of MR
- Color Doppler of LVOT and aortic valve for AI (use off axis views to ensure that all AI jets are demonstrated)
- Pulse Wave Doppler just apical to the valve frame as specified in apical 5 chamber view
- Note: record a full screen 2D image showing the pulsed wave sample position (either as moving image or still frame) as well as the Pulse Wave Spectral Doppler for each position
- Continuous Wave Doppler through the aortic valve



#### VIII. Right Parasternal view

• Continuous Wave Doppler through the aortic valve (Note: this view is particularly useful if you notice an anteriorly-directed transaortic jet from parasternal views)

#### IX. Suprasternal Notch view

- Pulsed Doppler of the descending thoracic aorta from the suprasternal notch should be obtained to assess for reversal of flow if significant (moderate or greater) aortic insufficiency is present (Note: sample volume is placed in the descending thoracic aorta below the take off of the subclavian artery).
- Continuous wave Doppler interrogation of the transaortic valvular flow should also be obtained using the pedoff transducer

#### X. Specific Comments on Imaging Planes

A. Parasternal long axis view is recorded with the transducer in the third or fourth intercostal space immediately to the left of the sternum. The transducer should be angled so that the aortic valve, mitral valve and left ventricle are in their long axis.

#### **IMAGING TIP 1: PARASTERNAL LONG AXIS VIEW**

It is important that the parasternal long axis view displays the true long axis of the ventricle with the left ventricle lying horizontally on the image. If it is impossible to obtain a single view which optimally displays the long axis of the aortic valve and aortic root as well as the long axis of the left ventricle, record 2 separate views. It is unacceptable to record an offaxis view in which the apex "points up" on the screen. If this type of image is obtained try moving the transducer up 1-2 intercostal spaces or having the subject take a breath in. Sometimes having the subject move to a more lateral decubitus position will help as well.

#### **IMAGING TIP 2: PARASTERNAL LONG AXIS VIEW**

Measurement of the left ventricular outflow tract and aortic annulus is a key component of the study. In pre-device imaging, it is important to note that the largest annulus may not be in a plane with valve opening centered in the aorta.

B. Parasternal short axis view is obtained by angling the probe 90° with respect to the parasternal long axis of the LV. The goal of this view is to obtain information about the aortic valve as well as the LV.

#### **IMAGING TIP 3: PARASTERNAL SHORT AXIS VIEW**

This is an essential view post-op to completely assess aortic regurgitation. This may be the only view in which prosthetic valve medial or lateral aortic regurgitant jets are imaged. Imaging at the level of as well as just below the leaflets may allow you to better image these jets.

- C. Apical four-chamber view provides considerable information including the relative sizes of the right and left ventricles and the regional function of the LV. The four chamber view is defined as a view which maximizes the LV long axis and the tricuspid and mitral annular dimensions. In this view, the full excursion of the mitral and tricuspid valves should be seen. The complete endocardial border of the LV will be traced for chamber volume assessment (method of discs) so all aspects including the apex should be visualized. In the apical four chamber view, color Doppler of mitral and tricuspid regurgitation should be recorded. The four chamber view should visualize the lateral, septal and apical walls.
- D. **Apical two-chamber** view should be obtained for the goal of assessment of LV size and function. The complete endocardial border of the LV will be traced for chamber volume assessment (method of discs) so all aspects including the apex should be visualized. The degree of MR by color Doppler will also be assessed. The two chamber view should visualize the anterior, inferior and apical walls.

#### **IMAGING TIP 4: APICAL 4 and 2 CHAMBER VIEWS**

Because we will measure volumes from the apical views as an important end-point of the study, please try to avoid apical foreshortening. If the view appears to be foreshortened, please bring the transducer down one intercostal space and have the subject take a breath in (particularly for the apical two-chamber view). Sometimes this will bring out a better (not foreshortened) view.

E. **Apical 5 chamber and 3 chamber** views are obtained to provide detailed information about the aortic valve color, spectral and continuous wave Doppler.

#### **IMAGING TIP 5: APICAL 5 and 3 CHAMBER VIEWS**

Both these views are essential in imaging post-device aortic regurgitant jets. Because we will be measuring jet vena contracta and jet length, a Res/Zoom view which includes imaging of the entire jet would be helpful. In addition, the 3Ch view may be used in the biplane Simpson's calculation of LV volume when the 2Ch view is inadequate. Thus, careful attention to endocardial definition is important.

#### XI. Abbreviations

2D=Two-dimensional

AI =Aortic Insufficiency

AR=Aortic Regurgitation

AV=Aortic Valve

AVA=Aortic valve area

BSA=Body Surface Area

CO=Cardiac Output

CSA=Cross sectional area

ED=End diastole

EF=Ejection fraction

ES=End systole

HR =Heart rate

LA=Left atrium

LV=Left Ventricle

LVED=Left ventricular end diastolic volume

LVEF=Left ventricular ejection fraction

LVES=Left ventricular end systolic volume

LVOT=Left ventricular outflow tract

MR=Mitral Regurgitation

MV=Mitral Valve

PI=Performance Index

PW=Pulse wave

SV=Stroke Volume

TR=Tricuspid Regurgitation

TVI or VTI=Time Velocity Integral

# 4. <u>Site Echocardiographer Checklist</u>

| Labeling ar | Labeling and Demographics: | | | | |
|---|---|---|---|---|---|
| Subject Stu | udy ID: | <u>.</u> | | | |
| Visit: | POD 390<br>6 yr | 2 yr<br>7 yr | | 4yr<br>9 yr | • |
| Height:<br>Weight: _<br>Heart Rate<br>Rhythm: _<br>Blood Pres<br>Systo | cm<br>kg<br>::bpm | | Ionth/Year) | | |
| 2D<br>Color<br>Color<br>Magn<br>High I | Doppler of MR<br>Doppler of LVC<br>lified views of L<br>Parasternal Vie | TLV, LVOT, Aorti<br>OT/aortic valve for<br>VOT and aortic valve for and aortic value (ascending aortic value) | or AR<br>valve<br>rta) | | |
| LV ap<br>LV<br>LV | mid-papillary r<br>base | | otional) | | |
| 2D<br>Color | rnal Short axis and Doppler of aor Doppler of TR | tic valve | | | |
| LV wi<br>Color<br>Color | | (with CW) | s | | |

| V. Apical 5 chamber view Pulsed Wave Doppler of LVOT (multiple levels) Continuous wave Doppler through the AV Color Doppler of LVOT and aortic valve |
|---|
| VI. Apical 2 chamber 2D optimizing LV endocardial borders LV with decreased depth Color Doppler of MR |
| VII. Apical long axis (3 chamber) view 2 D optimizing LV endocardial borders LV with decreased depth Pulsed Wave Doppler at the LVOT Continuous Wave Doppler through AV Color Doppler of LVOT and aortic valve for Al Color Doppler of MR |
| VIII. Right Parasternal view Continuous Wave Doppler through AV |
| IX. Suprasternal Notch view Pulsed Wave Doppler of the descending thoracic aorta for AI Continuous Wave Doppler through AV |

#### 5. Core Lab Echo Tracking Form

An Echo Tracking Form will be completed for each subject including the following information, and will be submitted along with the echo data via AG Mednet (vendor providing digital transfer of echo data) to the Core Lab:

- 1. Follow-up interval
- 2. Exam transfer date
- 3. Exam date
- 4. Subject number
- 5. Site number
- 6. Echo type: TTE/ TEE
- 7. Heart rate (bpm)
- 8. Cardiac rhythm
- 9. Site comments
- 10. Name and email of person completing form
- 11. Scan date
- 12. Date completed
- 13. DICOM scan date
- 14. Echo scanner manufacturer name and model
- 15. Subject height (cm) and weight (kg)

#### 6. Site Data Collection/ Entry into Oracle EDC (Echo Tracking Form)

Each echocardiogram should also be read by the sites and data should be entered on the appropriate case report form (CRF). Data to be reported in addition to what is requested in the Echo Tracking Form include the following measurements:

- Subject blood pressure (systolic and diastolic)
- LVOT assessment:
  - Peak velocity
  - Peak gradient
  - Mean gradient
  - ➤ VTI
- Aortic valve assessment:
  - Peak velocity
  - Peak gradient
  - Mean gradient
  - > VTI
  - Annulus size (cm)
  - > AV area (cm<sup>2</sup>)
- · Aortic regurgitation severity
  - > 0 None
  - > +1 Trivial/Trace

- > +2 Mild
- > +3 Moderate
- > +4 Severe
- > Indeterminate
- Mitral regurgitation severity
  - > 0 None
  - > +1 Trivial/Trace
  - > +2 Mild
  - > +3 Moderate
  - > +4 Severe
  - > Indeterminate
- LVEF
  - Range of LVEF
  - ➤ Method used to determine LVEF (single plane or biplane)
- Severity of paravalvular leak (PVL)
  - > 0 None
  - > +1 Trivial/Trace
  - > +2 Mild
  - > +3 Moderate
  - ➤ +4 Severe
  - > Indeterminate
- Assessment of RV function
  - Normal
  - Mildly reduced
  - > Severely reduced
  - > Indeterminate
- Method of delivery of echocardiographs to Core Lab
  - > Images uploaded, FedEx, UPS, DHL, Other
  - > Tracking number

#### 7. Shipping & Contact Information

A copy of all documents and data must be kept at your site. Documents and CD's must be labeled with the trial protocol number (Protocol # 2012-02), the site ID, subject ID, subject initials, exam date, and exam interval.

Though all data is preferred to be uploaded digitally via AG Mednet, if shipping CDs, please send us an e-mail at when you ship your package. Upon its receipt, an official e-mail notification will be sent from the Core Lab to your site coordinator. Please confirm that the e-mail notification correlates with your shipping records. You should contact the Core Lab immediately with any discrepancies or if you have shipped a study but you have not received an e-mail notification within 2 business days.

Please do not hesitate to contact us with any questions. For non-urgent communications, e-mail is typically the best means.

For echo-related urgent questions, please call

are looking forward to being your partners in this important clinical trial.

# Core Laboratory Procedure Manual (For Model 11000M)

ProspeCtive, nOn-randoMized, MulticENter Clinical evaluation of the Edwards Pericardial Aortic & Mitral Bioprostheses (Models 11000A & 11000M) with a new tissue treatment platform (COMMENCE TRIAL)

Clinical Protocol Number 2012-02

Revision F

# Table of Contents

# **Contents**

| 1. | Introduction and General Objectives | 3 |
|----|-----------------------------------------------------------|---|
| | Echo Timeline | |
| | Examination Protocol – Cardiac Echo-Doppler | |
| | Site Echocardiographer Checklist | |
| | Core Lab Echo Tracking Form | |
| | Site Data Collection/ Entry into EDC (Echo Tracking Form) | |
| | Shipping & Contact Information | |

#### 1. Introduction and General Objectives

Echocardiographic measures of aortic valve function, mitral valve function and left ventricular size and function are used as markers of success in this trial. The echocardiogram will be performed at specified time points. The majority of the echocardiograms will be transthoracic echocardiograms and this document focuses on this technique. The details of the image planes and the measurement conventions are described below.

#### 2. Echo Timeline

Each subject enrolled in the trial will have a completed echo at all of the following time points:

| Follow-up Visit | Visit Window |
|---|---|
| Screening | Day -60 to Day 0 |
| Operative (TEE) | Within 1 hr from cross clamp removal |
| Discharge | Prior to POD +10, or prior to Discharge, whichever is earlier |
| POD 105 | -15/+10 days |
| POD 390 | -25/+45 days |
| POD 730 | -25/+45 days |
| POD 1095 | -25/+45 days |
| POD 1460 | -25/+45 days |
| POD 1825 | -25/+45 days |
| POD 2190 (6 yr)* | -55/+75 days |
| POD 2555 (7 yr)* | -55/+75 days |
| POD 2920 (8 yr)* | -55/+75 days |
| POD 3285 (9 yr)* | -55/+75 days |
| POD 3650 (10yr)* | -55/+75 days |

<sup>\*</sup> Only required for subjects who have consented to continued follow-up with the Model 11000M valve at the 3 enrolling sites.

All echocardiograms should be full transthoracic echocardiograms (TTE) except at the operative interval, where a full transesophageal echocardiogram (TEE) should be performed. A TEE may also be accepted for the baseline/screening echocardiogram.

If applicable, always label the echo (or CD) with Subject ID, Visit Interval, and Exam Date and attach the Echo (Site) worksheet with vitals/ heart rhythm information. Please check to see that the demographic information on the images matches the data sheet.

#### 3. <u>Examination Protocol – Cardiac Echo-Doppler</u>

#### **OBJECTIVES:**

- The primary objective of the initial echo-Doppler examination is to establish baseline cardiac anatomy and function with an emphasis on the mitral valve and left ventricular size and function
- The primary goals of the follow-up post-implantation studies are to reassess the mitral valve prosthesis (structure and function) and to determine the impact of the implant on the parameters evaluated.
- Complete Echo-Doppler examinations are required at the time points specified in the table above.
- Two-dimensional ultrasound imaging systems with pulsed, continuous wave and color Doppler capability, and permanent recording capabilities are required.
- The only accepted storage format is DICOM standard digital.
- You should have transducers with both fundamental and harmonic capability with frequency ranges that are suitable for most adult subjects (approximately 2 to 7 mHz).

#### EXAMINATION PREPARATION, POSITIONING, AND GENERAL PROCEDURES:

- A qualified physician or sonographer must perform all ultrasound exams. If possible, participating sites should attempt to utilize the same person as well as the same machine for image acquisition throughout the trial.
- Prior to starting the study, the physician/sonographer should provide the subject with an overview of the study (duration, general procedure etc).
- Subjects will typically be studied while they are in the left lateral decubitus position although occasionally the best images will be obtained with the subject supine.
- EKG leads will be applied and the EKG control setting of the machine optimized to ensure a high quality EKG with adequate amplitude QRS complex for reliable digital capture (lead II equivalent preferred).
- All views will be acquired with 2 captures OF EACH VIEW as follows:
  - o Sinus rhythm (up to 90 bpm): 3 beat capture
  - Sinus rhythm (greater than 90 bpm): 5 beat capture
  - o Frequent atrial or ventricular ectopy: 3 second capture
  - o Atrial fibrillation or flutter, paced rhythm: 5 second capture
- It is essential that the view be optimized and stabilized before recording. Images are typically acquired during quiet respiration. Breath-holding during recording is not required unless necessary to ensure a stable high quality image.

- The spatial resolution of the images should be optimized using the highest frequencies capable of providing adequate penetration. For each view, the gain, compression and focus should be optimized so that the best echocardiographic image of the endocardial borders is obtained.
- Use echo contrast if available for images with suboptimal endocardial definition
- The sweep speed for all spectral Doppler and M-mode recordings should be 100 mm/sec. NOTE: at least 3 consecutive sinus beats and at least 5 consecutive "irregular rhythm" beats must be captured, so adjust the number of captures accordingly.
- As defined in the ASE Guidelines for the Quantification of Native Valve Regurgitation, Nyquist settings for color Doppler assessment of the cardiac valves should be 50-60 cm/sec.
- We encourage you to perform measurements as needed for clinical feedback to treating physicians. If you do perform on-line measurements, please do not obscure the flow profiles of subsequent beats. We suggest storing BOTH measured and unmeasured Doppler spectra and images.
- Once the data storage/file save operation is complete, transmit the data to the Core Lab, utilizing the instruction documentation provided in the AG Mednet Desktop Agent.
  - De-identify the images through the AG Mednet while uploading data. Enter the subject information as specified on the Echo Tracking Form. Importantly, the height and weight will have to be entered at every follow-up interval. Please measure and note the blood pressure on the subject ID screen or as an annotation on one or more images.

#### **EXAMINATION SEQUENCE:**

- 1. Parasternal Long Axis of LV, LVOT, and MV
- 2D (Image A below)
- Color Doppler of Aortic valve
- Color Doppler of Mitral Valve for mitral regurgitation
- Magnified views of LVOT and aortic valve to identify the true LVOT dimension
- Magnify Mitral valve
- Obtain an RV inflow view



#### II. Parasternal Short axis at LV level

- 2d should be obtained at 4 levels: apex, mid-papillary muscle, mitral valve, and LV outflow tract
- Color Doppler the Mitral valve for regurgitation at the mitral valve and LVOT level views.

#### III. Parasternal Short axis at aortic valve level

- 2D
- Zoom image of Aortic Valve
- Color Doppler of aortic valve
- Color Doppler of tricuspid valve



#### IV. Apical 4 chamber

- 2D optimizing LV endocardial borders: Need to see all aspects of the lateral wall, septum, and apex
- Zoom image of Mitral valve
- Show a loop with decreased depth such that LV occupies most of the imaging sector ensuring all walls are visualized
- Color Doppler of MR showing entire left atrium (to allow jet dimension/LA measurement)
- Provide components for PISA calculation
  - o CW of MR jet
  - o PW of MR jet
  - o Zoomed PISA display (baseline shift down to optimize hemispherical PISA shell)
  - The aliasing velocity of color scale should be shifted down or towards MR jet to around 40cm/sec
  - o If possible, provide split screen (color suppress) images (i.e. one side with color, one without)
  - o Pulse wave Doppler the mitral valve inflow. Maximize spectral Doppler wave form to provide a large enough tracing to make calculations.
  - o Continuous wave Doppler the mitral valve inflow. Maximize spectral Doppler wave form to provide a large enough tracing to make calculations.
- Color flow Doppler of tricuspid valve
- Continuous wave Doppler of TV



# V. Apical 5 chamber view

- 2D image of apical 5 chamber
- Pulse wave Doppler of LVOT (to avoid the region of flow acceleration sample volume should be positioned at valve level and then moved apically until valve noise or "clicks" are no longer detected and then recorded for the baseline study)
- Continuous wave Doppler through the aortic valve
- Note: record a full screen 2D image showing the pulse wave sample position (either as
  moving image or still frame) as well as the Pulse Wave Spectral Doppler for each position. It is
  very difficult to establish the sample volume position from the small image that is available
  when image and spectral display are provided simultaneously.

# VI. Apical 2 chamber

- 2D optimizing LV endocardial borders: Need to see all aspects of the anterior wall, inferior wall, and apex
- · Zoom image of Mitral valve
- Show a loop with decreased depth such that LV occupies most of the imaging sector ensuring all walls are visualized
- Color Doppler of MR



\* Image A shows the traditional 2 chamber while image B shows the 2 chamber with decreased depth

# VII. Apical long axis view (also known as 3 chamber view)

- 2D image of apical long axis
- Color Doppler of Mitral valve
- Zoom image of mitral valve
- Pulse Wave Doppler just **apical to the valve frame** as specified in apical 5 chamber view
- Note: record a full screen 2D image showing the pulsed wave sample position (either as moving image or still frame) as well as the Pulse Wave Spectral Doppler for each position
- Continuous Wave Doppler through the aortic valve



# VIII. Non imaging transducer in apical window

• Continuous wave Doppler interrogation of the mitral valvular flow should also be obtained using the pedoff transducer

#### IX. Specific Comments on Imaging Planes

A. Parasternal long axis view is recorded with the transducer in the third or fourth intercostal space immediately to the left of the sternum. The transducer should be angled so that the aortic valve, mitral valve and left ventricle are in their long axis.

# **IMAGING TIP 1: PARASTERNAL LONG AXIS VIEW**

It is important that the parasternal long axis view displays the true long axis of the ventricle with the left ventricle lying horizontally on the image. If it is impossible to obtain a single view which optimally displays the long axis of the aortic valve, mitral valve, and aortic root as well as the long axis of the left ventricle, record 2 separate views. It is unacceptable to record an off-axis view in which the apex "points up" on the screen. If this type of image is obtained try moving the transducer up 1-2 intercostal spaces or having the subject take a breath in. Sometimes having the subject move to a more lateral decubitus position will help as well.

#### **IMAGING TIP 2: PARASTERNAL LONG AXIS VIEW**

Measurement of the left ventricular outflow tract and aortic valve and mitral valve are the key components of the study.

B. Parasternal short axis view is obtained by angling the probe 90° with respect to the parasternal long axis of the LV. The goal of this view is to obtain information about the aortic valve, the mitral valve as well as the LV.

#### **IMAGING TIP 3: PARASTERNAL SHORT AXIS VIEW**

This is an essential view post-op to completely assess mitral regurgitation. This may be the only view in which prosthetic valve regurgitant jets are imaged. Imaging at the level of as well as just below the leaflets may allow you to better image these jets.

- C. Apical four-chamber view provides considerable information including the relative sizes of the right and left ventricles and the regional function of the LV. The four chamber view is defined as a view which maximizes the LV long axis and the tricuspid and mitral annular dimensions. In this view, the full excursion of the mitral and tricuspid valves should be seen. The complete endocardial border of the LV will be traced for chamber volume assessment (method of discs) so all aspects including the apex should be visualized. In the apical four chamber view, color Doppler of mitral and tricuspid regurgitation should be recorded. The four chamber view should visualize the lateral, septal and apical walls.
- D. **Apical two-chamber** view should be obtained for the goal of assessment of LV size and function. The complete endocardial border of the LV will be traced for chamber volume assessment (method of discs) so all aspects including the apex should be visualized. The degree of MR by color Doppler will also be assessed. The two chamber view should visualize the anterior, inferior and apical walls.

#### **IMAGING TIP 4: APICAL 4 and 2 CHAMBER VIEWS**

Because we will measure volumes from the apical views as an important end-point of the study, please try to avoid apical foreshortening. If the view appears to be foreshortened, please bring the transducer down one intercostal space and have the subject take a breath in (particularly for the apical two-chamber view). Sometimes this will bring out a better (not foreshortened) view.

E. **Apical 5 chamber and 3 chamber** views are obtained to provide detailed information about the aortic valve and mitral valve color, and the spectral and continuous wave Doppler.

# **IMAGING TIP 5: APICAL 5 and 3 CHAMBER VIEWS**

Both these views are essential in imaging post-device mitral regurgitant jets. Because we will be measuring jet vena contracta and jet length, a Res/Zoom view which includes imaging of the entire jet would be helpful. In addition, the 3Ch view may be used in the biplane Simpson's calculation of LV volume when the 2Ch view is inadequate. Thus, careful attention to endocardial definition is important.

#### XI. Abbreviations

2D=Two-dimensional

AI =Aortic Insufficiency

AR=Aortic Regurgitation

**AV=Aortic Valve** 

AVA=Aortic valve area

BSA=Body Surface Area

CO=Cardiac Output

CSA=Cross sectional area

ED=End diastole

EF=Ejection fraction

ES=End systole

HR =Heart rate

LA=Left atrium

LV=Left Ventricle

LVED=Left ventricular end diastolic volume

LVEF=Left ventricular ejection fraction

LVES=Left ventricular end systolic volume

LVOT=Left ventricular outflow tract

MR=Mitral Regurgitation

MV=Mitral Valve

PI=Performance Index

PW=Pulse wave

SV=Stroke Volume

TR=Tricuspid Regurgitation

TVI or VTI=Time Velocity Integral

# 4. Site Echocardiographer Checklist

| Labeling and | l Demographio | cs: | | | |
|---|---|---|---|---|---|
| Subject Stud | y ID: | | | | |
| Visit: | POD 390<br>6 yr | 2 yr<br>7 yr | Discharge<br>3yr<br>8 yr | 4yr<br>9 yr | • |
| Height:<br>Weight:<br>Heart Rate: _<br>Rhythm:<br>Blood Pressu<br>Systolic | cm<br>kg<br>bpm | | Ionth/Year) | | |
| 2D<br>Color D<br>Magnif | oppler of Mit | LV, LVOT, MV v<br>ral Valve for MF<br>VOT and aortic v<br>itral valve | 1 | | |
| LV apea<br>LV mid-<br>LV Mitr<br>LVOT | papillary mus<br>al valve | cle | regurgitation at | the mitral valv | e and LVOT level |
| 2D | nal Short axis a | | | | |
| LV with<br>Zoom I<br>Color D | | ral valve<br>with CW) | s | | |

| V. Apical 5 chamber view | Ja) | | | | | |
|---|---|---|---|---|---|---|
| Pulsed Wave Doppler of LVOT (multiple leve Continuous wave Doppler through the AV | 115) | | | | | |
| VI. Apical 2 chamber 2D optimizing LV endocardial borders LV with decreased depth Zoom Mitral valve Color Doppler of Mitral valve | | | | | | |
| VII. Apical long axis (3 chamber) view 2 D optimizing LV endocardial borders LV with decreased depth Zoom Mitral valve Pulsed Wave Doppler at the LVOT Continuous Wave Doppler through AV Color Doppler of Mitral valve for MR | | | | | | |
| VIII. Non imaging transducer in apical window | | | | | | |
| Continuous wave Doppler interrogation o obtained using the pedoff transducer | of the Mitr | al valvular | flow | should | also | be |

# 5. Core Lab Echo Tracking Form

An Echo Tracking Form will be completed for each subject including the following information, and will be submitted along with the echo data via AG Mednet (vendor providing digital transfer of echo data) to the Core Lab:

- 1. Follow-up interval
- 2. Exam transfer date
- 3. Exam date
- 4. Subject number
- 5. Site number
- 6. Echo type: TTE/ TEE
- 7. Heart rate (bpm)
- 8. Cardiac rhythm
- 9. Site comments
- 10. Name and email of person completing form
- 11. Scan date
- 12. Date completed
- 13. DICOM scan date
- 14. Echo scanner manufacturer name and model
- 15. Subject height (cm) and weight (kg)

# 6. Site Data Collection/ Entry into Oracle EDC (Echo Tracking Form)

Each echocardiogram should also be read by the sites and data should be entered on the appropriate case report form (CRF). Data to be reported in addition to what is requested in the Echo Tracking Form include the following measurements:

- Subject blood pressure (systolic and diastolic)
- LVOT assessment:
  - Peak velocity
  - Peak gradient
  - > Mean gradient
  - ➤ VTI
- Mitral valve assessment:
  - Peak velocity
  - Peak gradient
  - Mean gradient
  - ➤ VTI
  - Annulus size (cm)
  - ➤ MV area (cm²)
- Mitral regurgitation severity (Paravalvular, Transvalvular and Total Insufficiency/Regurgitation)

- > 0 None
- > +1 Trivial/Trace
- > +2 Mild
- > +3 Moderate
- > +4 Severe
- > Indeterminate
- Non-study valve regurgitation severity
  - > 0 None
  - > +1 Trivial/Trace
  - > +2 Mild
  - > +3 Moderate
  - > +4 Severe
  - > Indeterminate
- LVEF
  - Range of LVEF
  - ➤ Method used to determine LVEF (single plane or biplane)
- Assessment of RV function
  - Normal
  - > Mildly reduced
  - > Severely reduced
  - > Indeterminate
- Method of delivery of echocardiographs to Core Lab
  - > Images uploaded, FedEx, UPS, DHL, Other
  - > Tracking number

# 7. Shipping & Contact Information

A copy of all documents and data must be kept at your site. Documents and CD's must be labeled with the trial protocol number (Protocol # 2012-02), the site ID, subject initials, exam date, and exam interval.

Though all data is preferred to be uploaded digitally via AG Mednet, if shipping CDs, please send us an e-mail at when you ship your package. Upon its receipt, an official e-mail notification will be sent from the Core Lab to your site coordinator. Please confirm that the e-mail notification correlates with your shipping records. You should contact the Core Lab immediately with any discrepancies or if you have shipped a study but you have not received an e-mail notification within 2 business days.

Please do not hesitate to contact us with any questions. For non-urgent communications, email is typically the best means.

For echo-related urgent questions, please call

We are looking forward to being your partners in this important clinical trial.

EDWARDS LIFESCIENCES LLC
CLINICAL INVESTIGATIONAL PLAN


# ATTACHMENT F – SERUM GLYCEROL SAMPLE COLLECTION MANUAL

No Longer In Use

REVISION J: 03 MARCH 2021

# ATTACHMENT G – QUALITY OF LIFE QUESTIONNAIRE

(SF-12 V2)

No Longer In Use

REVISION J: 03 MARCH 2021

| CLINICAL INVESTIGATIONAL PLAN<br>PROTOCOL NUMBER: 2012-02 |
|-----------------------------------------------------------|
| ATTACHMENT H – ADVERSE EFFECT (CODES & DEFINITIONS) |

**ATTACHMENTS** 

REVISION J: 03 MARCH 2021

**EDWARDS LIFESCIENCES LLC** 

# Clinical Investigational Plan

Protocol Number: 2012-02

| | AE CODE LIST | |
|---|---|---|
| CODE | LABEL/NAME | DEFINITION |
| AE.1 | BLOOD AND LYMPHATIC (INCLUDING ALL BLEEDING COMPLICATIONS) | |
| AE101 | ANEMIA - NON-BLEEDING RELATED | A CONDITION IN WHICH RED BLOOD CELL COUNT AND/OR HEMOGLOBIN ARE LESS THAN NORMAL DUE TO LACK OF PRODUCTION OF RED BLOOD CELLS, AND THAT REQUIRES TREATMENT OR TRANSFUSION. |
| AE102 | ANEMIA - BLEEDING RELATED - MAJOR | A CONDITION IN WHICH RED BLOOD CELL COUNT AND/OR HEMOGLOBIN ARE LESS THAN NORMAL DUE TO BLOOD LOSS, AND THAT REQUIRES TREATMENT OR TRANSFUSION. |
| AE103 | ANEMIA - BLEEDING RELATED - MINOR | A CONDITION IN WHICH RED BLOOD CELL COUNT AND/OR HEMOGLOBIN ARE LESS THAN NORMAL DUE TO BLOOD LOSS, AND THAT REQUIRES TREATMENT OR TRANSFUSION. |
| AE104 | BLEEDING - CARDIOVASCULAR - MAJOR | ANY EPISODE OF MAJOR INTERNAL OR EXTERNAL BLEEDING THAT CAUSES DEATH, HOSPITALIZATION, OR PERMANENT INJURY (E.G., VISION LOSS) OR NECESSITATES TRANSFUSION, PERICARDIOCENTESIS, OR REOPERATION. MAJOR BLEEDING UNEXPECTEDLY ASSOCIATED WITH MINOR TRAUMA SHOULD BE REPORTED AS A BLEEDING EVENT, BUT BLEEDING ASSOCIATED WITH MAJOR TRAUMA OR A MAJOR OPERATION (INCLUDING THE INDEX PROCEDURE) SHOULD NOT. THE LOCATION OF THE BLEEDING (GASTROINTESTINAL, GENITOURINARY, ETC.) MUST BE REPORTED. FOR EACH REPORTED BLEEDING EVENT, INDICATE IF SUBJECT IS TAKING ANTICOAGULANTS OR ANTI-PLATELET AGENTS. |
| AE105 | BLEEDING - CARDIOVASCULAR - MINOR | " |
| AE106 | BLEEDING - GENITOURINARY - MAJOR | " |
| AE107 | BLEEDING - GENITOURINARY - MINOR | " |
| AE108 | BLEEDING - GASTROINTESTINAL UPPER -MAJOR | " |
| AE109 | BLEEDING - GASTROINTESTINAL UPPER -MINOR | " |
| AE110 | BLEEDING - GASTROINTESTINAL LOWER -MAJOR | " |
| AE111 | BLEEDING - GASTROINTESTINAL LOWER -MINOR | п |
| AE112 | BLEEDING - MUSCULOSKELETAL/DERMATOLOGICAL -MAJOR | " (E.G. ECCHYMOSIS) |
| AE113 | BLEEDING - MUSCULOSKELETAL/DERMATOLOGICAL -MINOR | " (E.G. ECCHYMOSIS) |
| AE114 | BLEEDING - NEUROLOGICAL - MAJOR | " (E.G. CEREBRAL VASCULAR ACCIDENT) |
| AE115 | BLEEDING - NEUROLOGICAL - MINOR | " (E.G. CEREBRAL VASCULAR ACCIDENT) |
| AE116 | BLEEDING - PERIPHERAL VASCULAR -MAJOR | " (E.G. NOSEBLEEDS; HEMATOMAS) |
| AE117 | BLEEDING - PERIPHERAL VASCULAR - MINOR | " (E.G. NOSEBLEEDS; HEMATOMAS) |
| AE118 | BLEEDING - PULMONARY/RESPIRATORY - MAJOR | " (E.G. HEMOTHORAX) |
| AE119 | BLEEDING - PULMONARY/RESPIRATORY MINOR | " (E.G. HEMOTHORAX) |
| AE120 | BLOOD SEPSIS | POSITIVE BLOOD CULTURE AND CLINICAL EVIDENCE OF INFECTION (E.G. FEVER, ELEVATED WBC COUNT, HYPOTENSION, END ORGAN DYSFUNCTION) EVENT MUST BE CONFIRMED BY 2 CONSECUTIVE POSITIVE BLOOD CULTURES, EXPLANT OR AUTOPSY. |

# Clinical Investigational Plan Protocol Number: 2012-02

| | AE CODE LIST | |
|---|---|---|
| CODE | LABEL/NAME | DEFINITION |
| AE.1 | BLOOD AND LYMPHATIC (INCLUDING ALL BLEEDING COMPLICATIONS) (CONTINUED) | |
| AE122 | HEMOLYSIS WITHOUT PARAVALVULAR LEAK | PLASMA -FREE HEMOGLOBIN > 40 MG/DL ON TWO CONSECUTIVE MEASUREMENTS WITHIN 48 HOURS; OR CLINICAL DIAGNOSIS OF HEMOLYSIS EVIDENCED BY LABORATORY TESTING SUCH AS SERUM HEMOGLOBIN, HEMATOCRIT, AND/OR PLASMA-FREE HEMOGLOBIN (NOT IMMUNOLOGICALLY BASED) |
| AE123 | DISSEMINATED INTRAVASCULAR COAGULATION (DIC) | DIFFUSE, NONSURGICAL, MICROVASCULAR HEMORRHAGE AND/OR THROMBOSES. |
| AE124 | THROMBOCYTOPENIA - HEPARIN INDUCED (HIT) | THROMBOCYTOPENIA (<150,000 PER CUBIC MILLIMETER), OR A RELATIVE DECREASE OF 50 PERCENT OR MORE FROM BASELINE, OR NEW THROMBOSIS IN A SUBJECT RECEIVING HEPARIN OR LMWH; CONFIRMED BY SEROLOGIC TESTING FOR PF4—HEPARIN ANTIBODIES. |
| AE125 | THROMBOCYTOPENIA - NON-HEPARIN INDUCED | THROMBOCYTOPENIA (<150,000 PER CUBIC MILLIMETER), OR A RELATIVE DECREASE OF 50 PERCENT OR MORE FROM BASELINE, ACCOMPANIED BY A LOW INDEX OF SUSPICION FOR HIT (I.E., NOT ASSOCIATED WITH HEPARIN USE, THE PRESENCE OF OTHER CAUSES OF THROMBOCYTOPENIA, SUCH AS DRUGS OTHER THAN HEPARIN, DIC OR OTHER CONSUMPTIVE PROCESSES, POST-TRANSFUSION PURPURA). |
| AE126 | BLOOD/ LYMPHATIC - OTHER | OTHER BLOOD OR LYMPHATIC EVENT THAT DOES NOT FIT IN ONE OF THE OTHER "BLOOD" CATEGORIES THAT REQUIRES HOSPITALIZATION OR MEDICAL INTERVENTION. |
| AE.2 | CARDIOVASCULAR - ARRHYTHMIA | |
| AE158 | ARRHYTHMIA - PERMANENT ATRIAL FIBRILLATION | AN ABNORMAL HEARTBEAT IN WHICH THE HEART RHYTHM IS FAST AND IRREGULARLY IRREGULAR. EVENT SHOULD BE DOCUMENTED AND CONFIRMED BY ECG TEST RESULTS. AF IS CONSIDERED PERMANENT WHEN IT HAS PERSISTED BEYOND 1 YEAR AND ATTEMPTS AT CARDIOVERSION HAVE FAILED OR COULD NOT BE ATTEMPTED. |
| AE149 | ARRHYTHMIA - PAROXYSMAL ATRIAL FIBRILLATION (PAF) | AN ABNORMAL HEARTBEAT IN WHICH THE HEART RHYTHM IS FAST AND IRREGULARLY IRREGULAR. EVENT SHOULD BE DOCUMENTED AND CONFIRMED BY ECG TEST RESULTS. AF IS CONSIDERED PAROXYSMAL WHEN EPISODES OF AF TERMINATE SPONTANEOUSLY WITHIN 7 DAYS (MOST EPISODES LAST LESS THAN 24 HOURS) |
| AE157 | ARRHYTHMIA - PERSISTENT ATRIAL FIBRILLATION | AN ABNORMAL HEARTBEAT IN WHICH THE HEART RHYTHM IS FAST AND IRREGULARLY IRREGULAR. EVENT SHOULD BE DOCUMENTED AND CONFIRMED BY ECG TEST RESULTS. AF IS CONSIDERED PERSISTENT WHEN EPISODES OF AF LAST MORE THAN 7 DAYS AND MAY REQUIRE EITHER PHARMACOLOGIC OR ELECTRICAL INTERVENTION TO TERMINATE |
| AE141 | ARRHYTHMIA - ATRIAL FLUTTER | WELL ORGANIZED BUT OVERLY RAPID CONTRACTIONS OF HEART ATRIUM (USUALLY AT A RATE OF 250-350 CONTRACTIONS PER MINUTE). EVENT SHOULD BE DOCUMENTED AND CONFIRMED BY ECG TEST RESULTS. |
| AE142 | ARRHYTHMIA - AV BLOCK - 1ST DEGREE | AV BLOCK I: A CONDUCTION DISORDER OF NERVOUS IMPULSE AT THE LEVEL OF THE ATRIOVENTRICULAR JUNCTION, I.E. BETWEEN ATRIUM AND VENTRICLE. |
| AE143 | ARRHYTHMIA - AV BLOCK - 2ND DEGREE | " AV BLOCK II: THERE ARE TWO TYPES: MOBITZ I PROGRESSIVE PROLONGATION OF PR INTERVAL WITH DROPPED BEATS (THE PR INTERVAL GETS LONGER AND LONGER; FINALLY ONE BEAT DROPS) MOBITZ II PR INTERVAL REMAINS UNCHANGED PRIOR TO THE P-WAVE WHICH SUDDENLY FAILS TO CONDUCT TO THE VENTRICLES; |
| AE144 | ARRHYTHMIA - AV BLOCK - 3RD DEGREE | " AV BLOCK III: , NO P-WAVES CONDUCT TO THE VENTRICLE AND AV DISSOCIATION IS COMPLETE. ANY LEVEL OF AV BLOCK EVENT SHOULD BE DOCUMENTED AND CONFIRMED BY ECG TEST RESULTS. |
| AE145 | ARRHYTHMIA - BUNDLE BRANCH BLOCK - LEFT | BUNDLE BRANCH BLOCK IS AN INTRAVENTRICULAR CONDUCTION DEFECT (IVCD) THAT DISRUPTS THE NORMAL FLOW OF ELECTRICAL IMPULSES THAT RESULT IN A NORMAL HEART BEAT. QRS DURATION OF GREATER THAN 110 MILLISECONDS IS A DIAGNOSTIC INDICATION OF BBB. EVENT SHOULD BE DOCUMENTED AND CONFIRMED BY ECG TEST RESULTS. |

# Clinical Investigational Plan Protocol Number: 2012-02

| | AE CODE LIST | |
|---|---|---|
| CODE | LABEL/NAME | DEFINITION |
| AE.2 | CARDIOVASCULAR – ARRHYTHMIA (CONTINUED) | |
| AE146 | ARRHYTHMIA - BUNDLE BRANCH BLOCK - RIGHT | " |
| AE147 | ARRHYTHMIA - SUPRAVENTRICULAR TACHYCARDIA (SVT) SUSTAINED TACHYARRHYTHMIA IN WHICH THE QRS APPEARS NORMAL AND HAS DURATION OF < 120 MSEC. EVENT SHOULD BE DOCUMENTED AND CONFIRMED BY ECG TEST RESULTS. | |
| AE148 | ARRHYTHMIA - PAROXYSMAL ATRIAL TACHYCARDIA (PAT) | A RAPID HEART RHYTHM ORIGINATING ABOVE THE VENTRICULAR TISSUE DUE TO AV NODAL REENTRANT TACHYCARDIA. EVENT SHOULD BE DOCUMENTED AND CONFIRMED BY ECG TEST RESULTS. |
| AE150 | ARRHYTHMIA - VENTRICULAR FIBRILLATION | A RAPID IRREGULAR VENTRICULAR RHYTHM DUE TO MULTIPLE REENTRANT ACTIVITIES ASSOCIATED WITH ESSENTIALLY ZERO CARDIAC OUTPUT. EVENT SHOULD BE DOCUMENTED AND CONFIRMED BY ECG TEST RESULTS. |
| AE151 | AN ABNORMALLY FAST HEART RATE (TYPICALLY DEFINED AS >100 BPM IN ADULTS) WHICH MAY REQUIRE IMPLANT OF A PACEMAKER TO MAINTAIN A NORMAL HEART RATE. EVENT SHOULD BE DOCUMENTED AND CONFIRMED BY ECG TEST RESULTS. VENTRICULAR TACHYCARDIA: DEFINED AS A REGULAR HEART RHYTHM ORIGINATING FROM THE VENTRICLE WITH A FREQUENCY OF 160 TO 200 BEATS PER MINUTE. EVENT SHOULD BE DOCUMENTED AND CONFIRMED BY ECG TEST RESULTS. | |
| AE152 | ARRHYTHMIA - TACHYCARDIA - NON-VENTRICULAR ASSUMED " | |
| AE153 | AN ABNORMALLY SLOW HEART RATE (TYPICALLY DEFINED AS <60 BPM IN ADULTS) EVENT SHOULD BE DOCUMENTE AND CONFIRMED BY ECG TEST RESULTS. | |
| AE154 | A VARIANT OF SICK SINUS SYNDROME IN WHICH SLOW ARRHYTHMIAS AND FAST ARRHYTHMIAS ALTERNATE. EVENT SHOULD BE DOCUMENTED AND CONFIRMED BY ECG TEST RESULTS. | |
| AE155 | ARRHYTHMIA - PACEMAKER/ICD MALFUNCTION | PACEMAKER/ICD DOES NOT FUNCTION AS INTENDED. |
| AE156 | ARRHYTHMIA - OTHER | ARRHYTHMIA THAT IS NOT COVERED BY ANY OF THE DEFINITIONS ABOVE. PLEASE SPECIFY |
| AE.3 | CARDIOVASCULAR - REGURGITATION | |
| | IF THE VALVE INVOLVED IS THE STUDY VALVE, THEN THIS DEFINITION SHOULD BE USED, BUT THE EVENT SHOULD BE REPORTED AS STRUCTURAL OR NON-STRUCTURAL VALVE DYSFUNCTION (AS APPROPRIATE) REGURGITATION, AORTIC: ALSO KNOWN AS AORTIC INSUFFICIENCY AND INCOMPETENCE OF THE AORTIC VALVE, IN WHICH A PORTION OF THE LEFT VENTRICULAR FORWARD STROKE VOLUME RETURNS TO THE CHAMBER DURING DIASTOLE. THIS CATEGORY DOES NOT INCLUDE PARAVALVULAR LEAK, WHICH SHOULD BE CAPTURED UNDER NON-STRUCTURAL VALVE DYSFUNCTION. REGURGITATION, CENTRAL: OCCURS WHEN THE VALVE LEAFLETS DO NOT COMPLETELY CLOSE AND ALLOW SOME BLOOD TO LEAK BACK INTO THE HEART. REGURGITATION, INDETERMINATE: OCCURS WHEN BLOOD LEAKS BACK INTO THE HEART AND CANNOT BE CATEGORIZED BY LOCATION AND OR SEVERITY. REGURGITATION, MITRAL: ALSO KNOWN AS MITRAL INCOMPETENCE AND MITRAL INSUFFICIENCY IN WHICH THE BLOOD FLOWS BACKWARDS THROUGH THE MITRAL VALVE EACH TIME THE LEFT VENTRICLE CONTRACTS. DIAGNOSED BY AUSCULTATION (MURMUR) OR ECHOCARDIOGRAPHY. REGURGITATION, TRICUSPID: INSUFFICIENCY OF THE TRICUSPID VALVE CAUSING BLOOD FLOW FROM THE RIGHT VENTRICLE TO THE RIGHT ATRIUM DURING SYSTOLE. | |
| AE160 | REGURGITATION - AORTIC-CENTRAL/TRANSVALVULAR-+1 TRIVIAL/TRACE | |
| AE161 | 1 REGURGITATION - AORTIC-CENTRAL/TRANSVALVULAR-+2 MILD | |
| AE162 | REGURGITATION - AORTIC-CENTRAL/TRANSVALVULAR-+3 | MODERATE |
| AE163 | REGURGITATION - AORTIC-CENTRAL/TRANSVALVULAR-+4 | SEVERE |
| AE168 | REGURGITATION - AORTIC-INDETERMINATE-+1 | TRIVIAL/TRACE |

# Clinical Investigational Plan Protocol Number: 2012-02

| | AE CODE LIST | |
|---|---|---|
| CODE | LABEL/NAME | DEFINITION |
| AE.3 | CARDIOVASCULAR - REGURGITATION (CONTINUED) | |
| AE169 | REGURGITATION - AORTIC-INDETERMINATE-+2 | MILD |
| AE170 | REGURGITATION - AORTIC-INDETERMINATE-+3 | MODERATE |
| AE171 | REGURGITATION - AORTIC-INDETERMINATE-+4 | SEVERE |
| AE172 | REGURGITATION - MITRAL-CENTRAL/TRANSVALVULAR-+1 | TRIVIAL/TRACE |
| AE173 | REGURGITATION - MITRAL-CENTRAL/TRANSVALVULAR-+2 | MILD |
| AE174 | REGURGITATION - MITRAL-CENTRAL/TRANSVALVULAR-+3 | MODERATE |
| AE175 | REGURGITATION - MITRAL-CENTRAL/TRANSVALVULAR-+4 | SEVERE |
| AE180 | REGURGITATION - MITRAL-INDETERMINATE-+1 | TRIVIAL/TRACE |
| AE181 | REGURGITATION - MITRAL-INDETERMINATE-+2 | MILD |
| AE182 | REGURGITATION - MITRAL-INDETERMINATE-+3 | MODERATE |
| AE183 | REGURGITATION - MITRAL-INDETERMINATE-+4 | SEVERE |
| AE190 | REGURGITATION - PULMONARY-CENTRAL/TRANSVALVULAR-+1 | TRIVIAL/TRACE |
| AE191 | REGURGITATION - PULMONARY-CENTRAL/TRANSVALVULAR-+2 | MILD |
| AE192 | REGURGITATION - PULMONARY-CENTRAL/TRANSVALVULAR-+3 | MODERATE |
| AE193 | REGURGITATION - PULMONARY-CENTRAL/TRANSVALVULAR-+4 | SEVERE |
| AE198 | REGURGITATION - PULMONARY-INDETERMINATE-+1 | TRIVIAL/TRACE |
| AE199 | REGURGITATION - PULMONARY-INDETERMINATE-+2 | MILD |
| AE200 | REGURGITATION - PULMONARY-INDETERMINATE-+3 | MODERATE |
| AE201 | REGURGITATION - PULMONARY-INDETERMINATE-+4 | SEVERE |
| AE202 | REGURGITATION - TRICUSPID-CENTRAL/TRANSVALVULAR-+1 | TRIVIAL/TRACE |
| AE203 | REGURGITATION - TRICUSPID-CENTRAL/TRANSVALVULAR-+2 | MILD |
| AE204 | REGURGITATION - TRICUSPID-CENTRAL/TRANSVALVULAR-+3 | MODERATE |
| AE205 | REGURGITATION - TRICUSPID-CENTRAL/TRANSVALVULAR-+4 | SEVERE |
| AE210 | REGURGITATION - TRICUSPID-INDETERMINATE-+1 | TRIVIAL/TRACE |
| AE211 | REGURGITATION - TRICUSPID-INDETERMINATE-+2 | MILD |
| AE212 | REGURGITATION - TRICUSPID-INDETERMINATE-+3 | MODERATE |
| AE213 | REGURGITATION - TRICUSPID-INDETERMINATE-+4 | SEVERE |

# Clinical Investigational Plan

Protocol Number: 2012-02

| AE CODE LIST | | |
|---|---|---|
| CODE | LABEL/NAME | DEFINITION |
| AE.5 | CARDIOVASCULAR - STENOSIS | *IF THE VALVE INVOLVED IS THE STUDY VALVE, THEN THIS DEFINITION SHOULD BE USED, BUT THE EVENT SHOULD BE REPORTED AS STRUCTURAL OR NON-STRUCTURAL VALVE DYSFUNCTION (AS APPROPRIATE) |
| AE220* | STENOSIS - AORTIC - MILD | AORTIC: FLOW OBSTRUCTION OF THE AORTIC VALVE DUE TO RESTRICTED LEAFLET OPENING. THE SEVERITY IS CATEGORIZED AS: MILD - JET VELOCITY (M/S) <3.0; MEAN GRADIENT (MMHG) <25; VALVE AREA (CM2) >1.5. MODERATE - JET VELOCITY (M/S) 3.0-4.0; MEAN GRADIENT (MMHG) 25-40; VALVE AREA (CM2) 1.0-1.5. OR SEVERE - JET VELOCITY (M/S) >4.0; MEAN GRADIENT (MMHG) >40; VALVE AREA (CM2) <1.0; VALVE AREA INDEX<0.6. MITRAL: MITRAL STENOSIS (MS) REFERS TO NARROWING OF THE MITRAL VALVE ORIFICE, RESULTING IN IMPEDANCE OF FILLING OF THE LEFT VENTRICLE IN DIASTOLE. THE SEVERITY OF MS IS CATEGORIZED AS: MILD - MEAN GRADIENT (MM HG) < 5, PULMONARY ARTERY SYSTOLIC PRESSURE (MM HG) <30, VALVE AREA (CM2) >1.5. MODERATE - MEAN GRADIENT (MM HG) 5-10, PULMONARY ARTERY SYSTOLIC PRESSURE (MM HG) 30-50, VALVE AREA (CM2) 1.0-1.5. SEVERE - MEAN GRADIENT (MM HG) > 10, PULMONARY ARTERY SYSTOLIC PRESSURE (MM HG)> 50, VALVE AREA (CM2) <1.0. TRICUSPID: A NARROWING OF THE TRICUSPID VALVE OPENING THAT INCREASES RESISTANCE TO BLOOD FLOW FROM THE RIGHT ATRIUM TO THE RIGHT VENTRICLE. SEVERE TRICUSPID STENOSIS IS DEFINED AS A VALVE AREA LESS THAN 1.0 CM2. |
| AE221* | STENOSIS - AORTIC - MODERATE | п |
| AE222* | STENOSIS - AORTIC - SEVERE | II . |
| AE223 | STENOSIS - MITRAL- MILD | " |
| AE224 | STENOSIS - MITRAL - MODERATE | " |
| AE225 | STENOSIS - MITRAL - SEVERE | " |
| AE226 | STENOSIS - PULMONARY- MILD | " |
| AE227 | STENOSIS - PULMONARY - MODERATE | n e e e e e e e e e e e e e e e e e e e |
| AE228 | STENOSIS - PULMONARY - SEVERE | " |
| AE229 | STENOSIS - TRICUSPID- MILD | " |
| AE230 | STENOSIS - TRICUSPID- MODERATE | " |
| AE231 | STENOSIS - TRICUSPID - SEVERE | " |

Clinical Investigational Plan Protocol Number: 2012-02

| AE CODE LIST | | |
|---|---|---|
| CODE | LABEL/NAME | DEFINITION |
| AE.6 | CARDIOVASCULAR - THROMBOEMBOLIC EVENT/VALVE THROMBOSIS | ANY EMBOLIC EVENT THAT OCCURS IN THE ABSENCE OF INFECTION AFTER THE IMMEDIATE PERIOPERATIVE PERIOD AND MAY BE MANIFESTED BY A NEUROLOGIC EVENT OR A NON-CEREBRAL EMBOLIC EVENT. EMBOLI CONSISTING OF NON-THROMBOTIC MATERIAL (E.G., ATHEROSCLEROSIS, MYXOMA) ARE NOT COUNTED. |
| AE250 | THROMBOEMBOLIC EVENT — STROKE | INCLUDES ANY CENTRAL, NEW NEUROLOGIC DEFICIT, WHETHER TEMPORARY OR PERMANENT AND WHETHER FOCAL OR GLOBAL, THAT OCCURS AFTER THE SUBJECT EMERGES FROM ANESTHESIA. POSTOPERATIVE NEUROLOGIC SYMPTOMS THAT MIMIC THOSE OF A PREOPERATIVELY DOCUMENTED NEUROLOGIC EVENT AND THAT ARE CONFIRMED RADIOGRAPHICALLY TO BE CONSISTENT WITH THE FORMER EVENT ARE NOT COUNTED. CENTRAL NEUROLOGIC EVENTS THAT ARE CLEARLY RELATED TO AORTIC, INTERNAL CAROTID ARTERY, OR VERTEBRAL ARTERY DISEASE ARE ALSO NOT COUNTED. PSYCHOMOTOR DEFICITS FOUND BY SPECIALIZED TESTING ARE NOT CONSIDERED NEUROLOGIC EVENTS RELATED TO OPERATED VALVES. SUBJECTS WHO DO NOT AWAKEN OR WHO AWAKEN AFTER OPERATION WITH A NEW STROKE ARE NOT CONSIDERED TO HAVE SUSTAINED VALVE-RELATED NEUROLOGIC EVENTS. STROKE: A PROLONGED (>72 HOURS) OR PERMANENT NEUROLOGIC DEFICIT THAT IS USUALLY ASSOCIATED WITH ABNORMAL RESULTS OF MRI OR CT SCANS. SUBJECTS WITH MINIMAL, ATYPICAL, OR PROTEAN SYMPTOMS THAT LEAD TO RADIOGRAPHIC IMAGING DEMONSTRATING AN ACUTE ISCHEMIC EVENT ARE CONSIDERED TO HAVE SUSTAINED A STROKE. TIA: CHARACTERIZED BY FULLY REVERSIBLE SYMPTOMS OF SHORT DURATION. IF RADIOGRAPHIC IMAGING DEMONSTRATES AN ACUTE CENTRAL NEUROLOGIC LESION, HOWEVER, SUCH SUBJECTS ARE RECLASSIFIED AS HAVING SUSTAINED A STROKE. |
| AE255 | THROMBOEMBOLIC EVENT – TRANSIENT ISCHEMIC ATTACK (TIA) | INCLUDES ANY CENTRAL, NEW NEUROLOGIC DEFICIT, WHETHER TEMPORARY OR PERMANENT AND WHETHER FOCAL OR GLOBAL, THAT OCCURS AFTER THE SUBJECT EMERGES FROM ANESTHESIA. POSTOPERATIVE NEUROLOGIC SYMPTOMS THAT MIMIC THOSE OF A PREOPERATIVELY DOCUMENTED NEUROLOGIC EVENT AND THAT ARE CONFIRMED RADIOGRAPHICALLY TO BE CONSISTENT WITH THE FORMER EVENT ARE NOT COUNTED. CENTRAL NEUROLOGIC EVENTS THAT ARE CLEARLY RELATED TO AORTIC, INTERNAL CAROTID ARTERY OR VERTEBRAL ARTERY DISEASE ARE ALSO NOT COUNTED. PSYCHOMOTOR DEFICITS FOUND BY SPECIALIZED TESTING ARE NOT CONSIDERED NEUROLOGIC EVENTS RELATED TO OPERATED VALVES. SUBJECTS WHO DO NOT AWAKEN OR WHO AWAKEN AFTER OPERATION WITH A NEW STROKE ARE NOT CONSIDERED TO HAVE SUSTAINED VALVE-RELATED NEUROLOGIC EVENTS. STROKE: A PROLONGED (>72 HOURS) OR PERMANENT NEUROLOGIC DEFICIT THAT IS USUALLY ASSOCIATED WITH ABNORMAL RESULTS OF MRI OR CT SCANS. SUBJECTS WITH MINIMAL, ATYPICAL, OR PROTEAN SYMPTOMS THAT LEAD TO RADIOGRAPHIC IMAGING DEMONSTRATING AN ACUTE ISCHEMIC EVENT ARE CONSIDERED TO HAVE SUSTAINED A STROKE. TIA: CHARACTERIZED BY FULLY REVERSIBLE SYMPTOMS OF SHORT DURATION. IF RADIOGRAPHIC IMAGING DEMONSTRATES AN ACUTE CENTRAL NEUROLOGIC LESION, HOWEVER, SUCH SUBJECTS ARE RECLASSIFIED AS HAVING SUSTAINED A STROKE. |
| AE256 | THROMBOEMBOLIC EVENT - OTHER - PERIPHERAL NO PARESIS | A PERIPHERAL EMBOLIC EVENT IS AN OPERATIVE, AUTOPSY, OR CLINICALLY DOCUMENTED EMBOLUS THAT PRODUCES SYMPTOMS FROM COMPLETE OR PARTIAL OBSTRUCTION OF A PERIPHERAL (NON-CEREBRAL) ARTERY. LOCATION SHOULD BE REPORTED. REPORT UNDER PULMONARY EMBOLISM IF EVENT OCCURS IN THE LUNG. |
| AE257 | THROMBOEMBOLIC EVENT - OTHER - PERIPHERAL | "HEMIPARESIS |
| AE258 | THROMBOEMBOLIC EVENT - OTHER - PERIPHERAL | " FULL PARESIS |
| AE259 | THROMBOEMBOLIC EVENT - OTHER - CENTRAL | " NO PARESIS |
| AE260 | THROMBOEMBOLIC EVENT - OTHER - CENTRAL | "HEMIPARESIS |
| AE.6 | CARDIOVASCULAR - THROMBOEMBOLIC EVENT/V | 'ALVE THROMBOSIS (CONTINUED) |

# Clinical Investigational Plan Protocol Number: 2012-02

| AE CODE LIST | | |
|---|---|---|
| CODE | LABEL/NAME | DEFINITION |
| AE261 | THROMBOEMBOLIC EVENT - OTHER - CENTRAL | " FULL PARESIS |
| AE262 | VALVE THROMBOSIS - AORTIC | ANY THROMBUS NOT CAUSED BY INFECTION ATTACHED TO OR NEAR AN OPERATED VALVE THAT OCCLUDES PART OF THE BLOOD FLOW PATH, INTERFERES WITH VALVE FUNCTION, OR IS SUFFICIENTLY LARGE TO WARRANT TREATMENT. VALVE THROMBUS FOUND AT AUTOPSY IN A SUBJECT WHOSE CAUSE OF DEATH WAS NOT VALVE RELATED OR FOUND AT OPERATION FOR AN UNRELATED INDICATION SHOULD ALSO BE COUNTED. |
| AE263 | VALVE THROMBOSIS - MITRAL | " |
| AE264 | VALVE THROMBOSIS - PULMONARY | " |
| AE265 | VALVE THROMBOSIS - TRICUSPID | " |
| AE.7 | CARDIOVASCULAR - MISC | |
| AE270 | ANGINA, STABLE | CHEST PAIN, TIGHT OR HEAVY FEELING IN THE CHEST, OR DISCOMFORT WHICH SPREADS FROM THE CHEST TO THE ARM, BACK, NECK, JAW, OR STOMACH, NUMBNESS OR TINGLING IN THE SHOULDERS, ARMS OR WRISTS, SHORTNESS OF BREATH, AND NAUSEA RELIEVED BY REST OR NITROGLYCERINE AND/OR CONFIRMED BY ECG. STABLE ANGINA IS ANGINA THAT IS CONTROLLED BY ORAL AND/OR TRANSCUTANEOUS MEDICATION. |
| AE271 | ANGINA, UNSTABLE | UNSTABLE ANGINA IS ANGINA, WHICH NECESSITATES THE INITIATION, CONTINUATION OR INCREASE OF ANGINA CONTROL THERAPIES THAT MAY INCLUDE: NITROGLYCERIN DRIP, HEPARIN DRIP, OR IABP PLACEMENT. THE TYPE OF ANGINA MAY INCLUDE, BUT IS NOT LIMITED TO: REST ANGINA, NEW ONSET EXERTIONAL ANGINA OF AT LEAST NEW YORK HEART ASSOCIATION (NYHA) CLASS III IN SEVERITY, RECENT ACCELERATION IN PATTERN AND INCREASE OF ONE NYHA CLASS TO AT LEAST NYHA CLASS III, VARIANT ANGINA, NON-Q WAVE MYOCARDIAL INFARCTION, OR POST-INFARCTION ANGINA. |
| AE272 | ANNULAR DISSECTION | DISSECTION OF THE VALVULAR ANNULUS EXTENDING INTO THE AORTA. ANNULAR DISSECTION OCCURRING WITHIN 30 DAYS OF THE INDEX PROCEDURE WILL BE CONSIDERED VALVE RELATED. SHOULD BE CONFIRMED BY IMAGING, OR DIRECT VISUAL INSPECTION. |
| AE273 | AORTIC DISSECTION | DISRUPTION OF THE MEDIA LAYER OF THE AORTA WITH BLEEDING WITHIN AND ALONG THE WALL OF THE AORTA. AORTIC DISSECTION MAY OCCUR IN THE ASCENDING THORACIC AORTA (TYPE A DISSECTION) OR IN THE DESCENDING THORACIC AORTA (TYPE B DISSECTION). DISSECTION SHOULD BE CONFIRMED BY IMAGING OR DIRECT VISUAL INSPECTION. |
| AE274 | ARTERIAL DISSECTION | DISRUPTION OF THE MEDIA LAYER OF AN ARTERY OTHER THAN THE AORTA WITH BLEEDING WITHIN AND ALONG THE WALL OF THE VESSEL. SHOULD BE CONFIRMED BY IMAGING OR DIRECT VISUAL INSPECTION. |
| AE275 | CARDIAC ARREST | CARDIAC ARREST DOCUMENTED BY ONE OF THE FOLLOWING: VENTRICULAR FIBRILLATION, RAPID VENTRICULAR TACHYCARDIA WITH HEMODYNAMIC INSTABILITY, ASYSTOLE. |
| AE276 | CARDIAC DECOMPENSATION | AN INABILITY OF THE HEART TO MAINTAIN ADEQUATE CIRCULATION; IT IS MARKED BY DYSPNEA, VENOUS ENGORGEMENT, CYANOSIS AND EDEMA. |
| AE277 | CARDIOGENIC SHOCK | A CLINICAL STATE OF HYPOPERFUSION SUSTAINED FOR GREATER THAN 30 MINUTES, WITH EITHER SYSTOLIC BLOOD PRESSURE < 80 MM HG, AND /OR CARDIAC INDEX < 1.8 DESPITE MAXIMAL TREATMENT (FLUIDS) OR REQUIRING INTRAVENOUS INOTROPES AND/OR PRESSOR AGENT OR AN INTRA-AORTIC BALLOON PUMP (IABP). |
| AE.7 | CARDIOVASCULAR - MISC (CONTINUED) | |

# Clinical Investigational Plan Protocol Number: 2012-02

| AE CODE LIST | | |
|---|---|---|
| CODE | CODE LABEL/NAME DEFINITION | |
| AE278 | CHORDAE TENDINEAE DAMAGE | |
| AE279 | CORONARY ARTERY OSTIAL OBSTRUCTION | OBSTRUCTION OF THE CORONARY OSTIA. SHOULD BE CONFIRMED BY IMAGING AND THE SOURCE OF THE OBSTRUCTION (AORTIC VALVE, THROMBUS, ETC. SHOULD BE REPORTED. |
| AE280 | ENDOCARDITIS | ANY INFECTION INVOLVING THE STUDY VALVE. THE DIAGNOSIS OF OPERATED VALVULAR ENDOCARDITIS IS BASED ON ONE OF THE FOLLOWING CRITERIA: (1) REOPERATION WITH EVIDENCE OF ABSCESS, PARAVALVULAR LEAK, PUS, OR VEGETATION CONFIRMED AS SECONDARY TO INFECTION BY HISTOLOGIC OR MICROBIOLOGIC STUDIES; (2) AUTOPSY FINDINGS OF ABSCESS, PUS, OR VEGETATION INVOLVING A REPAIRED OR REPLACED VALVE; OR (3) IN THE ABSENCE OF REOPERATION OR AUTOPSY, MEETING OF THE DUKE CRITERIA FOR ENDOCARDITIS [4]. MORBIDITIES ASSOCIATED WITH ACTIVE INFECTION, SUCH AS VALVE THROMBOSIS, THROMBOTIC EMBOLUS, BLEEDING EVENT, OR PARAVALVULAR LEAK, ARE INCLUDED UNDER THIS CATEGORY, BUT NOT COUNTED IN OTHER CATEGORIES OF MORBIDITY. |
| AE281 | HEART FAILURE - ACUTE | ACUTE HEART FAILURE DESCRIBES EXACERBATED OR DECOMPENSATED HEART FAILURE, REFERRING TO EPISODES IN WHICH A SUBJECT IS CHARACTERIZED AS HAVING A CHANGE IN HEART FAILURE SIGNS AND SYMPTOMS RESULTING IN A NEED FOR URGENT THERAPY OR HOSPITALIZATION. |
| AE282 | HEART FAILURE - CHRONIC (CHF) | AN EVENT IN WHICH THE HEART FAILS TO MEET THE CIRCULATORY REQUIREMENTS OF THE BODY UNDER DIFFERING PHYSIOLOGICAL CIRCUMSTANCES, AND/OR A STATE IN WHICH CARDIAC OUTPUT IS REDUCED RELATIVE TO THE DEMANDS OF THE BODY, ASSUMING THE EVIDENCE OF ADEQUATE VENOUS RETURN. EVENT IS CONFIRMED CLINICALLY OR BY DIAGNOSTIC TESTING. |
| AE283 | HYPERTENSION - SYSTEMIC | DEFINED AS BLOOD PRESSURE > 140 /90 MM HG FOR SUBJECT WITHOUT DIABETES OR KIDNEY DISEASE; >130/80 MMHG FOR SUBJECTS ON 2 OCCASIONS WITH DIABETES OR RENAL DISEASE. UNLESS DUE TO PRESENCE OF MEDICATION, E.G. BETA BLOCKERS FOR 10 YEARS |
| AE284 | HYPERTENSION — PULMONARY | MEAN PULMONARY ARTERY PRESSURE THAT IS GREATER THAN 25 MMHG AT REST AND/OR GREATER THAN 30 MMHG DURING EXERCISE CONFIRMED BY SWAN GANZ CATHETER OR DIAGNOSTIC PLACEMENT IN THE PULMONARY ARTERY BED AND CONDITION REQUIRES MEDICAL INTERVENTION TO RESOLVE OR TREAT THE CONDITION. |
| AE285 | HYPOTENSION | ABNORMALLY LOW BLOOD PRESSURE. FOR AN ADULT, HYPOTENSION IS DEFINED AS BLOOD PRESSURE LESS THAN 90/50 MMHG. |

# Clinical Investigational Plan

| Protocol | Numb | 30r. | 2012 | -02 |
|----------|------|--------|------|-----|
| Protocol | numi | ber: / | 2012 | -02 |

| | AE CODE LIST | |
|---|---|---|
| CODE | LABEL/NAME | DEFINITION |
| AE.7 | CARDIOVASCULAR - MISC (CONTINUED) | |
| AE286 | MYOCARDIAL INFARCTION | AN ACUTE MYOCARDIAL INFARCTION IS EVIDENCED BY ANY OF THE FOLLOWING: 1. A RISE AND FALL OF CARDIAC BIOMARKERS (PREFERABLY TROPONIN) WITH AT LEAST ONE OF THE VALUES IN THE ABNORMAL RANGE (CK ≥ 5X ULN) TOGETHER WITH AT LEAST ONE OF THE FOLLOWING MANIFESTATIONS OF MYOCARDIAL ISCHEMIA: A) ISCHEMIC SYMPTOMS; B) ECG CHANGES INDICATIVE OF NEW ISCHEMIA (NEW ST-T CHANGES, NEW LEFT BUNDLE BRANCH BLOCK, OR LOSS OF R WAVE VOLTAGE); C) DEVELOPMENT OF PATHOLOGICAL Q WAVES IN 2 OR MORE CONTIGUOUS LEADS IN THE ECG (OR EQUIVALENT FINDINGS FOR TRUE POSTERIOR MI); D. IMAGING EVIDENCE OF NEW LOSS OF VIABLE MYOCARDIUM OR NEW REGIONAL WALL MOTION ABNORMALITY. 2. DEVELOPMENT OF NEW PATHOLOGICAL Q WAVES IN 2 OR MORE CONTIGUOUS LEADS IN THE ECG, WITH OR WITHOUT SYMPTOMS. 3. IMAGING EVIDENCE OF A REGION WITH NEW LOSS OF VIABLE MYOCARDIUM AT REST IN THE ABSENCE OF A NON-ISCHEMIC CAUSE. THIS CAN BE MANIFEST AS: A. ECHOCARDIOGRAPHIC, CT, MR, VENTRICULOGRAPHIC OR NUCLEAR IMAGING EVIDENCE OF LEFT VENTRICULAR THINNING OR SCARRING AND FAILURE TO CONTRACT APPROPRIATELY (I.E., HYPOKINESIS, AKINESIS, OR DYSKINESIS); OR, B. FIXED (NON-REVERSIBLE) PERFUSION DEFECTS ON NUCLEAR RADIOISOTOPE IMAGING (E.G., MIBI, THALLIUM). |
| AE287 | MYOCARDITIS | AN INFECTION OF THE HEART MUSCLE |
| AE296 | PERFORATION - ATRIAL | AN ABNORMAL HOLE OR OPENING IN THE ATRIAL WALL CAUSED BY A DEVICE CAUSING PUNCTURE THROUGH THE WALL OR BY PRESSURE AGAINST A WEAKENED PORTION OF THE WALL. |
| AE297 | PERFORATION - VENTRICULAR | AN ABNORMAL HOLE OR OPENING IN THE VENTRICULAR WALL CAUSED BY A DEVICE CAUSING PUNCTURE THROUGH THE WALL OR BY PRESSURE AGAINST A WEAKENED PORTION OF THE WALL. |
| AE289 | PERFORATION - OTHER | n e e e e e e e e e e e e e e e e e e e |
| AE290 | PERICARDIAL EFFUSION - MAJOR | EXCESS FLUID ACCUMULATION IN THE PERICARDIAL SPACE THAT INTERFERES WITH NORMAL HEART FUNCTION AND REQUIRES MEDICAL INTERVENTION TO RESOLVE. IT SHOULD BE CONFIRMED BY ECHOCARDIOGRAPHY OR CT. |
| AE291 | PERICARDIAL EFFUSION - MINOR | " |
| AE292 | PERICARDIAL TAMPONADE - MAJOR | ABNORMAL FLUID ACCUMULATION WITHIN THE PERICARDIAL SPACE THAT CAUSES HEMODYNAMIC COMPROMISE. THIS SHOULD BE DOCUMENTED BY EITHER: 1. ECHO SHOWING PERICARDIAL FLUID AND SIGNS OF TAMPONADE SUCH AS RIGHT HEART COMPROMISE. 2. SYSTEMIC HYPOTENSION DUE TO PERICARDIAL FLUID COMPROMISING CARDIAC FUNCTION. |
| AE294 | PERICARDITIS | AN INFLAMMATION OF THE PERICARDIUM (THE FIBROUS SAC SURROUNDING THE HEART). |
| AE295 | CARDIOVASCULAR - OTHER | |

AE CODE LIST

# Clinical Investigational Plan

Protocol Number: 2012-02

| AE CODE LIST | | |
|---|---|---|
| CODE | LABEL/NAME | DEFINITION |
| AE.8 | GASTROINTESTINAL/HEPATIC | |
| AE350 | GASTROINTESTINAL - ESOPHAGEAL RUPTURE/TEAR | ANY EVIDENCE OF PUNCTURE/DISSECTION/PERFORATION, VARICES OR OTHER DAMAGE TO THE ESOPHAGUS REQUIRING INTERVENTION. |
| AE351 | GASTROINTESTINAL - INFECTION | SEVERE INFLAMMATION OF THE GASTROINTESTINAL TRACT INVOLVING BOTH THE STOMACH AND SMALL INTESTINE RESULTING IN ACUTE DIARRHEA AND VOMITING. SHOULD BE CONFIRMED BY CULTURE |
| AE352 | GASTROINTESTINAL - OTHER | OTHER GASTROINTESTINAL EVENT THAT DOES NOT FIT IN ONE OF THE OTHER GI/HEPATIC CATEGORIES. |
| AE353 | LIVER FAILURE - ACUTE | A SYNDROME DEFINED BY THE OCCURRENCE OF ENCEPHALOPATHY, COAGULOPATHY AND JAUNDICE IN AN INDIVIDUAL WITH A PREVIOUSLY NORMAL LIVER. |
| AE354 | LIVER FAILURE - CHRONIC | CHRONIC LIVER DISEASE CAUSES CAN BE ANY CONDITION THAT RESULTS IN THE GRADUAL DEGRADATION AND RENEWAL OF THE TISSUE CELLS WITH A BODY'S LIVER. THIS PROCESS USUALLY RESULTS IN FIBROSIS OR CIRRHOSIS. DIAGNOSIS MAY BE CONFIRMED BY ABNORMAL BLOOD ENZYMES AND/OR BIOPSY |
| AE355 | HEPATIC COMPLICATION - OTHER | OTHER LIVER EVENTS THAT DO NOT MEET THE DEFINITION OF LIVER FAILURE (E.G. LIVER DYSFUNCTION) REQUIRING HOSPITALIZATION OR MEDICAL INTERVENTION. |
| AE356 | PANCREATIC COMPLICATION (PANCREAS) | AN EVENT PERTAINING TO, CONNECTED WITH, OR AFFECTING THE PANCREAS REQUIRING HOSPITALIZATION OR MEDICAL INTERVENTION. |
| AE357 | SPLENIC COMPLICATION (SPLEEN) | AN EVENT PERTAINING TO, CONNECTED WITH, OR AFFECTING THE SPLEEN REQUIRING HOSPITALIZATION OR MEDICAL INTERVENTION. |
| AE358 | BILIARY (GALLBLADDER) | AN EVENT PERTAINING TO BILE OR TO THE GALLBLADDER AND BILE DUCTS, WHICH TRANSPORT BILE REQUIRING HOSPITALIZATION OR MEDICAL INTERVENTION. |
| AE359 | ENDOCRINE COMPLICATIONS | AN EVENT PERTAINING TO, CONNECTED WITH, OR AFFECTING THE ENDOCRINE SYSTEM REQUIRING HOSPITALIZATION OR MEDICAL INTERVENTION. |
| AE360 | METABOLIC COMPLICATIONS | AN EVENT PERTAINING TO, CONNECTED WITH, OR AFFECTING THE METABOLIC SYSTEM REQUIRING HOSPITALIZATION OR MEDICAL INTERVENTION. |
| AE.9 | GENITOURINARY/RENAL | |
| AE370 | URINARY TRACT INFECTION (UTI) | INFECTION THAT AFFECTS ANY PART OF THE URINARY TRACT THAT REQUIRE HOSPITALIZATION OR MEDICAL INTERVENTION. |
| AE371 | VAGINAL INFECTION | INFECTIONS AFFECTING THE VAGINAL AREA THAT REQUIRE HOSPITALIZATION OR MEDICAL INTERVENTION. |
| AE372 | GENITOURINARY - OTHER | OTHER GENITOURINARY EVENT NOT PREVIOUSLY DESCRIBED REQUIRING HOSPITALIZATION OR MEDICAL INTERVENTION. |
| AE373 | RENAL DYSFUNCTION | AN ACUTE EVENT OR WORSENING OF RENAL FUNCTION POST-OPERATIVELY (INCREASE OF SERUM CREATININE TO < 2.0, AND < 2X MOST RECENT PREOPERATIVE CREATININE LEVEL) AND DOES NOT REQUIRE DIALYSIS. |

# Clinical Investigational Plan Protocol Number: 2012-02

| AE CODE LIST | | |
|---|---|---|
| CODE | LABEL/NAME | DEFINITION |
| AE.9 | GENITOURINARY/RENAL (CONTINUED) | |
| AE374 | RENAL FAILURE - ACUTE | AN ACUTE EVENT OR WORSENING OF RENAL FUNCTION RESULTING IN ONE OR MORE OF THE FOLLOWING: 1) INCREASE OF SERUM CREATININE TO >2.0, AND 2X MOST RECENT PREOPERATIVE CREATININE LEVEL. 2) A NEW REQUIREMENT FOR DIALYSIS POSTOPERATIVELY. |
| AE375 | RENAL FAILURE - CHRONIC | A PROGRESSIVE LOSS IN RENAL FUNCTION OVER A PERIOD OF MONTHS OR YEARS RESULTING IN A DIAGNOSIS OF STAGE 5 - CHRONIC KIDNEY DISEASE. |
| AE376 | RENAL - OTHER | OTHER EVENT THAT IS NOT RENAL FAILURE OR RENAL DYSFUNCTION THAT REQUIRES HOSPITALIZATION OR MEDICAL INTERVENTION. |
| AE.10 | PULMONARY/RESPIRATORY | |
| AE380 | ATELECTASIS | COMPLETE OR PARTIAL COLLAPSE OF A PREVIOUSLY INFLATED LUNG; INABILITY OF LUNG TO FULLY EXPAND. |
| AE381 | НҮРОХЕМІА | DECREASED PARTIAL PRESSURE OF OXYGEN IN BLOOD SOMETIMES SPECIFICALLY AS LESS THAN 60 MMHG (8.0 KPA) OR CAUSING HEMOGLOBIN OXYGEN SATURATION OF LESS THAN 90%. |
| AE382 | PLEURAL EFFUSION - RIGHT | EXCESS ACCUMULATION OF FLUIDS, SOMETIMES BLOOD IN THE PLEURAL SPACE, WHICH IS COMMON AFTER CARDIAC SURGERY. REPORTABLE WHEN IT BECOMES SYMPTOMATIC AND REQUIRES FLUID TO BE INTERVENTIONALLY REMOVED. |
| AE383 | PLEURAL EFFUSION - LEFT | " |
| AE384 | PLEURAL EFFUSION - BILATERAL | " |
| AE385 | PNEUMOTHORAX | ACCUMULATION OF AIR OR GAS IN THE PLEURAL CAVITY, OCCURRING BECAUSE OF DISEASE OR INJURY AND REQUIRING SURGICAL INTERVENTION, HOSPITALIZATION OR MEDICAL INTERVENTION TO RESOLVE. |
| AE386 | PULMONARY EDEMA | AN ABNORMAL ACCUMULATION OF FLUID IN THE LUNGS REQUIRING HOSPITALIZATION OR MEDICAL INTERVENTION TO RESOLVE. |
| AE387 | PULMONARY HYPERTENSION | MEAN PULMONARY ARTERY PRESSURE THAT IS GREATER THAN 25 MMHG AT REST AND/OR GREATER THAN 30 MMHG DURING EXERCISE CONFIRMED BY SWAN GANZ CATHETER OR DIAGNOSTIC PLACEMENT IN THE PULMONARY ARTERY BED AND CONDITION REQUIRES HOSPITALIZATION OR MEDICAL INTERVENTION TO RESOLVE. |
| AE388 | PULMONARY REGURGITATION | THE BACKWARD FLOW OF BLOOD FROM THE PULMONARY ARTERY, THROUGH THE PULMONARY VALVE, AND INTO THE RIGHT VENTRICLE OF THE HEART DURING DIASTOLE. |
| AE389 | PULMONARY EMBOLISM - RIGHT | CLINICAL EVIDENCE OF NEW EMBOLISM WITH CONFIRMATION BY LUNG SCAN OR PULMONARY ANGIOGRAPHY. |
| AE390 | PULMONARY EMBOLISM - LEFT | " |
| AE391 | PULMONARY EMBOLISM - BILATERAL | " |
| AE392 | PULMONARY/RESPIRATORY - OTHER | OTHER RESPIRATORY EVENT THAT IS NOT RESPIRATORY FAILURE. |
| AE393 | RESPIRATORY DYSFUNCTION/INSUFFICIENCY | DETERIORATION OF SUBJECT'S RESPIRATORY EFFORTS LESS THAN 24 HRS AFTER COMPLETION OF THE INDEX PROCEDURE. |

# Clinical Investigational Plan

Protocol Number: 2012-02

| AE CODE LIST | | |
|---|---|---|
| CODE | LABEL/NAME | DEFINITION |
| AE.10 | PULMONARY/RESPIRATORY | |
| AE394 | RESPIRATORY FAILURE -ASTHMA | NEED FOR MECHANICAL VENTILATION REQUIRED GREATER THAN 24 HRS AFTER OF COMPLETION OF THE INDEX PROCEDURE (TIME 0 = WHEN THE SUBJECT LEAVES THE OR), OR NEED FOR RE-INTUBATION AND VENTILATOR SUPPORT OCCURRING ANY TIME WITHIN 30 DAY OF THE INDEX PROCEDURE WILL BE CONSIDERED RELATED TO THE INDEX PROCEDURE. |
| AE395 | RESPIRATORY FAILURE -EMPHYSEMA | п |
| AE396 | RESPIRATORY FAILURE -COPD | п |
| AE397 | RESPIRATORY FAILURE -PNEUMONIA | n e e e e e e e e e e e e e e e e e e e |
| AE398 | RESPIRATORY FAILURE -PNEUMOTHORAX | ı, |
| AE399 | RESPIRATORY FAILURE -HEMOTHORAX | · · |
| AE400 | RESPIRATORY FAILURE - ARDS | " ACUTE RESPIRATORY DISTRESS SYNDROME |
| AE401 | RESPIRATORY FAILURE -OTHER | ı, |
| AE402 | RESPIRATORY INFECTION - UPPER (URI) | THE ILLNESSES CAUSED BY AN ACUTE INFECTION WHICH INVOLVES THE UPPER RESPIRATORY TRACT: NOSE, SINUSES PHARYNX OR LARYNX. THIS COMMONLY INCLUDES: TONSILLITIS, PHARYNGITIS, LARYNGITIS, SINUSITIS, OTITIS MEDIA AND THE COMMON COLD. |
| AE403 | RESPIRATORY INFECTION - PNEUMONIA | LUNG INFECTION DOCUMENTED BY BLOOD STUDIES OR CHEST X-RAY, REQUIRING TREATMENT WITH ANTIBIOTICS, INHALATION THERAPY, INTUBATION OR SUCTIONING. |
| AE.11 | PERIPHERAL VASCULAR | |
| AE420 | VASCULAR - ACCESS SITE COMPLICATION | COMPLICATIONS OF BLEEDING OR INFECTION AT THE SITE OF CARDIOPULMONARY ACCESS AND OR PERCUTANEOUS CORONARY INTERVENTION OR DIAGNOSTICS THAT REQUIRE HOSPITALIZATION OR MEDICAL INTERVENTION. |
| AE421 | VASCULAR - DEEP VEIN THROMBOSIS (DVT) | FORMATION OF BLOOD CLOT (THROMBUS) IN THE LOWER EXTREMITIES (LEGS) CHARACTERIZED BY SWELLING, REDNESS, CLAUDICATION/PAIN IN AFFECTED LIMB. EVENT SHOULD BE CONFIRMED BY DOPPLER OR DUPLEX US STUDY, AND REQUIRES HOSPITALIZATION OR MEDICAL INTERVENTION TO RESOLVE. |
| AE423 | VASCULAR - OTHER | OTHER VASCULAR COMPLICATIONS GENERALLY RELATED TO A DISEASE PROCESS AND NOT TRAUMA THAT REQUIRE HOSPITALIZATION OR MEDICAL INTERVENTION. |
| AE.12 | PSYCHIATRIC | |
| AE431 | PSYCHIATRIC DISORDER | A PSYCHOLOGICAL OR BEHAVIORAL PATTERN GENERALLY ASSOCIATED WITH SUBJECTIVE DISTRESS OR DISABILITY THAT OCCURS IN AN INDIVIDUAL, AND WHICH IS NOT A PART OF NORMAL DEVELOPMENT OR CULTURE. SUCH A DISORDER MAY CONSIST OF A COMBINATION OF AFFECTIVE, BEHAVIORAL, COGNITIVE AND PERCEPTUAL COMPONENTS. |
| AE432 | SUICIDE | A PERSON WHO INTENTIONALLY TAKES HIS OR HER OWN LIFE. |
| AE433 | TRANSIENT PSYCHOTIC SYNDROME | A MENTAL STATE OFTEN DESCRIBED AS INVOLVING A "LOSS OF CONTACT WITH REALITY" THAT LASTS ONLY FOR A SHORT TIME. |
| AE.12 | PSYCHIATRIC (CONTINUED) | |

Clinical Investigational Plan Protocol Number: 2012-02

| AE CODE LIST | | |
|---|---|---|
| CODE | LABEL/NAME | DEFINITION |
| AE434 | PSYCHIATRIC - OTHER | OTHER NEUROLOGIC EVENT NOT PREVIOUSLY DESCRIBED THAT REQUIRES HOSPITALIZATION OR MEDICAL INTERVENTION. |
| AE.13 | MUSCULAR SKELETAL/ DERMATOLOGIC | |
| AE450 | STERNAL WOUND/THORACIC INFECTION | DEEP STERNAL INFECTION INVOLVING MUSCLE, BONE, AND/OR MEDIASTINUM. MUST INCLUDE ONE OF THE FOLLOWING: 1) WOUND OPENED WITH EXCISION OF TISSUE (I&D); 2) POSITIVE CULTURE; 3) TREATMENT WITH ANTIBIOTICS. (LAST SENTENCE REMOVED, WHICH IMPLIES THAT BACTERIAL PNEUMONIA AFFECTING PARTS OF THE LUNG ADJACENT TO THE STERNUM SHOULD BE COUNTED AS A STERNAL WOUND INFECTION.) |
| AE451 | BONE FRACTURE/BREAK | A BREAK IN BONE OR CARTILAGE. ALTHOUGH USUALLY THE RESULT OF TRAUMA, A FRACTURE CAN BE CAUSED BY AN ACQUIRED DISEASE OF BONE SUCH AS OSTEOPOROSIS OR BY ABNORMAL FORMATION OF BONE IN A DISEASE. |
| AE452 | WOUND INFECTION - OTHER | OTHER WOUND INFECTION THAT IS NOT RELATED TO THE SURGICAL ACCESS SITE. |
| AE454 | INFECTION /INFLAMMATION - OTHER | SOURCE OF INFECTION THAT IS CHARACTERIZED BY ELEVATED BLOOD LEVELS AND OR FEVER REQUIRING HOSPITALIZATION OR MEDICAL INTERVENTION (FEVER OF UNKNOWN ORIGIN FUO; CLINICALLY SIGNIFICANT ELEVATED WBC) |
| AE456 | MUSCULAR SKELETAL / DERMATOLOGIC - OTHER | OTHER SKIN/MUSCULAR/SKELETAL EVENT NOT PREVIOUSLY DESCRIBED THAT REQUIRES HOSPITALIZATION OR MEDICAL INTERVENTION. |
| AE.14 | NONSPECIFIC, UNKNOWN, OR OTHER BODY SYSTEM | |
| AE470 | ANAPHYLACTIC REACTION | AN ALLERGIC REACTION TO AN ANTIGEN THAT CAUSES CIRCULATORY COLLAPSE AND SUFFOCATION DUE TO BRONCHIAL AND TRACHEAL SWELLING. |
| AE471 | ALLERGIC REACTION - MEDICATION RELATED | A MILD TO MODERATE TO LIFE THREATENING REACTION TO A SUBSTANCE AND/OR MEDICATION. REPORT REACTIONS THAT REQUIRE HOSPITALIZATION OR MEDICAL INTERVENTION. |
| AE472 | ALLERGIC REACTION - OTHER | A MILD TO MODERATE TO LIFE-THREATENING REACTION TO AN ENVIRONMENTAL OR ANIMAL SUBSTANCE. REPORT REACTIONS THAT REQUIRE HOSPITALIZATION OR MEDICAL INTERVENTION. |
| AE473 | CANCER - PROGRESSION OF UNDERLYING DISEASE | AN EXACERBATION OR WORSENING OF A CANCER DIAGNOSED/KNOWN PRIOR TO THE INDEX PROCEDURE. |
| AE474 | CANCER - NEWLY DIAGNOSED | A NEWLY DIAGNOSED CANCER FOLLOWING INDEX PROCEDURE. |
| AE475 | HEARING DISORDER | ANY DISORDER RELATED TO HEARING IMPAIRMENT REQUIRING HOSPITALIZATION OR MEDICAL INTERVENTION. |
| AE476 | MULTI-SYSTEM ORGAN FAILURE | OCCURS WHEN MORE THAN ONE ORGAN OF THE BODY STOPS FUNCTIONING NORMALLY AND HOMEOSTASIS CANNOT BE MAINTAINED WITHOUT INTERVENTION. |
| AE477 | SPEECH DISORDER | ANY DISORDER RELATED TO A SPEECH IMPEDIMENT REQUIRING HOSPITALIZATION OR MEDICAL INTERVENTION. |
| AE479 | VISION DISORDER | ANY DISORDER RELATED TO VISION IMPAIRMENT REQUIRING HOSPITALIZATION OR MEDICAL INTERVENTION. |
| AE480 | FEVER - UNKNOWN ORIGIN | (1) A TEMPERATURE GREATER THAN 38.3°C (101°F) ON SEVERAL OCCASIONS, (2) MORE THAN 3 WEEKS' DURATION OF ILLNESS, AND (3) FAILURE TO REACH A DIAGNOSIS DESPITE 1 WEEK OF INSUBJECT INVESTIGATION. |
| AE481 | NONSPECIFIC, UNKNOWN, OR OTHER BODY SYSTEM - OTHER COMPLICATION | ANY COMPLICATION THAT CANNOT OTHERWISE BE CATEGORIZED REQUIRING HOSPITALIZATION OR MEDICAL INTERVENTION. |
| AE.15 | DEVICE DYSFUNCTION | |

# Clinical Investigational Plan Protocol Number: 2012-02

| AE CODE LIST | | |
|---|---|---|
| CODE | CODE LABEL/NAME DEFINITION | |
| AE500 | SVD - STUDY VALVE WEAR | INCLUDES DYSFUNCTION OR DETERIORATION INVOLVING THE OPERATED VALVE (EXCLUSIVE OF INFECTION OR THROMBOSIS). THE TERM STRUCTURAL VALVE DETERIORATION REFERS TO CHANGES INTRINSIC TO THE VALVE SUCH AS: WEAR, FRACTURE, CALCIFICATION, LEAFLET TEAR, MANUFACTURED SUTURE LINE DISRUPTION |
| AE501 | SVD - STUDY VALVE FRACTURE | " |
| AE502 | SVD - STUDY VALVE POPPET ESCAPE | " |
| AE503 | SVD - STUDY VALVE CALCIFICATION | " |
| AE504 | SVD - STUDY VALVE LEAFLET TEAR | " |
| AE505 | SVD - STUDY VALVE STENT CREEP | " |
| AE506 | SVD - STUDY VALVE SUTURE LINE DISRUPTION | " |
| AE507 | SVD - STRUCTURAL VALVE DETERIORATION, OTHER | " |
| AE508 | SVD - REPAIRED VALVE, NEW CHORDAL RUPTURE | |
| AE509 | SVD - REPAIRED VALVE, LEAFLET DISRUPTION | |
| AE510 | SVD - REPAIRED VALVE, LEAFLET RETRACTION | |
| AE511 | SVD- REPAIRED VALVE, OTHER | |
| AE525 | SVD - ANNULAR FRAME DAMAGE | " |
| AE526 | SVD - ANNULAR FRAME SEPARATION | " |
| AE <b>527</b> | SVD - STENT FRAME FRACTURE | " |
| AE528 | SVD - STENT FRAME DEFORMATION | " |
| AE <b>529</b> | SVD - STENT FRAME SEPARATION | " |
| AE512 | NSD - ENTRAPMENT BY PANNUS, TISSUE, OR SUTURE | ANY ABNORMALITY NOT INTRINSIC TO THE VALVE (DO NOT DIRECTLY INVOLVE VALVE COMPONENTS) ITSELF THAT RESULTS IN STENOSIS OR REGURGITATION OF THE OPERATED VALVE OR HEMOLYSIS (EXCLUDES THROMBOSIS AND INFECTION). EXAMPLES INCLUDE: ENTRAPMENT BY PANNUS, TISSUE, OR SUTURE, PARAVALVULAR LEAK, INAPPROPRIATE SIZING, INAPPROPRIATE POSITIONING, REGURGITATION AS A RESULT OF TECHNICAL ERROR, STJ DILATION, DILATION OF THE VALVE ANNULUS, OBSTRUCTION OF THE CORONARY OSTIA BY THE STUDY VALVE. |
| AE164 | NSD - PARAVALVULAR LEAK - +1 | LEAKAGE BETWEEN THE SEWING RING AND THE ANNULUS. |
| AE165 | NSD - PARAVALVULAR LEAK - +2 | п |
| AE166 | NSD - PARAVALVULAR LEAK - +3 | " |
| AE167 | NSD - PARAVALVULAR LEAK - +4 | " |
| AE176 | NSD - STUDY VALVE STENOSIS - MILD | NSD " |

Clinical Investigational Plan Protocol Number: 2012-02

| | AE CODE LIST | |
|---|---|---|
| CODE | CODE LABEL/NAME DEFINITION | |
| AE177 | NSD - STUDY VALVE STENOSIS - MODERATE | NSD " |
| AE178 | NSD - STUDY VALVE STENOSIS - SEVERE | NSD " |
| AE121 | NSD - PARAVALVULAR LEAK WITH HEMOLYSIS | NSD " |
| AE514 | NSD - INAPPROPRIATE SIZING | NSD" |
| AE516 | NSD - RESIDUAL LEAK OR OBSTRUCTION | NSD" |
| AE517 | NSD - INTRAVASCULAR HEMOLYTIC ANEMIA | NSD " CLINICALLY IMPORTANT |
| AE518 | NSD - DEVELOPMENT OF REGURGITATION | NSD " AS A RESULT OF TECHNICAL ERRORS |
| AE519 | NSD - DILATATION OF THE SINOTUBULAR JUNCTION | NSD" |
| AE520 | NSD - DILATION OF THE VALVE ANNULUS | NSD " |
| AE521 | NSD - CORONARY OSTIAL OBSTRUCTION | NSD " |
| AE522 | NSD - STUDY VALVE INSTABILITY | NSD" |
| AE <b>524</b> | NSD - LVOT DAMAGE | NSD " |
| AE530 | NSD - VALVE MALPOSITION | NSD" |
| AE531 | NSD - VALVE MIGRATION/EMBOLIZATION | NSD " |
| AE532 | NSD - VALVE DISLODGEMENT | NSD " |

**EDWARDS LIFESCIENCES LLC**CLINICAL INVESTIGATIONAL PLAN

# ATTACHMENT J – RESPONSIBILITIES INVESTIGATOR & SPONSOR

REVISION J: 03 MARCH 2021

#### **INVESTIGATORS' RESPONSIBILITIES**

# 1.0 Investigators' Responsibilities For Significant Risk Device Investigations (Nov. 1995)

This document is intended to assist investigators in identifying and complying with their responsibilities in connection with the conduct of clinical investigations involving medical devices. Although this guidance primarily addresses duties imposed upon clinical investigators by regulations of the Food and Drug Administration (FDA), investigators should be cognizant of additional responsibilities that may derive from other sources (such as the study protocol itself, the investigator agreement, any conditions of approval imposed by FDA or the governing Institutional Review Board, as well as institutional policy and state law).

# 2.0 General Responsibilities of Investigators (21 CFR 812.100)

- Ensuring that the investigation is conducted according to the signed agreement, the investigational plan and applicable FDA regulations.
- Protecting the rights, safety, and welfare of subjects under the investigator's care.
- Controlling devices under investigation.
- Ensuring that informed consent is obtained from each subject in accordance with 21 CFR Part 50, and that the study is not commenced until FDA and IRB approvals have been obtained.

# 3.0 Specific Responsibilities of Investigators (21 CFR 812.110)

- Awaiting IRB approval and any necessary FDA approval before requesting written informed consent or permitting subject participation.
- Conducting the investigation in accordance with:
  - the signed agreement with the sponsor
  - o the investigational plan
  - the regulations set forth in 21 CFR Part 812 and all other applicable FDA regulations
  - o any conditions of approval imposed by an IRB or FDA
- Supervising the use of the investigational device. An investigator shall permit an investigational
  device to be used only with subjects under the investigator's supervision. An investigator shall not
  supply an investigational device to any person not authorized under 21 CFR Part 812 to receive
  it.
- Disposing of the device properly. Upon completion or termination of a clinical investigation or the
  investigator's part of an investigation, or at the sponsor's request, an investigator shall return to
  the sponsor any remaining supply of the device or otherwise dispose of the device as the sponsor
  directs.

#### 4.0 Maintaining Records (21 CFR 812.140)

An investigator shall maintain the following accurate, complete, and current records relating to the investigator's participation in an investigation:

- Correspondence with another investigator, an IRB, the sponsor, a monitor, or FDA.
- Records of receipt, use or disposition of a device that relate to:
  - o the type and quantity of the device, dates of receipt, and batch numbers or code marks
  - o names of all persons who received, used, or disposed of each device
  - o the number of units of the device returned to the sponsor, repaired, or otherwise disposed of, and the reason(s) therefore
- Records of each subject's case history and exposure to the device, including:
  - documents evidencing informed consent and, for any use of a device by the investigator without informed consent, any written concurrence of a licensed physician and a brief description of the circumstances justifying the failure to obtain informed consent
  - all relevant observations, including records concerning adverse device effects (whether anticipated or not), information and data on the condition of each subject upon entering, and during the course of, the investigation, including information about relevant previous medical history and the results of all diagnostic tests
  - a record of the exposure of each subject to the investigational device, including the date and time of each use, and any other therapy
- The protocol, with documents showing the dates of and reasons for each deviation from the protocol.

#### **INVESTIGATORS' RESPONSIBILITIES**

• Any other records that FDA requires to be maintained by regulation or by specific requirement for a category of investigations or a particular investigation.

## 5.0 Inspections (21 CFR 812.145)

Investigators are required to permit FDA to inspect and copy any records pertaining to the investigation including, in certain situations, those which identify subjects.

# 6.0 Submitting Reports (21 CFR 812.150)

An investigator shall prepare and submit the following complete, accurate, and timely reports:

- To the sponsor and the IRB:
  - Any unanticipated adverse device effect occurring during an investigation. (Due no later than 10 working days after the investigator first learns of the effect.)
  - Progress reports on the investigation. (These reports must be provided at regular intervals, but in no event less often than yearly. If there is a study monitor, a copy of the report should also be sent to the monitor.)
  - Any deviation from the investigational plan made to protect the life or physical well-being of a subject in an emergency. (Report is due as soon as possible but no later than 5 working days after the emergency occurs. Except in emergency situations, a protocol deviation requires prior sponsor approval; and if the deviation may affect the scientific soundness of the plan or the rights, safety, or welfare of subjects, prior FDA and IRB approval are required.)
  - Any use of the device without obtaining informed consent. (Due within 5 working days after such use.)
  - A final report. (Due within 3 months following termination or completion of the investigation or the investigator's part of the investigation. For additional guidance, see the discussion under the section entitled "Annual Progress Reports and Final Reports.")
  - Any further information requested by FDA or the IRB about any aspect of the investigation.
- To the Sponsor: Withdrawal of IRB approval of the investigator's part of an investigation. (Due within 5 working days of such action)

# 7.0 Investigational Device Distribution and Tracking

The IDE regulations prohibit an investigator from providing an investigational device to any person not authorized to receive it [21 CFR 812.110(c)]. The best strategy for reducing the risk that an investigational device could be improperly dispensed (whether purposely or inadvertently) is for the sponsor and the investigators to closely monitor the shipping, use, and final disposal of the device(s). Upon completion or termination of a clinical investigation (or the investigator's part of an investigation), or at the sponsor's request, an investigator is required to return to the sponsor any remaining supply of the device or otherwise to dispose of the device as the sponsor directs [21 CFR 812.110(c)]. Investigators must also maintain complete, current and accurate records of the receipt, use, or disposition of investigational devices [21 CFR 812.140(a)(2)]. Specific recordkeeping requirements are set forth at 21 CFR 812.140(a).

# 8.0 Prohibition of Promotion and Other Practices (21 CFR 812.7)

The IDE regulations prohibit the promotion and commercialization of a device that has not been first cleared or approved for marketing by FDA. This prohibition is applicable to sponsors and investigators (or any person acting on behalf of a sponsor or investigator), and encompasses the following activities:

- Promotion or test marketing of the investigational device
- Charging subjects or investigators for the device a price larger than is necessary to recover the costs of manufacture, research, development, and handling
- Prolonging an investigation beyond the point needed to collect data required to determine whether the device is safe and effective
- Representing that the device is safe or effective for the purposes for which it is being investigated.

#### SPONSOR'S RESPONSIBILITIES

# 1.0 Sponsor's Responsibilities For Significant Risk Device Investigations (Nov. 1995)

This document is intended to assist sponsors in identifying and complying with their responsibilities in connection with the conduct of clinical investigations of medical devices that are deemed "significant risk" by the reviewing IRB or by FDA. For a complete description of their responsibilities, sponsors should refer to the actual text of the regulations cited below. In addition, sponsors should be aware that a clinical investigation must be conducted in accordance with any requirements imposed by the reviewing IRB, by institutional policies, or by state law.

# 2.0 General Duties (21 CFR 812.40)

- Submitting the IDE application to FDA
- Obtaining both FDA and IRB approvals for the investigation and submitting certification of IRB approval to FDA before shipping the device to any investigator
- Obtaining FDA approval and IRB approval for a supplemental application before beginning that portion of the investigation
- Selecting qualified investigators
- Ensuring proper monitoring
- Ensuring patient informed consent is obtained

# 3.0 Selection of Investigators (21 CFR 812.43)

- Assuring selection of investigators qualified by training and experience
- Shipping the investigational device only to participating investigators
- Obtaining a signed investigator's agreement containing:
  - o investigator's curriculum vitae
  - o statement of investigator's relevant experience, including dates
  - o location, extent, and type of experience
  - if an investigator was involved in an investigation or other research that was terminated, an explanation of the circumstances that led to the termination
  - statement of the investigator's commitment to:
    - conduct the investigation in accordance with the agreement, the investigational plan, Parts 50, 56, and 812, and any conditions of approval imposed by the IRB or FDA
    - supervise all testing of the device involving human subjects
    - ensure that the requirements for informed consent are met (21 CFR Part 50)
  - Providing investigators with the necessary information to conduct the investigation including, but not necessarily limited to:
  - o the investigational plan
  - the report of prior investigations

#### 4.0 Monitoring (21 CFR 812.46)

- Selecting monitor(s) qualified by training and experience to monitor the progress of the investigation
- Securing compliance of all investigators in accordance with the signed investigator's agreement, the
  investigational plan, the requirements of this part or other applicable FDA regulations, or any condition
  of approval imposed by the reviewing IRB or FDA. If compliance cannot be secured, shipment of the
  device to the investigator and the investigator's participation in the investigation must be discontinued
- Ensuring that significant new information about the investigation is provided to all reviewing IRBs, FDA, and investigators
- Evaluating all unanticipated adverse device effects and terminating the investigation, or portions of it, if that effect presents an unreasonable risk to subjects (reporting requirements are listed below.)
- · Resuming terminated investigations only after both FDA and IRB approvals are obtained.

# 5.0 Controlling Distribution and Disposition of Devices

Although investigators are responsible for ensuring that investigational devices are made available only to persons who are legally authorized to receive them (see 21 CFR 812.110(c)), sponsors also bear responsibility for taking proper measures to ensure that devices are not diverted outside of legally authorized channels. Sponsors may ship investigational devices only to qualified investigators participating in the clinical investigation (§ 812.43(b)). Sponsors must also maintain complete, current, and accurate records pertaining to

#### SPONSOR'S RESPONSIBILITIES

the shipment and disposition of the investigational device (§ 812.140(b)). Records of shipment shall include the name and address of the consignee, type and quantity of device, date of shipment, and batch number or code mark. Records of disposition shall describe the batch number or code marks of any devices returned to the sponsor, repaired, or disposed of in other ways by the investigator or another person, and the reasons for and method of disposal.

To further ensure compliance with these requirements, sponsors should take appropriate measures to instruct investigators regarding their responsibilities with respect to recordkeeping and device disposition. The specific recordkeeping requirements for investigators are set forth at § 812.140(a). Upon completion or termination of a clinical investigation (or the investigator's part of an investigation), or at the sponsor's request, an investigator is required to return to the sponsor any remaining supply of the device or otherwise to dispose of the device as the sponsor directs (§ 812.110(c)).

# 6.0 Prohibition of Promotion and Other Practices (21 CFR 812.7)

The IDE regulations prohibit the promotion and commercialization of a device that has not been first cleared or approved for marketing by FDA. This prohibition is applicable to sponsors and investigators (or any person acting on behalf of a sponsor or investigator), and encompasses the following activities:

- Promotion or test marketing of the investigational device
- Charging subjects or investigators for the device a price larger than is necessary to recover the costs
  of manufacture, research, development, and handling
- Prolonging an investigation beyond the point needed to collect data required to determine whether the
  device is safe and effective
- Representing that the device is safe or effective for the purposes for which it is being investigated.

# 7.0 Supplemental Applications [21 CFR 812.35(a) and (b)]

Supplemental applications are required to be submitted to, and approved by, FDA in the following situations:

- Changes in the investigational plan: FDA approval is required for any change that may affect the
  scientific soundness of the investigation or the rights, safety or welfare of the subjects. IRB approval is
  also required for changes that may affect the rights, safety or welfare of the subjects. The change in
  the investigational plan may not be implemented until FDA approval (and IRB approval, if required) is
  obtained.
- Addition of new institutions: IRB approval is also required for new institutions. The investigation at the new institution(s) may not begin until both FDA and IRB approval(s) are obtained, and certification of IRB approval is submitted to FDA.

# 8.0 Maintaining Records [21 CFR 812.140(b)]

A sponsor shall maintain the following accurate, complete, and current records relating to an investigation (also See Table I, next page):

- Correspondence (including reports) with another sponsor, monitor, investigators, an IRB or FDA
- Records of shipment, including:
  - o name and address of consignee
  - type and quantity of device
  - o date of shipment
  - batch numbers or code marks
- Records of disposition, describing:
  - Batch number or code mark of devices returned, repaired, or disposed of by the investigator or other persons
  - Reasons for and method of disposal
- Signed investigator agreements
- Adverse device effects (whether anticipated or unanticipated) and complaints
- Any other records that FDA requires by regulation or by specific requirement for a category of investigation or a particular investigation

#### SPONSOR'S RESPONSIBILITIES

Table I Responsibilities for Maintaining Records for a Significant Risk Device Study

| Records | Maintained by Investigator | Maintained by Sponsor |
|---|---|---|
| All Correspondence Pertaining to the Investigation | X | Х |
| Shipment, Receipt, Disposition | X | Х |
| Device Administration and Use | X | - |
| Subject Case Histories | X | - |
| Informed Consent | X | - |
| Protocols and Reasons for Deviations from Protocol | X | - |
| Adverse Device Effects and Complaints | X | Х |
| Signed Investigator Agreements | - | Х |
| Membership/Employment/Conflicts of Interest | - | Х |
| Minutes of Meetings | - | - |

# 9.0 Submitting Reports [21 CFR 812.150(b)]

A sponsor shall prepare and submit the following complete, accurate, and timely reports (see Table II).

- Unanticipated adverse device effects (with evaluation) to FDA, all IRBs, and investigators within 10 working days after notification by the investigator. Subsequent reports on the effect may be required by FDA.
- Withdrawal of IRB approval
- Withdrawal of FDA approval
- · Current 6month investigator list
- Annual progress report see format for IDE progress report
- Recall and device disposition (within 30 working days after the request was made)
- Final report see format for progress reports
- Use of device without obtaining patient informed consent
- Significant risk determinations by the IRB when proposed to be non-significant risk
- Other reports requested by the IRB or FDA

#### Table II Responsibilities for Preparing and Submitting Reports for Significant Risk Device Studies

| Type of Report | Prepared by Investigators for | Prepared by Sponsors for |
|---|---|---|
| Unanticipated Adverse Effect Evaluation | Sponsors & IRBs | FDA, IRBs & Investigators |
| Withdrawal of IDE Approval | Sponsors | FDA, IRBs, & Investigators |
| Progress Report | Sponsors, Monitors & IRBs | FDA & IRBs |
| Final Report | Sponsors & IRBs | FDA, IRBs, & Investigators |
| Emergencies (Protocol Deviations) | Sponsors & IRBs | FDA |
| Inability to Obtain Informed Consent | Sponsors & IRBs | FDA |
| Withdrawal of FDA Approval | N/A | IRBs & Investigators |
| Current Investigator List | N/A | FDA |
| Recall and Device Disposition | < N/A | FDA & IRBs |
| Records Maintenance Transfer | FDA | FDA |
| Significant Risk Determinations | N/A | FDA |

### 10.0 Inspections [21 CFR 812.145]

Sponsors are required to permit FDA to enter and inspect (at reasonable times and in a reasonable manner) any establishment where devices are held (including any establishment where devices are manufactured, processed, packed, installed, used, or implanted or where records or results from use of devices are kept). FDA may also inspect and copy all records relating to an investigation including, in certain situations, records which, identify subjects.

**EDWARDS LIFESCIENCES LLC**CLINICAL INVESTIGATIONAL PLAN

**ATTACHMENTS** 

# **ATTACHMENT K - SUBJECT IMPLANT CARD**

REVISION J: 03 MARCH 2021



Back (to have MR statement for USA)

Front

Inside of Card

The following aortic valve was implanted.

| | | Follow-Up Schedule | |
|---|---|---|---|
| | Please affix the self-adhesive label with the serial | 1 Month:/ | ☐ Office visit ☐ Telephone interview |
| | number for the aortic valve implanted in this patient. This label may be found in the original device package. | 3 Month:/ | 3 year:/ |
| IMPORTANT: | For all other questions or concerns, contact: | 1 year:/_<br>Month Year | 4 year:/_<br>Month Year |
| Physician Name | Contact Number | 2 year:/_<br>Month Year | 5 year:/_<br>Month Year |



Back (to have MR statement for USA)

Front

Inside of Card

The following mitral valve was implanted.

| | | | Follow-Up Schedule | | |
|---|---|---|---|---|---|
| | Please affix the self-adhesive label with the serial number for the mitral valve implanted in this | 1 Month: | /<br>Month Year | ☐ Office visit | |
| | patient. This label may be found in the original device package. | 3 Month: | Month Year | 3 year: _ | /<br>Month Year |
| IMPORTANT: For all other questions or concerns, contact: | | 1 year: | //<br>Ionth Year | 4 year: _ | /_<br>Month Year |
| Physician Name | Contact Number | 2 year: | /lonth Year | 5 year: <sub>-</sub> | /<br>Month Year |
**EDWARDS LIFESCIENCES LLC**CLINICAL INVESTIGATIONAL PLAN

## **ATTACHMENT L - PROTOCOL DEVIATION CODES**

REVISION J: 03 MARCH 2021

Clinical Investigational Plan Protocol Number: 2012-02

#### PROTOCOL DEVIATION CODES

#### SUBJECT SCREENING

- 1.01 SUBJECT DID NOT MEET INCLUSION CRITERION
- 1.02 SUBJECT MET EXCLUSION CRITERION
- 1.03 DATE OF INFORMED CONSENT IS AFTER DATE OF STUDY ENROLLMENT
- 1.04 INFORMED CONSENT WAS IMPROPERLY OBTAINED
- 1.05 PERSON OBTAINING INFORMED CONSENT DID NOT SIGN/DATE THE CONSENT FORM
- 1.06 OTHER SCREENING DEVIATION

#### BASELINE

- 2.01 BASELINE ECHOCARDIOGRAM NOT DONE
- 2.21 BASELINE ECHOCARDIOGRAM DONE > 60 DAYS PRIOR IMPLANT DATE
- 2.03 BASELINE BLOOD NOT DONE
- 2.22 BASELINE BLOOD DONE > 60 DAYS BEFORE IMPLANT
- 2.05 BASELINE BLOOD INCOMPLETE
- 2.06 BASELINE COAGULATION PROFILE NOT DONE
- 2.23 BASELINE COAGULATION PROFILE DONE > 60 DAYS BEFORE IMPLANT
- 2.08 BASELINE NYHA NOT DONE
- 2.09 BASELINE ELECTROCARDIOGRAM NOT DONE
- 2.24 BASELINE ELECTROCARDIOGRAM DONE > 60 DAYS BEFORE IMPLANT
- 2.11 BASELINE PHYSICAL ASSESSMENT / VITAL SIGNS NOT DONE
- 2.12 PREGNACY TEST NOT DONE
- 2.13 MEDICAL HISTORY NOT COLLECTED
- 2.10 BASELINE QUALITY OF LIFE NOT DONE
- 2.14 OTHER BASELINE DEVIATION

#### **IMPLANT SURGERY**

- 3.01 IMPLANTING SURGEON IS NOT ON APPROVED LIST
- 3.02 PROCEDURE DIAGNOSIS NOT DONE
- 3.28 INCORRECT SIZER USED
- 3.04 START SKIN INCISION TIME NOT RECORDED
- 3.05 START TIME OF ECC (PUMP) NOT RECORDED
- 3.06 START CROSS CLAMP TIME NOT RECORDED
- 3.07 START OF SIZING TIME NOT RECORDED
- 3.09 REMOVAL CROSS CLAMP TIME NOT RECORDED
- 3.10 END ECC (PUMP) TIME NOT RECORDED
- 3.11 END SKIN CLOSURE TIME NOT RECORDED
- 3.12 UNAPPROVED CONCOMITANT PROCEDURE PERFORMED
- 3.15 VALVE SERIAL NUMBER NOT RECORDED
- 3.18 MORE THAN 2 STUDY VALVES ATTEMPTED TO BE IMPLANTED
- 3.21 START TIME FOR STUDY PROCEDURE (FIST STITCH PLACED ON THE ANNULUS) NOT RECORDED
- 3.22 TIME FIST STITCH PLACED ON THE VALVE RING NOT RECORDED

Clinical Investigational Plan Protocol Number: 2012-02

- 3.26 COMPLETION TIME OF STUDY PROCEDURE (LAST STITCH TIED DOWN ON THE VALVE) NOT RECORDED
- 3.33 POST-IMPLANT ECHOCARDIOGRAM NOT DONE
- 3.30 POST-IMPLANT ECHOCARDIOGRAM NOT DONE WITHIN 1 HOUR OF REMOVING THE CROSS-CLAMP
- 3.31 PRE-IMPLANT BLOOD COLLECTION (SERUM GLYCEROL) NOT DONE (ONLY REQUIRED FOR 120 SUBJECTS)
- 3.19 POST-IMPLANT BLOOD COLLECTION (SERUM GLYCEROL) NOT DONE (ONLY REQUIRED FOR 120 SUBJECTS)
- 3.32 POST-IMPLANT BLOOD COLLECTION (SERUM GLYCEROL) NOT DONE WITHIN 120 MINUTES OF RESTARTING THE HEART (ONLY REQUIRED FOR 120 SUBJECTS)
- 3.27 OTHER PROCEDURE DEVIATION

#### DISCHARGE

- 4.01 DISCHARGE OR 10-DAY ECHOCARDIOGRAM NOT DONE
- 4.02 DISCHARGE OR 10-DAY ECHOCARDIOGRAM DONE > 10 DAYS POST IMPLANT DATE
- 4.03 DISCHARGE PHYSICAL ASSESSMENT / VITAL SIGNS NOT DONE
- 4.04 DISCHARGE ELECTROCARDIOGRAM NOT DONE
- 4.05 DISCHARGE COAGULATION PROFILE NOT DONE
- 4.07 DISCHARGE MEDICATIONS NOT ASSESSED
- 4.09 DISCHARGE HOSPITALIZATION TIMES NOT COLLECTED
- 4.08 OTHER DISCHARGE DEVIATION

#### 1 MONTH

- 5.01 1 MONTH- SUBJECT NOT CONTACTED
- 5.01 1 MONTH- MISSED VISIT- SUBJECT CONTACTED
- 5.02 1 MONTH- ASSESSMENT NOT DONE WITHIN FOLLOW-UP WINDOW
- 5.03 1 MONTH NYHA NOT DONE
- 5.04 1 MONTH MEDICATIONS NOT ASSESSED
- 5.05 1 MONTH OTHER DEVIATION

#### 3 MONTH

- 6.01 3 MONTH SUBJECT NOT CONTACTED
- 6.01 3 MONTH MISSED VISIT- SUBJECT CONTACTED
- 6.02 3 MONTH ASSESSMENT NOT DONE WITHIN FOLLOW-UP WINDOW
- 6.03 3 MONTH PHYSICAL ASSESSMENT / VITAL SIGNS NOT DONE
- 6.04 3 MONTH NYHA NOT DONE
- 3.05 3 MONTH ELECTROCARDIOGRAM NOT DONE
- 6.06 3 MONTH ELECTROCARDIOGRAM NOT DONE WITHIN FOLLOW-UP WINDOW
- 6.07 3 MONTH ECHOCARDIOGRAM NOT DONE
- 6.08 3 MONTH ECHOCARDIOGRAM NOT DONE WITHIN FOLLOW-UP WINDOW
- 6.09 3 MONTH BLOOD NOT DONE
- 6.10 3 MONTH BLOOD INCOMPLETE
- 6.11 3 MONTH COAGULATION PROFILE NOT DONE
- 6.12 3 MONTH BLOOD NOT DONE WITHIN FOLLOW-UP WINDOW
- 6.13 3 MONTH MEDICATIONS NOT ASSESSED
- 6.14 3 MONTH MEDICATIONS NOT ASSESSED WITHIN FOLLOW-UP WINDOW
- 6.15 3 MONTH OTHER DEVIATION

Clinical Investigational Plan Protocol Number: 2012-02

#### 1 YEAR

- 8.01 1 YEAR SUBJECT NOT CONTACTED
- 8.01 1 YEAR MISSED VISIT- SUBJECT CONTACTED
- 8.02 1 YEAR ASSESSMENT NOT DONE WITHIN FOLLOW-UP WINDOW
- 8.03 1 YEAR PHYSICAL ASSESSMENT / VITAL SIGNS NOT DONE
- 8.04 1 YEAR NYHA NOT DONE
- 8.05 1 YEAR ELECTROCARDIOGRAM NOT DONE
- 8.06 1 YEAR ELECTROCARDIOGRAM NOT DONE WITHIN FOLLOW-UP WINDOW
- 8.07 1 YEAR ECHOCARDIOGRAM NOT DONE
- 8.08 1 YEAR ECHOCARDIOGRAM NOT DONE WITHIN FOLLOW-UP WINDOW
- 8.09 1 YEAR BLOOD NOT DONE
- 8.10 1 YEAR BLOOD INCOMPLETE
- 8.11 1 YEAR COAGULATION PROFILE NOT DONE
- 8.12 1 YEAR BLOOD NOT DONE WITHIN FOLLOW-UP WINDOW
- 8.13 1 YEAR MEDICATIONS NOT ASSESSED
- 8.14 1 YEAR MEDICATIONS NOT ASSESSED WITHIN FOLLOW-UP WINDOW
- 8.16 1 YEAR- QUALITY OF LIFE NOT DONE
- 8.15 1 YEAR OTHER DEVIATION

#### 2 YEAR

- 9.01 2 YEAR SUBJECT NOT CONTACTED
- 9.01 2 YEAR -MISSED VISIT- SUBJECT CONTACTED
- 9.02 2 YEAR ASSESSMENT NOT DONE WITHIN FOLLOW-UP WINDOW
- 9.03 2 YEAR PHYSICAL ASSESSMENT / VITAL SIGNS NOT DONE
- 9.04 2 YEAR NYHA NOT DONE
- 9.05 2 YEAR ELECTROCARDIOGRAM NOT DONE
- 9.06 2 YEAR ELECTROCARDIOGRAM NOT DONE WITHIN FOLLOW-UP WINDOW
- 9.07 2 YEAR ECHOCARDIOGRAM NOT DONE
- 9.08 2 YEAR ECHOCARDIOGRAM NOT DONE WITHIN FOLLOW-UP WINDOW
- 9.09 2 YEAR BLOOD NOT DONE
- 9.10 2 YEAR BLOOD INCOMPLETE
- 9.11 2 YEAR COAGULATION PROFILE NOT DONE
- 9.12 2 YEAR- BLOOD NOT DONE WITHIN FOLLOW-UP WINDOW
- 9.13 2 YEAR MEDICATIONS NOT ASSESSED
- 9.14 2 YEAR MEDICATIONS NOT ASSESSED WITHIN FOLLOW-UP WINDOW
- 9.15 2 YEAR OTHER DEVIATION

Clinical Investigational Plan Protocol Number: 2012-02

#### 3 YEAR

- 10.01 3 YEAR SUBJECT NOT CONTACTED
- 10.01 3 YEAR MISSED VISIT- SUBJECT CONTACTED
- 10.02 3 YEAR ASSESSMENT NOT DONE WITHIN FOLLOW-UP WINDOW
- 10.03 3 YEAR PHYSICAL ASSESSMENT / VITAL SIGNS NOT DONE
- 10.04 3 YEAR NYHA NOT DONE
- 10.05 3 YEAR ELECTROCARDIOGRAM NOT DONE
- 10.06 3 YEAR ELECTROCARDIOGRAM NOT DONE WITHIN FOLLOW-UP WINDOW
- 10.07 3 YEAR ECHOCARDIOGRAM NOT DONE
- 10.08 3 YEAR ECHOCARDIOGRAM NOT DONE WITHIN FOLLOW-UP WINDOW
- 10.09 3 YEAR BLOOD NOT DONE
- 10.10 3 YEAR BLOOD INCOMPLETE
- 10.11 3 YEAR COAGULATION PROFILE NOT DONE
- 10.12 3 YEAR BLOOD NOT DONE WITHIN FOLLOW-UP WINDOW
- 10.13 3 YEAR MEDICATIONS NOT ASSESSED
- 10.14 3 YEAR MEDICATIONS NOT ASSESSED WITHIN FOLLOW-UP WINDOW
- 10.15 3 YEAR OTHER DEVIATION

#### 4 YEAR

- 11.01 4 YEAR SUBJECT NOT CONTACTED
- 11.01 4 YEAR MISSED VISIT- SUBJECT CONTACTED
- 11.02 4 YEAR ASSESSMENT NOT DONE WITHIN FOLLOW-UP WINDOW
- 11.03 4 YEAR PHYSICAL ASSESSMENT / VITAL SIGNS NOT DONE
- 11.04 4 YEAR NYHA NOT DONE
- 11.05 4 YEAR ELECTROCARDIOGRAM NOT DONE
- 11.06 4 YEAR ELECTROCARDIOGRAM NOT DONE WITHIN FOLLOW-UP WINDOW
- 11.07 4 YEAR ECHOCARDIOGRAM NOT DONE
- 11.08 4 YEAR ECHOCARDIOGRAM NOT DONE WITHIN FOLLOW-UP WINDOW
- 11.09 4 YEAR BLOOD NOT DONE
- 11.10 4 YEAR BLOOD INCOMPLETE
- 11.11 4 YEAR COAGULATION PROFILE NOT DONE
- 11.12 4 YEAR BLOOD NOT DONE WITHIN FOLLOW-UP WINDOW
- 11.13 4 YEAR MEDICATIONS NOT ASSESSED
- 11.14 4 YEAR MEDICATIONS NOT ASSESSED WITHIN FOLLOW-UP WINDOW
- 11.15 4 YEAR OTHER DEVIATION

Clinical Investigational Plan Protocol Number: 2012-02

#### 5 YEAR

- 12.01 5 YEAR SUBJECT NOT CONTACTED
- 12.01 5 YEAR MISSED VISIT SUBJECT CONTACTED
- 12.02 5 YEAR ASSESSMENT NOT DONE WITHIN FOLLOW-UP WINDOW
- 12.03 5 YEAR PHYSICAL ASSESSMENT / VITAL SIGNS NOT DONE
- 12.04 5 YEAR NYHA NOT DONE
- 12.05 5 YEAR ELECTROCARDIOGRAM NOT DONE
- 12.06 5 YEAR ELECTROCARDIOGRAM NOT DONE WITHIN FOLLOW-UP WINDOW
- 12.07 5 YEAR ECHOCARDIOGRAM NOT DONE
- 12.08 5 YEAR ECHOCARDIOGRAM NOT DONE WITHIN FOLLOW-UP WINDOW
- 12.09 5 YEAR BLOOD NOT DONE
- 12.10 5 YEAR BLOOD INCOMPLETE
- 12.11 5 YEAR COAGULATION PROFILE NOT DONE
- 12.12 5 YEAR BLOOD NOT DONE WITHIN FOLLOW-UP WINDOW
- 12.13 5 YEAR MEDICATIONS NOT ASSESSED
- 12.14 5 YEAR MEDICATIONS NOT ASSESSED WITHIN FOLLOW-UP WINDOW
- 12.15 5 YEAR OTHER DEVIATION

#### 6 year

- 16.01 6 YR SUBJECT NOT CONTACTED
- 16.01 6 YR MISSED VISIT SUBJECT CONTACTED
- 16.02 6 YR ASSESSMENT NOT DONE WITHIN FOLLOW-UP WINDOW
- 16.03 6 YR PHYSICAL ASSESSMENT / VITAL SIGNS NOT DONE
- 16.04 6 YR NYHA NOT DONE
- 16.05 6 YR ELECTROCARDIOGRAM NOT DONE
- 16.06 6 YR ELECTROCARDIOGRAM NOT DONE WITHIN FOLLOW-UP WINDOW
- 16.07 6 YR ECHOCARDIOGRAM NOT DONE
- 16.08 6 YR ECHOCARDIOGRAM NOT DONE WITHIN FOLLOW-UP WINDOW
- 16.09 6 YR BLOOD NOT DONE
- 16.10 6 YR BLOOD INCOMPLETE
- 16.11 6 YR COAGULATION PROFILE NOT DONE
- 16.12 6 YR BLOOD NOT DONE WITHIN FOLLOW-UP WINDOW
- 16.13 6 YR MEDICATIONS NOT ASSESSED
- 16.14 6 YR MEDICATIONS NOT ASSESSED WITHIN FOLLOW-UP WINDOW
- 16.15 6 YR OTHER DEVIATION

Clinical Investigational Plan Protocol Number: 2012-02

#### 7 year

- 17.01 7 YR SUBJECT NOT CONTACTED
- 17.01 7 YR MISSED VISIT SUBJECT CONTACTED
- 17.02 7 YR ASSESSMENT NOT DONE WITHIN FOLLOW-UP WINDOW
- 17.03 7 YR PHYSICAL ASSESSMENT / VITAL SIGNS NOT DONE
- 17.04 7 YR NYHA NOT DONE
- 17.05 7 YR ELECTROCARDIOGRAM NOT DONE
- 17.06 7 YR ELECTROCARDIOGRAM NOT DONE WITHIN FOLLOW-UP WINDOW
- 17.07 7 YR ECHOCARDIOGRAM NOT DONE
- 17.08 7 YR ECHOCARDIOGRAM NOT DONE WITHIN FOLLOW-UP WINDOW
- 17.09 7 YR BLOOD NOT DONE
- 17.10 7 YR BLOOD INCOMPLETE
- 17.11 7 YR COAGULATION PROFILE NOT DONE
- 17.12 7 YR BLOOD NOT DONE WITHIN FOLLOW-UP WINDOW
- 17.13 7 YR MEDICATIONS NOT ASSESSED
- 17.14 7 YR MEDICATIONS NOT ASSESSED WITHIN FOLLOW-UP WINDOW
- 17.15 7 YR OTHER DEVIATION

#### 8 year

- 18.01 8 YR SUBJECT NOT CONTACTED
- 18.01 8 YR MISSED VISIT SUBJECT CONTACTED
- 18.02 8 YR ASSESSMENT NOT DONE WITHIN FOLLOW-UP WINDOW
- 18.03 8 YR PHYSICAL ASSESSMENT / VITAL SIGNS NOT DONE
- 18.04 8 YR NYHA NOT DONE
- 18.05 8 YR ELECTROCARDIOGRAM NOT DONE
- 18.06 8 YR ELECTROCARDIOGRAM NOT DONE WITHIN FOLLOW-UP WINDOW
- 18.07 8 YR ECHOCARDIOGRAM NOT DONE
- 18.08 8 YR ECHOCARDIOGRAM NOT DONE WITHIN FOLLOW-UP WINDOW
- 18.09 8 YR BLOOD NOT DONE
- 18.10 8 YR BLOOD INCOMPLETE
- 18.11 8 YR COAGULATION PROFILE NOT DONE
- 18.12 8 YR BLOOD NOT DONE WITHIN FOLLOW-UP WINDOW
- 18.13 8 YR MEDICATIONS NOT ASSESSED
- 18.14 8 YR MEDICATIONS NOT ASSESSED WITHIN FOLLOW-UP WINDOW
- 18.15 8 YR OTHER DEVIATION

Clinical Investigational Plan Protocol Number: 2012-02

#### 9 year

- 19.01 9 YR SUBJECT NOT CONTACTED
- 19.01 9 YR MISSED VISIT SUBJECT CONTACTED
- 19.02 9 YR ASSESSMENT NOT DONE WITHIN FOLLOW-UP WINDOW
- 19.03 9 YR PHYSICAL ASSESSMENT / VITAL SIGNS NOT DONE
- 19.04 9 YR NYHA NOT DONE
- 19.05 9 YR ELECTROCARDIOGRAM NOT DONE
- 19.06 9 YR ELECTROCARDIOGRAM NOT DONE WITHIN FOLLOW-UP WINDOW
- 19.07 9 YR ECHOCARDIOGRAM NOT DONE
- 19.08 9 YR ECHOCARDIOGRAM NOT DONE WITHIN FOLLOW-UP WINDOW
- 19.09 9 YR BLOOD NOT DONE
- 19.10 9 YR BLOOD INCOMPLETE
- 19.11 9 YR COAGULATION PROFILE NOT DONE
- 19.12 9 YR BLOOD NOT DONE WITHIN FOLLOW-UP WINDOW
- 19.13 9 YR MEDICATIONS NOT ASSESSED
- 19.14 9 YR MEDICATIONS NOT ASSESSED WITHIN FOLLOW-UP WINDOW
- 19.15 9 YR OTHER DEVIATION

#### 10 year

- 20.01 10 YR SUBJECT NOT CONTACTED
- 20.01 10 YR MISSED VISIT SUBJECT CONTACTED
- 20.02 10 YR ASSESSMENT NOT DONE WITHIN FOLLOW-UP WINDOW
- 20.03 10 YR PHYSICAL ASSESSMENT / VITAL SIGNS NOT DONE
- 20.04 10 YR NYHA NOT DONE
- 20.05 10 YR ELECTROCARDIOGRAM NOT DONE
- 20.06 10 YR ELECTROCARDIOGRAM NOT DONE WITHIN FOLLOW-UP WINDOW
- 20.07 10 YR ECHOCARDIOGRAM NOT DONE
- 20.08 10 YR ECHOCARDIOGRAM NOT DONE WITHIN FOLLOW-UP WINDOW
- 20.09 10 YR BLOOD NOT DONE
- 20.10 10 YR BLOOD INCOMPLETE
- 20.11 10 YR COAGULATION PROFILE NOT DONE
- 20.12 10 YR BLOOD NOT DONE WITHIN FOLLOW-UP WINDOW
- 20.13 10 YR MEDICATIONS NOT ASSESSED
- 20.14 10 YR MEDICATIONS NOT ASSESSED WITHIN FOLLOW-UP WINDOW
- 20.15 10 YR OTHER DEVIATION

#### Adverse Event

- 14.01 UADE NOT REPORTED WITHIN 10 WORKING DAYS OF THE INVESTIGATOR AWARENESS DATE
- 14.02 OTHER ADVERSE EVENT DEVIATION

#### Miscellaneous

- 15.01 STUDY DEVICE USED IN A SUBJECT NOT ENROLLED IN THE STUDY
- 15.02 OTHER DEVIATION

**EDWARDS LIFESCIENCES LLC**CLINICAL INVESTIGATIONAL PLAN

## **ATTACHMENT M – DEVICE DEFICIENCY CODES**

REVISION J: 03 MARCH 2021

Clinical Investigational Plan Protocol Number: 2012-02

### **DEVICE DEFICIENCY CODES**

| Code | Label |
|---|---|
| DD.2 | Valve / Holder |
| DD.2.01 | Device function, packaging not intact |
| DD.2.02 | Device function, component contamination |
| DD.2.03 | Device function, unable to remove from jar |
| DD.2.04 | Device function, unable to place sutures through sewing ring |
| DD.2.05 | Device function, unable to position on the annulus |
| DD.2.06 | Device function, bioprosthesis and holder separate during procedure |
| DD.2.07 | Device function, other, specify |
| DD.2.08 | Device use, sizing technique |
| DD.2.09 | Device use, sterility compromised |
| DD.2.10 | Device use, used expired product |
| DD.2.11 | Device use, component damaged by operator |
| DD.2.12 | Device use, improper positioning |
| DD.2.13 | Device use, other specify |

EDWARDS LIFESCIENCES LLC
CLINICAL INVESTIGATIONAL PLAN


## **ATTACHMENT N – CLINICAL TRIAL AGREEMENT**

No Longer In Use

REVISION J: 03 MARCH 2021

# ATTACHMENT O – POWER SIMULATION CODE FOR PRIMARY SAFETY ENDPOINT

No Longer In Use